Replication of the EINSTEIN PE Anticoagulant Trial in

**Healthcare Claims Data** 

NCT04879407

**September 14, 2021** 

#### 1. RCT Details

This section provides a high-level overview of a **published** RCT that the described real-world evidence study is trying to replicate as closely as possible given the remaining limitations inherent in the healthcare databases.

#### 1.1 Title

Oral Rivaroxaban for the Treatment of Symptomatic Venous Thromboembolism (EINSTEIN PE)

#### 1.2 Intended aim(s)

To compare the risk of symptomatic, recurrent venous thromboembolism (VTE) in patients with acute, symptomatic pulmonary embolism (PE) with or without deep vein thrombosis for rivaroxaban versus standard therapy of warfarin.

#### 1.3 Primary endpoint for replication

The primary outcome of the study was symptomatic, recurrent VTE

#### 1.4 Required power for primary endpoint and noninferiority margin (if applicable)

Assuming a noninferiority margin of 2.0, it was determined that about 3,000 patients would be needed to achieve 90% power to conclude noninferiority of rivaroxaban over standard therapy at two-sided alpha of 0.05.

#### 1.5 Secondary endpoint for replication (assay sensitivity) and RCT finding

Major bleeding; RR = 0.90 (95% CI 0.76–1.07)

#### 1.6 Trial estimate

RR = 1.12 (95% CI 0.75-1.58) comparing rivaroxaban vs standard therapy (Agnelli et al., 2012)

### 2. Person responsible for implementation of replication in Aetion

Dureshahwar Jawaid, MPH implemented the study design in the Aetion Evidence Platform. She is not responsible for the validity of the design and analytic choices. All implementation steps are recorded and the implementation history is archived in the platform.

#### 3. Data Source(s)

Optum, MarketScan, Medicare

### 4. Study Design Diagram

The study design diagram visualizes key aspects of the longitudinal study design for expedited review.

Figure 1



#### 5. Cohort Identification

#### 5.1 Cohort Summary

This study will involve a new user, parallel group, propensity score-matched, retrospective cohort study design comparing rivaroxaban to warfarin users. The patients will be required to have continuous enrollment during a baseline period of 180 days before initiation of rivaroxaban or warfarin (index date). We will restrict the analyses to patients with a diagnosis of PE.

### 5.2 <u>Important steps for cohort formation</u>

New use of rivaroxaban, exposure, and warfarin, comparator, is defined as no use of either therapy in 180 days prior to index date.

#### 5.2.1 Eligible cohort entry dates

Market availability of rivaroxaban in the U.S. prevention of venous thromboembolism after orthopedic surgery started on July 01, 2011

- For Medicare: July 01, 2011– December 31, 2017 (end of available data)
- For Marketscan: July 01, 2011 December 31, 2018 (end of available data)
- For Optum: July 01, 2011 March 31, 2020 (end of available data)

### 5.2.2 Specify <u>inclusion/exclusion</u> criteria for cohort entry and define the index date.

Inclusion and exclusion criteria were adapted from the trial as closely as possible. Definitions for all inclusion/exclusion are provided in **Appendix A** and are summarized in the flowcharts below.

#### 5.3 Flowchart of the study cohort assembly

| | Optum | | Truven | | Medicare | |
|---|---|---|---|---|---|---|
| | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients |
| All patients | | 78,202,636 | | 200,203,908 | | 6,886,908 |
| Did not meet cohort entry criteria | -77,207,180 | 995,456 | -<br>199,008,369 | 1,195,539 | -1,964,276 | 4,922,632 |

| Excluded due to insufficient enrollment | -127,407 | 868,049 | -98,795 | 1,096,744 | -1,580,438 | 3,342,194 |
|---|---|---|---|---|---|---|
| Excluded due to prior use of referent | -508,219 | 359,830 | -676,683 | 420,061 | -2,158,638 | 1,183,556 |
| Excluded due to prior use of exposure and because patient qualified in >1 exposure category | -216,850 | 142,980 | -210,419 | 209,642 | -680,443 | 503,113 |
| Excluded based on Age < 65 (Medicare only) | - | - | - | - | -55358 | 447,755 |
| Excluded based on Age, Gender, and Use of other NOACs (dabigatran, apixaban, edoxaban) | -5393 | 137,587 | -4262 | 205,380 | -17641 | 430,114 |
| Excluded based on Inclusion 1 - Pulmonary embolism | -117,221 | 20,366 | -169,963 | 35,417 | -372,047 | 58,067 |
| Excluded based on Exclusion 1 - Age and Exclusion 2 - Thrombectomy or insertion of a caval filter | -196 | 20,170 | -274 | 35,143 | -546 | 57,521 |
| Excluded based on Exclusion 3 - Other Indications for VKA | -1836 | 18,334 | -1,617 | 33,526 | -6,213 | 51,308 |
| Excluded based on Exclusion 6 - KD stage 4/5/ESRD | -56 | 18,278 | -42 | 33,484 | -136 | 51,172 |
| Excluded based on Exclusion 7 - Significant liver disease | -426 | 17,852 | -505 | 32,979 | -900 | 50,272 |
| Excluded based on Exclusion 8 - Bacterial endocarditis and Exclusion 9 - CCI >= 10 | -154 | 17,698 | -114 | 32,865 | -398 | 49,874 |
| Excluded based on Exclusion 10 - Active bleeding or high risk for bleeding | -262 | 17,436 | -334 | 32,531 | -670 | 49,204 |
| Excluded based on Exclusion 11 - malignant hypertension | -33 | 17,403 | -42 | 32,489 | -57 | 49,147 |
| Excluded based on Exclusion 12 - Pregnancy and Exclusion 14 - strong CYP3A4 inhibitors or strong CYP3A4 inducers | -19 | 17,384 | -44 | 32,445 | -29 | 49,118 |
| Final cohort | | 17,384 | | 32,445 | | 49,118 |

### 6. Variables

## 6.1 Exposure-related variables:

### Study drug:

The study exposure of interest is initiation of rivaroxaban. New initiation will be defined by no use of rivaroxaban or warfarin in the prior 6 months before treatment initiation (washout period).

# **Comparator:**

Effectiveness research with Real World Data to support FDA's regulatory decision making

New initiators of warfarin, defined by no use of rivaroxaban or warfarin in the prior 6 months.

#### 6.2 Covariates:

- Age
- Sex
- Combined Comorbidity Index (CCI), measured over the baseline covariate assessment period, defined as 180 days prior to and including index date

Covariates listed above represent only a small subset of covariates that will ultimately be controlled for in the design and analysis. We use the covariates above only for initial feasibility analyses to judge whether there is likely to be sufficient overlap between treatment groups to proceed with the study. Remaining covariates are defined only after the study has passed the initial feasibility analysis and the initial power assessment and are listed in Table 1 (Appendix B).

### 6.3 Outcome variables and study follow-up:

#### 6.3.1 Outcome variables

Primary Effectiveness outcomes of interest: (definitions provided in **Appendix A**):

• Primary Outcome: VTE

Safety outcomes of interest:

1. Major bleeding

#### 6.3.2 Study follow-up

Both as-treated (AT) and intention-to-treat (ITT) analyses will be conducted with treatment defined as the index drug on the day of cohort entry. Because adherence in the real-world databases is expected to be much worse than in the trial, the AT analysis is the **primary** analysis, as it targets the relative hazard of outcomes on treatment.

For the AT analyses, the follow-up will start the day after initiation of rivaroxaban and comparator and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest, unless otherwise specified for selected outcomes,
- The date of end of continuous registration in the database,
- End of the study period,
- Measured death event occurs,
- Nursing home admission
  - Nursing home admissions are considered a censoring event because the data sources utilized typically provide little to no data on a patient, particularly on drug utilization, after admission. We will utilize this as an exclusion reason for cohorts for the same reason.
- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug
  (rivaroxaban and comparator) plus a defined grace period (i.e., 10 days after the end of the last prescription's days' supply in
  main analyses).
- The date of augmentation or switching from exposure to comparator or vice versa or augmentation/switching to any other NOAC (e.g. switching from rivaroxaban to apixaban would be a censoring event);
  - o A dosage change on the index treatment does not fulfill this criterion
  - o An added treatment that is not part of the exposure or comparator group does not fulfill this criterion

For the intention-to-treat (ITT) analyses, the censoring based on the augmentation/switching and treatment discontinuation will be replaced with a maximum allowed follow-up time of 365 days.

### 7. Initial Feasibility Analysis

#### Aetion report name:

Optum- https://bwh-dope.aetion.com/projects/details/1527/rwrs/66276

MarketScan- https://bwh-dope.aetion.com/projects/details/1653/rwrs/66277

Medicare- <a href="https://bwh-dope.aetion.com/projects/details/1525/rwrs/67892">https://bwh-dope.aetion.com/projects/details/1525/rwrs/67892</a>

Date conducted: 02/24/2021

Complete Aetion feasibility analysis using age, sex, and CCI as the only covariates and the primary endpoint (Section 6.3.1) as the outcome. No measures of association will be computed nor will incidence rates stratified by treatment group.

## • Report patient characteristics by treatment group

| Optum | | | Truven | | | Medicare | | | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | Reference-<br>warfarin | Exposure - rivaroxaban | Difference | Reference-<br>warfarin | Exposure - rivaroxaban | Difference | Reference-<br>warfarin | Exposure - rivaroxaban | Difference |
| Number of patients | 10,916 | 6,439 | - (-, -) | 22,999 | 9,389 | - (-, -) | 32,895 | 16,223 | - (-, -) |
| Age | | | | | | | | | |
| mean (sd) | 62.06<br>(15.66) | 60.27<br>(15.41) | 1.79 (1.31,<br>2.27) | 55.59<br>(15.02) | 53.62<br>(14.45) | 1.98 (1.63,<br>2.33) | 75.46<br>(7.25) | 74.46 (6.75) | 1.00 (0.87,<br>1.13) |
| median [IQR] | 65.00<br>[51.00,<br>74.00] | 62.00<br>[50.00,<br>72.00] | - (-, -) | 56.00<br>[46.00,<br>64.00] | 54.00<br>[44.00,<br>63.00] | - (-, -) | 74.00<br>[69.00,<br>80.00] | 73.00<br>[69.00,<br>79.00] | - (-, -) |
| Gender without unknown | | | | | | | | | |
| Male; n (%) | 4,950<br>(45.3%) | 3,030<br>(47.1%) | -1.7% (-<br>3.3%, -<br>0.2%) | 11,058<br>(48.1%) | 4,685<br>(49.9%) | -1.8% (-<br>3.0%, -<br>0.6%) | 12,293<br>(37.4%) | 6,712<br>(41.4%) | -4.0% (-<br>4.9%, -<br>3.1%) |
| Female; n (%) | 5,965<br>(54.6%) | 3,408<br>(52.9%) | 1.7%<br>(0.2%,<br>3.3%) | 11,941<br>(51.9%) | 4,704<br>(50.1%) | 1.8%<br>(0.6%,<br>3.0%) | 20,602<br>(62.6%) | 9,511<br>(58.6%) | 4.0%<br>(3.1%,<br>4.9%) |
| CCI (180 days)- ICD9 and ICD10 v2 | | | | | | | | | |
| mean (sd) | 3.04 (2.20) | 3.21 (2.00) | -0.18 (-<br>0.24, -0.11) | 2.11 (1.91) | 2.43 (1.82) | -0.32 (-<br>0.36, -<br>0.28) | 6.33 (3.30) | 6.24 (3.08) | 0.09 (0.03,<br>0.15) |
| median [IQR] | 3.00 [1.00,<br>4.00] | 3.00 [2.00,<br>4.00] | - (-, -) | 2.00 [1.00,<br>3.00] | 2.00 [1.00,<br>3.00] | - (-, -) | 6.00 [4.00,<br>8.00] | 6.00 [4.00,<br>8.00] | - (-, -) |

• Report summary parameters of study population **FEASIBILITY- FOR STUDY OUTCOME** 

| FEASIBILITY- FOR STUDY OUTCOME | | | |
|---|---|---|---|
| | Optum | Truven | Medicare |
| Variable | Value | Value | Value |
| Number of patients in full cohort | 17,384 | 32,445 | 49,118 |
| Number of patients dropped as incomplete cases | 0 | 0 | 0 |
| Number of patients that did not begin follow-up | 29 | 57 | 77 |
| Number of patients in analytic cohort | 17,355 | 32,388 | 49,041 |
| Number of events | 232 | 482 | 669 |
| Number of person-years | 6,152.63 | 12,258.57 | 20,258.62 |
| Number of patients in group: Reference- warfarin | 10,916 | 22,999 | 32,848 |
| Number of patients in group: Exposure - rivaroxaban | 6,439 | 9,389 | 16,193 |
| Risk per 1,000 patients | 13.37 | 14.88 | 13.64 |
| Rate per 1,000 person-years | 37.71 | 39.32 | 33.02 |

• Report median follow-up time by treatment group

| MEDIAN FOLLOW-UP TIME FOR STUDY OUTCOME | | | |
|-----------------------------------------|-------|--------|----------|
| Median Follow-Up Time (Days) [IQR] | | | |
| | Optum | Truven | Medicare |

| Patient Group | Median Follow-Up<br>Time (Days) [IQR] | Median Follow-Up<br>Time (Days) [IQR] | Median Follow-Up<br>Time (Days) [IQR] |
|---|---|---|---|
| <b>Overall Patient Population</b> | 76 [38, 174] | 93 [38, 183] | 98 [38, 196] |
| Referent | 82 [38, 177] | 96 [43, 184] | 103 [43, 201] |
| Exposure | 65 [38, 171] | 84 [38, 180] | 82 [38, 185] |

#### • Report reasons for censoring in the overall study population

| CENSORING REASONS FOR STUDY OUTCOME | | | |
|---|---|---|---|
| | Optum | Truven | Medicare |
| Outcome | 232 (1.3%) | 482 (1.5%) | 669 (1.4%) |
| Death | 118 (0.7%) | 63 (0.2%) | 1,199 (2.4%) |
| Start of an additional exposure | 606 (3.5%) | 1,277 (3.9%) | 2,077 (4.2%) |
| End of index exposure | 12,371<br>(71.3%) | 25,197<br>(77.8%) | 37,423<br>(76.3%) |
| Specified date reached | 476 (2.7%) | 709 (2.2%) | 3,194 (6.5%) |
| End of patient data | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) |
| End of patient enrollment | 1,340 (7.7%) | 4,035<br>(12.5%) | 833 (1.7%) |
| Censoring - Switch to other NOAC + nursing home Occurred | 2,212<br>(12.7%) | 625 (1.9%) | 3,646 (7.4%) |

### • Report overall risk of the primary outcome.

| | Optum | Marketscan | Medicare | Pooled |
|-------------------------|-------|------------|----------|--------|
| Risk per 1,000 patients | 13.37 | 14.88 | 13.64 | 13.98 |

#### 8. Initial Power Assessment

Aetion report name:

For rivaroxaban vs. warfarin

Optum- https://bwh-dope.aetion.com/projects/details/1527/rwrs/66281

MarketScan- https://bwh-dope.aetion.com/projects/details/1653/rwrs/66280

Mediare- https://bwh-dope.aetion.com/projects/details/1525/rwrs/67893

Date conducted: 02/24/2021

In order to complete the initial power analysis, the dummy outcome of a 90-day gap in database enrollment will be used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. Complete a 1:1 PS-matched comparative analysis using this outcome. PS should include only 2 covariates: age and combined comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

• Stop analyses until feasibility and power are reviewed by primary investigators and FDA. Reviewers evaluate the results of the analyses described above in Sections 7 and 8, including numbers of patients, patient characteristics, follow-up time, and reasons for censoring by treatment group, as well as overall rates of outcomes and study power. These parameters are re-evaluated and reported in the subsequent sections, after incorporating feedback and refining the protocol.

Pooled

| Non-inferiority Analysis | |
|----------------------------|-----------|
| Number of patients matched | 64,038 |
| Reference | 32,019 |
| Exposed | 32,019 |
| Risk per 1,000 patients | 13.98 |
| Assumed HR from RCT | 1.12 |
| Alpha (2-sided) | 0.05 |
| Non-inferiority margin | 2 |
| Number of events expected | 895.25124 |
| Power | 1 |

## o Optum

| Non-inferiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | 12,876 |
| Reference | 6,438 |
| Exposed | 6,438 |
| Risk per 1,000 patients | 13.37 |
| Assumed HR from RCT | 1.12 |
| Alpha (2-sided) | 0.05 |
| Non-inferiority margin | 2 |
| Number of events expected | 172.15212 |
| Power | 0.967396851 |

o MarketScan

| Non-inferiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | 18,776 |
| Reference | 9,388 |
| Exposed | 9,388 |
| Risk per 1,000 patients | 14.88 |
| Assumed HR from RCT | 1.12 |
| Alpha (2-sided) | 0.05 |
| Non-inferiority margin | 2 |
| Number of events expected | 279.38688 |
| Power | 0.998048094 |

### Medicare

| Non-inferiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | 32,386 |
| Reference | 16,193 |
| Exposed | 16,193 |
| Risk per 1,000 patients | 13.64 |
| Assumed HR from RCT | 1.12 |
| Alpha (2-sided) | 0.05 |
| Non-inferiority margin | 2 |
| Number of events expected | 441.74504 |
| Power | 0.999982118 |

Effectiveness research with Real World Data to support FDA's regulatory decision making

• Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Date revie | ewed: |
|-------------------------|------------|-------|
| Reviewed by FDA: | Date revie | ewed: |
| Reasons for stopping | | |
| analysis (if required): | | |

#### 9. Balance Assessment

#### **Aetion report links:**

Optum: https://bwh-dope.aetion.com/projects/details/1527/rwrs/67705

Marketscan: https://bwh-dope.aetion.com/projects/details/1653/rwrs/67706

Medicare: https://bwh-dope.aetion.com/projects/details/1525/rwrs/67894

Date conducted: 3/28/2021

After review of initial feasibility and power analyses, complete creation of the remaining covariates from Section 6.2. Again, using the dummy outcome of a 90-day gap in database enrollment, complete a 1:1 PS-matched analysis. The PS should include the complete list of covariates.

• Provide plot of PS distributions stratified by treatment group.

Note- Please refer to Appendix B.

Report covariate balance after matching.

Note- Please refer to Appendix B.

Report reasons for censoring by treatment group.

| | Overall | Referent | Exposure |
|---|---|---|---|
| Dummy outcome | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) |
| Death | 477 (1.50%) | 218 (1.37%) | 259 (1.63%) |
| Start of an additional exposure | 1,584 (4.98%) | 1,023 (6.44 %) | 561 (3.53%) |
| End of index exposure | 23,632 (74.35%) | 11,350 (71.42%) | 12,282 (77.28%) |
| Specified date reached | 1,617 (5.09%) | 875 (5.51%) | 742 (4.67%) |
| End of patient enrollment | 2,079 (6.54%) | 1,046 (6.58%) | 1,033 (6.50%) |
| Switch to other NOACs (for censoring) + nursing home admission | 2,397 (7.54%) | 1,381 (8.69%) | 1,016 (6.39%) |

• Report follow-up time by treatment group.

| Median Follow-Up Time (Days) [IQR] | | | |
|---|---|---|---|
| Patient Group Optum Marketscan Medicare | | | |
| Overall Patient Population | 70 [36-174] | 91 [38-184] | 97 [38-195] |
| Referent | 75 [38-173] | 92 [40-178] | 100 [41-199] |
| Exposure | 65 [33-175] | 91 [38-188] | 88 [38-190] |

#### 10. Final Power Assessment

Date conducted: 03/28/2021

• Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in Section 9. All other parameters in the table should be the same as in Section 8.

## Pooled

| Non-inferiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | 32,998 |
| Reference | 16,499 |
| Exposed | 16,499 |
| Risk per 1,000 patients | 13.87 |
| Assumed HR from RCT | 1.12 |
| Alpha (2-sided) | 0.05 |
| Non-inferiority margin | 2 |
| Number of events expected | 457.68226 |
| Power | 0.999988934 |

# Optum

| Non-inferiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | 4,306 |
| Reference | 2,153 |
| Exposed | 2,153 |
| Risk per 1,000 patients | 13.37 |
| Assumed HR from RCT | 1.12 |
| Alpha (2-sided) | 0.05 |
| Non-inferiority margin | 2 |
| Number of events expected | 57.57122 |
| Power | 0.594735156 |

## Marketscan

| Non-inferiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | 11,350 |
| Reference | 5,675 |
| Exposed | 5,675 |
| Risk per 1,000 patients | 14.88 |
| Assumed HR from RCT | 1.12 |
| Alpha (2-sided) | 0.05 |
| Non-inferiority margin | 2 |
| Number of events expected | 168.888 |
| Power | 0.964666171 |

## Medicare

| Non-inferiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | 17,342 |
| Reference | 8,671 |
| Exposed | 8,671 |
| Risk per 1,000 patients | 13.46 |
| Assumed HR from RCT | 1.12 |
| Alpha (2-sided) | 0.05 |
| Non-inferiority margin | 2 |
| Number of events expected | 233.42332 |
| Power | 0.993231623 |

• Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Date reviewed: |
|-------------------------|----------------|
| Reviewed by FDA: | Date reviewed: |
| Reasons for stopping | |
| analysis (if required): | |

#### 11. Study Confidence and Concerns

<u>Deadline for voting on study confidence and listing concerns:</u> Date votes and concerns are summarized:

- If final feasibility and power analyses are reviewed and approved, proceed to the remaining protocol steps.
- All study team and advisory board members that review this protocol should at this stage provide their level of confidence for the
  success of the RWD study in the <u>Google Form</u>. This form also provides space for reviewers to list any concerns that they feel may
  contribute to a failure to replicate the findings of the RCT, including differences in study populations, poor measurement of study
  variables, or residual confounding. All responses will be kept confidential and individual-level results will only be shared with the
  individual respondent.
- After the deadline for voting has passed, provide the distribution of responses and summarize all concerns here.

#### 12. Register study protocol on clinicalTrials.gov

#### Date conducted:

• Register the study on <u>clinicalTrials.gov</u> and upload this document.

#### 13. Comparative Analyses

Aetion report name:

Date conducted:

| Effectiveness | research with | Real World | Data to | support FDA | a's regulator | v decision | making |
|---|---|---|---|---|---|---|---|
| LITECUIVETICSS | i Cocai cii witti | INCUI VVOITA | Data to | Jupportible | 13 I Chalatol | y accision | THURSTIN |

## 13.1 For primary analysis:

# 13.2 <u>For sensitivity analyses:</u>

## 14. Requested Results

# 14.1 <u>Table 1: Baseline characteristics before and after adjustment</u>

| Variable | Before adjustment | | | After adjusti | ment | |
|---|---|---|---|---|---|---|
| | Referent | ferent Exposure Std. diff. | | Referent | Exposure | Std. diff. |
| Number of patients | | | - | | | - |
| Age categories | | | | | | |

## 14.2 <u>Table 2: Follow-up time</u>

| Patient Group Median Follow-Up Time (Days) [IQR] |
|--------------------------------------------------|
| Overall Patient Population |
| Referent |
| Exposure |

# 14.3 <u>Table 3: Censoring events</u>

| Overall | Referent | Exposure |
|---------|----------|----------|
| | | 1 |

Effectiveness research with Real World Data to support FDA's regulatory decision making

| Outcome |
|---------------------------------|
| Death |
| Start of an additional exposure |
| End of index exposure |
| Specified date reached |
| End of patient data |
| End of patient enrollment |

## 14.4 <u>Table 4: Results from primary analyses;</u>

| Analysis | No. exposed events | No. referent events | Exposed rate | Referent rate | HR (95% CI) |
|---|---|---|---|---|---|
| Crude | | | | | |
| Analysis 1 | | | | | |
| Analysis 2 | | | | | |

HR, Hazard Ratio; CI, Confidence Interval.

### 14.5 <u>Table 5: Results from secondary analyses;</u>

#### 15. References

Agnelli G, Berkowitz S, Bounameaux H, et al. Oral Rivaroxaban for the Treatment of Symptomatic Venous Thromboembolism. N Engl J Med. 2012; 366:1287-97

Chow S, Shao J, Wang H. 2008. Sample Size Calculations in Clinical Research. 2nd Ed. Chapman & Hall/CRC Biostatistics Series. page 177

| | T |
|---|---|
| Trial Name (with web links) | <u>FINSTEIN PE</u> |
| <u>Trial Name (with pdf links)</u> | <u>EINSTEIN PE</u> |
| NCT_ | NCT00439777 |
| Therapeutic Area | Cardiology/Vascular Diseases |
| Study batch | NOACs |
| Brand Name | Xarelto |
| Generic Name | Rivaroxaban |
| Sponsor | Bayer |
| Sholisol | Johnson & Johnson Pharmaceutical Research & Development, L.L.C |
| <u>Year</u> | 2012 |
| | Percentage of Participants With Symptomatic Recurrent Venous Thromboembolism [VTE] (i.e. the Composite of |
| Measurable endpoint | Recurrent Deep Vein Thrombosis [DVT] or Fatal or Non-fatal Pulmonary Embolism [PE]) Until the Intended End of |
| | Study Treatment |
| <u>Exposure</u> | Rivaroxaban |
| Comparator | Enoxaparin/VKA |
| Population | Patients of legal age who had acute symptomatic pulmonary embolism with or without deep-vein thrombosis |
| Trial finding | HR = 1.12 (95% CI 0.75 to 1.68) |
| No. of Patients | 4,832 (2,419 in exposed arm) |
| Non-inferiority margin | HR = 2.0 |
| Account Company To American Michigan | Percentage of Participants With the Composite Variable Comprising Recurrent DVT, Non-fatal PE and All Cause |
| Assay Sens. Endpoint (from trial) | Mortality Until the Intended End of Study Treatment |
| Finding for potential Assay Sens. Outcome from trial- | HR = 0.85 (95% CI 0.63 to 1.14) |
| | 0.90. Assuming equal efficacy, a total of 88 events was calculated to give a power of 90% to prove that rivaroxaban is at least as |
| <u>Power</u> | effective as the comparator, considering a non-inferiority upper CI margin for the hazard ratio of 2.0 (two-sided α=0.05). A mean |
| | incidence for the primary efficacy outcome of 3% was expected and an enrollment of at least 3000 patients was necessary |

### Title

Venous Thromboembolism (VTE)

## ICD-9 Dx inpatient primary position

| ne s ox inputient primary p | |
|---|---|
| PE | DUI MONADY EMPOLICA AND INCADCTION |
| 415.1 | PULMONARY EMBOLISM AND INFARCTION |
| 415.11 | IATROGENIC PULMONARY EMBOLISM AND INFARCTION |
| 415.19 | OTHER PULMONARY EMBOLISM AND INFARCTION |
| DVT | |
| 451.1 | PHLEBITIS AND THROMBOPHLEBITIS OF DEEP VEINS OF LOWER EXTREMITIES |
| 451.11 | PHLEBITIS AND THROMBOPHLEBITIS OF FEMORAL VEIN (DEEP) (SUPERFICIAL) |
| 451.19 | PHLEBITIS AND THROMBOPHLEBITIS OF OTHER |
| 451.2 | PHLEBITIS AND THROMBOPHLEBITIS OF LOWER EXTREMITIES UNSPECIFIED |
| 451.81 | PHLEBITIS AND THROMBOPHLEBITIS OF ILIAC VEIN |
| 451.9 | PHLEBITIS AND THROMBOPHLEBITIS OF UNSPECIFIED SITE |
| 453 | BUDD-CHIARI SYNDROME |
| 453.1 | THROMBOPHLEBITIS MIGRANS |
| 453.2 | EMBOLISM AND THROMBOSIS OF INFERIOR VENA CAVA |
| 453.4 | ACUTE VENOUS EMBOLISM AND THROMBOSIS OF DEEP VESSELS OF LOWER EXTREMITY |
| 453.4 | ACUTE VENOUS EMBOLISM AND THROMBOSIS OF UNSPECIFIED DEEP VESSELS OF LOWER EXTREMITY |
| 453.41 | ACUTE VENOUS EMBOLISM AND THROMBOSIS OF DEEP VESSELS OF PROXIMAL LOWER EXTREMITY |
| 453.42 | ACUTE VENOUS EMBOLISM AND THROMBOSIS OF DEEP VESSELS OF DISTAL LOWER EXTREMITY |
| 453.5 | CHRONIC VENOUS EMBOLISM AND THROMBOSIS OF DEEP VESSELS OF LOWER EXTREMITY |
| 453.5 | CHRONIC VENOUS EMBOLISM AND THROMBOSIS OF UNSPECIFIED DEEP VESSELS OF LOWER EXTREMITY |
| 453.51 | CHRONIC VENOUS EMBOLISM AND THROMBOSIS OF DEEP VESSELS OF PROXIMAL LOWER EXTREMITY |
| 453.52 | CHRONIC VENOUS EMBOLISM AND THROMBOSIS OF DEEP VESSELS OF DISTAL LOWER EXTREMITY |
| 453.8 | ACUTE VENOUS EMBOLISM AND THROMBOSIS OF OTHER SPECIFIED VEINS |
| 453.82 | ACUTE VENOUS EMBOLISM AND THROMBOSIS OF DEEP VEINS OF UPPER EXTREMITY |
| 453.83 | ACUTE VENOUS EMBOLISM AND THROMBOSIS OF UPPER EXTREMITY UNSPECIFIED |
| 453.84 | ACUTE VENOUS EMBOLISM AND THROMBOSIS OF AXILLARY VEINS |
| 453.85 | ACUTE VENOUS EMBOLISM AND THROMBOSIS OF SUBCLAVIAN VEINS |
| 453.86 | ACUTE VENOUS EMBOLISM AND THROMBOSIS OF INTERNAL JUGULAR VEINS |
| 453.87 | ACUTE VENOUS EMBOLISM AND THROMBOSIS OF OTHER THORACIC VEINS |
| 453.89 | ACUTE VENOUS EMBOLISM AND THROMBOSIS OF OTHER SPECIFIED VEINS |

#### 453.9 EMBOLISM AND THROMBOSIS OF UNSPECIFIED SITE

## ICD-10 Dx inpatient primary position

| PE | |
|---|---|
| 126.0 | Pulmonary embolism with acute cor pulmonale |
| 126.01 | Septic pulmonary embolism with acute cor pulmonale |
| 126.02 | Saddle embolus of pulmonary artery with acute cor pulmonale |
| 126.09 | Other pulmonary embolism with acute cor pulmonale |
| 126.9 | Pulmonary embolism without acute cor pulmonale |
| 126.99 | Other pulmonary embolism without acute cor pulmonale |
| DVT | |
| 180.1 | Phlebitis and thrombophlebitis of femoral vein |
| 180.10 | Phlebitis and thrombophlebitis of unspecified femoral vein |
| 180.11 | Phlebitis and thrombophlebitis of right femoral vein |
| 180.12 | Phlebitis and thrombophlebitis of left femoral vein |
| 180.13 | Phlebitis and thrombophlebitis of femoral vein, bilateral |
| 180.2 | Phlebitis and thrombophlebitis of other and unspecified deep vessels of lower extremities |
| 180.20 | Phlebitis and thrombophlebitis of unspecified deep vessels of lower extremities |
| 180.201 | Phlebitis and thrombophlebitis of unspecified deep vessels of right lower extremity |
| 180.202 | Phlebitis and thrombophlebitis of unspecified deep vessels of left lower extremity |
| 180.203 | Phlebitis and thrombophlebitis of unspecified deep vessels of lower extremities, bilateral |
| 180.209 | Phlebitis and thrombophlebitis of unspecified deep vessels of unspecified lower extremity |
| 180.21 | Phlebitis and thrombophlebitis of iliac vein |
| 180.211 | Phlebitis and thrombophlebitis of right iliac vein |
| 180.212 | Phlebitis and thrombophlebitis of left iliac vein |
| I80.213 | Phlebitis and thrombophlebitis of iliac vein, bilateral |
| 180.219 | Phlebitis and thrombophlebitis of unspecified iliac vein |
| 180.22 | Phlebitis and thrombophlebitis of popliteal vein |
| 180.221 | Phlebitis and thrombophlebitis of right popliteal vein |
| 180.222 | Phlebitis and thrombophlebitis of left popliteal vein |
| 180.223 | Phlebitis and thrombophlebitis of popliteal vein, bilateral |
| 180.229 | Phlebitis and thrombophlebitis of unspecified popliteal vein |
| 180.23 | Phlebitis and thrombophlebitis of tibial vein |
| 180.231 | Phlebitis and thrombophlebitis of right tibial vein |

| 180.232 | Phlebitis and thrombophlebitis of left tibial vein |
|---|---|
| 180.233 | Phlebitis and thrombophlebitis of tibial vein, bilateral |
| 180.239 | Phlebitis and thrombophlebitis of unspecified tibial vein |
| 180.29 | Phlebitis and thrombophlebitis of other deep vessels of lower extremities |
| 180.291 | Phlebitis and thrombophlebitis of other deep vessels of right lower extremity |
| 180.292 | Phlebitis and thrombophlebitis of other deep vessels of left lower extremity |
| 180.293 | Phlebitis and thrombophlebitis of other deep vessels of lower extremity, bilateral |
| 180.299 | Phlebitis and thrombophlebitis of other deep vessels of unspecified lower extremity |
| 180.3 | Phlebitis and thrombophlebitis of lower extremities, unspecified |
| 180.9 | Phlebitis and thrombophlebitis of unspecified site |
| 182.0 | Budd-Chiari syndrome |
| 182.1 | Thrombophlebitis migrans |
| 180.3 | Phlebitis and thrombophlebitis of lower extremities, unspecified |
| 182.4 | Acute embolism and thrombosis of deep veins of lower extremity |
| 182.40 | Acute embolism and thrombosis of unspecified deep veins of lower extremity |
| 182.401 | Acute embolism and thrombosis of unspecified deep veins of right lower extremity |
| 182.402 | Acute embolism and thrombosis of unspecified deep veins of left lower extremity |
| 182.403 | Acute embolism and thrombosis of unspecified deep veins of lower extremity, bilateral |
| 182.409 | Acute embolism and thrombosis of unspecified deep veins of unspecified lower extremity |
| 182.41 | Acute embolism and thrombosis of femoral vein |
| 182.411 | Acute embolism and thrombosis of right femoral vein |
| 182.412 | Acute embolism and thrombosis of left femoral vein |
| 182.413 | Acute embolism and thrombosis of femoral vein, bilateral |
| 182.419 | Acute embolism and thrombosis of unspecified femoral vein |
| 182.42 | Acute embolism and thrombosis of iliac vein |
| 182.421 | Acute embolism and thrombosis of right iliac vein |
| 182.422 | Acute embolism and thrombosis of left iliac vein |
| 182.423 | Acute embolism and thrombosis of iliac vein, bilateral |
| 182.429 | Acute embolism and thrombosis of unspecified iliac vein |
| 182.43 | Acute embolism and thrombosis of popliteal vein |
| 182.431 | Acute embolism and thrombosis of right popliteal vein |
| 182.432 | Acute embolism and thrombosis of left popliteal vein |
| 182.433 | Acute embolism and thrombosis of popliteal vein, bilateral |
| 182.439 | Acute embolism and thrombosis of unspecified popliteal vein |
| 182.44 | Acute embolism and thrombosis of tibial vein |

| 182.441 | Acute embolism and thrombosis of right tibial vein |
|---|---|
| 182.442 | Acute embolism and thrombosis of left tibial vein |
| 182.443 | Acute embolism and thrombosis of tibial vein, bilateral |
| 182.449 | Acute embolism and thrombosis of unspecified tibial vein |
| 182.49 | Acute embolism and thrombosis of other specified deep vein of lower extremity |
| 182.491 | Acute embolism and thrombosis of other specified deep vein of right lower extremity |
| 182.492 | Acute embolism and thrombosis of other specified deep vein of left lower extremity |
| 182.493 | Acute embolism and thrombosis of other specified deep vein of lower extremity, bilateral |
| 182.499 | Acute embolism and thrombosis of other specified deep vein of unspecified lower extremity |
| 182.4Y | Acute embolism and thrombosis of unspecified deep veins of proximal lower extremity |
| I82.4Y1 | Acute embolism and thrombosis of unspecified deep veins of right proximal lower extremity |
| 182.4Y2 | Acute embolism and thrombosis of unspecified deep veins of left proximal lower extremity |
| I82.4Y3 | Acute embolism and thrombosis of unspecified deep veins of proximal lower extremity, bilateral |
| I82.4Y9 | Acute embolism and thrombosis of unspecified deep veins of unspecified proximal lower extremity |
| 182.4Z | Acute embolism and thrombosis of unspecified deep veins of distal lower extremity |
| 182.471 | Acute embolism and thrombosis of unspecified deep veins of right distal lower extremity |
| 182.4Z2 | Acute embolism and thrombosis of unspecified deep veins of left distal lower extremity |
| 182.4Z3 | Acute embolism and thrombosis of unspecified deep veins of distal lower extremity, bilateral |
| 182.4Z9 | Acute embolism and thrombosis of unspecified deep veins of unspecified distal lower extremity |
| 182.5 | Chronic embolism and thrombosis of deep veins of lower extremity |
| 182.50 | Chronic embolism and thrombosis of unspecified deep veins of lower extremity |
| 182.501 | Chronic embolism and thrombosis of unspecified deep veins of right lower extremity |
| 182.502 | Chronic embolism and thrombosis of unspecified deep veins of left lower extremity |
| 182.503 | Chronic embolism and thrombosis of unspecified deep veins of lower extremity, bilateral |
| 182.509 | Chronic embolism and thrombosis of unspecified deep veins of unspecified lower extremity |
| 182.51 | Chronic embolism and thrombosis of femoral vein |
| 182.511 | Chronic embolism and thrombosis of right femoral vein |
| 182.512 | Chronic embolism and thrombosis of left femoral vein |
| 182.513 | Chronic embolism and thrombosis of femoral vein, bilateral |
| 182.519 | Chronic embolism and thrombosis of unspecified femoral vein |
| 182.52 | Chronic embolism and thrombosis of iliac vein |
| 182.521 | Chronic embolism and thrombosis of right iliac vein |
| 182.522 | Chronic embolism and thrombosis of left iliac vein |
| 182.523 | Chronic embolism and thrombosis of iliac vein, bilateral |
| 182.529 | Chronic embolism and thrombosis of unspecified iliac vein |

| 182.53 | Chronic embolism and thrombosis of popliteal vein |
|---|---|
| 182.531 | Chronic embolism and thrombosis of right popliteal vein |
| 182.532 | Chronic embolism and thrombosis of left popliteal vein |
| 182.533 | Chronic embolism and thrombosis of popliteal vein, bilateral |
| 182.539 | Chronic embolism and thrombosis of unspecified popliteal vein |
| 182.54 | Chronic embolism and thrombosis of tibial vein |
| 182.541 | Chronic embolism and thrombosis of right tibial vein |
| 182.542 | Chronic embolism and thrombosis of left tibial vein |
| 182.543 | Chronic embolism and thrombosis of tibial vein, bilateral |
| 182.549 | Chronic embolism and thrombosis of unspecified tibial vein |
| 182.59 | Chronic embolism and thrombosis of other specified deep vein of lower extremity |
| 182.591 | Chronic embolism and thrombosis of other specified deep vein of right lower extremity |
| 182.592 | Chronic embolism and thrombosis of other specified deep vein of left lower extremity |
| 182.593 | Chronic embolism and thrombosis of other specified deep vein of lower extremity, bilateral |
| 182.599 | Chronic embolism and thrombosis of other specified deep vein of unspecified lower extremity |
| 182.5Y | Chronic embolism and thrombosis of unspecified deep veins of proximal lower extremity |
| 182.5Y1 | Chronic embolism and thrombosis of unspecified deep veins of right proximal lower extremity |
| 182.5Y2 | Chronic embolism and thrombosis of unspecified deep veins of left proximal lower extremity |
| 182.5Y3 | Chronic embolism and thrombosis of unspecified deep veins of proximal lower extremity, bilateral |
| 182.5Y9 | Chronic embolism and thrombosis of unspecified deep veins of unspecified proximal lower extremity |
| 182.5Z | Chronic embolism and thrombosis of unspecified deep veins of distal lower extremity |
| I82.5Z1 | Chronic embolism and thrombosis of unspecified deep veins of right distal lower extremity |
| I82.5Z2 | Chronic embolism and thrombosis of unspecified deep veins of left distal lower extremity |
| 182.5Z3 | Chronic embolism and thrombosis of unspecified deep veins of distal lower extremity, bilateral |
| I82.5Z9 | Chronic embolism and thrombosis of unspecified deep veins of unspecified distal lower extremity |
| 182.6 | Acute embolism and thrombosis of veins of upper extremity |
| 182.60 | Acute embolism and thrombosis of unspecified veins of upper extremity |
| 182.601 | Acute embolism and thrombosis of unspecified veins of right upper extremity |
| 182.602 | Acute embolism and thrombosis of unspecified veins of left upper extremity |
| 182.603 | Acute embolism and thrombosis of unspecified veins of upper extremity, bilateral |
| 182.609 | Acute embolism and thrombosis of unspecified veins of unspecified upper extremity |
| 182.62 | Acute embolism and thrombosis of deep veins of upper extremity |
| 182.621 | Acute embolism and thrombosis of deep veins of right upper extremity |
| 182.622 | Acute embolism and thrombosis of deep veins of left upper extremity |
| 182.623 | Acute embolism and thrombosis of deep veins of upper extremity, bilateral |

| Acute embolism and thrombosis of deep veins of unspecified upper extremity |
|----------------------------------------------------------------------------|
| Acute embolism and thrombosis of other specified veins |
| Acute embolism and thrombosis of unspecified vein |
| Acute embolism and thrombosis of axillary vein |
| Acute embolism and thrombosis of right axillary vein |
| Acute embolism and thrombosis of left axillary vein |
| Acute embolism and thrombosis of axillary vein, bilateral |
| Acute embolism and thrombosis of unspecified axillary vein |
| Acute embolism and thrombosis of subclavian vein |
| Acute embolism and thrombosis of right subclavian vein |
| Acute embolism and thrombosis of left subclavian vein |
| Acute embolism and thrombosis of subclavian vein, bilateral |
| Acute embolism and thrombosis of unspecified subclavian vein |
| Acute embolism and thrombosis of internal jugular vein |
| Acute embolism and thrombosis of right internal jugular vein |
| Acute embolism and thrombosis of left internal jugular vein |
| Acute embolism and thrombosis of internal jugular vein, bilateral |
| Acute embolism and thrombosis of unspecified internal jugular vein |

### Title

Major Bleeding

### ICD-9 Dx inpatient any position

| icu-9 ux inpatient any positi | on |
|---|---|
| 423 | (ICD9) HEMOPERICARDIUM |
| 430 | (ICD9) SUBARACHNOID HEMORRHAGE |
| 431 | (ICD9) INTRACEREBRAL HEMORRHAGE |
| 432 | (ICD9) NONTRAUMATIC EXTRADURAL HEMORRHAGE |
| 432.1 | (ICD9) SUBDURAL HEMORRHAGE |
| 432.9 | (ICD9) UNSPECIFIED INTRACRANIAL HEMORRHAGE |
| 459 | (ICD9) HEMORRHAGE UNSPECIFIED |
| 531 | (ICD9) ACUTE GASTRIC ULCER WITH HEMORRHAGE |
| 531 | (ICD9) ACUTE GASTRIC ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| 531.01 | (ICD9) ACUTE GASTRIC ULCER WITH HEMORRHAGE WITH OBSTRUCTION |
| 531.2 | (ICD9) ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION |
| 531.2 | (ICD9) ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| 531.21 | (ICD9) ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| 531.4 | (ICD9) CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE |
| 531.4 | (ICD9) CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| 531.41 | (ICD9) CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE WITH OBSTRUCTION |
| 531.6 | (ICD9) CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION |
| 531.6 | (ICD9) CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| 531.61 | (ICD9) CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| 532 | (ICD9) ACUTE DUODENAL ULCER WITH HEMORRHAGE |
| 532 | (ICD9) ACUTE DUODENAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| 532.01 | (ICD9) ACUTE DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION |
| 532.2 | (ICD9) ACUTE DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION |
| 532.2 | (ICD9) ACUTE DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| 532.21 | (ICD9) ACUTE DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| 532.4 | (ICD9) CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE |
| 532.4 | (ICD9) CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION |

| (ICD9) CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION |
|---|
| (ICD9) CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION |
| (ICD9) CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| (ICD9) CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| (ICD9) ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE |
| (ICD9) ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| (ICD9) ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION |
| (ICD9) ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION |
| (ICD9) ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| (ICD9) ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| (ICD9) CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE |
| (ICD9) CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| (ICD9) CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION |
| (ICD9) CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION |
| (ICD9) CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| (ICD9) CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| (ICD9) ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE |
| (ICD9) ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| (ICD9) ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION |
| (ICD9) ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION |
| (ICD9) ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| (ICD9) ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| (ICD9) CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE |

| 534.4 | |
|---|---|
| | (ICD9) CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| 534.41 | (ICD9) CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION |
| 534.6 | (ICD9) CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION |
| 534.6 | (ICD9) CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| 534.61 | (ICD9) CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| 562.02 | (ICD9) DIVERTICULOSIS OF SMALL INTESTINE WITH HEMORRHAGE |
| 562.03 | (ICD9) DIVERTICULITIS OF SMALL INTESTINE WITH HEMORRHAGE |
| 562.12 | (ICD9) DIVERTICULOSIS OF COLON WITH HEMORRHAGE |
| 562.13 | (ICD9) DIVERTICULITIS OF COLON WITH HEMORRHAGE |
| 568.81 | (ICD9) HEMOPERITONEUM (NONTRAUMATIC) |
| 569.3 | (ICD9) HEMORRHAGE OF RECTUM AND ANUS |
| 569.83 | (ICD9) PERFORATION OF INTESTINE |
| 569.85 | (ICD9) ANGIODYSPLASIA OF INTESTINE WITH HEMORRHAGE |
| 569.86 | (ICD9) DIEULAFOY LESION (HEMORRHAGIC) OF INTESTINE |
| 578 | (ICD9) HEMATEMESIS |
| 578.1 | (ICD9) BLOOD IN STOOL |
| 578.9 | (ICD9) HEMORRHAGE OF GASTROINTESTINAL TRACT UNSPECIFIED |
| 719.1 | (ICD9) HEMARTHROSIS |
| 719.1 | (ICD9) HEMARTHROSIS SITE UNSPECIFIED |
| 719.11 | (ICD9) HERARTHROSIS INVOLVING SHOULDER REGION |
| 719.12 | (ICD9) HEMARTHORSIS INVOLVING UPPER ARM |
| 719.13 | (ICD9) HEMARTHROSIS INVOLVING FOREARM |
| 719.14 | (ICD9) HEMARTHROSIS INVOLVING HAND |
| 719.15 | (ICD9) HEMARTHROSIS INVOLVING PELVIC REGION AND THIGH |
| 719.16 | (ICD9) HEMARTHROSIS INVOLVING LOWER LEG |
| 719.17 | (ICD9) HEMARTHROSIS INVOLVING ANKLE AND FOOT |
| 719.18 | (ICD9) HEMARTHROSIS INVOLVING OTHER SPECIFIED SITES |
| 719.19 | (ICD9) HEMARTHROSIS INVOLVING MULTIPLE SITES |
| 784.7 | (ICD9) EPISTAXIS |
| 784.8 | (ICD9) HEMORRHAGE FROM THROAT |

| 599.7 | (ICD9) HEMATURIA |
|---|---|
| 599.7 | (ICD9) HEMATURIA UNSPECIFIED |
| 599.71 | (ICD9) GROSS HEMATURIA |
| 599.72 | (ICD9) MICROSCOPIC HEMATURIA |
| 786.3 | (ICD9) HEMOPTYSIS |
| 786.3 | (ICD9) HEMOPTYSIS UNSPECIFIED |
| 786.31 | (ICD9) ACUTE IDIOPATHIC PULMONARY HEMORRHAGE IN INFANTS |
| 786.39 | (ICD9) OTHER HEMOPTYSIS |
| ICD 40 Dulanations and all | ! |
| ICD-10 Dx inpatient any positi | |
| 131.2 | (ICD10) Hemopericardium, not elsewhere classified |
| 160.00 | (ICD10) Nontraumatic subarachnoid hemorrhage from unspecified carotid siphon and bifurcation |
| 160.01 | (ICD10) Nontraumatic subarachnoid hemorrhage from right carotid siphon and bifurcation |
| 160.02 | (ICD10) Nontraumatic subarachnoid hemorrhage from left carotid siphon and bifurcation |
| 160.10 | (ICD10) Nontraumatic subarachnoid hemorrhage from unspecified middle cerebral artery |
| 160.11 | (ICD10) Nontraumatic subarachnoid hemorrhage from right middle cerebral artery |
| 160.12 | (ICD10) Nontraumatic subarachnoid hemorrhage from left middle cerebral artery |
| 160.2 | (ICD10) Nontraumatic subarachnoid hemorrhage from anterior communicating artery |
| 160.30 | (ICD10) Nontraumatic subarachnoid hemorrhage from unspecified posterior communicating artery |
| 160.31 | (ICD10) Nontraumatic subarachnoid hemorrhage from right posterior communicating artery |
| 160.32 | (ICD10) Nontraumatic subarachnoid hemorrhage from left posterior communicating artery |
| 160.4 | (ICD10) Nontraumatic subarachnoid hemorrhage from basilar artery |
| 160.50 | (ICD10) Nontraumatic subarachnoid hemorrhage from unspecified vertebral artery |
| 160.51 | (ICD10) Nontraumatic subarachnoid hemorrhage from right vertebral artery |
| 160.52 | (ICD10) Nontraumatic subarachnoid hemorrhage from left vertebral artery |
| 160.6 | (ICD10) Nontraumatic subarachnoid hemorrhage from other intracranial arteries |
| 160.7 | (ICD10) Nontraumatic subarachnoid hemorrhage from unspecified intracranial artery |
| 160.8 | (ICD10) Other nontraumatic subarachnoid hemorrhage |
| 160.9 | (ICD10) Nontraumatic subarachnoid hemorrhage, unspecified |
| 161.0 | (ICD10) Nontraumatic intracerebral hemorrhage in hemisphere, subcortical |
| l61.1 | (ICD10) Nontraumatic intracerebral hemorrhage in hemisphere, cortical |
| l61.2 | (ICD10) Nontraumatic intracerebral hemorrhage in hemisphere, unspecified |
| I61.3 | (ICD10) Nontraumatic intracerebral hemorrhage in brain stem |

| 161.4 | (ICD10) Nontraumatic intracerebral hemorrhage in cerebellum |
|---|---|
| 161.5 | (ICD10) Nontraumatic intracerebral hemorrhage, intraventricular |
| 161.6 | (ICD10) Nontraumatic intracerebral hemorrhage, multiple localized |
| 161.8 | (ICD10) Other nontraumatic intracerebral hemorrhage |
| 161.9 | (ICD10) Nontraumatic intracerebral hemorrhage, unspecified |
| 162.00 | (ICD10) Nontraumatic subdural hemorrhage, unspecified |
| l62.01 | (ICD10) Nontraumatic acute subdural hemorrhage |
| 162.02 | (ICD10) Nontraumatic subacute subdural hemorrhage |
| 162.03 | (ICD10) Nontraumatic chronic subdural hemorrhage |
| 162.1 | (ICD10) Nontraumatic extradural hemorrhage |
| 162.9 | (ICD10) Nontraumatic intracranial hemorrhage, unspecified |
| K25.0 | (ICD10) Acute gastric ulcer with hemorrhage |
| K25.2 | (ICD10) Acute gastric ulcer with both hemorrhage and perforation |
| K25.4 | (ICD10) Chronic or unspecified gastric ulcer with hemorrhage |
| K25.6 | (ICD10) Chronic or unspecified gastric ulcer with both hemorrhage and perforation |
| K26.0 | (ICD10) Acute duodenal ulcer with hemorrhage |
| K26.2 | (ICD10) Acute duodenal ulcer with both hemorrhage and perforation |
| K26.4 | (ICD10) Chronic or unspecified duodenal ulcer with hemorrhage |
| K26.6 | (ICD10) Chronic or unspecified duodenal ulcer with both hemorrhage and perforation |
| K27.0 | (ICD10) Acute peptic ulcer, site unspecified, with hemorrhage |
| K27.2 | (ICD10) Acute peptic ulcer, site unspecified, with both hemorrhage and perforation |
| K27.4 | (ICD10) Chronic or unspecified peptic ulcer, site unspecified, with hemorrhage |
| K27.6 | (ICD10) Chronic or unspecified peptic ulcer, site unspecified, with both hemorrhage and perforation |
| K28.0 | (ICD10) Acute gastrojejunal ulcer with hemorrhage |
| K28.2 | (ICD10) Acute gastrojejunal ulcer with both hemorrhage and perforation |
| K28.4 | (ICD10) Chronic or unspecified gastrojejunal ulcer with hemorrhage |
| K28.6 | (ICD10) Chronic or unspecified gastrojejunal ulcer with both hemorrhage and perforation |
| K55.21 | (ICD10) Angiodysplasia of colon with hemorrhage |
| K56.60 | (ICD10) Unspecified intestinal obstruction |
| K57.01 | (ICD10) Diverticulitis of small intestine with perforation and abscess with bleeding |
| K57.11 | (ICD10) Diverticulosis of small intestine without perforation or abscess with bleeding |
| K57.13 | (ICD10) Diverticulitis of small intestine without perforation or abscess with bleeding |
| K57.21 | (ICD10) Diverticulitis of large intestine with perforation and abscess with bleeding |

| K57.31 | (ICD10) Diverticulosis of large intestine without perforation or abscess with bleeding |
|---|---|
| K57.33 | (ICD10) Diverticulitis of large intestine without perforation or abscess with bleeding |
| K57.41 | (ICD10) Diverticulitis of both small and large intestine with perforation and abscess with bleeding |
| K57.51 | (ICD10) Diverticulosis of both small and large intestine without perforation or abscess with bleeding |
| K57.53 | (ICD10) Diverticulitis of both small and large intestine without perforation or abscess with bleeding |
| K57.81 | (ICD10) Diverticulitis of intestine, part unspecified, with perforation and abscess with bleeding |
| K57.91 | (ICD10) Diverticulosis of intestine, part unspecified, without perforation or abscess with bleeding |
| K57.93 | (ICD10) Diverticulitis of intestine, part unspecified, without perforation or abscess with bleeding |
| K62.5 | (ICD10) Hemorrhage of anus and rectum |
| K63.1 | (ICD10) Perforation of intestine (nontraumatic) |
| K63.81 | (ICD10) Dieulafoy lesion of intestine |
| K66.1 | (ICD10) Hemoperitoneum |
| K92.0 | (ICD10) Hematemesis |
| K92.1 | (ICD10) Melena |
| K92.2 | (ICD10) Gastrointestinal hemorrhage, unspecified |
| M25.00 | (ICD10) Hemarthrosis, unspecified joint |
| M25.011 | (ICD10) Hemarthrosis, right shoulder |
| M25.012 | (ICD10) Hemarthrosis, left shoulder |
| M25.019 | (ICD10) Hemarthrosis, unspecified shoulder |
| M25.021 | (ICD10) Hemarthrosis, right elbow |
| M25.022 | (ICD10) Hemarthrosis, left elbow |
| M25.029 | (ICD10) Hemarthrosis, unspecified elbow |
| M25.031 | (ICD10) Hemarthrosis, right wrist |
| M25.032 | (ICD10) Hemarthrosis, left wrist |
| M25.039 | (ICD10) Hemarthrosis, unspecified wrist |
| M25.041 | (ICD10) Hemarthrosis, right hand |
| M25.042 | (ICD10) Hemarthrosis, left hand |
| M25.049 | (ICD10) Hemarthrosis, unspecified hand |
| M25.051 | (ICD10) Hemarthrosis, right hip |
| M25.052 | (ICD10) Hemarthrosis, left hip |
| M25.059 | (ICD10) Hemarthrosis, unspecified hip |
| M25.061 | (ICD10) Hemarthrosis, right knee |
| M25.062 | (ICD10) Hemarthrosis, left knee |

M25.069

| | (10020) Telliar all 0313) all specimed lines |
|---|---|
| M25.071 | (ICD10) Hemarthrosis, right ankle |
| M25.072 | (ICD10) Hemarthrosis, left ankle |
| M25.073 | (ICD10) Hemarthrosis, unspecified ankle |
| M25.074 | (ICD10) Hemarthrosis, right foot |
| M25.075 | (ICD10) Hemarthrosis, left foot |
| M25.076 | (ICD10) Hemarthrosis, unspecified foot |
| M25.08 | (ICD10) Hemarthrosis, other specified site |
| R58 | (ICD10) Hemorrhage, not elsewhere classified |
| R04 | (ICD10) Hemorrhage from respiratory passages |
| R04.0 | (ICD10) Epistaxis |
| R04.1 | (ICD10) Hemorrhage from throat |
| R04.2 | (ICD10) Hemoptysis |
| R04.8 | (ICD10) Hemorrhage from other sites in respiratory passages |
| R04.81 | (ICD10) Acute idiopathic pulmonary hemorrhage in infants |
| R04.89 | (ICD10) Hemorrhage from other sites in respiratory passages |
| R04.9 | (ICD10) Hemorrhage from respiratory passages, unspecified |
| R31 | (ICD10) Hematuria |
| R31.0 | (ICD10) Gross hematuria |
| R31.1 | (ICD10) Benign essential microscopic hematuria |
| R31.2 | (ICD10) Other microscopic hematuria |
| R31.21 | (ICD10) Asymptomatic microscopic hematuria |
| R31.29 | (ICD10) Other microscopic hematuria |
| R31.9 | (ICD10) Hematuria, unspecified |
| Px inpatient any position | |
| 44.43 | (ICD9) ENDOSCOPIC CONTROL OF GASTRIC OR DUODENAL BLEEDING |
| 0W3P8ZZ | (ICD10) Control Bleeding in Gastrointestinal Tract, Via Natural or Artificial Opening Endoscopic |
| | (HCPCS) Esophagogastroduodenoscopy, flexible, transoral; with control of bleeding, any method / Upper |
| 43255 | gastrointestinal endoscopy including esophagus, stomach, and either the duodenum and/or jejunum as |

appropriate; with control of bleeding, any method

(ICD10) Hemarthrosis, unspecified knee

## Title

Pregnancy

| ICD-9 Dx in | patient any position |
|---|---|
| 650 | Normal delivery |
| 660 | Obstructed labor |
| 661 | Abnormality of forces of labor |
| 662 | Longlabor |
| 663 | Umbilical cord complications during labor and delivery |
| 664 | Trauma to perneum and vulva during delivery |
| 665 | Other obstetrical trauma |
| 667 | Retained placenta or membranes without hemorrhage |
| 668 | Complications of the administration of anesthetic or other sedation in labor and delivery |
| 669.94 | Unspecified complication of labor and delivery postpartum condition or complication |
| V24 | Postpartum care and examination |
| V24.0 | Postpartum care and examination immediately after delivery |
| V24.1 | Postpartum care and examination of lactating mother |
| V24.2 | Routine postpartum follow |
| V27 | Outcome of delivery |
| V27.0 | Mother with single liveborn |
| V27.1 | Mother with single stillborn |
| V27.2 | Mother with twins both liveborn |
| V27.3 | Mother with twins one liveborn and one stillborn |
| V27.4 | Mother with twins both stillborn |
| V27.5 | Mother with other multiple birth all liveborn |
| V27.6 | Mother with other multiple birth some liveborn |
| V27.7 | Mother with other multiple birth all stillborn |
| V27.9 | Mother with unspecified outcome of delivery |
| ICD-9 Px in | patient any position |
| 72.0 | Low forceps operation |

| 72.0 | Low forceps operation |
|-------|---------------------------------------|
| 72.1 | Low forceps operation with episiotomy |
| 72.2 | Mid forceps operation |
| 72.21 | Mid forceps operation with episiotomy |
| 72.29 | Other mid forceps operation |

| 72.3 | High forceps operation |
|-------|------------------------------------------------------------|
| 72.31 | High forceps operation with episiotomy |
| 72.39 | Other high forceps operation |
| 72.4 | Forceps rotation of fetal head |
| 72.5 | Breech extraction |
| 72.51 | Partial breech extraction with forceps to aftercoming head |
| 72.52 | Other partial breech extraction |
| 72.53 | Total breech extraction with forceps to aftercoming head |
| 72.54 | Other total breech extraction |
| 72.6 | Forceps application to aftercoming head |
| 72.7 | Vacuum extraction |
| 72.71 | Vacuum extraction with episiotomy |
| 72.79 | Other vacuum extraction |
| 72.8 | Other specified instrumental delivery |
| 72.9 | Unspecified instrumental delivery |
| 73.0 | Artificial rupture of membranes |
| 73.01 | Induction of labor by artificial rupture of membranes |
| 73.09 | Other artificial rupture of membranes |
| 73.1 | Other surgical induction of labor |
| 73.2 | Internal and combined version and extraction |
| 73.21 | Internal and combined version without extraction |
| 73.22 | Internal and combined version with extraction |
| 73.3 | Failed forceps |
| 73.4 | Medical induction of labor |
| 73.5 | Manually assisted delivery |
| 73.51 | Manual rotation of fetal head |
| 73.59 | Other manually assisted delivery |
| 73.6 | Episiotomy |
| 73.8 | Operations on fetus to facilitate delivery |
| 73.9 | Other operations assisting delivery |
| 73.91 | External version assisting delivery |
| 73.92 | Replacement of prolapsed umbilical cord |
| 73.93 | Incision of cervix to assist delivery |
| 73.94 | Pubiotomy to assist delivery |
| 73.99 | Other operations assisting delivery |
# Appendix A

| 74.0 | Classical cesarean section |
|-------|--------------------------------------------------|
| 74.1 | Low cervical cesarean section |
| 74.2 | Extraperitoneal cesarean section |
| 74.3 | Removal of extratubal ectopic pregnancy |
| 74.4 | Cesarean section of other specified type |
| 74.9 | Cesarean section of unspecified type |
| 74.91 | Hysterotomy to terminate pregnancy |
| 74.99 | Other cesarean section of unspecified type |
| 75.4 | Manual removal of retained placenta |
| 75.5 | Repair of current obstetric laceration of uterus |
| 75.6 | Repair of other current obstetric laceration |
| 75.7 | Manual exploration of uterine cavity, postpartum |
| 75.9 | Other obstetric operations |



| | | | | | Unmatched | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Optu | | <u> </u> | Market: | Scan | | Medicare | | | | POOLED | |
| Variable | 2.6 | Exposure - rivaroxaban | C: D:# D | | | C: D:# D | | 5 | S: D:# D | | Exposure - rivaroxaban | St. Diff |
| Variable Number of patients | Reference- warfarin Copy<br>10.936 | (15 or 20 mg) Copy<br>6.448 | St. Diff. R | eference-warfarin Copy ()<br>23,040 | aban (15 or 20 mg) Copy<br>9.405 | St. Diff. Re | ference-warfarin Copy 1 | .5 or 20 mg) Copy<br>16.223 | St. Diff. R | eference- warfarin Copy<br>66,871 | (15 or 20 mg) Copy<br>32.076 | St. Diff. |
| Age | 10,930 | 0,448 | | 23,040 | 9,405 | | 32,895 | 16,223 | | 00,8/1 | 32,076 | |
| mean (sd) | 62.06 (15.66) | 60.27 (15.40) | 0.12 | 55.59 (15.02) | 53.61 (14.45) | 0.13 | 75.46 (7.25) | 74.46 (6.75) | 0.14 | 66.42 (11.99) | 65.49 (11.49) | 0.08 |
| median [IQR] | 65.00 [51.00, 74.00] | 62.00 [50.00, 72.00] | 0.19 | 56.00 [46.00, 64.00] | 54.00 [44.00, 63.00] | 0.14 | 74.00 [69.00, 80.00] 3 | | 0.14 | 66.33 (11.99) | 65.22 (11.49) | 0.09 |
| Age categories without zero category | 03.00 [31.00, 74.00] | 02.00 [30.00, 72.00] | 0.15 | 30.00 [40.00, 04.00] | 34.00 [44.00, 03.00] | 0.14 | 74.00 [05.00, 80.00] 5 | .00 [05.00, 75.00] | 0.14 | 00.33 (11.33) | 03.22 (11.43) | 0.05 |
| 18 - 54; n (%) | 3,304 (30.2%) | 2,172 (33.7%) | -0.08 | 10,427 (45.3%) | 4.739 (50.4%) | -0.10 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 13,731 (20.5%) | 6911 (21.5%) | -0.02 |
| 55 - 64: n (%) | 2,163 (19.8%) | 1,354 (21.0%) | -0.03 | 7,017 (30.5%) | 2,874 (30.6%) | 0.00 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 9,180 (13.7%) | 4,228 (13.2%) | 0.01 |
| 65 - 74; n (%) | 2,869 (26.2%) | 1,739 (27.0%) | -0.02 | 2,972 (12.9%) | 1,055 (11.2%) | 0.05 | 16,795 (51.1%) | 9,117 (56.2%) | -0.10 | 22,636 (33.9%) | 11,911 (37.1%) | -0.07 |
| >= 75; n (%) | 2,600 (23.8%) | 1,183 (18.3%) | 0.14 | 2,624 (11.4%) | 737 (7.8%) | 0.12 | 16,100 (48.9%) | 7,106 (43.8%) | 0.10 | 21,324 (31.9%) | 9,026 (28.1%) | 0.08 |
| Gender without zero category- United | | | | | | | | | | | | |
| Males; n (%) | 4,959 (45.3%) | 3,037 (47.1%) | -0.04 | 11,080 (48.1%) | 4,697 (49.9%) | -0.04 | 12,293 (37.4%) | 6,712 (41.4%) | -0.08 | 28,332 (42.4%) | 14,446 (45.0%) | -0.05 |
| Females; n (%) | 5,976 (54.6%) | 3,410 (52.9%) | 0.03 | 11,960 (51.9%) | 4,708 (50.1%) | 0.04 | 20,602 (62.6%) | 9,511 (58.6%) | 0.08 | 38,538 (57.6%) | 17,629 (55.0%) | 0.05 |
| Race | | | | | | | | | | | | |
| White; n (%) | | | | | | | 28,783 (87.5%) | 14,127 (87.1%) | 0.01 | 28,783 (87.5%) | 14,127 (87.1%) | 0.01 |
| Black; n (%) | | | | | | | 2,966 (9.0%) | 1,433 (8.8%) | 0.01 | 2,966 (9.0%) | 1,433 (8.8%) | 0.01 |
| Asian; n (%) | | | | | | | 194 (0.6%) | 121 (0.7%) | -0.01 | 194 (0.6%) | 121 (0.7%) | -0.01 |
| Hispanic; n (%) | | | | | | | 394 (1.2%) | 177 (1.1%) | 0.01 | 394 (1.2%) | 177 (1.1%) | 0.01 |
| North American Native; n (%) | | | | | | | 97 (0.3%) | 46 (0.3%) | 0.00 | 97 (0.3%) | 46 (0.3%) | 0.00 |
| Other/Unknown; n (%) | | | | | | | 461 (1.4%) | 319 (2.0%) | -0.05 | 461 (1.4%) | 319 (2.0%) | -0.05 |
| Region without zero category | | | | | | | | | | | | |
| Northeast; n (%) | 1,069 (9.8%) | 661 (10.3%) | -0.02 | 4,222 (18.3%) | 1,713 (18.2%) | 0.00 | 5,743 (17.5%) | 2.841 (17.5%) | 0.00 | 11034 (16.5%) | 5,215 (16.3%) | 0.01 |
| Northeast; n (%)<br>South; n (%) | 3,790 (34.7%) | 2,716 (42.1%) | -0.02 | 6,557 (28.5%) | 2,460 (26.2%) | 0.00 | 11,036 (33.5%) | 6,415 (39.5%) | -0.12 | 21.383 (32.0%) | 11,591 (36.1%) | -0.09 |
| Midwest; n (%) | 3,255 (29.8%) | 1,713 (26.6%) | 0.07 | 7,804 (33.9%) | 4,013 (42.7%) | -0.18 | 9,920 (30.2%) | 4,033 (24.9%) | 0.12 | 20,979 (31.4%) | 9,759 (30.4%) | 0.09 |
| West; n (%) | 2,822 (25.8%) | 1,358 (21.1%) | 0.11 | 4,149 (18.0%) | 1,125 (12.0%) | 0.17 | 6,157 (18.7%) | 2,922 (18.0%) | 0.02 | 13,128 (19.6%) | 5,405 (16.9%) | 0.02 |
| Unknown+missing; n (%) | N/A | N/A | #VALUE! | 308 (1.3%) | 94 (1.0%) | 0.03 | N/A | N/A | #VALUE! | 308 (1.3%) | 94 (1.0%) | 0.03 |
| CV Covariates | .4 | | | | (=) | | | | | | - () | |
| Ischemic heart disease; n (%) | 1,887 (17.3%) | 1.101 (17.1%) | 0.01 | 2.748 (11.9%) | 1.139 (12.1%) | -0.01 | 8.409 (25.6%) | 3,988 (24.6%) | 0.02 | 13.044 (19.5%) | 6,228 (19,4%) | 0.00 |
| Acute MI; n (%) | 396 (3.6%) | 245 (3.8%) | -0.01 | 680 (3.0%) | 297 (3.2%) | -0.01 | 1,323 (4.0%) | 646 (4.0%) | 0.00 | 2399 (3.6%) | 1188 (3.7%) | -0.01 |
| ACS/unstable angina; n (%) | 90 (0.8%) | 112 (1.7%) | -0.08 | 73 (0.3%) | 105 (1.1%) | -0.10 | 308 (0.9%) | 272 (1.7%) | -0.07 | 471 (0.7%) | 489 (1.5%) | -0.08 |
| Old MI; n (%) | 320 (2.9%) | 185 (2.9%) | 0.00 | 338 (1.5%) | 166 (1.8%) | -0.02 | 1,793 (5.5%) | 751 (4.6%) | 0.04 | 2451 (3.7%) | 1102 (3.4%) | 0.02 |
| Stable angina; n (%) | 216 (2.0%) | 137 (2.1%) | -0.01 | 333 (1.4%) | 160 (1.7%) | -0.02 | 801 (2.4%) | 409 (2.5%) | -0.01 | 1350 (2.0%) | 706 (2.2%) | -0.01 |
| Coronary atherosclerosis and other forms of chronic | | | | | | | | | | | | |
| ischemic heart disease; n (%) | 1,447 (13.2%) | 768 (11.9%) | 0.04 | 1,990 (8.6%) | 747 (7.9%) | 0.03 | 7,049 (21.4%) | 3,254 (20.1%) | 0.03 | 10,486 (15.7%) | 4,769 (14.9%) | 0.02 |
| Other atherosclerosis with ICD10 v2 Copy; n (%) | 106 (1.0%) | 43 (0.7%) | 0.03 | 134 (0.6%) | 43 (0.5%) | 0.01 | 418 (1.3%) | 163 (1.0%) | 0.03 | 658 (1.0%) | 249 (0.8%) | 0.02 |
| Previous cardiac procedure (CABG or PTCA or Stent) | | | | | | | | | | | | |
| v4; n (%) | 54 (0.5%) | 14 (0.2%) | 0.05 | 98 (0.4%) | 27 (0.3%) | 0.02 | 184 (0.6%) | 77 (0.5%) | 0.01 | 336 (0.5%) | 118 (0.4%) | 0.01 |
| History of CABG or PTCA; n (%) | 418 (3.8%) | 252 (3.9%) | -0.01 | 312 (1.4%) | 118 (1.3%) | 0.01 | 2,843 (8.6%) | 1,333 (8.2%) | 0.01 | 3,573 (5.3%) | 1,703 (5.3%) | 0.00 |
| Any stroke; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 000 (0.0%) | #DIV/0! |
| Ischemic stroke (w and w/o mention of cerebral | | | | | | | | | | | | |
| infarction); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 000 (0.0%) | #DIV/0! |
| Hemorrhagic stroke; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 000 (0.0%) | 0 (0.0%) | #DIV/0! |
| TIA; n (%) | 96 (0.9%) | 61 (0.9%) | 0.00 | 137 (0.6%) | 57 (0.6%) | 0.00 | 350 (1.1%) | 153 (0.9%) | 0.02 | 583 (0.9%) | 271 (0.8%) | 0.01 |
| Other cerebrovascular disease; n (%) Cerebrovascular procedure: n (%) | 173 (1.6%)<br>0 (0.0%) | 60 (0.9%)<br>0 (0.0%) | 0.06<br>#DIV/0! | 180 (0.8%)<br>** (0.0%) | 61 (0.6%)<br>0 (0.0%) | 0.02<br>#DIV/0! | 748 (2.3%)<br>0 (0.0%) | 273 (1.7%)<br>0 (0.0%) | 0.04<br>#DIV/0! | 1101 (1.6%)<br>#VALUE! | 394 (1.2%)<br>0 (0.0%) | #VALUE! |
| Heart failure (CHF); n (%) | ** (0.1%) | ** (0.0%) | #DIV/0!<br>0.04 | ** (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | #VALUE! | #VALUE! | #VALUE! |
| Peripheral Vascular Disease (PVD) or PVD Surgery v2; | ** (0.1%) | ** (0.0%) | 0.04 | ** (0.0%) | 0 (0.0%) | #DIV/U! | 0 (0.0%) | 0 (0.0%) | #DIV/U! | #VALUE! | #VALUE! | #VALUE! |
| n (%) | 513 (4.7%) | 289 (4.5%) | 0.01 | 690 (3.0%) | 266 (2.8%) | 0.01 | 2,261 (6.9%) | 996 (6.1%) | 0.03 | 3,464 (5.2%) | 1,551 (4.8%) | 0.02 |
| Atrial fibrillation; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 000 (0.0%) | #DIV/0! |
| Other cardiac dysrhythmia; n (%) | 1.679 (15.4%) | 849 (13.2%) | 0.06 | 3.124 (13.6%) | 1,204 (12,8%) | 0.02 | 5,727 (17.4%) | 2.406 (14.8%) | 0.07 | 10.530 (15.7%) | 4.459 (13.9%) | 0.05 |
| Cardiac conduction disorders; n (%) | 714 (6.5%) | 411 (6.4%) | 0.00 | 857 (3.7%) | 389 (4.1%) | -0.02 | 2.701 (8.2%) | 1.281 (7.9%) | 0.01 | 4272 (6.4%) | 2081 (6.5%) | 0.00 |
| Other CVD; n (%) | 2,738 (25.0%) | 1,629 (25.3%) | -0.01 | 4,454 (19.3%) | 1,993 (21.2%) | -0.05 | 7,925 (24.1%) | 4,007 (24.7%) | -0.01 | 15,117 (22.6%) | 7,629 (23.8%) | -0.03 |
| Diabetes-related complications | , , | , , | | , . , , | ,, | | , | ,, | | -, , , | ,, | |
| Occurrence of Diabetic Neuropathy v2 Copy; n (%) | 438 (4.0%) | 259 (4.0%) | 0.00 | 465 (2.0%) | 200 (2.1%) | -0.01 | 1,258 (3.8%) | 573 (3.5%) | 0.02 | 2161 (3.2%) | 1032 (3.2%) | 0.00 |
| Occurrence of diabetic nephropathy V3 with ICD10 | • • | , , | | | , , | | | , , | | , , | | |
| Copy; n (%) | 235 (2.1%) | 147 (2.3%) | -0.01 | 236 (1.0%) | 95 (1.0%) | 0.00 | 635 (1.9%) | 292 (1.8%) | 0.01 | 1,106 (1.7%) | 534 (1.7%) | 0.00 |
| Hypoglycemia v2; n (%) | 129 (1.2%) | 27 (0.4%) | 0.09 | 210 (0.9%) | 51 (0.5%) | 0.05 | 589 (1.8%) | 278 (1.7%) | 0.01 | 928 (1.4%) | 356 (1.1%) | 0.03 |
| Hyperglycemia; n (%) | 777 (7.1%) | 496 (7.7%) | -0.02 | 938 (4.1%) | 451 (4.8%) | -0.03 | 2,693 (8.2%) | 1,480 (9.1%) | -0.03 | 4408 (6.6%) | 2427 (7.6%) | -0.04 |
| Diabetic ketoacidosis; n (%) | 33 (0.3%) | 21 (0.3%) | 0.00 | 67 (0.3%) | 26 (0.3%) | 0.00 | 78 (0.2%) | 25 (0.2%) | 0.00 | 178 (0.3%) | 72 (0.2%) | 0.02 |
| Hypertension: 1 inpatient or 2 outpatient claims | | | | | | | | | | | | |
| within 365 days; n (%) | 6,750 (61.7%) | 3,702 (57.4%) | 0.09 | 11,057 (48.0%) | 4,458 (47.4%) | 0.01 | 26,870 (81.7%) | 12,798 (78.9%) | 0.07 | 44,677 (66.8%) | 20,958 (65.3%) | 0.03 |
| Hyperlipidemia v2; n (%) | 5,170 (47.3%) | 2,834 (44.0%) | 0.07 | 7,362 (32.0%) | 3,147 (33.5%) | -0.03 | 20,106 (61.1%) | 9,762 (60.2%) | 0.02 | 32,638 (48.8%) | 15,743 (49.1%) | -0.01 |
| Edema; n (%) | 1,721 (15.7%) | 1,080 (16.7%) | -0.03 | 2,586 (11.2%) | 1,243 (13.2%) | -0.06 | 4,315 (13.1%) | 1,982 (12.2%) | 0.03 | 8622 (12.9%) | 4305 (13.4%) | -0.01 |
| Renal Dysfunction (non-diabetic) v2; n (%) | 2,375 (21.7%) | 1,172 (18.2%) | 0.09 | 3,055 (13.3%) | 1,084 (11.5%) | 0.05 | 8,504 (25.9%) | 3,405 (21.0%) | 0.12 | 13,934 (20.8%) | 5,661 (17.6%) | 0.08 |
| Occurrence of acute renal disease v2; n (%) | 1,071 (9.8%) | 496 (7.7%) | 0.07 | 1,396 (6.1%) | 536 (5.7%) | 0.02 | 3,560 (10.8%) | 1,440 (8.9%) | 0.06 | 6027 (9.0%) | 2472 (7.7%) | 0.05 |
| Occurrence of chronic renal insufficiency; n (%) | 1,209 (11.1%) | 537 (8.3%) | 0.09 | 1,164 (5.1%) | 349 (3.7%) | 0.07 | 4,943 (15.0%) | 1,729 (10.7%) | 0.13 | 7,316 (10.9%) | 2,615 (8.2%) | 0.09 |
| Chronic kidney disease v2; n (%) | 1,170 (10.7%) | 512 (7.9%) | 0.10 | 1,088 (4.7%) | 323 (3.4%) | 0.07 | 4,739 (14.4%) | 1,645 (10.1%) | 0.13 | 6,997 (10.5%) | 2,480 (7.7%) | 0.10 |
| CKD Stage 3-4; n (%) | 714 (6.5%) | 311 (4.8%) | 0.07 | 599 (2.6%) | 178 (1.9%) | 0.05 | 2,836 (8.6%) | 999 (6.2%) | 0.09 | 4,149 (6.2%) | 1,488 (4.6%) | 0.07 |
| Occurrence of hypertensive nephropathy; n (%) | 792 (7.2%) | 325 (5.0%) | 0.09 | 706 (3.1%) | 213 (2.3%) | 0.05 | 3,862 (11.7%) | 1,288 (7.9%) | 0.13 | 5,360 (8.0%) | 1,826 (5.7%) | 0.09 |
| Occurrence of miscellaneous renal insufficiency v2; n | | | | | | | | | | | | |
| (%) | 927 (8.5%) | 463 (7.2%) | 0.05 | 1,292 (5.6%) | 439 (4.7%) | 0.04 | 3,000 (9.1%) | 1,209 (7.5%) | 0.06 | 5,219 (7.8%) | 2,111 (6.6%) | 0.05 |
| Other Covariates | | | | | | | | | | | | |

| Liver disease; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/01 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/01 | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Osteoarthritis; n (%) | 2,875 (26.3%) | 1,680 (26.1%) | 0.00 | 4,249 (18.4%) | 1,779 (18.9%) | -0.01 | 11,602 (35.3%) | 5,806 (35.8%) | -0.01 | 18726 (28.0%) | 9265 (28.9%) | -0.02 |
| Other arthritis, arthropathies and musculoskeletal | 2,073 (20.370) | 1,000 (20.1%) | 0.00 | 4,245 (20.470) | 1,773 (10.370) | 0.01 | 11,002 (33.370) | 3,000 (33.070) | 0.01 | 10720 (20.070) | 3203 (20.3%) | 0.02 |
| pain; n (%) | 7,107 (65.0%) | 4.067 (63.1%) | 0.04 | 13,537 (58.8%) | 5,724 (60.9%) | -0.04 | 19,911 (60.5%) | 9.597 (59.2%) | 0.03 | 40555 (60.6%) | 19388 (60.4%) | 0.00 |
| Dorsopathies; n (%) | 3,652 (33.4%) | 2,195 (34.0%) | -0.01 | 6,396 (27.8%) | 2,672 (28.4%) | -0.01 | 11,170 (34.0%) | 5,322 (32.8%) | 0.03 | 21218 (31.7%) | 10189 (31.8%) | 0.00 |
| Fractures; n (%) | 962 (8.8%) | 558 (8.7%) | 0.00 | 1,761 (7.6%) | 632 (6.7%) | 0.03 | 3,146 (9.6%) | 1,424 (8.8%) | 0.03 | 5869 (8.8%) | 2614 (8.1%) | 0.03 |
| Falls v2; n (%) | 771 (7.1%) | 477 (7.4%) | -0.01 | 434 (1.9%) | 267 (2.8%) | -0.06 | 1,170 (3.6%) | 542 (3.3%) | 0.02 | 2375 (3.6%) | 1286 (4.0%) | -0.02 |
| Osteoporosis; n (%) | 857 (7.8%) | 380 (5.9%) | 0.08 | 787 (3.4%) | 246 (2.6%) | 0.05 | 4,514 (13.7%) | 1,960 (12.1%) | 0.05 | 6158 (9.2%) | 2586 (8.1%) | 0.04 |
| Depression; n (%) | 2,091 (19.1%) | 1,156 (17.9%) | 0.03 | 3,206 (13.9%) | 1,262 (13.4%) | 0.01 | 6,138 (18.7%) | 2,809 (17.3%) | 0.04 | 11435 (17.1%) | 5227 (16.3%) | 0.02 |
| Anxiety; n (%) | 1,816 (16.6%) | 1,276 (19.8%) | -0.08 | 2,689 (11.7%) | 1,354 (14.4%) | -0.08 | 5,310 (16.1%) | 2,627 (16.2%) | 0.00 | 9815 (14.7%) | 5257 (16.4%) | -0.05 |
| Sleep_Disorder; n (%) | 1,580 (14.4%) | 476 (7.4%) | 0.23 | 2,974 (12.9%) | 935 (9.9%) | 0.09 | 4,052 (12.3%) | 1,350 (8.3%) | 0.13 | 8606 (12.9%) | 2761 (8.6%) | 0.14 |
| Dementia; n (%) | 660 (6.0%) | 344 (5.3%) | 0.03 | 481 (2.1%) | 195 (2.1%) | 0.00 | 3,564 (10.8%) | 1,522 (9.4%) | 0.05 | 4705 (7.0%) | 2061 (6.4%) | 0.02 |
| Delirium; n (%) | 341 (3.1%) | 154 (2.4%) | 0.04 | 378 (1.6%) | 152 (1.6%) | 0.00 | 1,162 (3.5%) | 469 (2.9%) | 0.03 | 1881 (2.8%) | 775 (2.4%) | 0.03 |
| Psychosis; n (%) | 264 (2.4%) | 120 (1.9%) | 0.03 | 262 (1.1%) | 94 (1.0%) | 0.01 | 893 (2.7%) | 364 (2.2%) | 0.03 | 1419 (2.1%) | 578 (1.8%) | 0.02 |
| Obesity; n (%) | 3,062 (28.0%) | 2,069 (32.1%) | -0.09 | 5,195 (22.5%) | 2,601 (27.7%) | -0.12 | 7,385 (22.5%) | 3,582 (22.1%) | 0.01 | 15642 (23.4%) | 8252 (25.7%) | -0.05 |
| Overweight; n (%) | 338 (3.1%) | 375 (5.8%) | -0.13 | 319 (1.4%) | 336 (3.6%) | -0.14 | 1,166 (3.5%) | 748 (4.6%) | -0.06 | 1823 (2.7%) | 1459 (4.5%) | -0.10 |
| Smoking; n (%) | 2,998 (27.4%) | 2,157 (33.5%) | -0.13 | 3,459 (15.0%) | 1,640 (17.4%) | -0.07 | 11,425 (34.7%) | 6,267 (38.6%) | -0.08 | 17882 (26.7%) | 10064 (31.4%) | -0.10 |
| Alcohol abuse or dependence; n (%) | 259 (2.4%) | 151 (2.3%) | 0.01 | 423 (1.8%) | 199 (2.1%) | -0.02 | 283 (0.9%) | 270 (1.7%) | -0.07 | 965 (1.4%) | 620 (1.9%) | -0.04 |
| Drug abuse or dependence; n (%) | 311 (2.8%) | 223 (3.5%) | -0.04<br>0.05 | 410 (1.8%) | 187 (2.0%) | -0.01<br>0.02 | 276 (0.8%) | 187 (1.2%) | -0.04<br>0.03 | 997 (1.5%) | 597 (1.9%) | -0.03<br>0.02 |
| COPD; n (%) | 1,833 (16.8%) | 973 (15.1%) | 0.05 | 2,312 (10.0%)<br>2,390 (10.4%) | 894 (9.5%) | -0.02 | 7,353 (22.4%) | 3,421 (21.1%)<br>1.853 (11.4%) | -0.01 | 11498 (17.2%)<br>7485 (11.2%) | 5288 (16.5%)<br>3676 (11.5%) | -0.02 |
| Asthma; n (%) Obstructive sleep apnea; n (%) | 1,395 (12.8%)<br>1,392 (12.7%) | 775 (12.0%)<br>846 (13.1%) | -0.01 | 2,390 (10.4%) | 1,048 (11.1%)<br>1,187 (12.6%) | -0.02 | 3,700 (11.2%)<br>3,411 (10.4%) | 1,853 (11.4%) | -0.01 | 7483 (11.2%) | 3745 (11.7%) | -0.01 |
| Pneumonia; n (%) | 1,796 (16.4%) | 989 (15.3%) | 0.03 | 3,434 (14.9%) | 1,343 (14.3%) | 0.02 | 5,572 (16.9%) | 2,491 (15.4%) | 0.04 | 10802 (16.2%) | 4823 (15.0%) | 0.03 |
| Other Medications | 1,750 (10.4%) | 505 (13.5%) | 0.03 | 3,434 (14.5%) | 1,343 (14.370) | 0.02 | 3,372 (10.5%) | 2,451 (13.470) | 0.04 | 10802 (10.2%) | 4823 (13.0%) | 0.03 |
| Use of ACE inhibitors; n (%) | 2.648 (24.2%) | 1.294 (20.1%) | 0.10 | 4,813 (20.9%) | 1,698 (18.1%) | 0.07 | 10,148 (30.8%) | 4,664 (28.7%) | 0.05 | 17609 (26.3%) | 7656 (23.9%) | 0.06 |
| Use of ARBs: n (%) | 1.386 (12.7%) | 923 (14.3%) | -0.05 | 2.855 (12.4%) | 1.146 (12.2%) | 0.01 | 6,221 (18,9%) | 3.261 (20.1%) | -0.03 | 10462 (15.6%) | 5330 (16.6%) | -0.03 |
| Use of Loop Diuretics - United; n (%) | 917 (8.4%) | 405 (6.3%) | 0.08 | 1,580 (6.9%) | 503 (5.3%) | 0.07 | 4,381 (13.3%) | 1,780 (11.0%) | 0.07 | 6878 (10.3%) | 2688 (8.4%) | 0.07 |
| Use of other diuretics- United; n (%) | 140 (1.3%) | 82 (1.3%) | 0.00 | 316 (1.4%) | 119 (1.3%) | 0.01 | 625 (1.9%) | 279 (1.7%) | 0.02 | 1081 (1.6%) | 480 (1.5%) | 0.01 |
| Use of nitrates-United; n (%) | 291 (2.7%) | 128 (2.0%) | 0.05 | 471 (2.0%) | 141 (1.5%) | 0.04 | 1,680 (5.1%) | 709 (4.4%) | 0.03 | 2442 (3.7%) | 978 (3.0%) | 0.04 |
| Use of other hypertension drugs; n (%) | 467 (4.3%) | 203 (3.1%) | 0.06 | 755 (3.3%) | 242 (2.6%) | 0.04 | 1,947 (5.9%) | 854 (5.3%) | 0.03 | 3169 (4.7%) | 1299 (4.0%) | 0.03 |
| Use of Anti-arrhythmics; n (%) | 24 (0.2%) | 13 (0.2%) | 0.00 | 70 (0.3%) | 19 (0.2%) | 0.02 | 118 (0.4%) | 49 (0.3%) | 0.02 | 212 (0.3%) | 81 (0.3%) | 0.00 |
| Use of COPD/asthma meds- United; n (%) | 1,985 (18.2%) | 1,117 (17.3%) | 0.02 | 4,137 (18.0%) | 1,708 (18.2%) | -0.01 | 7,383 (22.4%) | 3,707 (22.9%) | -0.01 | 13505 (20.2%) | 6532 (20.4%) | 0.00 |
| Use of statins; n (%) | 3,339 (30.5%) | 1,881 (29.2%) | 0.03 | 5,891 (25.6%) | 2,195 (23.3%) | 0.05 | 14,704 (44.7%) | 7,286 (44.9%) | 0.00 | 23934 (35.8%) | 11362 (35.4%) | 0.01 |
| Use of other lipid-lowering drugs; n (%) | 650 (5.9%) | 305 (4.7%) | 0.05 | 1,443 (6.3%) | 464 (4.9%) | 0.06 | 2,506 (7.6%) | 1,182 (7.3%) | 0.01 | 4599 (6.9%) | 1951 (6.1%) | 0.03 |
| Use of antiplatelet agents; n (%) | 402 (3.7%) | 251 (3.9%) | -0.01 | 974 (4.2%) | 341 (3.6%) | 0.03 | 2,429 (7.4%) | 1,076 (6.6%) | 0.03 | 3805 (5.7%) | 1668 (5.2%) | 0.02 |
| Use of heparin and other low-molecular weight | | | | | | | | | | | | |
| heparins; n (%) | 5,843 (53.4%) | 209 (3.2%) | 1.34 | 19 (0.1%) | ** (0.0%) | 0.04 | 15,058 (45.8%) | 487 (3.0%) | 1.15 | 20920 (31.3%) | #VALUE! | #VALUE! |
| Use of NSAIDs; n (%) | 2,235 (20.4%) | 1,367 (21.2%) | -0.02 | 4,992 (21.7%) | 2,348 (25.0%) | -0.08 | 6,301 (19.2%) | 3,269 (20.2%) | -0.03 | 13528 (20.2%) | 6984 (21.8%) | -0.04 |
| Use of oral corticosteroids; n (%) Use of bisphosphonate (United): n (%) | 2,937 (26.9%)<br>377 (3.4%) | 1,838 (28.5%)<br>131 (2.0%) | -0.04<br>0.09 | 6,039 (26.2%)<br>396 (1.7%) | 2,595 (27.6%)<br>101 (1.1%) | -0.03<br>0.05 | 10,634 (32.3%)<br>1.572 (4.8%) | 5,310 (32.7%)<br>625 (3.9%) | -0.01<br>0.04 | 19610 (29.3%)<br>2345 (3.5%) | 9743 (30.4%)<br>857 (2.7%) | -0.02<br>0.05 |
| Use of opioids- United; n (%) | 5,636 (51.5%) | 3,020 (46.8%) | 0.09 | 12,644 (54.9%) | 4,824 (51.3%) | 0.05 | 1,572 (4.8%) | 7,363 (45.4%) | 0.04 | 33810 (50.6%) | 857 (2.7%)<br>15207 (47.4%) | 0.05 |
| Use of antidepressants; n (%) | 2,945 (26.9%) | 1,722 (26.7%) | 0.00 | 5,760 (25.0%) | 2,242 (23.8%) | 0.07 | 9,959 (30.3%) | 4,877 (30.1%) | 0.00 | 18664 (27.9%) | 8841 (27.6%) | 0.01 |
| Use of antipsychotics; n (%) | 480 (4.4%) | 309 (4.8%) | -0.02 | 807 (3.5%) | 331 (3.5%) | 0.00 | 1,719 (5.2%) | 842 (5.2%) | 0.00 | 3006 (4.5%) | 1482 (4.6%) | 0.00 |
| Labs | 100 (1.170) | 303 (4.0%) | 0.02 | 007 (5.570) | 331 (3.370) | 0.00 | 1,713 (3.270) | 0.12 (3.270) | 0.00 | 3000 (4.370) | 1402 (4.0%) | 0.00 |
| Lab values- HbA1c (%) v3; n (%) | 881 (8.1%) | 779 (12.1%) | -0.13 | 205 (0.9%) | 83 (0.9%) | 0.00 | N/A | N/A | #VALUE! | 1.086 (3.2%) | 862 (5.4%) | -0.11 |
| Lab values-HbA1c (%) (within 3 months) v3; n (%) | 565 (5.2%) | 499 (7.7%) | -0.10 | 150 (0.7%) | 64 (0.7%) | 0.00 | N/A | N/A | #VALUE! | 715 (2.1%) | 563 (3.6%) | -0.09 |
| Lab values-HbA1c (%) (within 6 months) v3; n (%) | 881 (8.1%) | 779 (12.1%) | -0.13 | 205 (0.9%) | 83 (0.9%) | 0.00 | N/A | N/A | #VALUE! | 1,086 (3.2%) | 862 (5.4%) | -0.11 |
| Lab values- BNP; n (%) | 96 (0.9%) | 85 (1.3%) | -0.04 | ** (0.0%) | ** (0.1%) | -0.04 | N/A | N/A | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| Lab values- BNP (within 3 months); n (%) | 89 (0.8%) | 79 (1.2%) | -0.04 | ** (0.0%) | ** (0.0%) | #DIV/0! | N/A | N/A | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| Lab values- BNP (within 6 months); n (%) | 96 (0.9%) | 85 (1.3%) | -0.04 | ** (0.0%) | ** (0.1%) | -0.04 | N/A | N/A | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| Lab values- BUN (mg/dl); n (%) | 2,195 (20.1%) | 1,688 (26.2%) | -0.15 | 208 (0.9%) | 118 (1.3%) | -0.04 | N/A | N/A | #VALUE! | 2,403 (7.1%) | 1,806 (11.4%) | -0.15 |
| Lab values- BUN (mg/dl) (within 3 months); n (%) | 1,542 (14.1%) | 1,182 (18.3%) | -0.11 | 153 (0.7%) | 85 (0.9%) | -0.02 | N/A | N/A | #VALUE! | 1,695 (5.0%) | 1,267 (8.0%) | -0.12 |
| Lab values- BUN (mg/dl) (within 6 months); n (%) | 2,195 (20.1%) | 1,688 (26.2%) | -0.15 | 208 (0.9%) | 118 (1.3%) | -0.04 | N/A | N/A | #VALUE! | 2,403 (7.1%) | 1,806 (11.4%) | -0.15 |
| Lab values- Creatinine (mg/dl) v2; n (%) | 2,220 (20.3%) | 1,758 (27.3%) | -0.16 | 216 (0.9%) | 131 (1.4%) | -0.05 | N/A | N/A | #VALUE! | 2,436 (7.2%) | 1,889 (11.9%) | -0.16 |
| Lab values- Creatinine (mg/dl) (within 3 months) v2; | 1 5 (1 (14 30/) | 1 220 (10 20/) | -0.13 | 157 (0.70/) | 02 (1 00/) | -0.03 | N/A | N/A | #VALUE! | 1 710 (5 10/) | 1 220 (0 40/) | -0.13 |
| n (%) Lab values-Creatinine (mg/dl) (within 6 months) v2; | 1,561 (14.3%) | 1,238 (19.2%) | -0.13 | 157 (0.7%) | 92 (1.0%) | -0.03 | IN/A | N/A | #VALUE! | 1,718 (5.1%) | 1,330 (8.4%) | -0.13 |
| n (%) | 2,220 (20.3%) | 1,758 (27.3%) | -0.16 | 216 (0.9%) | 131 (1.4%) | -0.05 | N/A | N/A | #VALUE! | 2,436 (7.2%) | 1,889 (11.9%) | -0.16 |
| Lab values-HDL level (mg/dl); n (%) | 1,327 (12.1%) | 1,026 (15.9%) | -0.11 | 186 (0.8%) | 81 (0.9%) | -0.01 | N/A | N/A | #VALUE! | 1,513 (4.5%) | 1,107 (7.0%) | -0.11 |
| | , , , , , | , | | | , | | | | | , , | , . , . , | |
| Lab values-HDL level (mg/dl) (within 3 months); n (%) | 741 (6.8%) | 580 (9.0%) | -0.08 | 117 (0.5%) | 49 (0.5%) | 0.00 | N/A | N/A | #VALUE! | 858 (2.5%) | 629 (4.0%) | -0.08 |
| Lab values- HDL level (mg/dl) (within 6 months); n (%) | 1,327 (12.1%) | 1,026 (15.9%) | -0.11 | 186 (0.8%) | 81 (0.9%) | -0.01 | N/A | N/A | #VALUE! | 1,513 (4.5%) | 1,107 (7.0%) | -0.11 |
| Lab values-LDL level (mg/dl) v2; n (%) | 1,373 (12.6%) | 1,055 (16.4%) | -0.11 | 200 (0.9%) | 81 (0.9%) | 0.00 | N/A | N/A | #VALUE! | 1,573 (4.6%) | 1,136 (7.2%) | -0.11 |
| Lab values- LDL level (mg/dl) (within 3 months) v2; n | 762 (7.00() | 500 (0.20/) | 0.00 | 427 (0.00) | 40 (0 50() | 0.01 | **/* | | man until | 000 (2, 50() | C40 (4 40/) | 0.00 |
| (%) | 762 (7.0%) | 599 (9.3%) | -0.08 | 127 (0.6%) | 49 (0.5%) | 0.01 | N/A | N/A | #VALUE! | 889 (2.6%) | 648 (4.1%) | -0.08 |
| Lab values-LDL level (mg/dl) (within 6 months) v2; n<br>(%) | 1,373 (12.6%) | 1.055 (16.4%) | -0.11 | 200 (0.9%) | 81 (0.9%) | 0.00 | N/A | N/A | #VALUE! | 1,573 (4.6%) | 1,136 (7.2%) | -0.11 |
| Lab values- NT-proBNP: n (%) | 29 (0.3%) | 22 (0.3%) | 0.11 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | N/A | N/A | #VALUE! | 29 (0.1%) | 22 (0.1%) | 0.00 |
| Lab values- NT-proBNP (within 3 months); n (%) | 29 (0.3%) | 22 (0.3%) | 0.00 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | N/A | N/A | #VALUE! | 29 (0.1%) | 22 (0.1%) | - |
| Lab values- NT-proBNP (within 6 months); n (%) | 29 (0.3%) | 22 (0.3%) | 0.00 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | N/A | N/A | #VALUE! | 29 (0.1%) | 22 (0.1%) | _ |
| Lab values-Total cholesterol (mg/dl) v2; n (%) | 1,352 (12.4%) | 1,044 (16.2%) | -0.11 | 184 (0.8%) | 82 (0.9%) | -0.01 | N/A | N/A | #VALUE! | 1,536 (4.5%) | 1,126 (7.1%) | -0.11 |
| Lab values-Total cholesterol (mg/dl) (within 3 | | | | . , | , , | | * | • | | | | |
| months) v2; n (%) | 762 (7.0%) | 595 (9.2%) | -0.08 | 119 (0.5%) | 50 (0.5%) | 0.00 | N/A | N/A | #VALUE! | 881 (2.6%) | 645 (4.1%) | -0.08 |
| Lab values-Total cholesterol (mg/dl) (within 6 | | | | | | | | | | | | |
| months) v2; n (%) | 1,352 (12.4%) | 1,044 (16.2%) | -0.11 | 184 (0.8%) | 82 (0.9%) | -0.01 | N/A | N/A | #VALUE! | 1,536 (4.5%) | 1,126 (7.1%) | -0.11 |
| Lab values-Triglyceride level (mg/dl); n (%) | 1,335 (12.2%) | 1,038 (16.1%) | -0.11 | 177 (0.8%) | 80 (0.9%) | -0.01 | N/A | N/A | #VALUE! | 1,512 (4.5%) | 1,118 (7.1%) | -0.11 |

| Lab values-Triglyceride level (mg/dl) (within 3 | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| months); n (%) | 753 (6.9%) | 590 (9.2%) | -0.08 | 110 (0.5%) | 49 (0.5%) | 0.00 | N/A | N/A | #VALUE! | 863 (2.5%) | 639 (4.0%) | -0.08 |
| Lab values-Triglyceride level (mg/dl) (within 6 | | | | | | | | | | | | |
| months); n (%) | 1,335 (12.2%) | 1,038 (16.1%) | -0.11 | 177 (0.8%) | 80 (0.9%) | -0.01 | N/A | N/A | #VALUE! | 1,512 (4.5%) | 1,118 (7.1%) | -0.11 |
| Lab result number- HbA1c (%) mean (only 2 to 20 included) v4 | 876 | 776 | | 164 | 80 | | N/A | N/A | | 1.040 | 856 | |
| mean (sd) | 6.67 (1.48) | 6.52 (1.50) | 0.10 | 7.09 (1.41) | 7.06 (1.75) | 0.02 | N/A | N/A | #VALUE! | 6.74 (1.47) | 6.57 (1.53) | 0.11 |
| Missing; n (%) | 10,060 (92.0%) | 5,672 (88.0%) | 0.13 | 22,876 (99.3%) | 9,325 (99.1%) | 0.02 | N/A | N/A | #VALUE! | 32,936 (96.9%) | 14,997 (94.6%) | 0.11 |
| Lab result number- BNP mean v2 | 96 | 85 | | 8 | 6 | | N/A | N/A | | 104 | 91 | |
| mean (sd) | 83.18 (129.35) | 114.60 (175.32) | -0.20 | 70.15 (59.71) | 47.52 (53.77) | 0.40 | N/A | N/A | #VALUE! | 82.18 (126.43) | 110.18 (171.77) | -0.19 |
| Missing; n (%) | 10,840 (99.1%) | 6,363 (98.7%) | 0.04 | 23,032 (100.0%) | 9,399 (99.9%) | 0.04 | N/A | N/A | #VALUE! | 33,872 (99.7%) | 15,762 (99.4%) | 0.04 |
| Lab result number- BUN (mg/dl) mean v2 | 2,195 | 1,688 | | 208 | 118 | | N/A | N/A | | 2,403 | 1,806 | |
| mean (sd) | 17.31 (6.76) | 16.03 (5.52) | 0.21 | 1,651.89 (16,887.31) | 1,033.14 (11,045.39) | 0.04 | N/A | N/A | #VALUE! | 158.80 (4959.53) | 82.49 (2813.69) | 0.02 |
| Missing; n (%) | 8,741 (79.9%) | 4,760 (73.8%) | 0.15 | 22,832 (99.1%) | 9,287 (98.7%) | 0.04 | N/A | N/A | #VALUE! | 31,573 (92.9%) | 14,047 (88.6%) | 0.15 |
| Lab result number- Creatinine (mg/dl) mean (only 0.1 | 2.405 | 4 705 | | 206 | 420 | | N/A | | | 2 404 | 4.054 | |
| to 15 included) v3<br>mean (sd) | 2,195<br>0.97 (0.30) | 1,735<br>0.94 (0.23) | 0.11 | 1.00 (0.33) | 129<br>0.95 (0.24) | 0.17 | N/A<br>N/A | N/A<br>N/A | #VALUE! | 2,401<br>0.97 (0.30) | 1,864<br>0.94 (0.23) | 0.11 |
| Missing; n (%) | 8,741 (79.9%) | 4,713 (73.1%) | 0.11 | 22,834 (99.1%) | 9,276 (98.6%) | 0.05 | N/A | N/A | #VALUE! | 31,575 (92.9%) | 13,989 (88.2%) | 0.11 |
| Lab result number- HDL level (mg/dl) mean (only | 0,741 (75.570) | 4,713 (73.170) | 0.10 | 22,034 (33.170) | 3,270 (30.0%) | 0.03 | 14/1 | 19/0 | #VALUE: | 31,373 (32.370) | 13,303 (00.270) | 0.10 |
| =<5000 included) v2 | 1,327 | 1,026 | | 185 | 80 | | N/A | N/A | | 1,512 | 1,106 | |
| mean (sd) | 53.56 (16.61) | 52.84 (16.18) | 0.04 | 47.72 (21.06) | 49.04 (15.24) | -0.07 | N/A | N/A | #VALUE! | 52.85 (17.22) | 52.57 (16.12) | 0.02 |
| Missing; n (%) | 9,609 (87.9%) | 5,422 (84.1%) | 0.11 | 22,855 (99.2%) | 9,325 (99.1%) | 0.01 | N/A | N/A | #VALUE! | 32,464 (95.5%) | 14,747 (93.0%) | 0.11 |
| Lab result number- LDL level (mg/dl) mean (only | | | | | | | | | | | | |
| =<5000 included) v2 | 1,353 | 1,033 | | 176 | 76 | | N/A | N/A | | 1,529 | 1,109 | |
| mean (sd) | 102.31 (36.16) | 106.34 (37.86) | -0.11 | 94.29 (41.51) | 103.08 (42.40) | -0.21 | N/A | N/A | #VALUE! | 101.39 (36.82) | 106.12 (38.20) | -0.13 |
| Missing; n (%) | 9,583 (87.6%) | 5,415 (84.0%) | 0.10 | 22,864 (99.2%) | 9,329 (99.2%) | 0.00 | N/A | N/A | #VALUE! | 32,447 (95.5%) | 14,744 (93.0%) | 0.11 |
| Lab result number-Total cholesterol (mg/dl) mean<br>(only =<5000 included) v2 | 1,349 | 1.042 | | 183 | 81 | | N/A | N/A | | 1,532 | 1,123 | |
| mean (sd) | 185.42 (39.77) | 188.13 (42.80) | -0.07 | 178.14 (56.57) | 184.42 (43.66) | -0.12 | N/A | N/A | #VALUE! | 184.55 (42.13) | 187.86 (42.88) | -0.08 |
| Missing; n (%) | 9,587 (87.7%) | 5,406 (83.8%) | 0.11 | 22,857 (99.2%) | 9,324 (99.1%) | 0.01 | N/A | N/A | #VALUE! | 32,444 (95.5%) | 14,730 (92.9%) | 0.11 |
| Lab result number- Triglyceride level (mg/dl) mean | 0,000 (00000) | 0,100 (001011) | | ,, | -, (, | | | .4 | | , (, | | |
| (only =<5000 included) v2 | 1,335 | 1,038 | | 176 | 79 | | N/A | N/A | | 1,511 | 1,117 | |
| mean (sd) | 140.09 (77.34) | 141.14 (97.23) | -0.01 | 160.11 (109.08) | 146.12 (89.21) | 0.14 | N/A | N/A | #VALUE! | 142.42 (81.68) | 141.49 (96.73) | 0.01 |
| Missing; n (%) | 9,601 (87.8%) | 5,410 (83.9%) | 0.11 | 22,864 (99.2%) | 9,326 (99.2%) | 0.00 | N/A | N/A | #VALUE! | 32,465 (95.6%) | 14,736 (93.0%) | 0.11 |
| Lab result number- Hemoglobin mean (only >0 | | | | | | | | | | | | |
| included) | 1,839 | 1,402 | | 151 | 100 | | N/A | N/A | | 1,990 | 1,502 | |
| mean (sd) | 13.53 (1.77) | 13.58 (1.78) | -0.03 | 1,820.49 (15,673.46) | 1,503.13 (14,898.67) | 0.02 | N/A | N/A | #VALUE! | 150.64 (4306.37) | 112.75 (3828.81) | 0.01 |
| Missing; n (%) | 9,097 (83.2%) | 5,046 (78.3%) | 0.12 | 22,889 (99.3%) | 9,305 (98.9%) | 0.04 | N/A | N/A | #VALUE! | 31,986 (94.1%) | 14,351 (90.5%) | 0.14 |
| Lab result number- Serum sodium mean (only >90 and <190 included) | 2,155 | 1,663 | | 179 | 121 | | N/A | N/A | | 2,334 | 1,784 | |
| mean (sd) | 139.90 (2.72) | 140.21 (2.61) | -0.12 | 139.33 (2.67) | 139.44 (2.48) | -0.04 | N/A | N/A | #VALUE! | 139.86 (2.72) | 140.16 (2.60) | -0.11 |
| Missing; n (%) | 8,781 (80.3%) | 4,785 (74.2%) | 0.15 | 22,861 (99.2%) | 9,284 (98.7%) | 0.05 | N/A | N/A | #VALUE! | 31,642 (93.1%) | 14,069 (88.7%) | 0.15 |
| Lab result number- Albumin mean (only >0 and <=10 | ., . , , | ,, | | , , , | ., . , . , | | | | | | , ( , | |
| included) | 1,961 | 1,522 | | 153 | 97 | | N/A | N/A | | 2,114 | 1,619 | |
| mean (sd) | 4.09 (0.37) | 4.14 (0.37) | -0.14 | 3.86 (0.90) | 4.11 (0.56) | -0.33 | N/A | N/A | #VALUE! | 4.07 (0.43) | 4.14 (0.38) | -0.17 |
| Missing; n (%) | 8,975 (82.1%) | 4,926 (76.4%) | 0.14 | 22,887 (99.3%) | 9,308 (99.0%) | 0.03 | N/A | N/A | #VALUE! | 31,862 (93.8%) | 14,234 (89.8%) | 0.15 |
| Lab result number- Glucose (fasting or random) mean | 2445 | 1.640 | | 450 | 125 | | N/A | 21/2 | | 2 202 | 4.705 | |
| (only 10-1000 included) | 2,115<br>111.04 (41.01) | 1,640 | 0.01 | 168<br>134.34 (55.53) | | -0.09 | N/A<br>N/A | N/A<br>N/A | #VALUE! | 2,283<br>112.75 (42.25) | 1,765<br>112.86 (45.91) | 0.00 |
| mean (sd)<br>Missing; n (%) | 8,821 (80.7%) | 4,808 (74.6%) | 0.01 | 22,872 (99.3%) | 141.41 (91.92)<br>9,280 (98.7%) | 0.09 | N/A<br>N/A | N/A<br>N/A | #VALUE! | 31,693 (93.3%) | 14,088 (88.9%) | 0.00 |
| Lab result number- Potassium mean (only 1-7 | 8,821 (80.7%) | 4,000 (74.0%) | 0.13 | 22,072 (33.370) | 5,280 (58.7%) | 0.00 | N/A | N/A | #VALUE: | 31,093 (93.370) | 14,000 (00.5%) | 0.13 |
| included) | 2,197 | 1,722 | | 198 | 114 | | N/A | N/A | | 2,395 | 1,836 | |
| mean (sd) | 4.30 (0.42) | 4.35 (0.41) | -0.12 | 4.30 (0.36) | 4.28 (0.38) | 0.05 | N/A | N/A | #VALUE! | 4.30 (0.42) | 4.35 (0.41) | -0.12 |
| Missing; n (%) | 8,739 (79.9%) | 4,726 (73.3%) | 0.16 | 22,842 (99.1%) | 9,291 (98.8%) | 0.03 | N/A | N/A | #VALUE! | 31,581 (93.0%) | 14,017 (88.4%) | 0.16 |
| Comorbidity Scores | | | | | | | | | | | | |
| Combined comorbidity score, 365 days Copy | | | | | | | | | | | | |
| mean (sd) | 2.25 (2.33) | 2.73 (2.22) | -0.21 | 1.41 (1.99) | 1.88 (1.99) | -0.24 | 2.36 (2.34) | 2.51 (2.28) | -0.06 | 2.01 (2.22) | 2.37 (2.19) | -0.16 |
| Non-Frailty; n (%) | 5,267 (48.2%) | 3,125 (48.5%) | -0.01 | 9,522 (41.3%) | 4,016 (42.7%) | -0.03 | 1,353 (4.1%) | 507 (3.1%) | 0.05 | 16,142 (24.1%) | 7,648 (23.8%) | 0.01 |
| Frailty Score (mean): Empirical Version 365 days, v2mean (sd) | 0.18 (0.06) | 0.17 (0.06) | 0.17 | 0.16 (0.05) | 0.16 (0.05) | 0.00 | 0.10 (0.07) | 0.08 (0.06) | 0.31 | 0.13 (0.06) | 0.12 (0.06) | 0.17 |
| Healthcare Utilization | 0.18 (0.06) | 0.17 (0.06) | 0.17 | 0.16 (0.05) | 0.16 (0.05) | 0.00 | 0.10 (0.07) | 0.08 (0.06) | 0.31 | 0.13 (0.06) | 0.12 (0.06) | 0.17 |
| Any hospitalization; n (%) | 10,386 (95.0%) | 5,867 (91.0%) | 0.16 | 23.039 (100.0%) | 9,405 (100.0%) | #DIV/0! | 31,398 (95.4%) | 14.394 (88.7%) | 0.25 | 64,823 (96.9%) | 29,666 (92.5%) | 0.20 |
| Any hospitalization, it (%) Any hospitalization within prior 30 days; n (%) | 10,182 (93.1%) | 5,761 (89.3%) | 0.13 | 22,949 (99.6%) | 9,381 (99.7%) | -0.02 | 31,156 (94.7%) | 14,174 (87.4%) | 0.26 | 64287 (96.1%) | 29316 (91.4%) | 0.20 |
| Any hospitalization during prior 31-180 days; n (%) | 1,130 (10.3%) | 570 (8.8%) | 0.05 | 2,018 (8.8%) | 685 (7.3%) | 0.06 | 4,474 (13.6%) | 1,925 (11.9%) | 0.05 | 7622 (11.4%) | 3180 (9.9%) | 0.05 |
| Internal medicine/family medicine visits; n (%) | 9,617 (87.9%) | 5,557 (86.2%) | 0.05 | 17,146 (74.4%) | 7,369 (78.4%) | -0.09 | 31,976 (97.2%) | 15,692 (96.7%) | 0.03 | 58739 (87.8%) | 28618 (89.2%) | -0.04 |
| Internal medicine/family medicine visits (30 days | | | | | | | | | | | | |
| prior) v2; n (%) | 8,754 (80.0%) | 4,965 (77.0%) | 0.07 | 12,150 (52.7%) | 5,278 (56.1%) | -0.07 | 30,917 (94.0%) | 15,037 (92.7%) | 0.05 | 51821 (77.5%) | 25280 (78.8%) | -0.03 |
| Internal medicine/family medicine visits (31 to 180 | | | | | | | | | | | | |
| days prior) v2; n (%) | 6,709 (61.3%) | 3,740 (58.0%) | 0.07 | 13,848 (60.1%) | 5,879 (62.5%) | -0.05 | 23,994 (72.9%) | 11,647 (71.8%) | 0.02 | 44551 (66.6%) | 21266 (66.3%) | 0.01 |
| Cardiologist visit; n (%) | 7,333 (67.1%) | 4,602 (71.4%) | -0.09 | 5,677 (24.6%) | 2,412 (25.6%) | -0.02 | 23,928 (72.7%) | 11,816 (72.8%) | 0.00 | 36938 (55.2%) | 18830 (58.7%) | -0.07 |
| Number of Cardiologist visits (30 days prior); n (%)<br>Number of Cardiologist visits (31 to 180 days prior); | 6,782 (62.0%) | 4,321 (67.0%) | -0.10 | 3,914 (17.0%) | 1,712 (18.2%) | -0.03 | 21,746 (66.1%) | 10,824 (66.7%) | -0.01 | 32442 (48.5%) | 16857 (52.6%) | -0.08 |
| n (%) | 1,801 (16.5%) | 1,015 (15.7%) | 0.02 | 2,586 (11.2%) | 1,016 (10.8%) | 0.01 | 8,054 (24.5%) | 3.822 (23.6%) | 0.02 | 12441 (18.6%) | 5853 (18.2%) | 0.01 |
| Electrocardiogram v2; n (%) | 9,068 (82.9%) | 5,511 (85.5%) | -0.07 | 11,511 (50.0%) | 4,535 (48.2%) | 0.04 | 28,595 (86.9%) | 14,289 (88.1%) | -0.04 | 49174 (73.5%) | 24335 (75.9%) | -0.06 |
| Use of glucose test strips; n (%) | 137 (1.3%) | 75 (1.2%) | 0.01 | 213 (0.9%) | 65 (0.7%) | 0.02 | 393 (1.2%) | 196 (1.2%) | 0.00 | 743 (1.1%) | 336 (1.0%) | 0.01 |
| Dialysis; n (%) | ** (0.1%) | 0 (0.0%) | 0.04 | 15 (0.1%) | ** (0.0%) | 0.04 | 15 (0.0%) | ** (0.0%) | #DIV/0! | #VALUE! | #VALUE! | #VALUE! |

| t defendable and the second second | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| number of different/distinct medication<br>prescriptions | | | | | | | | | | | | |
| mean (sd) | 8.99 (5.19) | 8.21 (5.39) | 0.15 | 8.84 (5.26) | 8.08 (5.41) | 0.14 | 10.02 (4.85) | 9.34 (4.92) | 0.14 | 9.44 (5.05) | 8.74 (5.16) | 0.00 |
| Number of Hospitalizations | | | | | | | | | | | | |
| mean (sd) | 1.15 (0.58) | 1.08 (0.60) | 0.12 | 1.20 (0.54) | 1.17 (0.49) | 0.06 | 1.25 (0.69) | 1.13 (0.69) | 0.17 | 1.22 (0.62) | 1.13 (0.62) | 0.00 |
| Number of hospital days | | | | | | | | | | | | |
| mean (sd) | 5.90 (4.96) | 4.14 (4.04) | 0.39 | 6.36 (5.37) | 4.38 (4.12) | 0.41 | 6.79 (5.61) | 4.71 (4.84) | 0.40 | 6.50 (5.43) | 4.50 (4.48) | 0.00 |
| Number of Emergency Department (ED) visits v3 | | | | | | | | | | | | |
| mean (sd) | 1.48 (2.03) | 1.64 (2.60) | -0.07 | 2.38 (4.05) | 3.03 (4.79) | -0.15 | 1.67 (1.89) | 1.72 (1.95) | -0.03 | 1.88 (2.84) | 2.09 (3.16) | 0.00 |
| Number of Office visits | F 00 (4 C2) | F 06 (4 F0) | 0.01 | 4.01 (4.57) | 4 01 (4 40) | 0.02 | 42.07/42.50\ | 12 50 (14 24) | 0.05 | 0.00(40.07) | 0.26 (10.61) | 0.00 |
| mean (sd) Number of internal medicine/family medicine visits | 5.09 (4.63) | 5.06 (4.50) | 0.01 | 4.91 (4.57) | 4.81 (4.49) | 0.02 | 12.87 (13.58) | 13.50 (14.24) | -0.05 | 8.86 (10.07) | 9.26 (10.61) | 0.00 |
| mean (sd) | 10.30 (14.53) | 8.38 (11.56) | 0.15 | 5.49 (9.54) | 5.56 (8.69) | -0.01 | 12.43 (10.76) | 10.74 (10.42) | 0.16 | 9.69 (11.08) | 8.75 (10.19) | 0.00 |
| Number of Cardiologist visits | () | 0.00 (22.00) | | | () | | | | | () | (20.20) | |
| mean (sd) | 2.16 (3.37) | 2.17 (3.04) | 0.00 | 0.62 (1.75) | 0.62 (1.88) | 0.00 | 2.70 (3.86) | 2.65 (4.01) | 0.01 | 1.90 (3.20) | 1.96 (3.32) | 0.00 |
| Number electrocardiograms received v2 | | | | | | | | | | | | |
| mean (sd) | 1.86 (1.92) | 1.94 (1.89) | -0.04 | 0.85 (1.16) | 0.84 (1.31) | 0.01 | 1.98 (1.70) | 2.07 (1.69) | -0.05 | 1.57 (1.58) | 1.68 (1.63) | 0.00 |
| Number of HbA1c tests ordered | | | | | | | | | | | | |
| mean (sd) | 0.27 (0.59) | 0.31 (0.63) | -0.07 | 0.18 (0.49) | 0.21 (0.51) | -0.06 | 0.34 (0.66) | 0.36 (0.67) | -0.03 | 0.27 (0.59) | 0.31 (0.62) | 0.00 |
| Number of glucose tests ordered | 0.47 (0.05) | 0.20(4.74) | 0.02 | 0.43 (0.65) | 0.40 (0.70) | 0.00 | 0.44(0.57) | 0.44(0.55) | | 0.44(0.60) | 0.44(0.04) | 0.00 |
| mean (sd) Number of lipid tests ordered | 0.17 (0.96) | 0.20 (1.71) | -0.02 | 0.12 (0.65) | 0.10 (0.70) | 0.03 | 0.14 (0.57) | 0.14 (0.55) | 0.00 | 0.14 (0.68) | 0.14 (0.94) | 0.00 |
| mean (sd) | 0.46 (0.71) | 0.45 (0.88) | 0.01 | 0.34 (0.71) | 0.36 (0.78) | -0.03 | 0.54 (0.69) | 0.56 (0.73) | -0.03 | 0.46 (0.70) | 0.48 (0.78) | 0.00 |
| Total N distinct ICD9/ICD10 diagnoses at the 3rd | 0.40 (0.71) | 0.45 (0.00) | 0.01 | 0.54 (0.72) | 0.50 (0.70) | 0.03 | 0.54 (0.05) | 0.50 (0.75) | 0.03 | 0.40 (0.70) | 0.40 (0.70) | 0.00 |
| digit level Copy | | | | | | | | | | | | |
| mean (sd) | 7.42 (9.86) | 11.16 (11.73) | -0.35 | 5.13 (8.66) | 7.50 (9.39) | -0.26 | 11.08 (11.96) | 13.57 (12.42) | -0.20 | 8.43 (10.59) | 11.31 (11.47) | 0.00 |
| For PS | | | | | | | | | | | | |
| Hemorrhagic stroke+Other cerebrovascular | | | | | | | | | | | | |
| disease+Cerebrovascular procedure (for PS); n (%) | 173 (1.6%) | 60 (0.9%) | 0.06 | 180 (0.8%) | 61 (0.6%) | 0.02 | 748 (2.3%) | 273 (1.7%) | 0.04 | 1101 (1.6%) | 394 (1.2%) | 0.03 |
| immobilization; n (%) | 780 (7.1%) | 455 (7.1%) | #DIV/0! | 1,525 (6.6%) | 567 (6.0%) | #DIV/0! | 2,026 (6.2%) | 982 (6.1%) | #DIV/0! | 1,525 (6.6%) | 567 (6.0%) | 0.02 |
| Occurrence of creatinine tests ordered (for PS); n (%) | 840 (7.7%) | 422 (6.5%) | 0.05 | 1,609 (7.0%) | 497 (5.3%) | 0.07 | 3,658 (11.1%) | 1,608 (9.9%) | 0.04 | 6107 (9.1%) | 2527 (7.9%) | 0.04 |
| Occurrence of BUN tests ordered (for PS); n (%) | 426 (3.9%) | 179 (2.8%) | 0.06 | 852 (3.7%) | 261 (2.8%) | 0.05 | 1,920 (5.8%) | 811 (5.0%) | 0.04 | 3198 (4.8%) | 1251 (3.9%) | 0.04 |
| Occurrence of chronic renal insufficiency w/o CKD | , | | | , | . , , | | , , | , | | , | , | |
| (for PS) v2; n (%) | 635 (5.8%) | 227 (3.5%) | 0.11 | 613 (2.7%) | 177 (1.9%) | 0.05 | 2,501 (7.6%) | 749 (4.6%) | 0.13 | 3749 (5.6%) | 1153 (3.6%) | 0.10 |
| Chronic kidney disease Stage 1-2 (for PS); n (%) | 204 (1.9%) | 124 (1.9%) | 0.00 | 181 (0.8%) | 65 (0.7%) | 0.01 | 560 (1.7%) | 260 (1.6%) | 0.01 | 945 (1.4%) | 449 (1.4%) | 0.00 |
| Chronic kidney disease Stage 3-6 (for PS); n (%) | 714 (6.5%) | 311 (4.8%) | 0.07 | 599 (2.6%) | 178 (1.9%) | 0.05 | 2,836 (8.6%) | 999 (6.2%) | 0.09 | 4149 (6.2%) | 1488 (4.6%) | 0.07 |
| Acute kidney injury; n (%) | 1,115 (10.2%) | 505 (7.8%) | #DIV/0! | 1,462 (6.3%) | 549 (5.8%) | #DIV/0! | 3,684 (11.2%) | 1,487 (9.2%) | #DIV/0! | 1,462 (6.3%) | 549 (5.8%) | 0.02 |
| Bladder stones+Kidney stones (for PS); n (%) | 374 (3.4%) | 185 (2.9%) | 0.03 | 645 (2.8%) | 281 (3.0%) | -0.01 | 1,094 (3.3%) | 554 (3.4%) | -0.01 | 2113 (3.2%) | 1020 (3.2%) | 0.00 |
| Alcohol abuse or dependence+Drug abuse or<br>dependence (for PS); n (%) | 531 (4.9%) | 350 (5.4%) | -0.02 | 759 (3.3%) | 358 (3.8%) | -0.03 | 534 (1.6%) | 442 (2.7%) | -0.08 | 1824 (2.7%) | 1150 (3.6%) | -0.05 |
| Other atherosclerosis+Cardiac conduction | 332 (4.370) | 330 (3.470) | 0.02 | 755 (5.570) | 330 (3.670) | 0.03 | 334 (2.070) | 442 (2.770) | 0.00 | 1024 (2.770) | 1130 (3.074) | 0.03 |
| disorders+Other CVD (for PS) v2 Copy; n (%) | 3,257 (29.8%) | 1,919 (29.8%) | 0.00 | 5,127 (22.3%) | 2,292 (24.4%) | -0.05 | 9,987 (30.4%) | 4,973 (30.7%) | -0.01 | 18371 (27.5%) | 9184 (28.6%) | -0.02 |
| Previous cardiac procedure (CABG or PTCA or Stent) + | | | | | | | | | | | | |
| History of CABG or PTCA (for PS) v3; n (%) | 430 (3.9%) | 255 (4.0%) | -0.01 | 372 (1.6%) | 131 (1.4%) | 0.02 | 2,889 (8.8%) | 1,360 (8.4%) | 0.01 | 3691 (5.5%) | 1746 (5.4%) | 0.00 |
| Diabetes with complication; n (%) | 763 (7.0%) | 462 (7.2%) | #DIV/0! | 960 (4.2%) | 391 (4.2%) | #DIV/0! | 2,595 (7.9%) | 1,165 (7.2%) | #DIV/0! | 960 (4.2%) | 391 (4.2%) | 0.00 |
| Delirium + Psychosis (for PS); n (%) | 519 (4.7%) | 244 (3.8%) | 0.04 | 578 (2.5%) | 219 (2.3%) | 0.01 | 1,846 (5.6%) | 744 (4.6%) | 0.05<br>0.00 | 2943 (4.4%)<br>#VALUE! | 1207 (3.8%) | 0.03 |
| Any use of Meglitinides (for PS); n (%)<br>Any use of AGIs (for PS); n (%) | ** (0.1%)<br>** (0.1%) | ** (0.1%)<br>** (0.0%) | 0.00 | 26 (0.1%)<br>** (0.0%) | ** (0.1%)<br>** (0.0%) | #DIV/0! | 92 (0.3%)<br>12 (0.0%) | 46 (0.3%)<br>** (0.0%) | #DIV/0! | #VALUE! | #VALUE!<br>#VALUE! | #VALUE!<br>#VALUE! |
| CKD stage 3-6 + dialysis (for PS); n (%) | 725 (6.6%) | 313 (4.9%) | 0.04 | 612 (2.7%) | 179 (1.9%) | 0.05 | 2,844 (8.6%) | 1,001 (6.2%) | 0.09 | 4181 (6.3%) | 1493 (4.7%) | #VALUE: |
| Use of thiazide- United: n (%) | 1.000 (9.1%) | 520 (8.1%) | 0.04 | 1,829 (7.9%) | 626 (6.7%) | 0.05 | 4,263 (13.0%) | 1,863 (11.5%) | 0.05 | 7092 (10.6%) | 3009 (9.4%) | 0.04 |
| Use of beta blockers; n (%) | 2,546 (23.3%) | 1,195 (18.5%) | 0.12 | 4,775 (20.7%) | 1,650 (17.5%) | 0.08 | 11,795 (35.9%) | 5,207 (32.1%) | 0.08 | 19116 (28.6%) | 8052 (25.1%) | 0.08 |
| Use of calcium channel blockers; n (%) | 1,956 (17.9%) | 1,041 (16.1%) | 0.05 | 3,644 (15.8%) | 1,257 (13.4%) | 0.07 | 8,899 (27.1%) | 4,117 (25.4%) | 0.04 | 14499 (21.7%) | 6415 (20.0%) | 0.04 |
| All antidiabetic medications except Insulin; n (%) | 1,455 (13.3%) | 785 (12.2%) | 0.03 | 2,636 (11.4%) | 1,060 (11.3%) | 0.00 | 5,181 (15.8%) | 2,409 (14.8%) | 0.03 | 9272 (13.9%) | 4254 (13.3%) | 0.02 |
| DM Medications - Insulin Copy; n (%) | 492 (4.5%) | 257 (4.0%) | 0.02 | 963 (4.2%) | 323 (3.4%) | 0.04 | 1,236 (3.8%) | 539 (3.3%) | 0.03 | 2691 (4.0%) | 1119 (3.5%) | 0.03 |
| Use of Low Intensity Statins; n (%) | 2,224 (20.3%) | 1,095 (17.0%) | 0.08 | 3,726 (16.2%) | 1,295 (13.8%) | 0.07 | 10,072 (30.6%) | 4,682 (28.9%) | 0.04 | 16022 (24.0%) | 7072 (22.0%) | 0.05 |
| Use of High Intensity Statins; n (%) | 1,150 (10.5%)<br>730 (6.7%) | 813 (12.6%)<br>162 (2.5%) | -0.07<br>0.20 | 2,135 (9.3%)<br>9,082 (39.4%) | 897 (9.5%)<br>2,310 (24.6%) | -0.01<br>0.32 | 4,789 (14.6%)<br>15,204 (46.2%) | 2,689 (16.6%)<br>4,630 (28.5%) | -0.06<br>0.37 | 8074 (12.1%)<br>25016 (37.4%) | 4399 (13.7%)<br>7102 (22.1%) | -0.05<br>0.34 |
| Malignant hypertension; n (%)<br>Cardiovascular stress test; n (%) | 730 (6.7%)<br>78 (0.7%) | 162 (2.5%)<br>29 (0.4%) | 0.20 | 9,082 (39.4%) | 2,310 (24.6%)<br>44 (0.5%) | 0.32 | 15,204 (46.2%)<br>350 (1.1%) | 4,630 (28.5%)<br>201 (1.2%) | -0.01 | 25016 (37.4%)<br>563 (0.8%) | 7102 (22.1%)<br>274 (0.9%) | -0.01 |
| Echocardiogram; n (%) | 5,787 (52.9%) | 3,803 (59.0%) | -0.12 | 11,855 (51.5%) | 5,539 (58.9%) | -0.15 | 18,098 (55.0%) | 9,340 (57.6%) | -0.01 | 35740 (53.4%) | 18682 (58.2%) | -0.01 |
| Number of BNP tests | ., , | .,, | | ,, | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | | .,, | , | | , | | |
| mean (sd) | 0.10 (0.35) | 0.15 (0.44) | -0.13 | 0.09 (0.34) | 0.11 (0.36) | -0.06 | 0.14 (0.40) | 0.17 (0.44) | -0.07 | 0.12 (0.37) | 0.15 (0.42) | -0.08 |
| Number of Cardiac biomarkers tests (tropnin, CK-MBs, My | | | | | | | | | | g | | |
| mean (sd) | 0.42 (1.41) | 0.52 (1.28) | -0.07 | 0.35 (1.09) | 0.40 (1.24) | -0.04 | 0.30 (0.61) | 0.37 (0.67) | -0.11 | 0.34 (0.96) | 0.41 (1.00) | 0.00 |
| Number of Ambulatory Blood pressure monitoring tests | | | | | | | | | | | | |
| mean (sd) | 0.00 (0.04) | 0.00 (0.03) | 0.00 | 0.00 (0.04) | 0.00 (0.03) | 0.00 | 0.00 (0.02) | 0.00 (0.00) | 0.00 | 0.00 (0.03) | 0.00 (0.02) | 0.00 |
| | 0.00 (0.04) | 0.00 (0.03) | 5.50 | 0.00 (0.04) | 0.00 (0.03) | 0.00 | 3.55 (3.52) | 0.00 (0.00) | 0.00 | 0.00 (0.03) | 0.00 (0.02) | 0.00 |
| N of days on antihypertensive medications during baseline | 2 | | | | | | | | | | | |
| mean (sd) | 74.82 (79.61) | 70.24 (79.86) | 0.06 | 65.26 (78.27) | 58.82 (76.61) | 0.08 | 111.76 (76.90) | 108.30 (78.35) | 0.04 | 89.70 (77.82) | 86.14 (78.15) | 0.00 |
| N of days in database anytime prior | | | | | | | | | | | | |
| mean (sd) | 1,672.96 (1,192.85) | 1,774.82 (1,375.50) | -0.08 | 1,771.15 (1,221.31) | 2,056.97 (1,425.75) | -0.22 | 637.26 (351.73) | 659.79 (336.35) | -0.07 | 1197.31 (898.59) | 1293.60 (1016.64) | 0.00 |
| Moon Consular nor properiation and Johannesis 115 63/4 | 90 1 day aria-\ | | | | | | | | | | | |
| Mean Copay for per prescription cost (charges in U.S. \$) (1mean (sd) | 80-1 day prior)<br>23.14 (33.19) | 20.04 (30.76) | 0.10 | 16.79 (25.44) | 13.74 (31.23) | 0.11 | 110.77 (126.57) | 109.04 (134.46) | 0.01 | 64.06 (91.02) | 63.21 (98.08) | 0.00 |
| Missing; n (%) | 801 (7.3%) | 538 (8.3%) | -0.04 | 1,853 (8.0%) | 874 (9.3%) | -0.05 | 996 (3.0%) | 523 (3.2%) | -0.01 | 3650 (5.5%) | 1935 (6.0%) | -0.02 |
| ······0/ ·· · · · · / | 202 (7.370) | 250 (0.570) | 0.04 | _,555 (6.678) | 3, 4 (3.3,0) | 0.03 | 330 (3.370) | (5.270) | 0.01 | 2330 (3.370) | _333 (0.070) | 0.02 |

| Colonoscopy; n (%) | 409 (3.7%) | 230 (3.6%) | 0.01 | 966 (4.2%) | 347 (3.7%) | 0.03 | 1,620 (4.9%) | 772 (4.8%) | 0.00 | 2995 (4.5%) | 1349 (4.2%) | 0.01 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Fecal occult blood (FOB) test; n (%) | 340 (3.1%) | 183 (2.8%) | 0.02 | 886 (3.8%) | 308 (3.3%) | 0.03 | 937 (2.8%) | 436 (2.7%) | 0.01 | 2163 (3.2%) | 927 (2.9%) | 0.02 |
| Flu vaccine; n (%) | 1,631 (14.9%) | 967 (15.0%) | 0.00 | 2,149 (9.3%) | 1,007 (10.7%) | -0.05 | 10,466 (31.8%) | 5,207 (32.1%) | -0.01 | 14246 (21.3%) | 7181 (22.4%) | -0.03 |
| Mammogram; n (%) | 1,237 (11.3%) | 704 (10.9%) | 0.01 | 2,232 (9.7%) | 938 (10.0%) | -0.01 | 4,385 (13.3%) | 2,227 (13.7%) | -0.01 | 7854 (11.7%) | 3869 (12.1%) | -0.01 |
| Pap smear; n (%) | 651 (6.0%) | 384 (6.0%) | 0.00 | 1,873 (8.1%) | 773 (8.2%) | 0.00 | 963 (2.9%) | 514 (3.2%) | -0.02 | 3487 (5.2%) | 1671 (5.2%) | 0.00 |
| Pneumonia vaccine; n (%) | 1,134 (10.4%) | 1,158 (18.0%) | -0.22 | 988 (4.3%) | 793 (8.4%) | -0.17 | 6,053 (18.4%) | 4,358 (26.9%) | -0.20 | 8175 (12.2%) | 6309 (19.7%) | -0.21 |
| PSA test or Prostate exam for DRE; n (%) | 1,083 (9.9%) | 690 (10.7%) | -0.03 | 1,944 (8.4%) | 818 (8.7%) | -0.01 | 3,705 (11.3%) | 2,058 (12.7%) | -0.04 | 6732 (10.1%) | 3566 (11.1%) | -0.03 |
| Bone mineral density; n (%) | 317 (2.9%) | 200 (3.1%) | -0.01 | 396 (1.7%) | 143 (1.5%) | 0.02 | 1,608 (4.9%) | 809 (5.0%) | 0.00 | 2321 (3.5%) | 1152 (3.6%) | -0.01 |
| Use of CNS stimulants; n (%) | 85 (0.8%) | 70 (1.1%) | -0.03 | 335 (1.5%) | 129 (1.4%) | 0.01 | 133 (0.4%) | 72 (0.4%) | 0.00 | 553 (0.8%) | 271 (0.8%) | 0.00 |
| Use of estrogens, progestins, androgens; n (%) | 1,084 (9.9%) | 683 (10.6%) | -0.02 | 3,192 (13.9%) | 1,414 (15.0%) | -0.03 | 1,380 (4.2%) | 655 (4.0%) | 0.01 | 5656 (8.5%) | 2752 (8.6%) | 0.00 |
| Use of Angiogenesis inhibitors; n (%) | ** (0.1%) | ** (0.0%) | 0.04 | 18 (0.1%) | ** (0.0%) | 0.04 | 21 (0.1%) | ** (0.0%) | 0.04 | #VALUE! | #VALUE! | #VALUE! |
| Use of Oral Immunosuppressants; n (%) | 24 (0.2%) | ** (0.2%) | 0.00 | 75 (0.3%) | 18 (0.2%) | 0.02 | 20 (0.1%) | ** (0.1%) | 0.00 | 119 (0.2%) | #VALUE! | #VALUE! |
| Use of fondaparinux or Bivalirudin; n (%) | 137 (1.3%) | ** (0.1%) | 0.14 | 430 (1.9%) | 15 (0.2%) | 0.17 | 250 (0.8%) | ** (0.1%) | 0.10 | 817 (1.2%) | #VALUE! | #VALUE! |
| Use of other direct thrombin inhibitors (lepirudin, | | | | | | | | | | | | |
| desirudin, argatroban); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Use of Ticagrelor ON CED; n (%) | ** (0.0%) | ** (0.1%) | -0.04 | ** (0.0%) | ** (0.0%) | #DIV/0! | 0 (0.0%) | ** (0.0%) | #DIV/0! | #VALUE! | #VALUE! | #VALUE! |
| Use of Ticagrelor; n (%) | ** (0.0%) | ** (0.1%) | -0.04 | ** (0.0%) | ** (0.1%) | -0.04 | 22 (0.1%) | 19 (0.1%) | 0.00 | #VALUE! | #VALUE! | #VALUE! |
| Number of D-dimer tests | | | | | | | | | | | | |
| mean (sd) | 0.12 (0.36) | 0.16 (0.42) | -0.10 | 0.13 (0.38) | 0.14 (0.39) | -0.03 | 0.14 (0.36) | 0.17 (0.40) | -0.08 | 0.13 (0.37) | 0.16 (0.40) | 0.00 |
| Numbe of CRP, high-sensitivity CRP tests | | , | | | | | () | () | | (, | | |
| mean (sd) | 0.10 (0.47) | 0.12 (0.53) | -0.04 | 0.09 (0.48) | 0.09 (0.45) | 0.00 | 0.13 (0.55) | 0.14 (0.57) | -0.02 | 0.11 (0.51) | 0.12 (0.53) | 0.00 |
| | 0.10 (0.47) | 0.12 (0.55) | -0.04 | 0.05 (0.46) | 0.03 (0.43) | 0.00 | 0.13 (0.33) | 0.14 (0.37) | -0.02 | 0.11(0.31) | 0.12 (0.33) | 0.00 |
| Number of PT or aPTTt tests | 0.66 (4.77) | 0.50(4.30) | 0.05 | 0.50(4.40) | 0.47 (4.22) | 0.00 | 0.20 (0.04) | 0.25 (0.74) | 0.04 | 0.40 (4.20) | 0.43 (4.05) | 0.00 |
| mean (sd) | 0.66 (1.77) | 0.58 (1.39) | 0.05 | 0.58 (1.48) | 0.47 (1.22) | 0.08 | 0.38 (0.91) | 0.35 (0.74) | 0.04 | 0.49 (1.29) | 0.43 (1.05) | 0.00 |
| Number of Bleeding time tests | | | | | | | | | | | | |
| mean (sd) | 0.00 (0.02) | 0.00 (0.01) | 0.00 | 0.00 (0.02) | 0.00 (0.01) | 0.00 | 0.00 (0.03) | 0.00 (0.02) | 0.00 | 0.00 (0.03) | 0.00 (0.02) | 0.00 |
| HAS-BLED Score (ICD-9 and ICD-10), 180 days | | | | | | | | | | | | |
| mean (sd) | 2.68 (1.05) | 2.55 (1.03) | 0.12 | 2.28 (0.98) | 2.21 (0.95) | 0.07 | 3.43 (0.79) | 3.39 (0.80) | 0.05 | 2.91 (0.90) | 2.88 (0.90) | 0.00 |
| N of Generic name drugs | | | | | | | | | | | | |
| mean (sd) | 15.36 (13.41) | 13.47 (14.05) | 0.14 | 13.18 (11.45) | 11.66 (11.95) | 0.13 | 18.30 (13.64) | 16.35 (14.30) | 0.14 | 16.06 (12.89) | 14.40 (13.60) | 0.00 |
| N of Brand name drugs | , , | | | | , , | | , , | | | | , , | |
| mean (sd) | 2.98 (4.53) | 3.58 (3.90) | -0.14 | 3.30 (4.45) | 3.75 (3.79) | -0.11 | 3.22 (4.77) | 3.92 (4.27) | -0.15 | 3.21 (4.62) | 3.80 (4.06) | 0.00 |
| Use of clopidogrel ; n (%) | 259 (2.4%) | 122 (1.9%) | 0.03 | 499 (2.2%) | 145 (1.5%) | 0.05 | 1,670 (5.1%) | 716 (4.4%) | 0.03 | 2428 (3.6%) | 983 (3.1%) | 0.03 |
| Systemic embolism; n (%) | 221 (2.0%) | 112 (1.7%) | 0.03 | 404 (1.8%) | 141 (1.5%) | 0.03 | 462 (1.4%) | 200 (1.2%) | 0.03 | 1087 (1.6%) | 453 (1.4%) | 0.02 |
| DVT; n (%) | 5,150 (47.1%) | 3,078 (47.7%) | -0.01 | 10,806 (46.9%) | 4,578 (48.7%) | -0.04 | 14,349 (43.6%) | 6,958 (42.9%) | 0.01 | 30305 (45.3%) | 14614 (45.6%) | -0.01 |
| Post-thrombotic syndrome; n (%) | ** (0.1%) | ** (0.1%) | #DIV/0! | 14 (0.1%) | ** (0.1%) | #DIV/0! | 21 (0.1%) | 12 (0.1%) | #DIV/0! | 14 (0.1%) | ** (0.1%) | 0.00 |
| PE; n (%) | 10,931 (100.0%) | 6,448 (100.0%) | #DIV/0! | 23,030 (100.0%) | 9,398 (99.9%) | 0.04 | | 16,217 (100.0%) | -0.04 | 66826 (99.9%) | 32063 (100.0%) | -0.04 |
| Coagulation defects; n (%) | 285 (2.6%) | 123 (1.9%) | #DIV/0! | 654 (2.8%) | 211 (2.2%) | #DIV/0! | 579 (1.8%) | 213 (1.3%) | #DIV/0! | 654 (2.8%) | 211 (2.2%) | 0.04 |
| Diabatas, 1 innations of 2 cutantians daine, within | | | | | | | | | | | | |
| Diabetes: 1 inpatient or 2 outpatient claims within | | | | | | | | | | | | |
| 183 days; n (%) | 2,243 (20.5%) | 1,185 (18.4%) | 0.05 | 3,626 (15.7%) | 1,408 (15.0%) | 0.02 | 8,179 (24.9%) | 3,686 (22.7%) | 0.05 | 14048 (21.0%) | 6279 (19.6%) | 0.03 |
| 183 days ; n (%) | 2,243 (20.5%) | 1,185 (18.4%) | 0.05 | 3,626 (15.7%) | 1,408 (15.0%) | 0.02 | 8,179 (24.9%) | 3,686 (22.7%) | 0.05 | 14048 (21.0%) | 6279 (19.6%) | 0.03 |
| | , | 1,185 (18.4%) | 0.05 | 3,626 (15.7%) | 1,408 (15.0%) | 0.02 | 8,179 (24.9%) | 3,686 (22.7%) | 0.05 | 14048 (21.0%) | 6279 (19.6%) | 0.03 |
| 183 days ; n (%)<br>Intracranial or retroperitoneal hemorrhage: 1 | , | 1,185 (18.4%)<br>** (0.0%) | 0.05<br>#DIV/0! | 3,626 (15.7%)<br>** (0.0%) | 1,408 (15.0%)<br>** (0.0%) | 0.02<br>#DIV/0! | 8,179 (24.9%)<br>15 (0.0%) | 3,686 (22.7%)<br>** (0.0%) | 0.05<br>#DIV/0! | 14048 (21.0%)<br>#VALUE! | 6279 (19.6%)<br>#VALUE! | 0.03<br>#VALUE! |
| 183 days; n (%)<br>Intracranial or retroperitoneal hemorrhage: 1<br>inpatient or 2 outpatient claims within 183 days; n<br>(%) | ** (0.0%) | ** (0.0%) | | ** (0.0%) | ** (0.0%) | #DIV/0! | 15 (0.0%) | ** (0.0%) | #DIV/0! | #VALUE! | #VALUE! | |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease; n (%) | ** (0.0%)<br>2,932 (26.8%) | ** (0.0%)<br>1,734 (26.9%) | #DIV/0!<br>0.00 | ** (0.0%)<br>4,029 (17.5%) | ** (0.0%)<br>1,736 (18.5%) | #DIV/0!<br>-0.03 | 15 (0.0%)<br>11,261 (34.2%) | ** (0.0%)<br>5,399 (33.3%) | #DIV/0!<br>0.02 | #VALUE!<br>18222 (27.2%) | #VALUE!<br>8869 (27.6%) | #VALUE!<br>-0.01 |
| 183 days; n (%)<br>Intracranial or retroperitoneal hemorrhage: 1<br>Inpatient or 2 outpatient claims within 183 days; n<br>(%)<br>Peptic Ulcer Disease; n (%)<br>Major Surgery; n (%) | ** (0.0%)<br>2,932 (26.8%)<br>739 (6.8%) | ** (0.0%)<br>1,734 (26.9%)<br>491 (7.6%) | #DIV/0!<br>0.00<br>#DIV/0! | ** (0.0%)<br>4,029 (17.5%)<br>1,391 (6.0%) | ** (0.0%)<br>1,736 (18.5%)<br>507 (5.4%) | #DIV/0!<br>-0.03<br>#DIV/0! | 15 (0.0%)<br>11,261 (34.2%)<br>2,747 (8.4%) | ** (0.0%)<br>5,399 (33.3%)<br>1,625 (10.0%) | #DIV/0!<br>0.02<br>#DIV/0! | #VALUE!<br>18222 (27.2%)<br>1,391 (6.0%) | #VALUE!<br>8869 (27.6%)<br>507 (5.4%) | #VALUE!<br>-0.01<br>0.03 |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper G bleed; n (%) | ** (0.0%)<br>2,932 (26.8%)<br>739 (6.8%)<br>0 (0.0%) | ** (0.0%)<br>1,734 (26.9%)<br>491 (7.6%)<br>0 (0.0%) | #DIV/0!<br>0.00<br>#DIV/0!<br>#DIV/0! | ** (0.0%)<br>4,029 (17.5%)<br>1,391 (6.0%)<br>0 (0.0%) | ** (0.0%)<br>1,736 (18.5%)<br>507 (5.4%)<br>0 (0.0%) | #DIV/0!<br>-0.03<br>#DIV/0!<br>#DIV/0! | 15 (0.0%)<br>11,261 (34.2%)<br>2,747 (8.4%)<br>0 (0.0%) | ** (0.0%)<br>5,399 (33.3%)<br>1,625 (10.0%)<br>0 (0.0%) | #DIV/0!<br>0.02<br>#DIV/0!<br>#DIV/0! | #VALUE!<br>18222 (27.2%)<br>1,391 (6.0%)<br>0 (0.0%) | #VALUE!<br>8869 (27.6%)<br>507 (5.4%)<br>0 (0.0%) | #VALUE!<br>-0.01<br>0.03<br>#DIV/0! |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Lower/ unspecified Gi bleed; n (%) | ** (0.0%)<br>2,932 (26.8%)<br>739 (6.8%)<br>0 (0.0%)<br>0 (0.0%) | ** (0.0%)<br>1,734 (26.9%)<br>491 (7.6%)<br>0 (0.0%)<br>0 (0.0%) | #DIV/0!<br>0.00<br>#DIV/0!<br>#DIV/0!<br>#DIV/0! | ** (0.0%)<br>4,029 (17.5%)<br>1,391 (6.0%)<br>0 (0.0%)<br>0 (0.0%) | ** (0.0%)<br>1,736 (18.5%)<br>507 (5.4%)<br>0 (0.0%)<br>0 (0.0%) | #DIV/0!<br>-0.03<br>#DIV/0!<br>#DIV/0!<br>#DIV/0! | 15 (0.0%)<br>11,261 (34.2%)<br>2,747 (8.4%)<br>0 (0.0%) | ** (0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) 0 (0.0%) | #DIV/0!<br>0.02<br>#DIV/0!<br>#DIV/0!<br>#DIV/0! | #VALUE!<br>18222 (27.2%)<br>1,391 (6.0%)<br>0 (0.0%)<br>0 (0.0%) | #VALUE!<br>8869 (27.6%)<br>507 (5.4%)<br>0 (0.0%)<br>0 (0.0%) | #VALUE!<br>-0.01<br>0.03<br>#DIV/0!<br>#DIV/0! |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 Inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Lower/ unspecified Gi bleed; n (%) Urogenital bleed; n (%) | ** (0.0%)<br>2,932 (26.8%)<br>739 (6.8%)<br>0 (0.0%)<br>0 (0.0%)<br>73 (0.7%) | ** (0.0%)<br>1,734 (26.9%)<br>491 (7.6%)<br>0 (0.0%)<br>0 (0.0%)<br>49 (0.8%) | #DIV/0!<br>0.00<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>-0.01 | ** (0.0%)<br>4,029 (17.5%)<br>1,391 (6.0%)<br>0 (0.0%)<br>0 (0.0%)<br>171 (0.7%) | ** (0.0%)<br>1,736 (18.5%)<br>507 (5.4%)<br>0 (0.0%)<br>0 (0.0%)<br>81 (0.9%) | #DIV/0!<br>-0.03<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>-0.02 | 15 (0.0%)<br>11,261 (34.2%)<br>2,747 (8.4%)<br>0 (0.0%)<br>0 (0.0%)<br>** (0.0%) | **(0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) 0 (0.0%) **(0.0%) | #DIV/0!<br>0.02<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>#DIV/0! | #VALUE!<br>18222 (27.2%)<br>1,391 (6.0%)<br>0 (0.0%)<br>0 (0.0%)<br>#VALUE! | #VALUE!<br>8869 (27.6%)<br>507 (5.4%)<br>0 (0.0%)<br>0 (0.0%)<br>#VALUE! | #VALUE!<br>-0.01<br>0.03<br>#DIV/0!<br>#DIV/0!<br>#VALUE! |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gl bleed; n (%) Lower/ unspecified Gl bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) | ** (0.0%)<br>2,932 (26.8%)<br>739 (6.8%)<br>0 (0.0%)<br>0 (0.0%)<br>73 (0.7%)<br>504 (4.6%) | ** (0.0%)<br>1,734 (26.9%)<br>491 (7.6%)<br>0 (0.0%)<br>0 (0.0%)<br>49 (0.8%)<br>232 (3.6%) | #DIV/0!<br>0.00<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>-0.01<br>0.05 | ** (0.0%)<br>4,029 (17.5%)<br>1,391 (6.0%)<br>0 (0.0%)<br>0 (0.0%)<br>171 (0.7%)<br>819 (3.6%) | ** (0.0%)<br>1,736 (18.5%)<br>507 (5.4%)<br>0 (0.0%)<br>0 (0.0%)<br>81 (0.9%)<br>301 (3.2%) | #DIV/0!<br>-0.03<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>-0.02<br>0.02 | 15 (0.0%)<br>11,261 (34.2%)<br>2,747 (8.4%)<br>0 (0.0%)<br>0 (0.0%)<br>**(0.0%)<br>1,521 (4.6%) | ** (0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) ** (0.0%) 607 (3.7%) | #DIV/0!<br>0.02<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>0.05 | #VALUE! 18222 (27.2%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) #VALUE! 2844 (4.3%) | #VALUE!<br>8869 (27.6%)<br>507 (5.4%)<br>0 (0.0%)<br>0 (0.0%)<br>#VALUE!<br>1140 (3.6%) | #VALUE!<br>-0.01<br>0.03<br>#DIV/0!<br>#DIV/0!<br>#VALUE!<br>0.04 |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Lower/ unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) | ** (0.0%)<br>2,932 (26.8%)<br>739 (6.8%)<br>0 (0.0%)<br>0 (0.0%)<br>73 (0.7%)<br>504 (4.6%)<br>1,356 (12.4%) | ** (0.0%)<br>1,734 (26.9%)<br>491 (7.6%)<br>0 (0.0%)<br>0 (0.0%)<br>49 (0.8%)<br>232 (3.6%)<br>1,060 (16.4%) | #DIV/0!<br>0.00<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>-0.01<br>0.05 | ** (0.0%)<br>4,029 (17.5%)<br>1,391 (6.0%)<br>0 (0.0%)<br>171 (0.7%)<br>819 (3.6%)<br>1,964 (8.5%) | ** (0.0%)<br>1,736 (18.5%)<br>507 (5.4%)<br>0 (0.0%)<br>81 (0.9%)<br>301 (3.2%)<br>1,011 (10.7%) | #DIV/0!<br>-0.03<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>-0.02<br>0.02 | 15 (0.0%)<br>11,261 (34.2%)<br>2,747 (8.4%)<br>0 (0.0%)<br>0 (0.0%)<br>**(0.0%)<br>1,521 (4.6%)<br>5,398 (16.4%) | ** (0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) ** (0.0%) 607 (3.7%) 3,537 (21.8%) | #DIV/0!<br>0.02<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>0.05<br>-0.14 | #VALUE!<br>18222 (27.2%)<br>1,391 (6.0%)<br>0 (0.0%)<br>0 (0.0%)<br>#VALUE!<br>2844 (4.3%)<br>8718 (13.0%) | #VALUE!<br>8869 (27.6%)<br>507 (5.4%)<br>0 (0.0%)<br>0 (0.0%)<br>#VALUE!<br>1140 (3.6%)<br>5608 (17.5%) | #VALUE!<br>-0.01<br>0.03<br>#DIV/0!<br>#DIV/0!<br>#VALUE!<br>0.04 |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Lower/ unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Antibiotics; n (%) | **(0.0%) 2,932 (26.8%) 739 (6.8%) 0 (0.0%) 0 (0.0%) 73 (0.7%) 504 (4.6%) 1,356 (12.4%) 5,272 (48.2%) | ** (0.0%)<br>1,734 (26.9%)<br>491 (7.6%)<br>0 (0.0%)<br>0 (0.0%)<br>49 (0.8%)<br>232 (3.6%)<br>1,060 (16.4%) | #DIV/0!<br>0.00<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>-0.01<br>0.05<br>-0.11<br>#DIV/0! | ** (0.0%)<br>4,029 (17.5%)<br>1,391 (6.0%)<br>0 (0.0%)<br>0 (0.0%)<br>171 (0.7%)<br>819 (3.6%)<br>1,964 (8.5%)<br>11,518 (50.0%) | ** (0.0%) 1,736 (18.5%) 507 (5.4%) 0 (0.0%) 0 (0.0%) 81 (0.9%) 301 (3.2%) 1,011 (10.7%) 4,633 (49.3%) | #DIV/0!<br>-0.03<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>-0.02<br>-0.07<br>#DIV/0! | 15 (0.0%) 11,261 (34.2%) 2,747 (8.4%) 0 (0.0%) 0 (0.0%) ** (0.0%) 1,521 (4.6%) 17,994 (54.7%) | ** (0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) ** (0.0%) 607 (3.7%) 3,537 (21.8%) 8,891 (54.8%) | #DIV/0!<br>0.02<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>0.05<br>-0.14<br>#DIV/0! | #VALUE! 18222 (27.2%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) #VALUE! 2844 (4.3%) 8718 (13.0%) | #VALUE!<br>8869 (27.6%)<br>507 (5.4%)<br>0 (0.0%)<br>0 (0.0%)<br>#VALUE!<br>1140 (3.6%)<br>5608 (17.5%)<br>4,633 (49.3%) | #VALUE! -0.01 0.03 #DIV/0! #DIV/0! #VALUE! 0.04 -0.13 |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Lower/ unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) | ** (0.0%) 2,932 (26.8%) 739 (6.8%) 0 (0.0%) 0 (0.0%) 73 (0.7%) 504 (4.6%) 1,356 (12.4%) 5,272 (48.2%) 63 (0.6%) | ** (0.0%)<br>1,734 (26.9%)<br>491 (7.6%)<br>0 (0.0%)<br>0 (0.0%)<br>49 (0.8%)<br>232 (3.6%)<br>1,060 (16.4%)<br>95 (48.0%)<br>71 (1.1%) | #DIV/0!<br>0.00<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>-0.01<br>0.05<br>-0.11<br>#DIV/0!<br>-0.05 | ** (0.0%)<br>4,029 (17.5%)<br>1,391 (6.0%)<br>0 (0.0%)<br>171 (0.7%)<br>819 (3.6%)<br>1,964 (8.5%)<br>11,518 (50.0%)<br>254 (1.1%) | ** (0.0%)<br>1,736 (18.5%)<br>507 (5.4%)<br>0 (0.0%)<br>0 (0.0%)<br>81 (0.9%)<br>301 (3.2%)<br>1,011 (10.7%)<br>4,633 (49.3%) | #DIV/0! -0.03 #DIV/0! #DIV/0! #DIV/0! -0.02 -0.07 #DIV/0! | 15 (0.0%)<br>11,261 (34.2%)<br>2,747 (8.4%)<br>0 (0.0%)<br>0 (0.0%)<br>** (0.0%)<br>1,521 (4.6%)<br>5,398 (16.4%)<br>17,994 (54.7%) | ** (0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) ** (0.0%) 607 (3.7%) 3,537 (21.8%) 46 (0.3%) | #DIV/0! 0.02 #DIV/0! #DIV/0! #DIV/0! #DIV/0! 0.05 -0.14 #DIV/0! 0.03 | #VALUE! 18222 (27.2%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) #VALUE! 2844 (4.3%) 8718 (13.0%) 11,518 (50.0%) 475 (0.7%) | #VALUE!<br>8869 (27.6%)<br>507 (5.4%)<br>0 (0.0%)<br>0 (0.0%)<br>#VALUE!<br>1140 (3.6%)<br>5608 (17.5%)<br>4,633 (49.3%)<br>254 (0.8%) | #VALUEI<br>-0.01<br>0.03<br>#DIV/0!<br>#DIV/0!<br>#VALUEI<br>0.04<br>-0.13<br>0.01<br>-0.01 |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 Inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gl bleed; n (%) Lower/ unspecified Gl bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cance; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) | **(0.0%) 2,932 (26.8%) 739 (6.8%) 0 (0.0%) 0 (0.0%) 73 (0.7%) 504 (4.6%) 1,356 (12.4%) 5,272 (48.2%) 3,05 | ** (0.0%) 1,734 (26.9%) 491 (7.6%) 0 (0.0%) 0 (0.0%) 49 (0.8%) 232 (3.6%) 1,060 (16.4%) 95 (48.0%) 71 (1.1%) ** (0.1%) | #DIV/0! 0.00 #DIV/0! #DIV/0! #DIV/0! 0.01 0.05 -0.11 #DIV/0! -0.05 0.05 | ** (0.0%)<br>4,029 (17.5%)<br>1,391 (6.0%)<br>0 (0.0%)<br>171 (0.7%)<br>819 (3.6%)<br>1,964 (8.5%)<br>11,518 (50.0%)<br>254 (1.1%)<br>36 (0.2%) | ** (0.0%)<br>1,736 (18.5%)<br>507 (5.4%)<br>0 (0.0%)<br>0 (0.0%)<br>81 (0.9%)<br>301 (3.2%)<br>1,011 (10.7%)<br>4,633 (49.3%)<br>137 (1.5%)<br>** (0.1%) | #DIV/0!<br>-0.03<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>-0.02<br>-0.07<br>#DIV/0! | 15 (0.0%) 11,261 (34.2%) 2,747 (8.4%) 0 (0.0%) 0 (0.0%) ** (0.0%) 1,521 (4.6%) 5,398 (16.4%) 17,994 (54.7%) 158 (0.5%) | ** (0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) ** (0.0%) 607 (3.7%) 3,537 (21.8%) 8,891 (54.8%) 46 (0.3%) 33 (0.2%) | #DIV/0!<br>0.02<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>0.05<br>-0.14<br>#DIV/0!<br>0.03<br>0.02 | #VALUE! 18222 (27.2%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) #VALUE! 2844 (4.3%) 8718 (13.0%) 11,518 (50.0%) 475 (0.7%) | #VALUE!<br>8869 (27.6%)<br>507 (5.4%)<br>0 (0.0%)<br>0 (0.0%)<br>#VALUE!<br>1140 (3.6%)<br>5608 (17.5%)<br>4,633 (49.3%)<br>254 (0.8%)<br>#VALUE! | #VALUE! -0.01 0.03 #DIV/0! #DIV/0! #VALUE! 0.04 -0.13 0.01 -0.01 #VALUE! |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Lower/ unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) | ** (0.0%) 2,932 (26.8%) 739 (6.8%) 0 (0.0%) 0 (0.0%) 73 (0.7%) 504 (4.6%) 1,356 (12.4%) 5,272 (48.2%) 63 (0.6%) ** (0.1%) 22 (0.2%) | ** (0.0%) 1,734 (26.9%) 491 (7.6%) 0 (0.0%) 49 (0.8%) 232 (3.6%) 1,060 (16.4%) 95 (48.0%) 71 (1.1%) ** (0.1%) 13 (0.2%) | #DIV/0! 0.00 #DIV/0! #DIV/0! #DIV/0! -0.01 0.05 -0.11 #DIV/0! -0.05 0.00 | ** (0.0%)<br>4,029 (17.5%)<br>1,391 (6.0%)<br>0 (0.0%)<br>171 (0.7%)<br>819 (3.6%)<br>1,964 (8.5%)<br>11,518 (50.0%)<br>254 (1.1%)<br>36 (0.2%) | ** (0.0%)<br>1,736 (18.5%)<br>507 (5.4%)<br>0 (0.0%)<br>0 (0.0%)<br>81 (0.9%)<br>301 (3.2%)<br>1,011 (10.7%)<br>4,633 (49.3%)<br>137 (1.5%)<br>** (0.1%)<br>** (0.1%) | #DIV/01 -0.03 #DIV/01 #DIV/01 #DIV/01 -0.02 -0.07 #DIV/01 -0.04 -0.03 -0.03 | 15 (0.0%) 11,261 (34.2%) 2,747 (8.4%) 0 (0.0%) 0 (0.0%) **(0.0%) 1,521 (4.6%) 5,398 (16.4%) 17,994 (54.7%) 158 (0.5%) 199 (0.3%) 139 (0.4%) | **(0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) **(0.0%) 607 (3.7%) 3,537 (21.8%) 8,891 (54.8%) 46 (0.3%) 33 (0.2%) 57 (0.4%) | #DIV/01<br>0.02<br>#DIV/01<br>#DIV/01<br>#DIV/01<br>0.05<br>-0.14<br>#DIV/01<br>0.03<br>0.02<br>0.00 | #VALUE! 18222 (27.2%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) #VALUE! 2844 (4.3%) 8718 (13.0%) 11,518 (50.0%) #VALUE! 197 (0.3%) | #VALUEI<br>8869 (27.6%)<br>507 (5.4%)<br>0 (0.0%)<br>0 (0.0%)<br>#VALUEI<br>1140 (3.6%)<br>5608 (17.5%)<br>4,633 (49.3%)<br>#VALUEI<br>#VALUEI | #VALUE! -0.01 0.03 #DIV/0! #DIV/0! #VALUE! 0.04 -0.13 0.01 -0.01 #VALUE! |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 Inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gl bleed; n (%) Lower/ unspecified Gl bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cance; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) | **(0.0%) 2,932 (26.8%) 739 (6.8%) 0 (0.0%) 0 (0.0%) 73 (0.7%) 504 (4.6%) 1,356 (12.4%) 5,272 (48.2%) 3,05 | ** (0.0%) 1,734 (26.9%) 491 (7.6%) 0 (0.0%) 0 (0.0%) 49 (0.8%) 232 (3.6%) 1,060 (16.4%) 95 (48.0%) 71 (1.1%) ** (0.1%) | #DIV/0! 0.00 #DIV/0! #DIV/0! #DIV/0! 0.01 0.05 -0.11 #DIV/0! -0.05 0.05 | ** (0.0%)<br>4,029 (17.5%)<br>1,391 (6.0%)<br>0 (0.0%)<br>171 (0.7%)<br>819 (3.6%)<br>1,964 (8.5%)<br>11,518 (50.0%)<br>254 (1.1%)<br>36 (0.2%) | ** (0.0%)<br>1,736 (18.5%)<br>507 (5.4%)<br>0 (0.0%)<br>0 (0.0%)<br>81 (0.9%)<br>301 (3.2%)<br>1,011 (10.7%)<br>4,633 (49.3%)<br>137 (1.5%)<br>** (0.1%) | #DIV/0! -0.03 #DIV/0! #DIV/0! #DIV/0! -0.02 -0.07 #DIV/0! -0.04 -0.03 | 15 (0.0%) 11,261 (34.2%) 2,747 (8.4%) 0 (0.0%) 0 (0.0%) ** (0.0%) 1,521 (4.6%) 5,398 (16.4%) 17,994 (54.7%) 158 (0.5%) | ** (0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) ** (0.0%) 607 (3.7%) 3,537 (21.8%) 8,891 (54.8%) 46 (0.3%) 33 (0.2%) | #DIV/0!<br>0.02<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>0.05<br>-0.14<br>#DIV/0!<br>0.03<br>0.02 | #VALUE! 18222 (27.2%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) #VALUE! 2844 (4.3%) 8718 (13.0%) 11,518 (50.0%) 475 (0.7%) | #VALUE!<br>8869 (27.6%)<br>507 (5.4%)<br>0 (0.0%)<br>0 (0.0%)<br>#VALUE!<br>1140 (3.6%)<br>5608 (17.5%)<br>4,633 (49.3%)<br>254 (0.8%)<br>#VALUE! | #VALUE! -0.01 0.03 #DIV/0! #DIV/0! #VALUE! 0.04 -0.13 0.01 -0.01 #VALUE! |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Lower/ unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) | ** (0.0%) 2,932 (26.8%) 739 (6.8%) 0 (0.0%) 0 (0.0%) 73 (0.7%) 504 (4.6%) 1,356 (12.4%) 5,272 (48.2%) 63 (0.6%) ** (0.1%) 22 (0.2%) | ** (0.0%) 1,734 (26.9%) 491 (7.6%) 0 (0.0%) 49 (0.8%) 232 (3.6%) 1,060 (16.4%) 95 (48.0%) 71 (1.1%) ** (0.1%) 13 (0.2%) | #DIV/0! 0.00 #DIV/0! #DIV/0! #DIV/0! -0.01 0.05 -0.11 #DIV/0! -0.05 0.00 | ** (0.0%)<br>4,029 (17.5%)<br>1,391 (6.0%)<br>0 (0.0%)<br>171 (0.7%)<br>819 (3.6%)<br>1,964 (8.5%)<br>11,518 (50.0%)<br>254 (1.1%)<br>36 (0.2%) | ** (0.0%)<br>1,736 (18.5%)<br>507 (5.4%)<br>0 (0.0%)<br>0 (0.0%)<br>81 (0.9%)<br>301 (3.2%)<br>1,011 (10.7%)<br>4,633 (49.3%)<br>137 (1.5%)<br>** (0.1%)<br>** (0.1%) | #DIV/01 -0.03 #DIV/01 #DIV/01 #DIV/01 -0.02 -0.07 #DIV/01 -0.04 -0.03 -0.03 | 15 (0.0%) 11,261 (34.2%) 2,747 (8.4%) 0 (0.0%) 0 (0.0%) **(0.0%) 1,521 (4.6%) 5,398 (16.4%) 17,994 (54.7%) 158 (0.5%) 199 (0.3%) 139 (0.4%) | **(0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) **(0.0%) 607 (3.7%) 3,537 (21.8%) 8,891 (54.8%) 46 (0.3%) 33 (0.2%) 57 (0.4%) | #DIV/01<br>0.02<br>#DIV/01<br>#DIV/01<br>#DIV/01<br>0.05<br>-0.14<br>#DIV/01<br>0.03<br>0.02<br>0.00 | #VALUE! 18222 (27.2%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) #VALUE! 2844 (4.3%) 8718 (13.0%) 11,518 (50.0%) #VALUE! 197 (0.3%) | #VALUEI<br>8869 (27.6%)<br>507 (5.4%)<br>0 (0.0%)<br>0 (0.0%)<br>#VALUEI<br>1140 (3.6%)<br>5608 (17.5%)<br>4,633 (49.3%)<br>#VALUEI<br>#VALUEI | #VALUE! -0.01 0.03 #DIV/0! #DIV/0! #VALUE! 0.04 -0.13 0.01 -0.01 #VALUE! |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper GI bleed; n (%) Lower/ unspecified GI bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) | ** (0.0%) 2,932 (26.8%) 739 (6.8%) 0 (0.0%) 0 (0.0%) 73 (0.7%) 504 (4.6%) 1,356 (12.4%) 5,272 (48.2%) 63 (0.6%) ** (0.1%) 22 (0.2%) 2,367 (21.6%) | ** (0.0%) 1,734 (26.9%) 491 (7.6%) 0 (0.0%) 49 (0.8%) 232 (3.6%) 1,060 (16.4%) 95 (48.0%) 71 (1.1%) ** (0.1%) 13 (0.2%) 1,341 (20.8%) | #DIV/01 0.00 #DIV/01 #DIV/01 #DIV/01 -0.01 0.05 -0.11 #DIV/01 -0.05 0.00 0.00 | ** (0.0%)<br>4,029 (17.5%)<br>1,391 (6.0%)<br>0 (0.0%)<br>0 (0.0%)<br>171 (0.7%)<br>819 (3.6%)<br>1,964 (8.5%)<br>11,518 (50.0%)<br>254 (1.1%)<br>36 (0.2%)<br>36 (0.2%)<br>5,284 (22.9%) | ** (0.0%) 1,736 (18.5%) 507 (5.4%) 0 (0.0%) 0 (0.0%) 81 (0.9%) 301 (3.2%) 1,011 (10.7%) 4,633 (49.3%) 137 (1.5%) ** (0.1%) (0.1%) 1,997 (21.2%) | #DIV/0! -0.03 #DIV/0! #DIV/0! #DIV/0! -0.02 -0.02 -0.07 #DIV/0! -0.04 -0.03 -0.03 | 15 (0.0%) 11,261 (34.2%) 2,747 (8.4%) 0 (0.0%) 0 (0.0%) 1,521 (4.6%) 5,398 (16.4%) 17,994 (54.7%) 158 (0.5%) 109 (0.3%) 139 (0.4%) 8,671 (26.4%) | **(0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) 0 (0.0%) **(0.0%) 607 (3.7%) 3,537 (21.8%) 46 (0.3%) 33 (0.2%) 57 (0.4%) 4,164 (25.7%) | #DIV/01 0.02 #DIV/01 #DIV/01 #DIV/01 #DIV/01 #DIV/01 0.05 -0.14 #DIV/01 0.03 0.02 0.00 0.00 | #VALUE! 18222 (27.2%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) #VALUE! 2844 (4.3%) 8718 (13.0%) 11,518 (50.0%) #VALUE! 197 (0.3%) 16322 (24.4%) | #VALUE!<br>8869 (27.6%)<br>507 (5.4%)<br>0 (0.0%)<br>0 (0.0%)<br>#VALUE!<br>1140 (3.6%)<br>5608 (17.5%)<br>4,633 (49.3%)<br>254 (0.8%)<br>#VALUE!<br>#VALUE!<br>7502 (23.4%) | #VALUE! -0.01 0.03 #DIV/01 #VALUE! 0.04 -0.13 0.01 -0.01 #VALUE! |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Lower/ unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests ordered | **(0.0%) 2,932 (26.8%) 739 (6.8%) 0 (0.0%) 0 (0.0%) 3 (0.7%) 504 (4.6%) 1,356 (12.4%) 5,272 (48.2%) 63 (0.6%) **(0.1%) 22 (0.2%) 2,367 (21.6%) 128 (1.2%) | ** (0.0%) 1,734 (26.9%) 491 (7.6%) 0 (0.0%) 49 (0.8%) 232 (3.6%) 1,060 (16.4%) 95 (48.0%) 71 (1.1%) ** (0.1%) 13 (0.2%) 1,341 (20.8%) | #DIV/01 0.00 #DIV/01 #DIV/01 #DIV/01 -0.01 0.05 -0.11 #DIV/01 -0.05 0.00 0.00 | ** (0.0%)<br>4,029 (17.5%)<br>1,391 (6.0%)<br>0 (0.0%)<br>0 (0.0%)<br>171 (0.7%)<br>819 (3.6%)<br>1,964 (8.5%)<br>11,518 (50.0%)<br>254 (1.1%)<br>36 (0.2%)<br>36 (0.2%)<br>5,284 (22.9%) | ** (0.0%) 1,736 (18.5%) 507 (5.4%) 0 (0.0%) 0 (0.0%) 81 (0.9%) 301 (3.2%) 1,011 (10.7%) 4,633 (49.3%) 137 (1.5%) ** (0.1%) 1,997 (21.2%) 101 (1.1%) | #DIV/0! -0.03 #DIV/0! #DIV/0! #DIV/0! -0.02 -0.02 -0.07 #DIV/0! -0.04 -0.03 -0.03 | 15 (0.0%) 11,261 (34.2%) 2,747 (8.4%) 0 (0.0%) 0 (0.0%) **(0.0%) 1,521 (4.6%) 5,398 (16.4%) 17,994 (54.7%) 198 (0.5%) 109 (0.3%) 139 (0.4%) 8,671 (26.4%) 581 (1.8%) | **(0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) 0 (0.0%) **(0.0%) 607 (3.7%) 3,537 (21.8%) 46 (0.3%) 33 (0.2%) 57 (0.4%) 4,164 (25.7%) | #DIV/01 0.02 #DIV/01 #DIV/01 #DIV/01 #DIV/01 #DIV/01 0.05 -0.14 #DIV/01 0.03 0.02 0.00 0.00 | #VALUE! 18222 (27.2%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) #VALUE! 2844 (4.3%) 8718 (13.0%) 11,518 (50.0%) #VALUE! 197 (0.3%) 16322 (24.4%) | #VALUE!<br>8869 (27.6%)<br>507 (5.4%)<br>0 (0.0%)<br>0 (0.0%)<br>#VALUE!<br>1140 (3.6%)<br>5608 (17.5%)<br>4,633 (49.3%)<br>254 (0.8%)<br>#VALUE!<br>#VALUE!<br>7502 (23.4%) | #VALUE! -0.01 0.03 #DIV/01 #VALUE! 0.04 -0.13 0.01 -0.01 #VALUE! |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Upper Gi bleed; n (%) Urogenital bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) Other gastroprotective agents; n (%) Other gastroprotective agents; n (%) Other gastroprotective agents; n (%)mean (sd) | ** (0.0%) 2,932 (26.8%) 739 (6.8%) 0 (0.0%) 0 (0.0%) 73 (0.7%) 504 (4.6%) 1,356 (12.4%) 5,272 (48.2%) 63 (0.6%) ** (0.1%) 22 (0.2%) 2,367 (21.6%) 128 (1.2%) | ** (0.0%) 1,734 (26.9%) 491 (7.6%) 0 (0.0%) 0 (0.0%) 49 (0.8%) 232 (3.6%) 1,060 (16.4%) 95 (48.0%) 71 (1.1%) ** (0.1%) 13 (0.2%) 1,341 (20.8%) 85 (1.3%) 0.45 (0.88) | #DIV/0! 0.00 #DIV/0! #DIV/0! #DIV/0! -0.01 0.05 -0.11 #DIV/0! -0.05 0.00 0.00 0.00 0.00 0.00 | ** (0.0%)<br>4,029 (17.5%)<br>1,391 (6.0%)<br>0 (0.0%)<br>171 (0.7%)<br>819 (3.6%)<br>1,964 (8.5%)<br>11,518 (50.0%)<br>254 (1.1%)<br>36 (0.2%)<br>36 (0.2%)<br>284 (22.9%)<br>287 (1.2%) | ** (0.0%) 1,736 (18.5%) 507 (5.4%) 0 (0.0%) 0 (0.0%) 81 (0.9%) 301 (3.2%) 1,011 (10.7%) 4,633 (49.3%) 137 (1.5%) ** (0.1%) (0.1%) 1,997 (21.2%) 101 (1.1%) | #DIV/0! -0.03 #DIV/0! #DIV/0! #DIV/0! -0.02 -0.07 #DIV/0! -0.04 0.03 0.03 0.04 0.01 | 15 (0.0%) 11,261 (34.2%) 2,747 (8.4%) 0 (0.0%) 0 (0.0%) 1,521 (4.6%) 5,398 (16.4%) 17,994 (54.7%) 158 (0.5%) 109 (0.3%) 139 (0.4%) 8,671 (26.4%) 581 (1.8%) | ** (0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) 0 (0.0%) ** (0.0%) (67 (3.7%) 3,537 (21.8%) 46 (0.3%) 33 (0.2%) 57 (0.4%) 4,164 (25.7%) 248 (1.5%) 0.58 (0.82) | #DIV/01 0.02 #DIV/01 #DIV/01 #DIV/01 #DIV/01 #DIV/01 0.05 -0.14 #DIV/01 0.03 0.02 0.00 0.02 -0.02 | #VALUE! 18222 (27.2%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) #VALUE! 2844 (4.3%) 8718 (13.0%) 11,518 (50.0%) 475 (0.7%) #VALUE! 197 (0.3%) 16322 (24.4%) 996 (1.5%) | #VALUE! 8869 (27.6%) 507 (5.4%) 0 (0.0%) 0 (0.0%) #VALUE! 1140 (3.6%) 5608 (17.5%) 4,633 (49.3%) 254 (0.8%) #VALUE! #VALUE! #7ALUE! 7502 (23.4%) 434 (1.4%) | #VALUE! -0.01 0.03 #DIV/0! #DIV/0! #VALUE! 0.04 -0.13 0.01 -0.01 #VALUE! 0.02 0.01 |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 Inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease: n (%) Major Surgery; n (%) Upper Gl bleed; n (%) Lower/ unspecified Gl bleed; n (%) Urogenital bleed; n (%) Urogenital bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) | ** (0.0%) 2,932 (26.8%) 739 (6.8%) 0 (0.0%) 0 (0.0%) 73 (0.7%) 504 (4.6%) 1,356 (12.4%) 5,272 (48.2%) 3,05 4 (0.1%) 22 (0.2%) 2,367 (21.6%) 128 (1.2%) 0.46 (0.71) 2,563 (23.4%) | ** (0.0%) 1,734 (26.9%) 491 (7.6%) 0 (0.0%) 0 (0.0%) 49 (0.8%) 232 (3.6%) 1,060 (16.4%) 95 (48.0%) 71 (1.1%) ** (0.1%) 13 (0.2%) 1,341 (20.8%) 85 (1.3%) 0.45 (0.88) 1,362 (21.1%) | #DIV/01 0.00 #DIV/01 #DIV/01 -0.01 0.05 -0.11 #DIV/01 -0.05 0.00 0.00 0.00 0.00 0.02 -0.01 0.01 | ** (0.0%) 4,029 (17.5%) 1,391 (6.0%) 0 (0.0%) 171 (0.7%) 819 (3.6%) 1,964 (8.5%) 11,518 (50.0%) 254 (1.1%) 36 (0.2%) 36 (0.2%) 5,284 (22.9%) 287 (1.2%) 0.34 (0.71) 5,093 (22.1%) | ** (0.0%) 1,736 (18.5%) 507 (5.4%) 0 (0.0%) 0 (0.0%) 81 (0.9%) 301 (3.2%) 1,011 (10.7%) 4,633 (49.3%) 137 (1.5%) ** (0.1%) ** (0.1%) 1,997 (21.2%) 101 (1.1%) 0.36 (0.78) 1,943 (20.7%) | #DIV/01 -0.03 #DIV/01 #DIV/01 -0.02 -0.07 #DIV/01 -0.04 -0.03 -0.04 -0.01 -0.03 -0.04 -0.01 | 15 (0.0%) 11,261 (34.2%) 2,747 (8.4%) 0 (0.0%) 0 (0.0%) ** (0.0%) 1,521 (4.6%) 5,398 (16.4%) 17,994 (54.7%) 158 (0.5%) 109 (0.3%) 139 (0.4%) 8,671 (26.4%) 581 (1.8%) 0.56 (0.76) 10,854 (33.0%) | ** (0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) ** (0.0%) 607 (3.7%) 3,537 (21.8%) 8,891 (54.8%) 46 (0.3%) 33 (0.2%) 57 (0.4%) 4,164 (25.7%) 248 (1.5%) 0.58 (0.82) 4,940 (30.5%) | #DIV/01 0.02 #DIV/01 #DIV/01 #DIV/01 #DIV/01 #DIV/01 #DIV/01 0.05 -0.14 #DIV/01 0.03 0.02 0.00 0.02 0.02 -0.02 | #VALUE! 18222 (27.2%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) #VALUE! 2844 (4.3%) 8718 (13.0%) 11,518 (50.0%) #VALUE! 197 (0.3%) 16322 (24.4%) 996 (1.5%) 0.47 (0.74) 18510 (27.7%) | #VALUE! 8869 (27.6%) 507 (5.4%) 0 (0.0%) 0 (0.0%) #WALUE! 1140 (3.6%) 5608 (17.5%) 4,633 (49.3%) 254 (0.8%) #VALUE! #VALUE! #VALUE! 7502 (23.4%) 434 (1.4%) 0.49 (0.82) 8245 (25.7%) | #VALUE! -0.01 0.03 #DIV/0! #DIV/0! #VALUE! 0.04 -0.13 0.01 -0.01 #VALUE! #VALUE! 0.02 0.01 0.00 0.05 |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Lower/ unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Ofher antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) | **(0.0%) 2,932 (26.8%) 739 (6.8%) 0 (0.0%) 0 (0.0%) 504 (4.6%) 1,356 (12.4%) 5,272 (48.2%) 63 (0.6%) **(0.1%) 22 (0.2%) 2,367 (21.6%) 128 (1.2%) 0.46 (0.71) 2,563 (23.4%) 385 (3.5%) | ** (0.0%) 1,734 (26.9%) 491 (7.6%) 0 (0.0%) 0 (0.0%) 49 (0.8%) 232 (3.6%) 1,060 (16.4%) 95 (48.0%) 71 (1.1%) ** (0.1%) 13 (0.2%) 1,341 (20.8%) 85 (1.3%) 0.45 (0.88) 1,362 (21.1%) 201 (3.1%) | #DIV/0! 0.00 #DIV/0! #DIV/0! #DIV/0! #DIV/0! -0.01 0.05 -0.11 #DIV/0! -0.05 0.00 0.00 0.02 -0.01 | ** (0.0%) 4,029 (17.5%) 1,391 (6.0%) 0 (0.0%) 171 (0.7%) 819 (3.6%) 1,964 (8.5%) 11,518 (50.0%) 254 (1.1%) 36 (0.2%) 36 (0.2%) 5,284 (22.9%) 287 (1.2%) 0.34 (0.71) 5,093 (22.1%) 774 (3.4%) | ** (0.0%) 1,736 (18.5%) 507 (5.4%) 0 (0.0%) 0 (0.0%) 81 (0.9%) 301 (3.2%) 1,011 (10.7%) 4,633 (49.3%) 137 (1.5%) ** (0.1%) 1,997 (21.2%) 101 (1.1%) 0.36 (0.78) 1,943 (20.7%) 305 (3.2%) | #DIV/0! -0.03 #DIV/0! #DIV/0! #DIV/0! #DIV/0! -0.02 -0.07 #DIV/0! -0.04 -0.03 -0.04 -0.01 | 15 (0.0%) 11,261 (34.2%) 2,747 (8.4%) 0 (0.0%) 0 (0.0%) **(0.0%) 1,521 (4.6%) 5,398 (16.4%) 17,994 (54.7%) 109 (0.3%) 139 (0.4%) 8,671 (26.4%) 581 (1.8%) 0.56 (0.76) 10,854 (33.0%) 2,080 (6.3%) | **(0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) 0 (0.0%) **(0.0%) 607 (3.7%) 3,537 (21.8%) 8,891 (54.8%) 46 (0.3%) 33 (0.2%) 57 (0.4%) 4,164 (25.7%) 248 (1.5%) 0.58 (0.82) 4,940 (30.5%) 891 (5.5%) | #DIV/0! 0.02 #DIV/0! #DIV/0! #DIV/0! #DIV/0! #DIV/0! 0.05 -0.14 #DIV/0! 0.03 0.02 0.02 0.02 -0.03 0.05 | #VALUE! 18222 (27.2%) 1,391 (6.0%) 0 (0.0%) #VALUE! 2844 (4.3%) 8718 (13.0%) 11,518 (50.0%) #VALUE! 197 (0.3%) #O.3%) 16322 (24.4%) 996 (1.5%) 0.47 (0.74) 18510 (27.7%) 3239 (4.8%) | #VALUEI 8869 (27.6%) 507 (5.4%) 0 (0.0%) 0 (0.0%) #VALUEI 1140 (3.6%) 5608 (17.5%) 4,633 (49.3%) 254 (0.8%) #VALUEI #VALUEI 7502 (23.4%) 434 (1.4%) 0.49 (0.82) 8245 (25.7%) 1397 (4.4%) | #VALUE! -0.01 0.03 #DIV/0! #DIV/0! #DIV/0! #VALUE! 0.04 -0.13 0.01 -0.01 #VALUE! #VALUE! 0.02 0.01 |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 Inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Lower/ unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests or deredmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) | ** (0.0%) 2,932 (26.8%) 739 (6.8%) 0 (0.0%) 0 (0.0%) 73 (0.7%) 504 (4.6%) 1,356 (12.4%) 5,272 (48.2%) 3,05 4 (0.1%) 22 (0.2%) 2,367 (21.6%) 128 (1.2%) 0.46 (0.71) 2,563 (23.4%) | ** (0.0%) 1,734 (26.9%) 491 (7.6%) 0 (0.0%) 0 (0.0%) 49 (0.8%) 232 (3.6%) 1,060 (16.4%) 95 (48.0%) 71 (1.1%) ** (0.1%) 13 (0.2%) 1,341 (20.8%) 85 (1.3%) 0.45 (0.88) 1,362 (21.1%) | #DIV/01 0.00 #DIV/01 #DIV/01 -0.01 0.05 -0.11 #DIV/01 -0.05 0.00 0.00 0.00 0.00 0.02 -0.01 0.01 | ** (0.0%) 4,029 (17.5%) 1,391 (6.0%) 0 (0.0%) 171 (0.7%) 819 (3.6%) 1,964 (8.5%) 11,518 (50.0%) 254 (1.1%) 36 (0.2%) 36 (0.2%) 5,284 (22.9%) 287 (1.2%) 0.34 (0.71) 5,093 (22.1%) | ** (0.0%) 1,736 (18.5%) 507 (5.4%) 0 (0.0%) 0 (0.0%) 81 (0.9%) 301 (3.2%) 1,011 (10.7%) 4,633 (49.3%) 137 (1.5%) ** (0.1%) ** (0.1%) 1,997 (21.2%) 101 (1.1%) 0.36 (0.78) 1,943 (20.7%) | #DIV/01 -0.03 #DIV/01 #DIV/01 -0.02 -0.07 #DIV/01 -0.04 -0.03 -0.04 -0.01 -0.03 -0.04 -0.01 | 15 (0.0%) 11,261 (34.2%) 2,747 (8.4%) 0 (0.0%) 0 (0.0%) ** (0.0%) 1,521 (4.6%) 5,398 (16.4%) 17,994 (54.7%) 158 (0.5%) 109 (0.3%) 139 (0.4%) 8,671 (26.4%) 581 (1.8%) 0.56 (0.76) 10,854 (33.0%) | ** (0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) ** (0.0%) 607 (3.7%) 3,537 (21.8%) 8,891 (54.8%) 46 (0.3%) 33 (0.2%) 57 (0.4%) 4,164 (25.7%) 248 (1.5%) 0.58 (0.82) 4,940 (30.5%) | #DIV/01 0.02 #DIV/01 #DIV/01 #DIV/01 #DIV/01 #DIV/01 #DIV/01 0.05 -0.14 #DIV/01 0.03 0.02 0.00 0.02 0.02 -0.02 | #VALUE! 18222 (27.2%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) #VALUE! 2844 (4.3%) 8718 (13.0%) 11,518 (50.0%) #VALUE! 197 (0.3%) 16322 (24.4%) 996 (1.5%) 0.47 (0.74) 18510 (27.7%) | #VALUE! 8869 (27.6%) 507 (5.4%) 0 (0.0%) 0 (0.0%) #WALUE! 1140 (3.6%) 5608 (17.5%) 4,633 (49.3%) 254 (0.8%) #VALUE! #VALUE! #VALUE! 7502 (23.4%) 434 (1.4%) 0.49 (0.82) 8245 (25.7%) | #VALUE! -0.01 0.03 #DIV/0! #DIV/0! #VALUE! 0.04 -0.13 0.01 -0.01 #VALUE! #VALUE! 0.02 0.01 0.00 0.05 |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease: n (%) Major Surgery; n (%) Upper Gl bleed; n (%) Lower/ unspecified Gl bleed; n (%) Urogenital bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of liNR (prothrombin) tests ordered | **(0.0%) 2,932 (26.8%) 739 (6.8%) 0 (0.0%) 0 (0.0%) 73 (0.7%) 504 (4.6%) 1,356 (12.4%) 5,272 (48.2%) 63 (0.6%) **(0.1%) 22 (0.2%) 2,367 (21.6%) 128 (1.2%) 0.46 (0.71) 2,563 (23.4%) 385 (3.5%) **(0.0%) | ** (0.0%) 1,734 (26.9%) 491 (7.6%) 0 (0.0%) 0 (0.0%) 49 (0.8%) 232 (3.6%) 1,060 (16.4%) 95 (48.0%) 71 (1.1%) ** (0.1%) 13 (0.2%) 1,341 (20.8%) 85 (13.3%) 0.45 (0.88) 1,362 (21.1%) 0 (0.0%) | #DIV/0! 0.00 #DIV/0! #DIV/0! -0.01 0.05 -0.11 #DIV/0! -0.05 0.00 0.00 0.00 0.02 -0.01 0.01 0.06 0.02 #DIV/0! | ** (0.0%) 4,029 (17.5%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) 171 (0.7%) 819 (3.6%) 1,964 (8.5%) 11,518 (50.0%) 254 (1.1%) 36 (0.2%) 36 (0.2%) 5,284 (22.9%) 287 (1.2%) 0.34 (0.71) 5,093 (22.1%) 774 (3.4%) 24 (0.1%) | ** (0.0%) 1,736 (18.5%) 507 (5.4%) 0 (0.0%) 0 (0.0%) 31 (0.9%) 301 (3.2%) 1,011 (10.7%) 4,633 (49.3%) 137 (1.5%) ** (0.1%) 1,997 (21.2%) 0.36 (0.78) 1,943 (20.7%) 305 (3.2%) 0 (0.0%) | #DIV/01 -0.03 #DIV/01 #DIV/01 -0.02 -0.07 #DIV/01 -0.04 -0.03 -0.04 -0.01 -0.03 -0.04 -0.01 | 15 (0.0%) 11,261 (34.2%) 2,747 (8.4%) 0 (0.0%) 0 (0.0%) **(0.0%) 1,521 (4.6%) 5,398 (16.4%) 17,994 (54.7%) 158 (0.5%) 139 (0.3%) 8,671 (26.4%) 0.56 (0.76) 10,854 (33.0%) 2,080 (6.3%) **(0.0%) | ** (0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) 0 (0.0%) ** (0.0%) 607 (3.7%) 3,537 (21.8%) 8,891 (54.8%) 46 (0.3%) 33 (0.2%) 57 (0.4%) 4,164 (25.7%) 248 (1.5%) 0.58 (0.82) 4,940 (30.5%) 891 (5.5%) 0 (0.0%) | #DIV/01 0.02 #DIV/01 #DIV/01 #DIV/01 #DIV/01 #DIV/01 0.05 -0.14 #DIV/01 0.03 0.02 0.00 0.02 0.02 0.02 0.03 #DIV/01 | #VALUE! 18222 (27.2%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) #VALUE! 2844 (4.3%) 8718 (13.0%) 11,518 (50.0%) 475 (0.7%) #VALUE! 197 (0.3%) 0.47 (0.74) 18510 (27.7%) 3239 (4.8%) #VALUE! | #VALUEI 8869 (27.6%) 507 (5.4%) 0 (0.0%) 0 (0.0%) #VALUEI 1140 (3.6%) 5608 (17.5%) 4,633 (49.3%) 254 (0.8%) #VALUEI 7502 (23.4%) 434 (1.4%) 0.49 (0.82) 8245 (25.7%) 1397 (4.4%) 0 (0.0%) | #VALUE! -0.01 0.03 #DIV/0! #DIV/0! #VALUE! 0.04 -0.13 0.01 -0.01 #VALUE! #VALUE! #VALUE! 0.02 0.01 0.00 0.05 0.02 #VALUE! |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Lower/ unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of lipid tests orderedmean (sd) | ** (0.0%) 2,932 (26.8%) 739 (6.8%) 0 (0.0%) 0 (0.0%) 504 (4.6%) 1,356 (12.4%) 5,272 (48.2%) 63 (0.6%) ** (0.1%) 22 (0.2%) 2,367 (21.6%) 128 (1.2%) 0.46 (0.71) 2,563 (23.4%) 385 (3.5%) ** (0.0%) | ** (0.0%) 1,734 (26.9%) 491 (7.6%) 0 (0.0%) 49 (0.8%) 232 (3.6%) 1,060 (16.4%) 95 (48.0%) 71 (1.1%) ** (0.1%) 13 (0.2%) 1,341 (20.8%) 85 (1.3%) 0.45 (0.88) 1,362 (21.1%) 201 (3.1%) 0 (0.0%) 0.31 (0.75) | #DIV/0! 0.00 #DIV/0! #DIV/0! #DIV/0! #DIV/0! -0.01 0.05 -0.11 #DIV/0! -0.05 0.00 0.00 0.02 -0.01 0.01 0.06 0.02 #DIV/0! | ** (0.0%) 4,029 (17.5%) 1,391 (6.0%) 0 (0.0%) 171 (0.7%) 819 (3.6%) 1,964 (8.5%) 11,518 (50.0%) 36 (0.2%) 36 (0.2%) 5,284 (22.9%) 287 (1.2%) 0.34 (0.71) 5,093 (22.1%) 774 (3.4%) 24 (0.1%) | ** (0.0%) 1,736 (18.5%) 507 (5.4%) 0 (0.0%) 0 (0.0%) 81 (0.9%) 301 (3.2%) 1,011 (10.7%) 4,633 (49.3%) 137 (1.5%) ** (0.1%) 1,019 (1.1%) 1,019 (1.1%) 0.36 (0.78) 1,943 (20.7%) 305 (3.2%) 0 (0.0%) | #DIV/0! -0.03 #DIV/0! #DIV/0! #DIV/0! #DIV/0! -0.02 -0.07 #DIV/0! -0.04 -0.03 -0.04 -0.01 -0.03 -0.04 -0.01 | 15 (0.0%) 11,261 (34.2%) 2,747 (8.4%) 0 (0.0%) 0 (0.0%) **(0.0%) **(0.0%) 1,521 (4.6%) 5,398 (16.4%) 17,994 (54.7%) 109 (0.3%) 139 (0.4%) 8,671 (26.4%) 581 (1.8%) 0.56 (0.76) 10,854 (33.0%) 2,080 (6.3%) ***(0.0%) | **(0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) 0 (0.0%) **(0.0%) 607 (3.7%) 3,537 (21.8%) 8,891 (54.8%) 46 (0.3%) 33 (0.2%) 57 (0.4%) 4,164 (25.7%) 248 (1.5%) 0.58 (0.82) 4,940 (30.5%) 891 (5.5%) 0 (0.0%) | #DIV/0! 0.02 #DIV/0! #DIV/0! #DIV/0! #DIV/0! #DIV/0! 0.05 -0.14 #DIV/0! 0.03 0.02 0.02 0.02 0.02 0.02 -0.03 #DIV/0! 0.03 | #VALUE! 18222 (27.2%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) #VALUE! 2844 (4.3%) 8718 (13.0%) 11,518 (50.0%) 475 (0.7%) #VALUE! 197 (0.3%) 16322 (24.4%) 996 (1.5%) 0.47 (0.74) 18510 (27.7%) 3239 (4.8%) #VALUE! | #VALUEI 8869 (27.6%) 507 (5.4%) 0 (0.0%) 0 (0.0%) #VALUEI 1140 (3.6%) 5608 (17.5%) 4,633 (49.3%) 254 (0.8%) #VALUEI #VALUEI 7502 (23.4%) 434 (1.4%) 0.49 (0.82) 8245 (25.7%) 1397 (4.4%) 0 (0.0%) | #VALUE! -0.01 0.03 #DIV/0! #DIV/0! #DIV/0! #VALUE! 0.04 -0.13 0.01 -0.01 #VALUE! #VALUE! 0.02 0.01 0.05 0.02 #VALUE! |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Lower ( unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of INR (prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) | ** (0.0%) 2,932 (26.8%) 739 (6.8%) 0 (0.0%) 0 (0.0%) 3 (0.7%) 504 (4.6%) 1,356 (12.4%) 5,272 (48.2%) 63 (0.6%) ** (0.1%) 22 (0.2%) 2,367 (21.6%) 128 (1.2%) 0.46 (0.71) 2,563 (23.4%) 385 (3.5%) ** (0.0%) 0.45 (1.24) 6,854 (62.7%) | ** (0.0%) 1,734 (26.9%) 491 (7.6%) 0 (0.0%) 49 (0.8%) 232 (3.6%) 1,060 (16.4%) 95 (48.0%) 71 (1.1%) 13 (0.2%) 1,341 (20.8%) 85 (1.3%) 0.45 (0.88) 1,362 (21.1%) 201 (3.1%) 0 (0.0%) 0.31 (0.75) 4,359 (67.6%) | #DIV/0! 0.00 #DIV/0! #DIV/0! #DIV/0! -0.01 0.05 -0.11 #DIV/0! -0.05 0.00 0.00 0.00 0.00 0.01 0.01 0.06 0.02 #DIV/0! 0.14 -0.10 | ** (0.0%) 4,029 (17.5%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) 171 (0.7%) 819 (3.6%) 1,964 (8.5%) 11,518 (50.0%) 254 (1.1%) 36 (0.2%) 36 (0.2%) 36 (0.2%) 287 (1.2%) 0.34 (0.71) 5,093 (22.1%) 774 (3.4%) 24 (0.1%) 0.43 (1.02) 12,270 (53.3%) | ** (0.0%) 1,736 (18.5%) 507 (5.4%) 0 (0.0%) 0 (0.0%) 81 (0.9%) 301 (3.2%) 1,011 (10.7%) 4,633 (49.3%) 137 (1.5%) ** (0.1%) 0.10 (1.1%) 0.36 (0.78) 1,943 (20.7%) 305 (3.2%) 0 (0.0%) 0.31 (0.74) 5,766 (61.3%) | #DIV/0! -0.03 #DIV/0! #DIV/0! -0.02 -0.07 #DIV/0! -0.04 -0.03 -0.03 -0.04 -0.01 -0.03 -0.03 -0.01 -0.04 | 15 (0.0%) 11,261 (34.2%) 2,747 (8.4%) 0 (0.0%) 0 (0.0%) 15,21 (4.6%) 5,398 (16.4%) 17,994 (54.7%) 158 (0.5%) 109 (0.3%) 139 (0.4%) 8,671 (26.4%) 581 (1.8%) 0.56 (0.76) 10,854 (33.0%) 2,080 (6.3%) **(0.0%) | ** (0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) 0 (0.0%) ** (0.0%) (507 (3.7%) 3,537 (21.8%) 46 (0.3%) 33 (0.2%) 57 (0.4%) 4,164 (25.7%) 248 (1.5%) 0.58 (0.82) 4,940 (30.5%) 891 (5.5%) 0 (0.0%) 0.31 (0.63) 10.824 (66.7%) | #DIV/0! 0.02 #DIV/0! #DIV/0! #DIV/0! #DIV/0! #DIV/0! #DIV/0! 0.05 -0.14 #DIV/0! 0.03 0.02 0.00 0.02 0.02 0.02 0.03 0.05 #DIV/0! 0.06 -0.01 | #VALUE! 18222 (27.2%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) #VALUE! 2844 (4.3%) 8718 (13.0%) 11,518 (50.0%) 475 (0.7%) #VALUE! 197 (0.3%) 16322 (24.4%) 996 (1.5%) 0.47 (0.74) 18510 (27.7%) 3239 (4.8%) #VALUE! 0.39 (0.95) 40870 (61.1%) | #VALUE! 8869 (27.6%) 507 (5.4%) 0 (0.0%) 0 (0.0%) #VALUE! 1140 (3.6%) 5608 (17.5%) 4,633 (49.3%) 254 (0.8%) #VALUE! #VALUE! #VALUE! 7502 (23.4%) 434 (1.4%) 0.49 (0.82) 8245 (25.7%) 1397 (4.4%) 0 (0.0%) 0.31 (0.69) 20949 (55.3%) | #VALUE! -0.01 0.03 #DIV/01 #DIV/01 #VALUE! 0.04 -0.13 0.01 -0.01 #VALUE! 0.02 0.01 0.00 0.05 0.02 #VALUE! 0.00 -0.09 |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gl bleed; n (%) Lower/ unspecified Gl bleed; n (%) Urogenital bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of iNR (prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Primary Care Physician; n (%) | **(0.0%) 2,932 (26.8%) 739 (6.8%) 0 (0.0%) 0 (0.0%) 73 (0.7%) 504 (4.6%) 1,356 (12.4%) 5,272 (48.2%) 63 (0.6%) **(0.1%) 22 (0.2%) 2,367 (21.6%) 128 (1.2%) 0.46 (0.71) 2,563 (23.4%) 385 (3.5%) **(0.0%) | ** (0.0%) 1,734 (26.9%) 491 (7.6%) 0 (0.0%) 49 (0.8%) 49 (0.8%) 232 (3.6%) 1,060 (16.4%) 95 (48.0%) 71 (1.1%) ** (0.1%) 13 (0.2%) 1,341 (20.8%) 85 (1.3%) 0.45 (0.88) 1,362 (21.1%) 0 (0.0%) 0.31 (0.75) 4,359 (67.6%) 5,708 (88.5%) | #DIV/01 0.00 #DIV/01 #DIV/01 #DIV/01 #DIV/01 -0.01 0.05 -0.11 #DIV/01 -0.05 0.00 0.00 0.02 -0.01 0.06 0.02 #DIV/01 0.14 -0.10 0.09 | ** (0.0%) 4,029 (17.5%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) 171 (0.7%) 819 (3.6%) 1,964 (8.5%) 11,518 (50.0%) 36 (0.2%) 36 (0.2%) 36 (0.2%) 5,284 (22.9%) 287 (1.2%) 0.34 (0.71) 5,093 (22.1%) 774 (3.4%) 24 (0.1%) 0.43 (1.02) 12,270 (53.3%) 9,641 (41.8%) | ** (0.0%) 1,736 (18.5%) 507 (5.4%) 0 (0.0%) 0 (0.0%) 81 (0.9%) 301 (3.2%) 1,011 (10.7%) 4,633 (49.3%) 137 (1.5%) ** (0.1%) ** (0.1%) 1,997 (21.2%) 0.36 (0.78) 1,943 (20.7%) 305 (3.2%) 0 (0.0%) 0.31 (0.74) 5,766 (61.3%) 4,170 (44.3%) | #DIV/0! -0.03 #DIV/0! #DIV/0! #DIV/0! #DIV/0! -0.02 -0.07 #DIV/0! -0.04 -0.03 -0.04 -0.01 -0.03 -0.04 -0.01 -0.03 -0.01 -0.03 -0.01 -0.03 -0.01 -0.05 | 15 (0.0%) 11,261 (34.2%) 2,747 (8.4%) 0 (0.0%) 0 (0.0%) **(0.0%) 1,521 (4.6%) 5,398 (16.4%) 17,994 (54.7%) 158 (0.5%) 139 (0.3%) 139 (0.4%) 8,671 (26.4%) 581 (1.8%) 0.56 (0.76) 10,854 (33.0%) 2,080 (6.3%) **(0.0%) | **(0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) 0 (0.0%) **(0.0%) 607 (3.7%) 3,537 (21.8%) 8,891 (54.8%) 46 (0.3%) 33 (0.2%) 57 (0.4%) 4,164 (25.7%) 248 (1.5%) 0.58 (0.82) 4,940 (30.5%) 891 (5.5%) 0 (0.0%) 0.31 (0.63) 10,824 (66.7%) 6,722 (41.4%) | #DIV/01 0.02 #DIV/01 #DIV/01 #DIV/01 #DIV/01 #DIV/01 0.05 -0.14 #DIV/01 0.03 0.02 0.00 0.02 0.02 -0.03 #DIV/01 0.05 0.03 #DIV/01 0.06 -0.01 0.03 | #VALUE! 18222 (27.2%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) #VALUE! 2844 (4.3%) 8718 (13.0%) 11,518 (50.0%) #VALUE! 197 (0.3%) 16322 (24.4%) 996 (1.5%) 0.47 (0.74) 18510 (27.7%) 3239 (4.8%) #VALUE! 0.39 (0.95) 40870 (61.1%) 33733 (50.4%) | #VALUEI 8869 (27.6%) 507 (5.4%) 0 (0.0%) 0 (0.0%) #VALUEI 1140 (3.6%) 5608 (17.5%) 4,633 (49.3%) 4,633 (49.3%) #VALUEI #VALUEI #VALUEI 7502 (23.4%) 434 (1.4%) 0.49 (0.82) 8245 (25.7%) 1397 (4.4%) 0 (0.0%) 0.31 (0.69) 20949 (65.3%) 16600 (51.8%) | #VALUE! -0.01 0.03 #DIV/0! #DIV/0! #VALUE! 0.04 -0.13 0.01 -0.01 +VALUE! #VALUE! #VALUE! 0.02 0.01 0.00 0.05 0.02 #VALUE! |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Lower ( unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of INR (prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) | ** (0.0%) 2,932 (26.8%) 739 (6.8%) 0 (0.0%) 0 (0.0%) 3 (0.7%) 504 (4.6%) 1,356 (12.4%) 5,272 (48.2%) 63 (0.6%) ** (0.1%) 22 (0.2%) 2,367 (21.6%) 128 (1.2%) 0.46 (0.71) 2,563 (23.4%) 385 (3.5%) ** (0.0%) 0.45 (1.24) 6,854 (62.7%) | ** (0.0%) 1,734 (26.9%) 491 (7.6%) 0 (0.0%) 49 (0.8%) 232 (3.6%) 1,060 (16.4%) 95 (48.0%) 71 (1.1%) 13 (0.2%) 1,341 (20.8%) 85 (1.3%) 0.45 (0.88) 1,362 (21.1%) 201 (3.1%) 0 (0.0%) 0.31 (0.75) 4,359 (67.6%) | #DIV/0! 0.00 #DIV/0! #DIV/0! #DIV/0! -0.01 0.05 -0.11 #DIV/0! -0.05 0.00 0.00 0.00 0.00 0.01 0.01 0.06 0.02 #DIV/0! 0.14 -0.10 | ** (0.0%) 4,029 (17.5%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) 171 (0.7%) 819 (3.6%) 1,964 (8.5%) 11,518 (50.0%) 254 (1.1%) 36 (0.2%) 36 (0.2%) 36 (0.2%) 287 (1.2%) 0.34 (0.71) 5,093 (22.1%) 774 (3.4%) 24 (0.1%) 0.43 (1.02) 12,270 (53.3%) | ** (0.0%) 1,736 (18.5%) 507 (5.4%) 0 (0.0%) 0 (0.0%) 81 (0.9%) 301 (3.2%) 1,011 (10.7%) 4,633 (49.3%) 137 (1.5%) ** (0.1%) 0.10 (1.1%) 0.36 (0.78) 1,943 (20.7%) 305 (3.2%) 0 (0.0%) 0.31 (0.74) 5,766 (61.3%) | #DIV/0! -0.03 #DIV/0! #DIV/0! -0.02 -0.07 #DIV/0! -0.04 -0.03 -0.03 -0.04 -0.01 -0.03 -0.03 -0.01 -0.04 | 15 (0.0%) 11,261 (34.2%) 2,747 (8.4%) 0 (0.0%) 0 (0.0%) 15,21 (4.6%) 5,398 (16.4%) 17,994 (54.7%) 158 (0.5%) 109 (0.3%) 139 (0.4%) 8,671 (26.4%) 581 (1.8%) 0.56 (0.76) 10,854 (33.0%) 2,080 (6.3%) **(0.0%) | ** (0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) 0 (0.0%) ** (0.0%) (507 (3.7%) 3,537 (21.8%) 46 (0.3%) 33 (0.2%) 57 (0.4%) 4,164 (25.7%) 248 (1.5%) 0.58 (0.82) 4,940 (30.5%) 891 (5.5%) 0 (0.0%) 0.31 (0.63) 10.824 (66.7%) | #DIV/0! 0.02 #DIV/0! #DIV/0! #DIV/0! #DIV/0! #DIV/0! #DIV/0! 0.05 -0.14 #DIV/0! 0.03 0.02 0.00 0.02 0.02 0.02 0.03 0.05 #DIV/0! 0.06 -0.01 | #VALUE! 18222 (27.2%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) #VALUE! 2844 (4.3%) 8718 (13.0%) 11,518 (50.0%) #VALUE! 197 (0.3%) 16322 (24.4%) 996 (1.5%) 0.47 (0.74) 18510 (27.7%) 3239 (4.8%) 473 (0.9%) 473 (0.9%) 6347 (61.1%) 33733 (50.4%) 65477 (97.9%) | #VALUEI 8869 (27.6%) 507 (5.4%) 0 (0.0%) 0 (0.0%) #VALUEI 1140 (3.6%) 5608 (17.5%) 4,633 (49.3%) 254 (0.8%) #VALUEI #VALUEI 7502 (23.4%) 434 (1.4%) 0.49 (0.82) 8245 (25.7%) 1397 (4.4%) 0 (0.0%) 0.31 (0.69) 20949 (65.3%) 16600 (51.8%) 31393 (97.9%) | #VALUE! -0.01 0.03 #DIV/01 #DIV/01 #VALUE! 0.04 -0.13 0.01 -0.01 #VALUE! 0.02 0.01 0.00 0.05 0.02 #VALUE! 0.00 -0.09 |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gl bleed; n (%) Lower/ unspecified Gl bleed; n (%) Urogenital bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of iNR (prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Primary Care Physician; n (%) | **(0.0%) 2,932 (26.8%) 739 (6.8%) 0 (0.0%) 0 (0.0%) 73 (0.7%) 504 (4.6%) 1,356 (12.4%) 5,272 (48.2%) 63 (0.6%) **(0.1%) 22 (0.2%) 2,367 (21.6%) 128 (1.2%) 0.46 (0.71) 2,563 (23.4%) 385 (3.5%) **(0.0%) | ** (0.0%) 1,734 (26.9%) 491 (7.6%) 0 (0.0%) 49 (0.8%) 49 (0.8%) 232 (3.6%) 1,060 (16.4%) 95 (48.0%) 71 (1.1%) ** (0.1%) 13 (0.2%) 1,341 (20.8%) 85 (1.3%) 0.45 (0.88) 1,362 (21.1%) 0 (0.0%) 0.31 (0.75) 4,359 (67.6%) 5,708 (88.5%) | #DIV/01 0.00 #DIV/01 #DIV/01 #DIV/01 #DIV/01 -0.01 0.05 -0.11 #DIV/01 -0.05 0.00 0.00 0.02 -0.01 0.06 0.02 #DIV/01 0.14 -0.10 0.09 | ** (0.0%) 4,029 (17.5%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) 171 (0.7%) 819 (3.6%) 1,964 (8.5%) 11,518 (50.0%) 36 (0.2%) 36 (0.2%) 36 (0.2%) 5,284 (22.9%) 287 (1.2%) 0.34 (0.71) 5,093 (22.1%) 774 (3.4%) 24 (0.1%) 0.43 (1.02) 12,270 (53.3%) 9,641 (41.8%) | ** (0.0%) 1,736 (18.5%) 507 (5.4%) 0 (0.0%) 0 (0.0%) 81 (0.9%) 301 (3.2%) 1,011 (10.7%) 4,633 (49.3%) 137 (1.5%) ** (0.1%) ** (0.1%) 1,997 (21.2%) 0.36 (0.78) 1,943 (20.7%) 305 (3.2%) 0 (0.0%) 0.31 (0.74) 5,766 (61.3%) 4,170 (44.3%) | #DIV/0! -0.03 #DIV/0! #DIV/0! #DIV/0! #DIV/0! -0.02 -0.07 #DIV/0! -0.04 -0.03 -0.04 -0.01 -0.03 -0.04 -0.01 -0.03 -0.01 -0.03 -0.01 -0.03 -0.01 -0.05 | 15 (0.0%) 11,261 (34.2%) 2,747 (8.4%) 0 (0.0%) 0 (0.0%) **(0.0%) 1,521 (4.6%) 5,398 (16.4%) 17,994 (54.7%) 158 (0.5%) 139 (0.3%) 139 (0.4%) 8,671 (26.4%) 581 (1.8%) 0.56 (0.76) 10,854 (33.0%) 2,080 (6.3%) **(0.0%) | **(0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) 0 (0.0%) **(0.0%) 607 (3.7%) 3,537 (21.8%) 8,891 (54.8%) 46 (0.3%) 33 (0.2%) 57 (0.4%) 4,164 (25.7%) 248 (1.5%) 0.58 (0.82) 4,940 (30.5%) 891 (5.5%) 0 (0.0%) 0.31 (0.63) 10,824 (66.7%) 6,722 (41.4%) | #DIV/01 0.02 #DIV/01 #DIV/01 #DIV/01 #DIV/01 #DIV/01 0.05 -0.14 #DIV/01 0.03 0.02 0.00 0.02 0.02 -0.03 #DIV/01 0.05 0.03 #DIV/01 0.06 -0.01 0.03 | #VALUE! 18222 (27.2%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) #VALUE! 2844 (4.3%) 8718 (13.0%) 11,518 (50.0%) #VALUE! 197 (0.3%) 16322 (24.4%) 996 (1.5%) 0.47 (0.74) 18510 (27.7%) 3239 (4.8%) #VALUE! 0.39 (0.95) 40870 (61.1%) 33733 (50.4%) | #VALUEI 8869 (27.6%) 507 (5.4%) 0 (0.0%) 0 (0.0%) #VALUEI 1140 (3.6%) 5608 (17.5%) 4,633 (49.3%) 4,633 (49.3%) #VALUEI #VALUEI #VALUEI 7502 (23.4%) 434 (1.4%) 0.49 (0.82) 8245 (25.7%) 1397 (4.4%) 0 (0.0%) 0.31 (0.69) 20949 (65.3%) 16600 (51.8%) | #VALUE! -0.01 0.03 #DIV/0! #DIV/0! #VALUE! 0.04 -0.13 0.01 -0.01 +VALUE! #VALUE! #VALUE! 0.02 0.01 0.00 0.05 0.02 #VALUE! |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Lower/ unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of link (prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Primary Care Physician; n (%) Treating prescriber - Primary Care Physician; n (%) | **(0.0%) 2,932 (26.8%) 739 (6.8%) 0 (0.0%) 0 (0.0%) 504 (4.6%) 1,356 (12.4%) 5,272 (48.2%) 63 (0.6%) **(0.1%) 22 (0.2%) 2,367 (21.6%) 128 (1.2%) 0.46 (0.71) 2,563 (23.4%) 385 (3.5%) ***(0.0%) 0.45 (1.24) 6,884 (62.7%) 9,965 (91.1%) 10,881 (91.5%) | ** (0.0%) 1,734 (26.9%) 491 (7.6%) 0 (0.0%) 0 (0.0%) 49 (0.8%) 232 (3.6%) 1,060 (16.4%) 95 (48.0%) 71 (1.1%) ** (0.1%) 13 (0.2%) 1,341 (20.8%) 85 (1.3%) 0.45 (0.88) 1,362 (21.1%) 201 (3.1%) 201 (3.1%) 0 (0.0%) 0.31 (0.75) 4,359 (67.6%) 5,708 (88.5%) 6,428 (99.7%) | #DIV/0! 0.00 #DIV/0! #DIV/0! #DIV/0! #DIV/0! -0.01 0.05 -0.11 #DIV/0! -0.05 0.00 0.00 0.02 -0.01 0.01 0.06 0.02 #DIV/0! 0.14 -0.10 0.09 -0.03 | ** (0.0%) 4,029 (17.5%) 1,391 (6.0%) 0 (0.0%) 171 (0.7%) 819 (3.6%) 1,964 (8.5%) 11,518 (50.0%) 36 (0.2%) 36 (0.2%) 36 (0.2%) 287 (1.2%) 0.34 (0.71) 5,093 (22.1%) 774 (3.4%) 24 (0.1%) 0.43 (1.02) 12,270 (53.3%) 9,641 (41.8%) 21,748 (94.4%) | ** (0.0%) 1,736 (18.5%) 507 (5.4%) 0 (0.0%) 0 (0.0%) 81 (0.9%) 301 (3.2%) 1,011 (10.7%) 4,633 (49.3%) 137 (1.5%) ** (0.1%) 1,019 (1.1%) 0.36 (0.78) 1,997 (21.2%) 101 (1.1%) 0.36 (0.78) 1,943 (20.7%) 305 (3.2%) 0 (0.0%) 0.31 (0.74) 5,766 (61.3%) 4,170 (44.3%) 8,758 (93.1%) | #DIV/0! -0.03 #DIV/0! #DIV/0! #DIV/0! #DIV/0! -0.02 -0.07 #DIV/0! -0.04 -0.03 -0.04 -0.01 -0.03 -0.04 -0.01 -0.03 -0.04 -0.05 -0.05 | 15 (0.0%) 11,261 (34.2%) 2,747 (8.4%) 0 (0.0%) 0 (0.0%) 1,521 (4.6%) 5,398 (16.4%) 17,994 (54.7%) 139 (0.3%) 139 (0.4%) 8,671 (26.4%) 581 (1.8%) 0.56 (0.76) 10,854 (33.0%) 2,080 (6.3%) **(0.0%) 0.35 (0.77) 21,746 (66.1%) 14,127 (42.9%) 32,848 (99.9%) | **(0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) 0 (0.0%) **(0.0%) 607 (3.7%) 3,537 (21.8%) 46 (0.3%) 33 (0.2%) 57 (0.4%) 4,164 (25.7%) 248 (1.5%) 0.58 (0.82) 4,940 (30.5%) 891 (5.5%) 0 (0.0%) 0.31 (0.63) 10,824 (66.7%) 6,722 (41.4%) 16,207 (99.9%) | #DIV/0! 0.02 #DIV/0! #DIV/0! #DIV/0! #DIV/0! #DIV/0! 0.05 -0.14 #DIV/0! 0.03 0.02 0.02 0.02 0.02 0.03 #DIV/0! 0.03 #DIV/0! 0.03 0.05 0.03 #DIV/0! | #VALUE! 18222 (27.2%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) #VALUE! 2844 (4.3%) 8718 (13.0%) 11,518 (50.0%) #VALUE! 197 (0.3%) 16322 (24.4%) 996 (1.5%) 0.47 (0.74) 18510 (27.7%) 3239 (4.8%) 473 (0.9%) 473 (0.9%) 6347 (61.1%) 33733 (50.4%) 65477 (97.9%) | #VALUEI 8869 (27.6%) 507 (5.4%) 0 (0.0%) 0 (0.0%) #VALUEI 1140 (3.6%) 5608 (17.5%) 4,633 (49.3%) 254 (0.8%) #VALUEI #VALUEI 7502 (23.4%) 434 (1.4%) 0.49 (0.82) 8245 (25.7%) 1397 (4.4%) 0 (0.0%) 0.31 (0.69) 20949 (65.3%) 16600 (51.8%) 31393 (97.9%) | #VALUE! -0.01 0.03 #DIV/0! #DIV/0! #DIV/0! #VALUE! 0.04 -0.13 0.01 -0.01 #VALUE! #VALUE! 0.02 0.01 0.05 0.02 #VALUE! 0.00 -0.09 -0.03 0.00 |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 Inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Lower ( unspecified Gi bleed; n (%) Urogenital bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP Inhibitors; n (%) Other astroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Number of INR (prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Primary Care Physician; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) | **(0.0%) 2,932 (26.8%) 739 (6.8%) 0 (0.0%) 0 (0.0%) 504 (4.6%) 1,356 (12.4%) 5,272 (48.2%) 63 (0.6%) **(0.1%) 22 (0.2%) 2,367 (21.6%) 128 (1.2%) 0.46 (0.71) 2,563 (23.4%) 385 (3.5%) ***(0.0%) 0.45 (1.24) 6,884 (62.7%) 9,965 (91.1%) 10,881 (91.5%) | ** (0.0%) 1,734 (26.9%) 491 (7.6%) 0 (0.0%) 0 (0.0%) 49 (0.8%) 232 (3.6%) 1,060 (16.4%) 95 (48.0%) 71 (1.1%) ** (0.1%) 13 (0.2%) 1,341 (20.8%) 85 (1.3%) 0.45 (0.88) 1,362 (21.1%) 201 (3.1%) 201 (3.1%) 0 (0.0%) 0.31 (0.75) 4,359 (67.6%) 5,708 (88.5%) 6,428 (99.7%) | #DIV/0! 0.00 #DIV/0! #DIV/0! #DIV/0! #DIV/0! -0.01 0.05 -0.11 #DIV/0! -0.05 0.00 0.00 0.02 -0.01 0.01 0.06 0.02 #DIV/0! 0.14 -0.10 0.09 -0.03 | ** (0.0%) 4,029 (17.5%) 1,391 (6.0%) 0 (0.0%) 171 (0.7%) 819 (3.6%) 1,964 (8.5%) 11,518 (50.0%) 36 (0.2%) 36 (0.2%) 36 (0.2%) 287 (1.2%) 0.34 (0.71) 5,093 (22.1%) 774 (3.4%) 24 (0.1%) 0.43 (1.02) 12,270 (53.3%) 9,641 (41.8%) 21,748 (94.4%) | ** (0.0%) 1,736 (18.5%) 507 (5.4%) 0 (0.0%) 0 (0.0%) 81 (0.9%) 301 (3.2%) 1,011 (10.7%) 4,633 (49.3%) 137 (1.5%) ** (0.1%) 1,019 (1.1%) 0.36 (0.78) 1,997 (21.2%) 101 (1.1%) 0.36 (0.78) 1,943 (20.7%) 305 (3.2%) 0 (0.0%) 0.31 (0.74) 5,766 (61.3%) 4,170 (44.3%) 8,758 (93.1%) | #DIV/0! -0.03 #DIV/0! #DIV/0! #DIV/0! #DIV/0! -0.02 -0.07 #DIV/0! -0.04 -0.03 -0.04 -0.01 -0.03 -0.04 -0.01 -0.03 -0.04 -0.05 -0.05 | 15 (0.0%) 11,261 (34.2%) 2,747 (8.4%) 0 (0.0%) 0 (0.0%) 1,521 (4.6%) 5,398 (16.4%) 17,994 (54.7%) 139 (0.3%) 139 (0.4%) 8,671 (26.4%) 581 (1.8%) 0.56 (0.76) 10,854 (33.0%) 2,080 (6.3%) **(0.0%) 0.35 (0.77) 21,746 (66.1%) 14,127 (42.9%) 32,848 (99.9%) | **(0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) 0 (0.0%) **(0.0%) 607 (3.7%) 3,537 (21.8%) 46 (0.3%) 33 (0.2%) 57 (0.4%) 4,164 (25.7%) 248 (1.5%) 0.58 (0.82) 4,940 (30.5%) 891 (5.5%) 0 (0.0%) 0.31 (0.63) 10,824 (66.7%) 6,722 (41.4%) 16,207 (99.9%) | #DIV/0! 0.02 #DIV/0! #DIV/0! #DIV/0! #DIV/0! #DIV/0! 0.05 -0.14 #DIV/0! 0.03 0.02 0.02 0.02 0.02 0.03 #DIV/0! 0.03 #DIV/0! 0.03 0.05 0.03 #DIV/0! | #VALUE! 18222 (27.2%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) #VALUE! 2844 (4.3%) 8718 (13.0%) 11,518 (50.0%) #VALUE! 197 (0.3%) 16322 (24.4%) 996 (1.5%) 0.47 (0.74) 18510 (27.7%) 3239 (4.8%) 473 (0.9%) 473 (0.9%) 6347 (61.1%) 33733 (50.4%) 65477 (97.9%) | #VALUEI 8869 (27.6%) 507 (5.4%) 0 (0.0%) 0 (0.0%) #VALUEI 1140 (3.6%) 5608 (17.5%) 4,633 (49.3%) 254 (0.8%) #VALUEI #VALUEI 7502 (23.4%) 434 (1.4%) 0.49 (0.82) 8245 (25.7%) 1397 (4.4%) 0 (0.0%) 0.31 (0.69) 20949 (65.3%) 16600 (51.8%) 31393 (97.9%) | #VALUE! -0.01 0.03 #DIV/0! #DIV/0! #DIV/0! #VALUE! 0.04 -0.13 0.01 -0.01 #VALUE! #VALUE! 0.02 0.01 0.05 0.02 #VALUE! 0.00 -0.09 -0.03 0.00 |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Uoper Gi bleed; n (%) Urogenital bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Ytamin K therapy; n (%) Number of INR (prothrombin) tests orderedmean (sd) Treating prescriber - Primary Care Physician; n (%) Treating prescriber - Pramary Care Physician; n (%) Treating prescriber - Pramary Care Physician; n (%) Treating prescriber - Primary Care Physician; n (%) Treating prescriber - Gen (%) Alpha blockers; n (%) CHA2DS2 VASc score, 180 days, Vmean (sd) | **(0.0%) 2,932 (26.8%) 739 (6.8%) 0 (0.0%) 0 (0.0%) 3 (0.7%) 504 (4.6%) 1,356 (12.4%) 5,272 (48.2%) 63 (0.6%) **(0.1%) 22 (0.2%) 2,367 (21.6%) 128 (1.2%) 0.46 (0.71) 2,563 (23.4%) 385 (3.5%) **(0.0%) 0.45 (1.24) 6,854 (62.7%) 9,965 (91.1%) 10,881 (99.5%) 747 (6.8%) | ** (0.0%) 1,734 (26.9%) 491 (7.6%) 0 (0.0%) 49 (0.8%) 232 (3.6%) 1,060 (16.4%) 95 (48.0%) 71 (1.1%) 13 (0.2%) 1,341 (20.8%) 85 (1.3%) 0.45 (0.88) 1,362 (21.1%) 201 (3.1%) 0 (0.0%) 0.31 (0.75) 4,359 (7.6%) 5,708 (88.5%) 6,428 (99.7%) 400 (6.2%) | #DIV/0! 0.00 #DIV/0! #DIV/0! #DIV/0! #DIV/0! -0.01 0.05 -0.11 #DIV/0! -0.05 0.00 0.02 -0.01 0.06 0.02 #DIV/0! 0.14 -0.10 0.09 -0.03 0.02 | ** (0.0%) 4,029 (17.5%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) 171 (0.7%) 819 (3.6%) 1,964 (8.5%) 11,518 (50.0%) 254 (1.1%) 36 (0.2%) 36 (0.2%) 36 (0.2%) 0.34 (0.71) 5,093 (22.1%) 774 (3.4%) 24 (0.1%) 0.43 (1.02) 12,270 (53.3%) 9,641 (41.8%) 21,748 (94.4%) 1,170 (5.1%) | ** (0.0%) 1,736 (18.5%) 507 (5.4%) 0 (0.0%) 0 (0.0%) 81 (0.9%) 301 (3.2%) 1,011 (10.7%) 4,633 (49.3%) 137 (1.5%) ** (0.1%) ** (0.1%) 1,997 (21.2%) 0.36 (0.78) 1,943 (20.7%) 305 (3.2%) 0 (0.0%) 0.31 (0.74) 5,766 (61.3%) 4,170 (44.3%) 8,758 (93.1%) 438 (4.7%) | #DIV/0! -0.03 #DIV/0! #DIV/0! #DIV/0! #DIV/0! -0.02 -0.07 #DIV/0! -0.04 -0.03 -0.04 -0.01 -0.03 -0.04 -0.01 -0.03 -0.05 -0.05 -0.05 | 15 (0.0%) 11,261 (34.2%) 2,747 (8.4%) 0 (0.0%) 0 (0.0%) **(0.0%) 1,521 (4.6%) 5,398 (16.4%) 17,994 (54.7%) 198 (0.3%) 139 (0.4%) 8,671 (26.4%) 581 (1.8%) 0.56 (0.76) 10,854 (33.0%) 2,080 (6.3%) **(0.0%) 0.35 (0.77) 21,746 (66.1%) 14,127 (42.9%) 32,848 (99.9%) 3,271 (9.9%) | **(0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) 0 (0.0%) **(0.0%) 607 (3.7%) 3,537 (21.8%) 46 (0.3%) 33 (0.2%) 57 (0.4%) 4,164 (25.7%) 248 (1.5%) 0.58 (0.82) 4,940 (30.5%) 891 (5.5%) 0 (0.0%) 0.31 (0.63) 10.824 (66.7%) 6,722 (41.4%) 16,207 (99.9%) 1,719 (10.6%) | #DIV/0! 0.02 #DIV/0! #DIV/0! #DIV/0! #DIV/0! #DIV/0! 0.05 -0.14 #DIV/0! 0.03 0.02 0.02 -0.03 0.05 0.03 #DIV/0! 0.06 -0.01 0.03 0.05 0.03 | #VALUE! 18222 (27.2%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) #VALUE! 2844 (4.3%) 8718 (13.0%) 11,518 (50.0%) #VALUE! 197 (0.3%) 16322 (24.4%) 996 (1.5%) 0.47 (0.74) 18510 (27.7%) #VALUE! 0.39 (0.95) 40870 (61.1%) 33733 (50.4%) 65477 (97.9%) 5188 (7.8%) | #VALUEI 8869 (27.6%) 507 (5.4%) 0 (0.0%) 10 (0.0%) #VALUEI 1140 (3.6%) 5608 (17.5%) 4,633 (49.3%) 254 (0.8%) #VALUEI 17502 (23.4%) 434 (1.4%) 0.49 (0.82) 8245 (25.7%) 1397 (4.4%) 0 (0.0%) 0.31 (0.69) 20949 (65.3%) 16600 (51.8%) 31393 (97.9%) 2557 (8.0%) | #VALUE! -0.01 0.03 #DIV/0! #DIV/0! #DIV/0! #VALUE! 0.04 -0.13 0.01 -0.01 #VALUE! #VALUE! 0.02 0.01 0.00 0.05 0.02 #VALUE! 0.00 -0.09 -0.03 0.00 -0.01 |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease: n (%) Major Surgery; n (%) Upper Gl bleed; n (%) Lower/ unspecified Gl bleed; n (%) Urogenital bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of INR (prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Cardiologist; n (%) Treating prescriber - Primary Care Physician; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHA2DS2 VASc score, 180 days, V | ** (0.0%) 2,932 (26.8%) 739 (6.8%) 0 (0.0%) 0 (0.0%) 504 (4.6%) 1,356 (12.4%) 5,272 (48.2%) 63 (0.6%) ** (0.1%) 22 (0.2%) 2,367 (21.6%) 128 (1.2%) 0.46 (0.71) 2,563 (23.4%) 385 (3.5%) ** (0.0%) 0.45 (1.24) 6,854 (62.7%) 9,965 (91.1%) 10,881 (95.5%) 747 (6.8%) 3.62 (1.72) | ** (0.0%) 1,734 (26.9%) 491 (7.6%) 0 (0.0%) 49 (0.8%) 1,060 (16.4%) 95 (48.0%) 71 (1.1%) ** (0.1%) 13 (0.2%) 1,341 (20.8%) 85 (1.3%) 0.45 (0.88) 1,362 (21.1%) 201 (3.1%) 0 (0.0%) 0.31 (0.75) 4,359 (67.6%) 5,708 (88.5%) 6,428 (99.7%) 400 (6.2%) | #DIV/0! 0.00 #DIV/0! #DIV/0! #DIV/0! #DIV/0! -0.01 0.05 -0.11 #DIV/0! -0.05 0.00 0.00 0.02 -0.01 0.01 0.06 0.02 #DIV/0! 0.14 -0.10 0.09 -0.03 0.02 | ** (0.0%) 4,029 (17.5%) 1,391 (6.0%) 0 (0.0%) 171 (0.7%) 819 (3.6%) 1,964 (8.5%) 11,518 (50.0%) 36 (0.2%) 36 (0.2%) 36 (0.2%) 287 (1.2%) 0.34 (0.71) 5,093 (22.1%) 774 (3.4%) 24 (0.1%) 0.43 (1.02) 12,270 (53.3%) 9,641 (41.8%) 21,748 (94.4%) 1,170 (5.1%) | ** (0.0%) 1,736 (18.5%) 507 (5.4%) 0 (0.0%) 0 (0.0%) 81 (0.9%) 301 (3.2%) 1,011 (10.7%) 4,633 (49.3%) 137 (1.5%) ** (0.1%) 1,099 (21.2%) 101 (1.1%) 0.36 (0.78) 1,997 (21.2%) 010 (1.1%) 0.36 (0.78) 305 (3.2%) 0 (0.0%) 0.31 (0.74) 5,766 (61.3%) 4,170 (44.3%) 8,758 (93.1%) 438 (4.7%) | #DIV/0! -0.03 #DIV/0! #DIV/0! #DIV/0! #DIV/0! -0.02 -0.07 #DIV/0! -0.04 -0.03 -0.04 -0.01 -0.03 -0.03 -0.04 -0.01 -0.03 -0.04 -0.05 -0.05 -0.02 | 15 (0.0%) 11,261 (34.2%) 2,747 (8.4%) 0 (0.0%) 0 (0.0%) 1,521 (4.6%) 5,398 (16.4%) 17,994 (54.7%) 158 (0.5%) 109 (0.3%) 139 (0.4%) 8,671 (26.4%) 581 (1.8%) 0.56 (0.76) 10,854 (33.0%) 2,080 (6.3%) 2,080 (6.3%) 2,1746 (66.1%) 11,27 (42.9%) 3,271 (9.9%) 4.52 (1.74) | **(0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) 0 (0.0%) **(0.0%) 607 (3.7%) 3,537 (21.8%) 46 (0.3%) 33 (0.2%) 57 (0.4%) 4,164 (25.7%) 248 (1.5%) 0.58 (0.82) 4,940 (30.5%) 891 (5.5%) 0 (0.0%) 0.31 (0.63) 10,824 (66.7%) 6,722 (41.4%) 16,207 (99.9%) 1,719 (10.6%) | #DIV/0I 0.02 #DIV/0I #DIV/0I #DIV/0I #DIV/0I #DIV/0I #DIV/0I #DIV/0I 0.05 -0.14 #DIV/0I 0.03 0.02 0.02 0.02 0.02 0.02 0.02 -0.03 #DIV/0I 0.03 0.05 -0.03 #DIV/0I 0.06 -0.01 0.03 0.00 -0.02 | #VALUE! 18222 (27.2%) 1,391 (6.0%) 0 (0.0%) #VALUE! 2844 (4.3%) 8718 (13.0%) 11,518 (50.0%) #VALUE! 197 (0.3%) #O.3%) 16322 (24.4%) 996 (1.5%) 0.47 (0.74) 18510 (27.7%) 3239 (4.8%) 9329 (4.8%) 40870 (61.1%) 3733 (50.4%) 55477 (97.9%) 5188 (7.8%) | #VALUEI 8869 (27.6%) 507 (5.4%) 0 (0.0%) 0 (0.0%) #VALUEI 1140 (3.6%) 5608 (17.5%) 4,633 (49.3%) 254 (0.8%) #VALUEI 7502 (23.4%) 434 (1.4%) 0.49 (0.82) 8245 (25.7%) 1397 (4.4%) 0 (0.0%) 0.31 (0.69) 20949 (65.3%) 16600 (51.8%) 31393 (97.9%) 2557 (8.0%) | #VALUEI -0.01 0.03 #DIV/01 #DIV/01 #DIV/01 #VALUEI 0.04 -0.13 0.01 -0.01 #VALUEI #VALUEI #VALUEI 0.02 0.01 0.05 0.02 #VALUEI 0.00 -0.09 -0.03 0.00 -0.01 |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gl bleed; n (%) Lower/unspecified Gl bleed; n (%) Urogenital bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) Vitamin K therapy; n (%) Vitamin K therapy; n (%) Treating prescriber - Cardiologist; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHA2DS2 VASc soore, 180 days, Vmean (sd) Use of Prasugrel; n (%) Use of Prasugrel; n (%) Use of Loop Diuretics+other diuretics+other | ** (0.0%) 2,932 (26.8%) 739 (6.8%) 0 (0.0%) 0 (0.0%) 3 (0.0%) 504 (4.6%) 1,356 (12.4%) 5,272 (48.2%) 63 (0.6%) ** (0.1%) 22 (0.2%) 2,367 (21.6%) 128 (1.2%) 0.46 (0.71) 2,563 (23.4%) 385 (3.5%) ** (0.0%) 0.45 (1.24) 6,854 (62.7%) 9,965 (91.1%) 10,881 (99.5%) 747 (6.8%) 3.62 (1.72) ** (0.1%) | ** (0.0%) 1,734 (26.9%) 491 (7.6%) 0 (0.0%) 49 (0.8%) 232 (3.6%) 1,060 (16.4%) 95 (48.0%) 71 (1.1%) 13 (0.2%) 1,341 (20.8%) 85 (13.3%) 0.45 (0.88) 1,362 (21.1%) 201 (3.1%) 0 (0.0%) 0.31 (0.75) 4,359 (67.6%) 5,708 (88.5%) 6,428 (99.7%) 400 (6.2%) 2.28 (1.64) ** (0.2%) | #DIV/0! 0.00 #DIV/0! #DIV/0! #DIV/0! #DIV/0! -0.01 0.05 -0.11 #DIV/0! -0.05 0.00 0.00 0.02 -0.01 0.01 0.06 0.02 #DIV/0! 0.14 -0.10 0.09 -0.03 0.02 | ** (0.0%) 4,029 (17.5%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) 171 (0.7%) 819 (3.6%) 1,964 (8.5%) 11,518 (50.0%) 254 (1.1%) 36 (0.2%) 36 (0.2%) 5,284 (22.9%) 287 (1.2%) 0.34 (0.71) 5,093 (22.1%) 774 (3.4%) 24 (0.1%) 0.43 (1.02) 12,270 (53.3%) 9,641 (41.8%) 21,748 (94.4%) 1,170 (5.1%) 3.42 (1.47) 30 (0.1%) | ** (0.0%) 1,736 (18.5%) 507 (5.4%) 0 (0.0%) 0 (0.0%) 81 (0.9%) 301 (3.2%) 1,011 (10.7%) 4,633 (49.3%) 137 (1.5%) ** (0.1%) ** (0.1%) 1,097 (21.2%) 0.36 (0.78) 1,943 (20.7%) 0 (0.0%) 0.31 (0.74) 5,766 (61.3%) 4,770 (44.3%) 4,780 (4.3%) 4,780 (4.3%) 4,780 (4.3%) 4,770 (4.3%) 4,770 (4.3%) 4,780 (4.3%) 4,780 (4.3%) 4,780 (4.5%) | #DIV/0! -0.03 #DIV/0! #DIV/0! #DIV/0! #DIV/0! -0.02 -0.07 #DIV/0! -0.04 -0.03 -0.04 -0.01 -0.03 -0.03 -0.04 -0.01 -0.03 -0.04 -0.05 -0.05 -0.02 | 15 (0.0%) 11,261 (34.2%) 2,747 (8.4%) 0 (0.0%) 0 (0.0%) 1,521 (4.6%) 5,398 (16.4%) 17,994 (54.7%) 139 (0.4%) 8,671 (26.4%) 581 (1.8%) 0.56 (0.76) 10,854 (33.0%) 2,080 (6.3%) **(0.0%) 14,127 (42.9%) 32,848 (99.9%) 3,271 (9.9%) 4.52 (1.74) **(0.0%) | **(0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) 0 (0.0%) **(0.0%) 607 (3.7%) 3,537 (21.8%) 8,891 (54.8%) 46 (0.3%) 33 (0.2%) 57 (0.4%) 4,164 (25.7%) 248 (1.5%) 0.58 (0.82) 4,940 (30.5%) 891 (5.5%) 0 (0.0%) 0.31 (0.63) 10,824 (66.7%) 6,722 (41.4%) 16,207 (99.9%) 1,719 (10.6%) 3.51 (1.84) **(0.0%) | #DIV/0I 0.02 #DIV/0I #DIV/0I #DIV/0I #DIV/0I #DIV/0I #DIV/0I #DIV/0I 0.05 -0.14 #DIV/0I 0.03 0.02 0.02 0.02 0.02 0.02 0.02 -0.03 #DIV/0I 0.03 0.05 -0.03 #DIV/0I 0.06 -0.01 0.03 0.00 -0.02 | #VALUE! 18222 (27.2%) 1,391 (6.0%) 0 (0.0%) **VALUE! 2844 (4.3%) 8718 (13.0%) 11,518 (50.0%) #VALUE! 197 (0.3%) 16322 (24.4%) 996 (1.5%) 0.47 (0.74) 18510 (27.7%) #VALUE! 0.39 (0.95) 40870 (61.1%) 32733 (50.4%) 65477 (97.9%) 5188 (7.8%) 3.99 (1.65) #VALUE! | #VALUEI 8869 (27.6%) 507 (5.4%) 0 (0.0%) 0 (0.0%) 4/VALUEI 1140 (3.6%) 5608 (17.5%) 4,633 (49.3%) 254 (0.8%) #VALUEI 17502 (23.4%) 434 (1.4%) 0.49 (0.82) 8245 (25.7%) 1397 (4.4%) 0 (0.0%) 0.31 (0.69) 20949 (65.3%) 16600 (51.8%) 31933 (97.9%) 2557 (8.0%) | #VALUEI -0.01 0.03 #DIV/01 #DIV/01 #DIV/01 #VALUEI 0.04 -0.13 0.01 -0.01 #VALUEI #VALUEI #VALUEI 0.02 0.01 0.05 0.02 #VALUEI 0.00 -0.09 -0.03 0.00 -0.01 |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 Inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Lower (unspecified Gi bleed; n (%) Urogenital bleed; n (%) Urogenital bleed; n (%) Prior cance; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of INR (prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) Lapper Surger; n (%) Lapper Surger; n (%) Use of Prasugrel; n (%) Use of Loop Diuretics-other diuretics+other hypertension drugs; n (%) | ** (0.0%) 2,932 (26.8%) 739 (6.8%) 0 (0.0%) 0 (0.0%) 504 (4.6%) 1,356 (12.4%) 5,272 (48.2%) 63 (0.6%) ** (0.1%) 22 (0.2%) 2,367 (21.6%) 128 (1.2%) 0.46 (0.71) 2,563 (23.4%) 385 (3.5%) ** (0.0%) 0.45 (1.24) 6,854 (62.7%) 9,965 (91.1%) 10,881 (95.5%) 747 (6.8%) 3.62 (1.72) | ** (0.0%) 1,734 (26.9%) 491 (7.6%) 0 (0.0%) 49 (0.8%) 1,060 (16.4%) 95 (48.0%) 71 (1.1%) ** (0.1%) 13 (0.2%) 1,341 (20.8%) 85 (1.3%) 0.45 (0.88) 1,362 (21.1%) 201 (3.1%) 0 (0.0%) 0.31 (0.75) 4,359 (67.6%) 5,708 (88.5%) 6,428 (99.7%) 400 (6.2%) | #DIV/0! 0.00 #DIV/0! #DIV/0! #DIV/0! #DIV/0! -0.01 0.05 -0.11 #DIV/0! -0.05 0.00 0.02 -0.01 0.01 0.06 0.02 #DIV/0! 0.14 -0.10 0.09 -0.03 0.02 | ** (0.0%) 4,029 (17.5%) 1,391 (6.0%) 0 (0.0%) 171 (0.7%) 819 (3.6%) 1,964 (8.5%) 11,518 (50.0%) 36 (0.2%) 36 (0.2%) 36 (0.2%) 287 (1.2%) 0.34 (0.71) 5,093 (22.1%) 774 (3.4%) 24 (0.1%) 0.43 (1.02) 12,270 (53.3%) 9,641 (41.8%) 21,748 (94.4%) 1,170 (5.1%) | ** (0.0%) 1,736 (18.5%) 507 (5.4%) 0 (0.0%) 0 (0.0%) 81 (0.9%) 301 (3.2%) 1,011 (10.7%) 4,633 (49.3%) 137 (1.5%) ** (0.1%) 1,099 (21.2%) 101 (1.1%) 0.36 (0.78) 1,997 (21.2%) 010 (1.1%) 0.36 (0.78) 305 (3.2%) 0 (0.0%) 0.31 (0.74) 5,766 (61.3%) 4,170 (44.3%) 8,758 (93.1%) 438 (4.7%) | #DIV/0! -0.03 #DIV/0! #DIV/0! #DIV/0! #DIV/0! -0.02 -0.07 #DIV/0! -0.04 -0.03 -0.04 -0.01 -0.03 -0.04 -0.01 -0.03 -0.05 -0.05 -0.05 -0.02 | 15 (0.0%) 11,261 (34.2%) 2,747 (8.4%) 0 (0.0%) 0 (0.0%) 1,521 (4.6%) 5,398 (16.4%) 17,994 (54.7%) 158 (0.5%) 109 (0.3%) 139 (0.4%) 8,671 (26.4%) 581 (1.8%) 0.56 (0.76) 10,854 (33.0%) 2,080 (6.3%) 2,080 (6.3%) 2,1746 (66.1%) 11,27 (42.9%) 3,271 (9.9%) 4.52 (1.74) | **(0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) 0 (0.0%) **(0.0%) 607 (3.7%) 3,537 (21.8%) 46 (0.3%) 33 (0.2%) 57 (0.4%) 4,164 (25.7%) 248 (1.5%) 0.58 (0.82) 4,940 (30.5%) 891 (5.5%) 0 (0.0%) 0.31 (0.63) 10,824 (66.7%) 6,722 (41.4%) 16,207 (99.9%) 1,719 (10.6%) | #DIV/0! 0.02 #DIV/0! #DIV/0! #DIV/0! #DIV/0! #DIV/0! #DIV/0! 0.05 -0.14 #DIV/0! 0.03 0.02 0.02 0.02 -0.03 #DIV/0! 0.06 -0.01 0.03 0.05 0.03 #DIV/0! | #VALUE! 18222 (27.2%) 1,391 (6.0%) 0 (0.0%) #VALUE! 2844 (4.3%) 8718 (13.0%) 11,518 (50.0%) #VALUE! 197 (0.3%) #O.3%) 16322 (24.4%) 996 (1.5%) 0.47 (0.74) 18510 (27.7%) 3239 (4.8%) 9329 (4.8%) 40870 (61.1%) 3733 (50.4%) 55477 (97.9%) 5188 (7.8%) | #VALUEI 8869 (27.6%) 507 (5.4%) 0 (0.0%) 0 (0.0%) #VALUEI 1140 (3.6%) 5608 (17.5%) 4,633 (49.3%) 254 (0.8%) #VALUEI 7502 (23.4%) 434 (1.4%) 0.49 (0.82) 8245 (25.7%) 1397 (4.4%) 0 (0.0%) 0.31 (0.69) 20949 (65.3%) 16600 (51.8%) 31393 (97.9%) 2557 (8.0%) | #VALUE! -0.01 0.03 #DIV/0! #DIV/0! #DIV/0! #VALUE! 0.04 -0.13 0.01 -0.01 #VALUE! #VALUE! 0.02 0.01 0.05 0.02 #VALUE! 0.00 -0.09 -0.03 0.00 -0.01 0.01 #VALUE! |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease: n (%) Major Surgery; n (%) Upper Gl bleed; n (%) Lower ( unspecified Gl bleed; n (%) Urogenital bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other astroprotective agents; n (%) PGP inhibitors; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of INR (prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Other; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHA2DS2 VASc score, 180 days, Vmean (sd) Use of Prasugrel; n (%) Commercial vs Medicare Advantage-Business Type | ** (0.0%) 2,932 (26.8%) 739 (6.8%) 0 (0.0%) 0 (0.0%) 3 (0.0%) 504 (4.6%) 1,356 (12.4%) 5,272 (48.2%) 63 (0.6%) ** (0.1%) 22 (0.2%) 2,367 (21.6%) 128 (1.2%) 0.46 (0.71) 2,563 (23.4%) 385 (3.5%) ** (0.0%) 0.45 (1.24) 6,854 (62.7%) 9,965 (91.1%) 10,881 (99.5%) 747 (6.8%) 3.62 (1.72) ** (0.1%) | ** (0.0%) 1,734 (26.9%) 491 (7.6%) 0 (0.0%) 49 (0.8%) 232 (3.6%) 1,060 (16.4%) 95 (48.0%) 71 (1.1%) 13 (0.2%) 1,341 (20.8%) 85 (13.3%) 0.45 (0.88) 1,362 (21.1%) 201 (3.1%) 0 (0.0%) 0.31 (0.75) 4,359 (67.6%) 5,708 (88.5%) 6,428 (99.7%) 400 (6.2%) 2.28 (1.64) ** (0.2%) | #DIV/0! 0.00 #DIV/0! #DIV/0! #DIV/0! #DIV/0! -0.01 0.05 -0.11 #DIV/0! -0.05 0.00 0.02 -0.01 0.01 0.06 0.02 #DIV/0! 0.14 -0.10 0.09 -0.03 0.02 | ** (0.0%) 4,029 (17.5%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) 171 (0.7%) 819 (3.6%) 1,964 (8.5%) 11,518 (50.0%) 254 (1.1%) 36 (0.2%) 36 (0.2%) 5,284 (22.9%) 287 (1.2%) 0.34 (0.71) 5,093 (22.1%) 774 (3.4%) 24 (0.1%) 0.43 (1.02) 12,270 (53.3%) 9,641 (41.8%) 21,748 (94.4%) 1,170 (5.1%) 3.42 (1.47) 30 (0.1%) | ** (0.0%) 1,736 (18.5%) 507 (5.4%) 0 (0.0%) 0 (0.0%) 81 (0.9%) 301 (3.2%) 1,011 (10.7%) 4,633 (49.3%) 137 (1.5%) ** (0.1%) ** (0.1%) 1,097 (21.2%) 0.36 (0.78) 1,943 (20.7%) 0 (0.0%) 0.31 (0.74) 5,766 (61.3%) 4,770 (44.3%) 4,780 (4.3%) 4,780 (4.3%) 4,780 (4.3%) 4,770 (4.3%) 4,770 (4.3%) 4,780 (4.3%) 4,780 (4.3%) 4,780 (4.5%) | #DIV/0! -0.03 #DIV/0! #DIV/0! #DIV/0! #DIV/0! -0.02 -0.07 #DIV/0! -0.04 -0.03 -0.04 -0.01 -0.03 -0.04 -0.01 -0.03 -0.05 -0.05 -0.05 -0.02 | 15 (0.0%) 11,261 (34.2%) 2,747 (8.4%) 0 (0.0%) 0 (0.0%) 1,521 (4.6%) 5,398 (16.4%) 17,994 (54.7%) 139 (0.4%) 8,671 (26.4%) 581 (1.8%) 0.56 (0.76) 10,854 (33.0%) 2,080 (6.3%) **(0.0%) 14,127 (42.9%) 32,848 (99.9%) 3,271 (9.9%) 4.52 (1.74) **(0.0%) | **(0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) 0 (0.0%) **(0.0%) 607 (3.7%) 3,537 (21.8%) 8,891 (54.8%) 46 (0.3%) 33 (0.2%) 57 (0.4%) 4,164 (25.7%) 248 (1.5%) 0.58 (0.82) 4,940 (30.5%) 891 (5.5%) 0 (0.0%) 0.31 (0.63) 10,824 (66.7%) 6,722 (41.4%) 16,207 (99.9%) 1,719 (10.6%) 3.51 (1.84) **(0.0%) | #DIV/0! 0.02 #DIV/0! #DIV/0! #DIV/0! #DIV/0! #DIV/0! #DIV/0! 0.05 -0.14 #DIV/0! 0.03 0.02 0.02 0.02 -0.03 #DIV/0! 0.06 -0.01 0.03 0.05 0.03 #DIV/0! | #VALUE! 18222 (27.2%) 1,391 (6.0%) 0 (0.0%) **VALUE! 2844 (4.3%) 8718 (13.0%) 11,518 (50.0%) #VALUE! 197 (0.3%) 16322 (24.4%) 996 (1.5%) 0.47 (0.74) 18510 (27.7%) #VALUE! 0.39 (0.95) 40870 (61.1%) 32733 (50.4%) 65477 (97.9%) 5188 (7.8%) 3.99 (1.65) #VALUE! | #VALUEI 8869 (27.6%) 507 (5.4%) 0 (0.0%) 0 (0.0%) 4/VALUEI 1140 (3.6%) 5608 (17.5%) 4,633 (49.3%) 254 (0.8%) #VALUEI 17502 (23.4%) 434 (1.4%) 0.49 (0.82) 8245 (25.7%) 1397 (4.4%) 0 (0.0%) 0.31 (0.69) 20949 (65.3%) 16600 (51.8%) 31933 (97.9%) 2557 (8.0%) | #VALUE! -0.01 0.03 #DIV/0! #DIV/0! #DIV/0! #VALUE! 0.04 -0.13 0.01 -0.01 #VALUE! #VALUE! 0.02 0.01 0.05 0.02 #VALUE! 0.00 -0.09 -0.03 0.00 -0.01 0.01 #VALUE! |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Upper Gi bleed; n (%) Upper Gi bleed; n (%) Urogenital bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) Vitamin K therapy; n (%) Number of iNR (prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Cardiologist; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) Ch42DS2 VASc score, 180 days, Vmean (sd) Useo f Prasugrel; n (%) Useo f Loop Diuretic-swher diuretics+other hypertension drugs; n (%) Commercial vs Medicare Advantage-Business Type Code - CORRECT ONE - OPTUM | **(0.0%) 2,932 (26.8%) 739 (6.8%) 0 (0.0%) 0 (0.0%) 5,078 (1.6%) 1,356 (12.4%) 5,272 (48.2%) 63 (0.6%) 128 (1.2%) 2,367 (21.6%) 128 (1.2%) 0.46 (0.71) 2,563 (23.4%) 385 (3.5%) **(0.0%) 0.45 (1.24) 6,854 (62.7%) 9,965 (91.1%) 10,881 (99.5%) 747 (6.8%) 3.62 (1.72) **(0.1%) | ** (0.0%) 1,734 (26.9%) 491 (7.6%) 0 (0.0%) 0 (0.0%) 49 (0.8%) 232 (3.6%) 1,060 (16.4%) 95 (48.0%) 71 (1.1%) 13 (0.2%) 1,341 (20.8%) 85 (1.3%) 0.45 (0.88) 1,362 (21.1%) 201 (3.1%) 201 (3.1%) 0 (0.0%) 0.31 (0.75) 4,359 (67.6%) 5,708 (88.5%) 6,428 (99.7%) 400 (6.2%) 2.28 (1.64) ** (0.2%) 633 (9.8%) | #DIV/0! 0.00 #DIV/0! #DIV/0! #DIV/0! #DIV/0! -0.01 0.05 -0.11 #DIV/0! -0.05 0.00 0.02 -0.01 0.01 0.06 0.02 #DIV/0! 0.14 -0.10 0.09 -0.03 0.02 | ** (0.0%) 4,029 (17.5%) 1,391 (6.0%) 0 (0.0%) 171 (0.7%) 819 (3.6%) 1,964 (8.5%) 11,518 (50.0%) 36 (0.2%) 36 (0.2%) 36 (0.2%) 287 (1.2%) 0.34 (0.71) 5,093 (22.1%) 774 (3.4%) 24 (0.1%) 0.43 (1.02) 12,270 (53.3%) 9,641 (41.8%) 1,170 (5.1%) 3.42 (1.47) 30 (0.1%) | ** (0.0%) 1,736 (18.5%) 507 (5.4%) 0 (0.0%) 0 (0.0%) 81 (0.9%) 301 (3.2%) 1,011 (10.7%) 4,633 (49.3%) 137 (1.5%) ** (0.1%) 1,019 (10.1%) 1,019 (10.1%) 0.36 (0.78) 1,943 (20.7%) 305 (3.2%) 0 (0.0%) 0.31 (0.74) 5,766 (61.3%) 4,170 (44.3%) 8,758 (93.1%) 438 (4.7%) 2.40 (1.69) ** (0.1%) | #DIV/0! -0.03 #DIV/0! #DIV/0! #DIV/0! #DIV/0! -0.02 -0.07 #DIV/0! -0.04 -0.03 -0.04 -0.01 -0.03 -0.04 -0.01 -0.03 -0.05 -0.05 -0.05 -0.02 -0.06 | 15 (0.0%) 11,261 (34.2%) 2,747 (8.4%) 0 (0.0%) 0 (0.0%) 1,521 (4.6%) 5,398 (16.4%) 17,994 (54.7%) 139 (0.4%) 8,671 (26.4%) 581 (1.8%) 0.56 (0.76) 10,854 (33.0%) 2,080 (6.3%) **(0.0%) 14,127 (42.9%) 32,848 (99.9%) 3,271 (9.9%) 4.52 (1.74) **(0.0%) | **(0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) 0 (0.0%) **(0.0%) 607 (3.7%) 3,537 (21.8%) 8,891 (54.8%) 46 (0.3%) 33 (0.2%) 57 (0.4%) 4,164 (25.7%) 248 (1.5%) 0.58 (0.82) 4,940 (30.5%) 891 (5.5%) 0 (0.0%) 0.31 (0.63) 10,824 (66.7%) 6,722 (41.4%) 16,207 (99.9%) 1,719 (10.6%) 3.51 (1.84) **(0.0%) | #DIV/0! 0.02 #DIV/0! #DIV/0! #DIV/0! #DIV/0! #DIV/0! #DIV/0! 0.05 -0.14 #DIV/0! 0.03 0.02 0.02 0.02 -0.03 #DIV/0! 0.06 -0.01 0.03 0.05 0.03 #DIV/0! | #VALUE! 18222 (27.2%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) #VALUE! 2844 (4.3%) 8718 (13.0%) 11,518 (50.0%) 475 (0.7%) #VALUE! 197 (0.3%) 16322 (24.4%) 996 (1.5%) 0.47 (0.74) 18510 (27.7%) 3239 (4.8%) #VALUE! 0.39 (0.95) 40870 (61.1%) 33733 (50.4%) 65477 (97.9%) 5188 (7.8%) 3.99 (1.65) #VALUE! | #VALUEI 8869 (27.6%) 507 (5.4%) 0 (0.0%) 0 (0.0%) 4 (0.0%) 6 (0.0% | #VALUE! -0.01 0.03 #DIV/0! #DIV/0! #DIV/0! #VALUE! 0.04 -0.13 0.01 -0.01 #VALUE! #VALUE! 0.02 0.01 0.05 0.02 #VALUE! 0.00 -0.09 -0.03 0.00 -0.01 #VALUE! |
| 183 days; n (%) Intracranial or retroperitoneal hemorrhage: 1 inpatient or 2 outpatient claims within 183 days; n (%) Peptic Ulcer Disease: n (%) Major Surgery; n (%) Upper Gl bleed; n (%) Lower ( unspecified Gl bleed; n (%) Urogenital bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other astroprotective agents; n (%) PGP inhibitors; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of INR (prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Other; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHA2DS2 VASc score, 180 days, Vmean (sd) Use of Prasugrel; n (%) Commercial vs Medicare Advantage-Business Type | ** (0.0%) 2,932 (26.8%) 739 (6.8%) 0 (0.0%) 0 (0.0%) 3 (0.0%) 504 (4.6%) 1,356 (12.4%) 5,272 (48.2%) 63 (0.6%) ** (0.1%) 22 (0.2%) 2,367 (21.6%) 128 (1.2%) 0.46 (0.71) 2,563 (23.4%) 385 (3.5%) ** (0.0%) 0.45 (1.24) 6,854 (62.7%) 9,965 (91.1%) 10,881 (99.5%) 747 (6.8%) 3.62 (1.72) ** (0.1%) | ** (0.0%) 1,734 (26.9%) 491 (7.6%) 0 (0.0%) 49 (0.8%) 232 (3.6%) 1,060 (16.4%) 95 (48.0%) 71 (1.1%) 13 (0.2%) 1,341 (20.8%) 85 (13.3%) 0.45 (0.88) 1,362 (21.1%) 201 (3.1%) 0 (0.0%) 0.31 (0.75) 4,359 (67.6%) 5,708 (88.5%) 6,428 (99.7%) 400 (6.2%) 2.28 (1.64) ** (0.2%) | #DIV/0! 0.00 #DIV/0! #DIV/0! #DIV/0! #DIV/0! -0.01 0.05 -0.11 #DIV/0! -0.05 0.00 0.02 -0.01 0.01 0.06 0.02 #DIV/0! 0.14 -0.10 0.09 -0.03 0.02 0.02 0.03 0.09 | ** (0.0%) 4,029 (17.5%) 1,391 (6.0%) 0 (0.0%) 0 (0.0%) 171 (0.7%) 819 (3.6%) 1,964 (8.5%) 11,518 (50.0%) 254 (1.1%) 36 (0.2%) 36 (0.2%) 5,284 (22.9%) 287 (1.2%) 0.34 (0.71) 5,093 (22.1%) 774 (3.4%) 24 (0.1%) 0.43 (1.02) 12,270 (53.3%) 9,641 (41.8%) 21,748 (94.4%) 1,170 (5.1%) 3.42 (1.47) 30 (0.1%) | ** (0.0%) 1,736 (18.5%) 507 (5.4%) 0 (0.0%) 0 (0.0%) 81 (0.9%) 301 (3.2%) 1,011 (10.7%) 4,633 (49.3%) 137 (1.5%) ** (0.1%) ** (0.1%) 1,097 (21.2%) 0.36 (0.78) 1,943 (20.7%) 0 (0.0%) 0.31 (0.74) 5,766 (61.3%) 4,770 (44.3%) 4,780 (4.3%) 4,780 (4.3%) 4,780 (4.3%) 4,770 (4.3%) 4,770 (4.3%) 4,780 (4.3%) 4,780 (4.3%) 4,780 (4.5%) | #DIV/0! -0.03 #DIV/0! #DIV/0! #DIV/0! #DIV/0! -0.02 -0.07 #DIV/0! -0.04 -0.03 -0.04 -0.01 -0.03 -0.04 -0.01 -0.03 -0.05 -0.05 -0.05 -0.02 | 15 (0.0%) 11,261 (34.2%) 2,747 (8.4%) 0 (0.0%) 0 (0.0%) 1,521 (4.6%) 5,398 (16.4%) 17,994 (54.7%) 139 (0.4%) 8,671 (26.4%) 581 (1.8%) 0.56 (0.76) 10,854 (33.0%) 2,080 (6.3%) **(0.0%) 14,127 (42.9%) 32,848 (99.9%) 3,271 (9.9%) 4.52 (1.74) **(0.0%) | **(0.0%) 5,399 (33.3%) 1,625 (10.0%) 0 (0.0%) 0 (0.0%) **(0.0%) 607 (3.7%) 3,537 (21.8%) 8,891 (54.8%) 46 (0.3%) 33 (0.2%) 57 (0.4%) 4,164 (25.7%) 248 (1.5%) 0.58 (0.82) 4,940 (30.5%) 891 (5.5%) 0 (0.0%) 0.31 (0.63) 10,824 (66.7%) 6,722 (41.4%) 16,207 (99.9%) 1,719 (10.6%) 3.51 (1.84) **(0.0%) | #DIV/0! 0.02 #DIV/0! #DIV/0! #DIV/0! #DIV/0! #DIV/0! 0.05 -0.14 #DIV/0! 0.03 0.02 0.02 0.02 0.02 0.02 -0.03 #DIV/0! 0.05 -0.01 0.05 -0.05 0.03 #DIV/0! 0.06 -0.01 0.03 0.00 -0.02 0.02 | #VALUE! 18222 (27.2%) 1,391 (6.0%) 0 (0.0%) **VALUE! 2844 (4.3%) 8718 (13.0%) 11,518 (50.0%) #VALUE! 197 (0.3%) 16322 (24.4%) 996 (1.5%) 0.47 (0.74) 18510 (27.7%) #VALUE! 0.39 (0.95) 40870 (61.1%) 32733 (50.4%) 65477 (97.9%) 5188 (7.8%) 3.99 (1.65) #VALUE! | #VALUEI 8869 (27.6%) 507 (5.4%) 0 (0.0%) 0 (0.0%) 4/VALUEI 1140 (3.6%) 5608 (17.5%) 4,633 (49.3%) 254 (0.8%) #VALUEI 17502 (23.4%) 434 (1.4%) 0.49 (0.82) 8245 (25.7%) 1397 (4.4%) 0 (0.0%) 0.31 (0.69) 20949 (65.3%) 16600 (51.8%) 31933 (97.9%) 2557 (8.0%) | #VALUE! -0.01 0.03 #DIV/0! #DIV/0! #DIV/0! #VALUE! 0.04 -0.13 0.01 -0.01 #VALUE! #VALUE! 0.02 0.01 0.05 0.02 #VALUE! 0.00 -0.09 -0.03 0.00 -0.01 0.01 #VALUE! |

| Commercial vs Medicare Advantage- Business Type | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Code | | | | | | | | | | | | |
| COM = COMMERCIAL; n (%) | 5,252 (48.0%) | 3,352 (52.0%) | -0.08 | - | - | | - | - | #VALUE! | 5,252 (48.0%) | 3,352 (52.0%) | -0.08 |
| MCR = MEDICARE; n (%) | 5,684 (52.0%) | 3,096 (48.0%) | 0.08 | - | - | | - | - | #VALUE! | 5,684 (52.0%) | 3,096 (48.0%) | 0.08 |
| MCD = MEDICAID; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| NONE = NO BUSINESS LINE CODE (added in 2015); n | | | | | | | | | | | | |
| (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| UNK = UNKNOWN (added in 2015); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Commercial vs Medicare Advantage- Data Type | | | | | | | | | | | | |
| 1 - Fee For Service; n (%) | - | - | | 15,188 (65.9%) | 6,798 (72.3%) | -0.14 | - | - | | 15,188 (65.9%) | 6,798 (72.3%) | -0.14 |
| 2 - Encounter; n (%) | - | - | | 2,210 (9.6%) | 785 (8.3%) | 0.05 | - | - | | 2,210 (9.6%) | 785 (8.3%) | 0.05 |
| 3 - Medicare; n (%) | - | - | | 4,938 (21.4%) | 1,622 (17.2%) | 0.11 | - | - | | 4,938 (21.4%) | 1,622 (17.2%) | 0.11 |
| 4 - Medicare Encounter; n (%) | - | - | | 704 (3.1%) | 200 (2.1%) | 0.06 | - | - | | 704 (3.1%) | 200 (2.1%) | 0.06 |
| Metropolitan Statistical Area - Urban (any MSA) vs | | | | | | | | | | | | |
| Rural (non-MSA) | | | | | | | | | | 0 | 0 | 0.00 |
| Urban; n (%) | - | - | | 18,451 (80.1%) | 6,998 (74.4%) | 0.14 | - | - | | 18,451 (80.1%) | 6,998 (74.4%) | 0.14 |
| Rural; n (%) | - | - | | 290 (1.3%) | 433 (4.6%) | -0.20 | - | - | | 290 (1.3%) | 433 (4.6%) | -0.20 |
| Unknown/Missing; n (%) | - | - | | 4,299 (18.7%) | 1,974 (21.0%) | -0.06 | - | - | | 4,299 (18.7%) | 1,974 (21.0%) | -0.06 |
| Due to CMS cell suppression policy, all values less than 11 | are denoted with ** | | | | | | | | | | | |

| | | | | | PS-matched | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Optur | n | | Markets | ican | | Medica | re | | POOLED | |
| Variable | Reference- warfarin Copy 'or | vahan (15 or 20 mg) Conv | St Diff | Reference-warfarin Copy o | rahan (15 or 20 mg) Conv | St Diff | Reference- warfarin Copy 'ox | ahan (15 or 20 mg) Conv. I | Reference-warfarin Conv | Exposure - rivaroxaban<br>(15 or 20 mg) Copy | St. Diff. |
| Number of patients | 2.153 | 2,153 | Jt. Dill. | 5,675 | 5.675 | St. Dill. | 8.065 | 8.065 | 15,893 | 15,893 | Jt. Dill. |
| Age | -, | -, | | -, | -, | | 2,222 | -, | , | , | |
| mean (sd) | 62.79 (15.74) | 63.58 (14.79) | -0.05 | 54.36 (14.93) | 54.95 (14.55) | -0.04 | 75.04 (7.11) | 75.35 (7.03) | 66.00 (11.78) | 66.47 (11.41) | -0.04 |
| median [IQR] | 65.00 [53.00, 75.00] | 66.00 [54.00, 74.00] | -0.07 | 55.00 [45.00, 63.00] | 56.00 [45.00, 64.00] | -0.07 | 74.00 [69.00, 80.00] | 74.00 [70.00, 80.00] | 66.00 (11.78) | 66.49 (11.41) | -0.04 |
| Age categories without zero category | | | | | | | | | , | , | |
| 18 - 54; n (%) | 601 (27.9%) | 564 (26.2%) | 0.04 | 2,732 (48.1%) | 2,665 (47.0%) | 0.02 | 0 (0.0%) | 0 (0.0%) | 3333 (21.0%) | 3229 (20.3%) | 0.02 |
| 55 -64; n (%) | 445 (20.7%) | 406 (18.9%) | 0.05 | 1,749 (30.8%) | 1,755 (30.9%) | 0.00 | 0 (0.0%) | 0 (0.0%) | 2,194 (13.8%) | 2,161 (13.6%) | 0.01 |
| 65 - 74; n (%) | 558 (25.9%) | 649 (30.1%) | -0.09 | 666 (11.7%) | 709 (12.5%) | -0.02 | 4,295 (53.3%) | 4,133 (51.2%) | 5,519 (34.7%) | 5,491 (34.5%) | 0.00 |
| >= 75; n (%) | 549 (25.5%) | 534 (24.8%) | 0.02 | 528 (9.3%) | 546 (9.6%) | -0.01 | 3,770 (46.7%) | 3,932 (48.8%) | 4,847 (30.5%) | 5,012 (31.5%) | -0.02 |
| Gender without zero category- United | | | | | | | | | | | |
| Males; n (%) | 938 (43.6%) | 900 (41.8%) | 0.04 | 2,751 (48.5%) | 2,745 (48.4%) | 0.00 | 3,089 (38.3%) | 2,987 (37.0%) | 6,778 (42.6%) | 6,632 (41.7%) | 0.02 |
| Females; n (%) | 1,215 (56.4%) | 1,253 (58.2%) | -0.04 | 2,924 (51.5%) | 2,930 (51.6%) | 0.00 | 4,976 (61.7%) | 5,078 (63.0%) | 9,115 (57.4%) | 9,261 (58.3%) | -0.02 |
| Race | | | | | | | | | | | |
| White; n (%) | | | | | | | 7,031 (87.2%) | 7,010 (86.9%) | 7,031 (87.2%) | 7,010 (86.9%) | 0.01 |
| Black; n (%) | | | | | | | 726 (9.0%) | 767 (9.5%) | 726 (9.0%) | 767 (9.5%) | -0.02<br>0.00 |
| Asian; n (%) | | | | | | | 58 (0.7%) | 53 (0.7%) | 58 (0.7%) | 53 (0.7%) | -0.01 |
| Hispanic; n (%)<br>North American Native; n (%) | | | | | | | 95 (1.2%)<br>29 (0.4%) | 101 (1.3%)<br>24 (0.3%) | 95 (1.2%)<br>29 (0.4%) | 101 (1.3%)<br>24 (0.3%) | 0.01 |
| Other/Unknown; n (%) | | | | | | | 126 (1.6%) | 110 (1.4%) | 126 (1.6%) | 110 (1.4%) | 0.02 |
| Gener/Onknown, ii (/o) | | | | | | | 120 (1.0%) | 110 (1.4%) | 120 (1.0%) | 110 (1.4%) | 0.02 |
| Region without zero category | | | | | | | | | | | |
| Northeast; n (%) | 226 (10.5%) | 223 (10.4%) | 0.00 | 1,034 (18.2%) | 1,037 (18.3%) | 0.00 | 1,407 (17.4%) | 1,427 (17.7%) | 2,667 (16.8%) | 2,687 (16.9%) | 0.00 |
| South; n (%) | 885 (41.1%) | 881 (40.9%) | 0.00 | 1,616 (28.5%) | 1,653 (29.1%) | -0.01 | 3,171 (39.3%) | 3,105 (38.5%) | 5,672 (35.7%) | 5,639 (35.5%) | 0.00 |
| Midwest; n (%) | 587 (27.3%) | 582 (27.0%) | 0.01 | 2,148 (37.9%) | 2,057 (36.2%) | 0.04 | 2,171 (26.9%) | 2,267 (28.1%) | 4,906 (30.9%) | 4,906 (30.9%) | 0.00 |
| West; n (%) | 455 (21.1%) | 467 (21.7%) | -0.01 | 794 (14.0%) | 853 (15.0%) | -0.03 | 1,316 (16.3%) | 1,266 (15.7%) | 2,565 (16.1%) | 2,586 (16.3%) | -0.01 |
| Unknown+missing; n (%) | N/A | N/A | #VALUE! | 83 (1.5%) | 75 (1.3%) | 0.02 | N/A | N/A | 83 (1.5%) | 75 (1.3%) | 0.02 |
| CV Covariates | | | | | | | | | | | |
| Ischemic heart disease; n (%) | 416 (19.3%) | 410 (19.0%) | 0.01 | 675 (11.9%) | 696 (12.3%) | -0.01 | 2,065 (25.6%) | 2,108 (26.1%) | 3,156 (19.9%) | 3,214 (20.2%) | -0.01 |
| Acute MI; n (%) | 105 (4.9%) | 99 (4.6%) | 0.01 | 181 (3.2%) | 186 (3.3%) | -0.01 | 360 (4.5%) | 359 (4.5%) | 646 (4.1%) | 644 (4.1%) | 0.00 |
| ACS/unstable angina; n (%) | 37 (1.7%) | 37 (1.7%) | 0.00 | 54 (1.0%) | 51 (0.9%) | 0.01 | 115 (1.4%) | 93 (1.2%) | 206 (1.3%) | 181 (1.1%) | 0.02 |
| Old MI; n (%) | 83 (3.9%) | 71 (3.3%) | 0.03 | 87 (1.5%) | 87 (1.5%) | 0.00 | 384 (4.8%) | 453 (5.6%) | 554 (3.5%) | 611 (3.8%) | -0.02 |
| Stable angina; n (%) | 48 (2.2%) | 48 (2.2%) | 0.00 | 79 (1.4%) | 79 (1.4%) | 0.00 | 206 (2.6%) | 224 (2.8%) | 333 (2.1%) | 351 (2.2%) | -0.01 |
| Coronary atherosclerosis and other forms of chronic ischemic heart disease: n (%) | 289 (13.4%) | 298 (13.8%) | -0.01 | 454 (8.0%) | 461 (8.1%) | 0.00 | 1,692 (21.0%) | 1,759 (21.8%) | 2,435 (15.3%) | 2,518 (15.8%) | -0.01 |
| Other atherosclerosis with ICD10 v2 Copy; n (%) | 18 (0.8%) | 18 (0.8%) | 0.00 | 27 (0.5%) | 23 (0.4%) | 0.01 | 95 (1.2%) | 84 (1.0%) | 140 (0.9%) | 125 (0.8%) | 0.01 |
| Previous cardiac procedure (CABG or PTCA or Stent) | 18 (0.8%) | 10 (0.070) | 0.00 | 27 (0.5%) | 23 (0.470) | 0.01 | 33 (1.270) | 04 (1.070) | 140 (0.570) | 123 (0.070) | 0.01 |
| v4; n (%) | 16 (0.7%) | ** (0.2%) | 0.07 | 22 (0.4%) | 18 (0.3%) | 0.02 | 38 (0.5%) | 47 (0.6%) | 76 (0.5%) | #VALUE! | #VALUE! |
| History of CABG or PTCA; n (%) | 91 (4.2%) | 91 (4.2%) | 0.00 | 77 (1.4%) | 68 (1.2%) | 0.02 | 686 (8.5%) | 719 (8.9%) | 854 (5.4%) | 878 (5.5%) | 0.00 |
| Any stroke; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Ischemic stroke (w and w/o mention of cerebral | | | | | | | | | | | |
| infarction); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Hemorrhagic stroke; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| TIA; n (%) | 25 (1.2%) | 21 (1.0%) | 0.02 | 39 (0.7%) | 42 (0.7%) | 0.00 | 83 (1.0%) | 86 (1.1%) | 147 (0.9%) | 149 (0.9%) | 0.00 |
| Other cerebrovascular disease; n (%) | 33 (1.5%) | 29 (1.3%) | 0.02 | 44 (0.8%) | 39 (0.7%) | 0.01 | 157 (1.9%) | 172 (2.1%) | 234 (1.5%) | 240 (1.5%) | 0.00 |
| Cerebrovascular procedure; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Heart failure (CHF); n (%) | ** (0.0%) | ** (0.1%) | -0.04 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #VALUE! | #VALUE! | #VALUE! |
| $Peripheral\ Vascular\ Disease\ (PVD)\ or\ PVD\ Surgery\ v2;$ | | | | | | | | | | | |
| n (%) | 110 (5.1%) | 117 (5.4%) | -0.01 | 158 (2.8%) | 170 (3.0%) | -0.01 | 562 (7.0%) | 582 (7.2%) | 830 (5.2%) | 869 (5.5%) | -0.01 |
| Atrial fibrillation; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Other cardiac dysrhythmia; n (%) | 340 (15.8%) | 346 (16.1%) | -0.01 | 765 (13.5%) | 774 (13.6%) | 0.00 | 1,354 (16.8%) | 1,380 (17.1%) | 2,459 (15.5%) | 2,500 (15.7%) | -0.01 |
| Cardiac conduction disorders; n (%) Other CVD; n (%) | 160 (7.4%)<br>562 (26.1%) | 143 (6.6%)<br>566 (26.3%) | 0.03 | 253 (4.5%)<br>1,205 (21.2%) | 242 (4.3%)<br>1,196 (21.1%) | 0.01 | 687 (8.5%)<br>1,992 (24.7%) | 625 (7.7%)<br>2,067 (25.6%) | 1100 (6.9%)<br>3,759 (23.7%) | 1010 (6.4%)<br>3,829 (24.1%) | 0.02<br>-0.01 |
| | 302 (20.1%) | 300 (20.3%) | 0.00 | 1,205 (21.2%) | 1,190 (21.1%) | 0.00 | 1,992 (24.7%) | 2,067 (23.6%) | 3,/39 (23.7%) | 3,829 (24.1%) | -0.01 |
| Diabetes-related complications Occurrence of Diabetic Neuropathy v2 Copy; n (%) | 122 (5.7%) | 102 (4.7%) | 0.05 | 129 (2.3%) | 126 (2.2%) | 0.01 | 296 (3.7%) | 329 (4.1%) | 547 (3.4%) | 557 (3.5%) | -0.01 |
| Occurrence of diabetic nephropathy V3 with ICD10 | 122 (3.7%) | 102 (4.7%) | 0.03 | 125 (2.5%) | 120 (2.270) | 0.01 | 250 (3.7%) | 325 (4.176) | 347 (3.470) | 337 (3.370) | -0.01 |
| Copy: n (%) | 64 (3.0%) | 68 (3.2%) | -0.01 | 67 (1.2%) | 59 (1.0%) | 0.02 | 166 (2.1%) | 160 (2.0%) | 297 (1.9%) | 287 (1.8%) | 0.01 |
| Hypoglycemia v2; n (%) | 19 (0.9%) | 20 (0.9%) | 0.00 | 34 (0.6%) | 42 (0.7%) | -0.01 | 159 (2.0%) | 160 (2.0%) | 212 (1.3%) | 222 (1.4%) | -0.01 |
| Hyperglycemia; n (%) | 184 (8.5%) | 165 (7.7%) | 0.03 | 254 (4.5%) | 279 (4.9%) | -0.02 | 684 (8.5%) | 723 (9.0%) | 1122 (7.1%) | 1167 (7.3%) | -0.01 |
| Diabetic ketoacidosis; n (%) | ** (0.2%) | ** (0.4%) | -0.04 | 13 (0.2%) | 18 (0.3%) | -0.02 | 17 (0.2%) | 12 (0.1%) | #VALUE! | #VALUE! | #VALUE! |
| Hypertension: 1 inpatient or 2 outpatient claims | ( | , | | - (- /-/ | / | | · | · · · · · · · | | | |
| within 365 days; n (%) | 1,369 (63.6%) | 1,422 (66.0%) | -0.05 | 2,732 (48.1%) | 2,786 (49.1%) | -0.02 | 6,580 (81.6%) | 6,669 (82.7%) | 10,681 (67.2%) | 10,877 (68.4%) | -0.03 |
| Hyperlipidemia v2; n (%) | 1,052 (48.9%) | 1,086 (50.4%) | -0.03 | 1,897 (33.4%) | 1,933 (34.1%) | -0.01 | 4,942 (61.3%) | 5,001 (62.0%) | 7,891 (49.7%) | 8,020 (50.5%) | -0.02 |
| Edema; n (%) | 388 (18.0%) | 395 (18.3%) | -0.01 | 733 (12.9%) | 731 (12.9%) | 0.00 | 1,048 (13.0%) | 1,096 (13.6%) | 2169 (13.6%) | 2222 (14.0%) | -0.01 |
| Renal Dysfunction (non-diabetic) v2; n (%) | 501 (23.3%) | 506 (23.5%) | 0.00 | 698 (12.3%) | 725 (12.8%) | -0.02 | 1,871 (23.2%) | 2,002 (24.8%) | 3070 (19.3%) | 3233 (20.3%) | -0.03 |
| Occurrence of acute renal disease v2; n (%) | 229 (10.6%) | 224 (10.4%) | 0.01 | 340 (6.0%) | 354 (6.2%) | -0.01 | 799 (9.9%) | 858 (10.6%) | 1368 (8.6%) | 1436 (9.0%) | -0.01 |
| Occurrence of chronic renal insufficiency; n (%) | 241 (11.2%) | 271 (12.6%) | -0.04 | 257 (4.5%) | 267 (4.7%) | -0.01 | 988 (12.3%) | 1,094 (13.6%) | 1486 (9.4%) | 1632 (10.3%) | -0.03 |
| Chronic kidney disease v2; n (%) | 236 (11.0%) | 258 (12.0%) | -0.03 | 226 (4.0%) | 246 (4.3%) | -0.02 | 951 (11.8%) | 1,039 (12.9%) | 1413 (8.9%) | 1543 (9.7%) | -0.03 |
| CKD Stage 3-4; n (%) | 154 (7.2%) | 158 (7.3%) | 0.00 | 121 (2.1%) | 139 (2.4%) | -0.02 | 595 (7.4%) | 649 (8.0%) | 870 (5.5%) | 946 (6.0%) | -0.02 |
| Occurrence of hypertensive nephropathy; n (%) | 154 (7.2%) | 170 (7.9%) | -0.03 | 154 (2.7%) | 165 (2.9%) | -0.01 | 758 (9.4%) | 839 (10.4%) | 1066 (6.7%) | 1174 (7.4%) | -0.03 |
| Occurrence of miscellaneous renal insufficiency v2; n | | | | | | | | | | | |
| (%) | 187 (8.7%) | 182 (8.5%) | 0.01 | 286 (5.0%) | 286 (5.0%) | 0.00 | 681 (8.4%) | 697 (8.6%) | 1154 (7.3%) | 1165 (7.3%) | 0.00 |

| Liver disease; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Osteoarthritis; n (%) Other arthritis, arthropathies and musculoskeletal | 665 (30.9%) | 642 (29.8%) | 0.02 | 1,107 (19.5%) | 1,110 (19.6%) | 0.00 | 3,006 (37.3%) | 2,998 (37.2%) | 4778 (30.1%) | 4750 (29.9%) | 0.00 |
| pain; n (%) | 1,448 (67.3%) | 1,425 (66.2%) | 0.02 | 3,489 (61.5%) | 3,441 (60.6%) | 0.02 | 4,956 (61.5%) | 4.958 (61.5%) | 9893 (62.2%) | 9824 (61.8%) | 0.01 |
| Dorsopathies; n (%) | 797 (37.0%) | 772 (35.9%) | 0.02 | 1,632 (28.8%) | 1,652 (29.1%) | -0.01 | 2,750 (34.1%) | 2,772 (34.4%) | 5179 (32.6%) | 5196 (32.7%) | 0.00 |
| Fractures; n (%) | 230 (10.7%) | 225 (10.5%) | 0.01 | 430 (7.6%) | 402 (7.1%) | 0.02 | 838 (10.4%) | 816 (10.1%) | 1498 (9.4%) | 1443 (9.1%) | 0.01 |
| Falls v2; n (%) | 186 (8.6%) | 186 (8.6%) | 0.00 | 166 (2.9%) | 152 (2.7%) | 0.01 | 313 (3.9%) | 308 (3.8%) | 665 (4.2%) | 646 (4.1%) | 0.01 |
| Osteoporosis; n (%) | 137 (6.4%) | 178 (8.3%) | -0.07 | 153 (2.7%) | 165 (2.9%) | -0.01 | 1,050 (13.0%) | 1,096 (13.6%) | 1340 (8.4%) | 1439 (9.1%) | -0.02 |
| Depression; n (%) | 428 (19.9%) | 441 (20.5%) | -0.01 | 810 (14.3%) | 802 (14.1%) | 0.01 | 1,481 (18.4%) | 1,528 (18.9%) | 2719 (17.1%) | 2771 (17.4%) | -0.01 |
| Anxiety; n (%) | 409 (19.0%) | 425 (19.7%) | -0.02 | 797 (14.0%) | 791 (13.9%) | 0.00 | 1,388 (17.2%) | 1,389 (17.2%) | 2594 (16.3%) | 2605 (16.4%) | 0.00 |
| Sleep_Disorder; n (%) | 245 (11.4%) | 259 (12.0%) | -0.02 | 651 (11.5%) | 697 (12.3%) | -0.02 | 827 (10.3%) | 851 (10.6%) | 1723 (10.8%) | 1807 (11.4%) | -0.02 |
| Dementia; n (%) | 160 (7.4%) | 171 (7.9%) | -0.02 | 134 (2.4%) | 135 (2.4%) | 0.00 | 842 (10.4%) | 913 (11.3%) | 1136 (7.1%) | 1219 (7.7%) | -0.02 |
| Delirium; n (%) | 74 (3.4%) | 87 (4.0%) | -0.03 | 104 (1.8%) | 92 (1.6%) | 0.02 | 306 (3.8%) | 299 (3.7%) | 484 (3.0%) | 478 (3.0%) | 0.00 |
| Psychosis; n (%) | 59 (2.7%) | 66 (3.1%) | -0.02 | 65 (1.1%) | 64 (1.1%) | 0.00 | 219 (2.7%) | 224 (2.8%) | 343 (2.2%) | 354 (2.2%) | 0.00 |
| Obesity; n (%) | 704 (32.7%) | 715 (33.2%) | -0.01 | 1,534 (27.0%) | 1,531 (27.0%) | 0.00 | 1,869 (23.2%) | 1,896 (23.5%) | 4107 (25.8%) | 4142 (26.1%) | -0.01 |
| Overweight; n (%) | 111 (5.2%) | 99 (4.6%) | 0.03 | 156 (2.7%) | 136 (2.4%) | 0.02 | 369 (4.6%) | 368 (4.6%) | 636 (4.0%) | 603 (3.8%) | 0.01 |
| Smoking; n (%) | 690 (32.0%)<br>62 (2.9%) | 677 (31.4%)<br>57 (2.6%) | 0.01<br>0.02 | 934 (16.5%)<br>129 (2.3%) | 920 (16.2%)<br>111 (2.0%) | 0.01<br>0.02 | 3,048 (37.8%)<br>106 (1.3%) | 2,933 (36.4%)<br>91 (1.1%) | 4672 (29.4%)<br>297 (1.9%) | 4530 (28.5%)<br>259 (1.6%) | 0.02 |
| Alcohol abuse or dependence; n (%) | | | | | | | . , | , , | | , , | 0.02 |
| Drug abuse or dependence; n (%)<br>COPD; n (%) | 78 (3.6%)<br>382 (17.7%) | 79 (3.7%)<br>428 (19.9%) | -0.01<br>-0.06 | 110 (1.9%)<br>582 (10.3%) | 111 (2.0%)<br>567 (10.0%) | -0.01<br>0.01 | 90 (1.1%)<br>1,887 (23.4%) | 80 (1.0%)<br>1,932 (24.0%) | 278 (1.7%)<br>2851 (17.9%) | 270 (1.7%)<br>2927 (18.4%) | -0.01 |
| Asthma: n (%) | 276 (12.8%) | 297 (13.8%) | -0.03 | 628 (11.1%) | 632 (11.1%) | 0.01 | 900 (11.2%) | 931 (11.5%) | 1804 (11.4%) | 1860 (11.7%) | -0.01 |
| Obstructive sleep apnea; n (%) | 309 (14.4%) | 310 (14.4%) | 0.00 | 689 (12.1%) | 706 (12.4%) | -0.01 | 825 (10.2%) | 824 (10.2%) | 1823 (11.5%) | 1840 (11.6%) | 0.00 |
| Pneumonia; n (%) | 378 (17.6%) | 411 (19.1%) | -0.04 | 856 (15.1%) | 841 (14.8%) | 0.01 | 1,435 (17.8%) | 1,421 (17.6%) | 2669 (16.8%) | 2673 (16.8%) | 0.00 |
| Other Medications | 370 (17.070) | 411 (13.170) | 0.04 | 050 (15.170) | 041 (14.0%) | 0.01 | 1,455 (17.070) | 1,421 (17.070) | 2003 (20.070) | 2073 (20.070) | 0.00 |
| Use of ACE inhibitors; n (%) | 487 (22.6%) | 520 (24.2%) | -0.04 | 1,094 (19.3%) | 1,090 (19.2%) | 0.00 | 2,376 (29.5%) | 2,459 (30.5%) | 3957 (24.9%) | 4069 (25.6%) | -0.02 |
| Use of ARBs: n (%) | 323 (15.0%) | 332 (15.4%) | -0.01 | 691 (12.2%) | 745 (13.1%) | -0.03 | 1.583 (19.6%) | 1.624 (20.1%) | 2597 (16.3%) | 2701 (17.0%) | -0.02 |
| Use of Loop Diuretics - United; n (%) | 189 (8.8%) | 195 (9.1%) | -0.01 | 333 (5.9%) | 336 (5.9%) | 0.00 | 967 (12.0%) | 1,047 (13.0%) | 1489 (9.4%) | 1578 (9.9%) | -0.02 |
| Use of other diuretics- United; n (%) | 36 (1.7%) | 37 (1.7%) | 0.00 | 84 (1.5%) | 80 (1.4%) | 0.01 | 136 (1.7%) | 166 (2.1%) | 256 (1.6%) | 283 (1.8%) | -0.02 |
| Use of nitrates-United; n (%) | 53 (2.5%) | 53 (2.5%) | 0.00 | 98 (1.7%) | 96 (1.7%) | 0.00 | 393 (4.9%) | 401 (5.0%) | 544 (3.4%) | 550 (3.5%) | -0.01 |
| Use of other hypertension drugs; n (%) | 85 (3.9%) | 83 (3.9%) | 0.00 | 151 (2.7%) | 159 (2.8%) | -0.01 | 474 (5.9%) | 436 (5.4%) | 710 (4.5%) | 678 (4.3%) | 0.01 |
| Use of Anti-arrhythmics; n (%) | ** (0.3%) | ** (0.1%) | 0.04 | 17 (0.3%) | ** (0.2%) | 0.02 | 28 (0.3%) | 27 (0.3%) | #VALUE! | #VALUE! | #VALUE! |
| Use of COPD/asthma meds- United; n (%) | 418 (19.4%) | 417 (19.4%) | 0.00 | 941 (16.6%) | 1,113 (19.6%) | -0.08 | 1,885 (23.4%) | 1,847 (22.9%) | 3244 (20.4%) | 3377 (21.2%) | -0.02 |
| Use of statins; n (%) | 707 (32.8%) | 726 (33.7%) | -0.02 | 1,422 (25.1%) | 1,416 (25.0%) | 0.00 | 3,609 (44.7%) | 3,654 (45.3%) | 5738 (36.1%) | 5796 (36.5%) | -0.01 |
| Use of other lipid-lowering drugs; n (%) | 115 (5.3%) | 133 (6.2%) | -0.04 | 293 (5.2%) | 306 (5.4%) | -0.01 | 606 (7.5%) | 620 (7.7%) | 1014 (6.4%) | 1059 (6.7%) | -0.01 |
| Use of antiplatelet agents; n (%) | 91 (4.2%) | 95 (4.4%) | -0.01 | 223 (3.9%) | 210 (3.7%) | 0.01 | 597 (7.4%) | 586 (7.3%) | 911 (5.7%) | 891 (5.6%) | 0.00 |
| Use of heparin and other low-molecular weight | | | | | | | | | | | |
| heparins; n (%) | 243 (11.3%) | 207 (9.6%) | 0.06 | ** (0.0%) | ** (0.0%) | #DIV/0! | 650 (8.1%) | 484 (6.0%) | #VALUE! | #VALUE! | #VALUE! |
| Use of NSAIDs; n (%) | 489 (22.7%) | 440 (20.4%) | 0.06 | 1,388 (24.5%) | 1,337 (23.6%) | 0.02 | 1,650 (20.5%) | 1,599 (19.8%) | 3527 (22.2%) | 3376 (21.2%) | 0.02 |
| Use of oral corticosteroids; n (%) Use of bisphosphonate (United); n (%) | 619 (28.8%)<br>58 (2.7%) | 619 (28.8%)<br>63 (2.9%) | 0.00<br>-0.01 | 1,372 (24.2%)<br>48 (0.8%) | 1,678 (29.6%)<br>72 (1.3%) | -0.12<br>-0.05 | 2,737 (33.9%)<br>352 (4.4%) | 2,708 (33.6%)<br>348 (4.3%) | 4728 (29.7%)<br>458 (2.9%) | 5005 (31.5%)<br>483 (3.0%) | -0.04<br>-0.01 |
| Use of opioids- United; n (%) | 1,105 (51.3%) | 1,065 (49.5%) | 0.04 | 3,029 (53.4%) | 3,012 (53.1%) | 0.01 | 3,819 (47.4%) | 3,797 (47.1%) | 7953 (50.0%) | 7874 (49.5%) | 0.01 |
| Use of antidepressants; n (%) | 614 (28.5%) | 621 (28.8%) | -0.01 | 1,416 (25.0%) | 1,411 (24.9%) | 0.00 | 2,513 (31.2%) | 2,528 (31.3%) | 4543 (28.6%) | 4560 (28.7%) | 0.00 |
| Use of antipsychotics; n (%) | 109 (5.1%) | 120 (5.6%) | -0.02 | 211 (3.7%) | 204 (3.6%) | 0.01 | 453 (5.6%) | 461 (5.7%) | 773 (4.9%) | 785 (4.9%) | 0.00 |
| Labs | 103 (3.170) | 120 (5.0%) | -0.02 | 211 (3.770) | 204 (3.0%) | 0.01 | 455 (5.0%) | 401 (3.770) | 773 (4.570) | 705 (4.570) | 0.00 |
| Lab values- HbA1c (%) v3; n (%) | 259 (12.0%) | 263 (12.2%) | -0.01 | 42 (0.7%) | 49 (0.9%) | -0.02 | N/A | N/A | 301 (3.8%) | 312 (4.0%) | -0.01 |
| Lab values-HbA1c (%) (within 3 months) v3: n (%) | 164 (7.6%) | 161 (7.5%) | 0.00 | 27 (0.5%) | 41 (0.7%) | -0.03 | N/A | N/A | 191 (2.4%) | 202 (2.6%) | -0.01 |
| Lab values-HbA1c (%) (within 6 months) v3; n (%) | 259 (12.0%) | 263 (12.2%) | -0.01 | 42 (0.7%) | 49 (0.9%) | -0.02 | N/A | N/A | 301 (3.8%) | 312 (4.0%) | -0.01 |
| Lab values- BNP; n (%) | 23 (1.1%) | 29 (1.3%) | -0.02 | ** (0.0%) | ** (0.1%) | -0.04 | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| Lab values-BNP (within 3 months); n (%) | 23 (1.1%) | 27 (1.3%) | -0.02 | ** (0.0%) | ** (0.1%) | -0.04 | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| Lab values- BNP (within 6 months); n (%) | 23 (1.1%) | 29 (1.3%) | -0.02 | ** (0.0%) | ** (0.1%) | -0.04 | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| Lab values- BUN (mg/dl); n (%) | 508 (23.6%) | 589 (27.4%) | -0.09 | 51 (0.9%) | 68 (1.2%) | -0.03 | N/A | N/A | 559 (7.1%) | 657 (8.4%) | -0.05 |
| Lab values-BUN (mg/dl) (within 3 months); n (%) | 358 (16.6%) | 415 (19.3%) | -0.07 | 36 (0.6%) | 53 (0.9%) | -0.03 | N/A | N/A | 394 (5.0%) | 468 (6.0%) | -0.04 |
| Lab values-BUN (mg/dl) (within 6 months); n (%) | 508 (23.6%) | 589 (27.4%) | -0.09 | 51 (0.9%) | 68 (1.2%) | -0.03 | N/A | N/A | 559 (7.1%) | 657 (8.4%) | -0.05 |
| Lab values- Creatinine (mg/dl) v2; n (%) | 512 (23.8%) | 608 (28.2%) | -0.10 | 52 (0.9%) | 74 (1.3%) | -0.04 | N/A | N/A | 564 (7.2%) | 682 (8.7%) | -0.06 |
| Lab values- Creatinine (mg/dl) (within 3 months) v2; | | | | | / /- | | | | | | |
| n (%)<br>Lab values-Creatinine (mg/dl) (within 6 months) v2; | 359 (16.7%) | 431 (20.0%) | -0.09 | 37 (0.7%) | 57 (1.0%) | -0.03 | N/A | N/A | 396 (5.1%) | 488 (6.2%) | -0.05 |
| n (%) | 512 (23.8%) | 608 (28.2%) | -0.10 | 52 (0.9%) | 74 (1.3%) | -0.04 | N/A | N/A | 564 (7.2%) | 682 (8.7%) | -0.06 |
| Lab values- HDL level (mg/dl); n (%) | 314 (14.6%) | 352 (16.3%) | -0.05 | 35 (0.6%) | 44 (0.8%) | -0.02 | N/A | N/A | 349 (4.5%) | 396 (5.1%) | -0.03 |
| tab values ristricter (ing/ai/, ii (/a/ | 324 (24.070) | 332 (20.370) | 0.03 | 33 (0.070) | 44 (0.0%) | 0.02 | 14/11 | .,,, | 343 (4.370) | 330 (3.170) | 0.03 |
| Lab values- HDL level (mg/dl) (within 3 months); n (%) | 179 (8.3%) | 191 (8.9%) | -0.02 | 21 (0.4%) | 28 (0.5%) | -0.01 | N/A | N/A | 200 (2.6%) | 219 (2.8%) | -0.01 |
| | | () | | | | | | | | **** | |
| Lab values- HDL level (mg/dl) (within 6 months); n (%) | 314 (14.6%) | 352 (16.3%) | -0.05 | 35 (0.6%) | 44 (0.8%) | -0.02 | N/A | N/A | 349 (4.5%) | 396 (5.1%) | -0.03 |
| Lab values- LDL level (mg/dl) v2; n (%) | 324 (15.0%) | 363 (16.9%) | -0.05 | 38 (0.7%) | 44 (0.8%) | -0.01 | N/A | N/A | 362 (4.6%) | 407 (5.2%) | -0.03 |
| Lab values-LDL level (mg/dl) (within 3 months) v2; n<br>(%) | 181 (8.4%) | 197 (9.2%) | -0.03 | 24 (0.4%) | 28 (0.5%) | -0.01 | N/A | N/A | 205 (2.6%) | 225 (2.9%) | -0.02 |
| Lab values-LDL level (mg/dl) (within 6 months) v2; n | 101 (0.470) | 137 (3.270) | -0.03 | 24 (0.470) | 20 (0.5%) | -0.01 | 14/15 | 11/15 | 203 (2.0%) | 223 (2.370) | -0.02 |
| (%) | 324 (15.0%) | 363 (16.9%) | -0.05 | 38 (0.7%) | 44 (0.8%) | -0.01 | N/A | N/A | 362 (4.6%) | 407 (5.2%) | -0.03 |
| Lab values- NT-proBNP; n (%) | ** (0.2%) | ** (0.3%) | -0.02 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| Lab values- NT-proBNP (within 3 months); n (%) | ** (0.2%) | ** (0.3%) | -0.02 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| Lab values- NT-proBNP (within 6 months); n (%) | ** (0.2%) | ** (0.3%) | -0.02 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| Lab values-Total cholesterol (mg/dl) v2; n (%) | 321 (14.9%) | 355 (16.5%) | -0.04 | 35 (0.6%) | 45 (0.8%) | -0.02 | N/A | N/A | 356 (4.5%) | 400 (5.1%) | -0.03 |
| Lab values-Total cholesterol (mg/dl) (within 3 | | | | | | | | | | | |
| months) v2; n (%) | 183 (8.5%) | 192 (8.9%) | -0.01 | 21 (0.4%) | 29 (0.5%) | -0.01 | N/A | N/A | 204 (2.6%) | 221 (2.8%) | -0.01 |
| Lab values-Total cholesterol (mg/dl) (within 6 | | | | | | | | | | | |
| months) v2; n (%) | 321 (14.9%) | 355 (16.5%) | -0.04 | 35 (0.6%) | 45 (0.8%) | -0.02 | N/A | N/A | 356 (4.5%) | 400 (5.1%) | -0.03 |
| Lab values-Triglyceride level (mg/dl); n (%) | 316 (14.7%) | 351 (16.3%) | -0.04 | 34 (0.6%) | 43 (0.8%) | -0.02 | N/A | N/A | 350 (4.5%) | 394 (5.0%) | -0.02 |

| Lab values-Triglyceride level (mg/dl) (within 3 | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| months); n (%) | 181 (8.4%) | 190 (8.8%) | -0.01 | 20 (0.4%) | 28 (0.5%) | -0.01 | N/A | N/A | 201 (2.6%) | 218 (2.8%) | -0.01 |
| Lab values-Triglyceride level (mg/dl) (within 6 | | | | | | | | | | | |
| months); n (%) | 316 (14.7%) | 351 (16.3%) | -0.04 | 34 (0.6%) | 43 (0.8%) | -0.02 | N/A | N/A | 350 (4.5%) | 394 (5.0%) | -0.02 |
| Lab result number- HbA1c (%) mean (only 2 to 20 included) v4 | 258 | 259 | | 41 | 47 | | N/A | N/A | 299 | 306 | |
| mean (sd) | 6.67 (1.56) | 6.63 (1.56) | 0.03 | 7.09 (1.30) | 7.13 (1.71) | -0.03 | N/A<br>N/A | N/A<br>N/A | 6.73 (1.53) | 6.71 (1.59) | 0.01 |
| Missing; n (%) | 1,895 (88.0%) | 1,894 (88.0%) | 0.00 | 5,634 (99.3%) | 5,628 (99.2%) | 0.01 | N/A | N/A | 7,529 (96.2%) | 7,522 (96.1%) | 0.01 |
| Lab result number- BNP mean v2 | 23 | 29 | | 2 | 3 | | N/A | N/A | 25 | 32 | |
| mean (sd) | 65.94 (82.23) | 155.95 (239.40) | -0.50 | 38.70 (3.11) | 75.00 (68.46) | -0.75 | N/A | N/A | 63.76 (82.23) | 148.36 (235.92) | -0.48 |
| Missing; n (%) | 2,130 (98.9%) | 2,124 (98.7%) | 0.02 | 5,673 (100.0%) | 5,672 (99.9%) | 0.04 | N/A | N/A | 7,803 (99.7%) | 7,796 (99.6%) | 0.02 |
| Lab result number- BUN (mg/dl) mean v2 | 508 | 589 | | 51 | 68 | | N/A | N/A | 559 | 657 | |
| mean (sd) | 16.85 (6.32) | 16.63 (6.05) | 0.04 | 3,939.06 (28,003.10) | 1,780.81 (14,550.16) | 0.10 | N/A | N/A | 374.69 (8397.57) | 199.22 (4657.11) | 0.03 |
| Missing; n (%) | 1,645 (76.4%) | 1,564 (72.6%) | 0.09 | 5,624 (99.1%) | 5,607 (98.8%) | 0.03 | N/A | N/A | 7,269 (92.9%) | 7,171 (91.6%) | 0.05 |
| Lab result number- Creatinine (mg/dl) mean (only 0.1 to 15 included) v3 | 508 | 601 | | 49 | 72 | | N/A | N/A | 557 | 673 | |
| mean (sd) | 0.97 (0.31) | 0.94 (0.24) | 0.11 | 1.01 (0.26) | 0.96 (0.26) | 0.19 | N/A | N/A | 0.97 (0.31) | 0.94 (0.24) | 0.11 |
| Missing; n (%) | 1,645 (76.4%) | 1,552 (72.1%) | 0.10 | 5,626 (99.1%) | 5,603 (98.7%) | 0.04 | N/A | N/A | 7,271 (92.9%) | 7,155 (91.4%) | 0.06 |
| Lab result number- HDL level (mg/dl) mean (only | | | | | | | | | | | |
| =<5000 included) v2 | 314 | 352 | | 35 | 43 | | N/A | N/A | 349 | 395 | |
| mean (sd) | 53.71 (16.56) | 52.98 (16.30) | 0.04 | 46.42 (18.95) | 48.02 (16.23) | -0.09 | N/A | N/A | 52.98 (16.83) | 52.44 (16.31) | 0.03 |
| Missing; n (%) | 1,839 (85.4%) | 1,801 (83.7%) | 0.05 | 5,640 (99.4%) | 5,632 (99.2%) | 0.02 | N/A | N/A | 7,479 (95.5%) | 7,433 (95.0%) | 0.02 |
| Lab result number- LDL level (mg/dl) mean (only<br>=<5000 included) v2 | 318 | 351 | | 32 | 41 | | N/A | N/A | 350 | 392 | |
| mean (sd) | 102.29 (35.24) | 102.76 (39.24) | -0.01 | 100.14 (43.88) | 102.63 (43.57) | -0.06 | N/A | N/A | 102.09 (36.15) | 102.75 (39.76) | -0.02 |
| Missing; n (%) | 1,835 (85.2%) | 1,802 (83.7%) | 0.04 | 5,643 (99.4%) | 5,634 (99.3%) | 0.01 | N/A | N/A | 7,478 (95.5%) | 7,436 (95.0%) | 0.02 |
| Lab result number-Total cholesterol (mg/dl) mean | ,, | , | | ., , , | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | | | | , , | , , | |
| (only =<5000 included) v2 | 320 | 354 | | 35 | 44 | | N/A | N/A | 355 | 398 | |
| mean (sd) | 186.00 (39.30) | 186.53 (44.31) | -0.01 | 179.03 (51.44) | 184.27 (47.29) | -0.11 | N/A | N/A | 185.31 (40.69) | 186.28 (44.70) | -0.02 |
| Missing; n (%) | 1,833 (85.1%) | 1,799 (83.6%) | 0.04 | 5,640 (99.4%) | 5,631 (99.2%) | 0.02 | N/A | N/A | 7,473 (95.5%) | 7,430 (94.9%) | 0.03 |
| Lab result number-Triglyceride level (mg/dl) mean | 316 | 351 | | 34 | 42 | | N/A | N/A | 350 | 393 | |
| (only =<5000 included) v2<br>mean (sd) | 141.37 (80.85) | 145.40 (97.12) | -0.05 | 161.92 (102.42) | 148.55 (81.44) | 0.14 | N/A | N/A | 143.37 (83.26) | 145.74 (95.72) | -0.03 |
| Missing; n (%) | 1,837 (85.3%) | 1,802 (83.7%) | 0.04 | 5,641 (99.4%) | 5,633 (99.3%) | 0.01 | N/A | N/A | 7,478 (95.5%) | 7,435 (95.0%) | 0.02 |
| Lab result number- Hemoglobin mean (only >0 | _,, | _, | | 0,012 (001111) | -, (, | | .4 | | ., | ., (, | |
| included) | 427 | 464 | | 42 | 56 | | N/A | N/A | 469 | 520 | |
| mean (sd) | 13.45 (1.77) | 13.33 (1.82) | 0.07 | 3,417.04 (22,063.44) | 2,673.48 (19,909.23) | 0.04 | N/A | N/A | 318.25 (6544.44) | 299.81 (6493.68) | 0.00 |
| Missing; n (%) | 1,726 (80.2%) | 1,689 (78.4%) | 0.04 | 5,633 (99.3%) | 5,619 (99.0%) | 0.03 | N/A | N/A | 7,359 (94.0%) | 7,308 (93.4%) | 0.02 |
| Lab result number- Serum sodium mean (only > 90 | 495 | | | 47 | 67 | | N/A | *** | 542 | 641 | |
| and < 190 included)<br>mean (sd) | 140.20 (2.66) | 574<br>140.06 (2.68) | 0.05 | 139.22 (3.38) | 139.19 (2.55) | 0.01 | N/A<br>N/A | N/A<br>N/A | 140.12 (2.73) | 139.97 (2.67) | 0.06 |
| Missing; n (%) | 1,658 (77.0%) | 1,579 (73.3%) | 0.09 | 5,628 (99.2%) | 5,608 (98.8%) | 0.04 | N/A | N/A | 7,286 (93.1%) | 7,187 (91.8%) | 0.05 |
| Lab result number- Albumin mean (only >0 and <=10 | 2,030 (77.070) | 1,575 (75.570) | 0.03 | 3,020 (33.270) | 3,000 (30.0%) | 0.04 | 14/11 | .,,,, | 7,200 (33.270) | 7,107 (51.070) | 0.03 |
| included) | 472 | 522 | | 42 | 55 | | N/A | N/A | 514 | 577 | |
| mean (sd) | 4.08 (0.39) | 4.10 (0.36) | -0.05 | 3.91 (0.93) | 4.02 (0.66) | -0.14 | N/A | N/A | 4.07 (0.46) | 4.09 (0.40) | -0.05 |
| Missing; n (%) | 1,681 (78.1%) | 1,631 (75.8%) | 0.05 | 5,633 (99.3%) | 5,620 (99.0%) | 0.03 | N/A | N/A | 7,314 (93.4%) | 7,251 (92.6%) | 0.03 |
| Lab result number-Glucose (fasting or random) mean | 491 | 500 | | 50 | 71 | | N/A | N/A | 541 | 639 | |
| (only 10-1000 included)<br>mean (sd) | 113.45 (43.92) | 568<br>110.67 (37.41) | 0.07 | 142.44 (59.71) | 144.25 (99.21) | -0.02 | N/A<br>N/A | N/A<br>N/A | 116.13 (45.62) | 114.40 (48.28) | 0.04 |
| Missing; n (%) | 1,662 (77.2%) | 1,585 (73.6%) | 0.07 | 5,625 (99.1%) | 5,604 (98.7%) | 0.04 | N/A | N/A | 7,287 (93.1%) | 7,189 (91.8%) | 0.04 |
| Lab result number- Potassium mean (only 1-7 | 2,002 (77.270) | 1,505 (75.070) | 0.00 | 3,023 (33.270) | 3,004 (30.770) | 0.04 | 14/11 | .,,,, | 7,207 (33.270) | 7,103 (31.070) | 0.03 |
| included) | 507 | 592 | | 48 | 64 | | N/A | N/A | 555 | 656 | |
| mean (sd) | 4.33 (0.42) | 4.32 (0.42) | 0.02 | 4.30 (0.44) | 4.24 (0.40) | 0.14 | N/A | N/A | 4.33 (0.42) | 4.31 (0.42) | 0.05 |
| Missing; n (%) | 1,646 (76.5%) | 1,561 (72.5%) | 0.09 | 5,627 (99.2%) | 5,611 (98.9%) | 0.03 | N/A | N/A | 7,273 (92.9%) | 7,172 (91.6%) | 0.05 |
| Comorbidity Scores | | | | | | | | | | | |
| CCI (180 days)-ICD9 and ICD10 v2 | 2 70 (2 24) | 2 70 (2 47) | 0.00 | 1.74 (2.00) | 1 (0 (2 04) | 0.03 | 2.57/2.24) | 2 52 (2 20) | 2 20 (2 22) | 2.26 (2.28) | 0.03 |
| mean (sd)<br>Non-Frailty; n (%) | 2.79 (2.31)<br>1,041 (48.4%) | 2.78 (2.47)<br>1,027 (47.7%) | 0.00<br>0.01 | 1.74 (2.00)<br>2,447 (43.1%) | 1.69 (2.04)<br>2,383 (42.0%) | 0.02<br>0.02 | 2.57 (2.34)<br>310 (3.8%) | 2.53 (2.39)<br>252 (3.1%) | 2.30 (2.22)<br>3,798 (23.9%) | 2.26 (2.28)<br>3,662 (23.0%) | 0.02<br>0.02 |
| Frailty Score (mean): Empirical Version 365 days, v2 | 2,0-1 (40.4/0) | 2,02/(47.7/0) | 0.01 | 2,447 (43.1/0) | 2,303 (42.070) | 0.02 | 313 (3.070) | 232 (3.170) | 5,, 50 (23.570) | 3,002 (23.070) | 0.02 |
| mean (sd) | 0.19 (0.06) | 0.19 (0.07) | 0.00 | 0.16 (0.05) | 0.16 (0.05) | 0.00 | 0.09 (0.07) | 0.10 (0.07) | 0.13 (0.06) | 0.13 (0.06) | 0.00 |
| Healthcare Utilization | | | | | | | | | | | |
| Any hospitalization; n (%) | 2,034 (94.5%) | 2,011 (93.4%) | 0.05 | 5,674 (100.0%) | 5,675 (100.0%) | #DIV/0! | 7,678 (95.2%) | 7,733 (95.9%) | 15,386 (96.8%) | 15,419 (97.0%) | -0.01 |
| Any hospitalization within prior 30 days; n (%) | 1,966 (91.3%) | 1,967 (91.4%) | 0.00 | 5,661 (99.8%) | 5,658 (99.7%) | 0.02 | 7,617 (94.4%) | 7,655 (94.9%) | 15244 (95.9%) | 15280 (96.1%) | -0.01 |
| Any hospitalization during prior 31-180 days; n (%) | 262 (12.2%) | 247 (11.5%) | 0.02 | 448 (7.9%) | 415 (7.3%) | 0.02 | 1,216 (15.1%) | 1,052 (13.0%) | 1926 (12.1%) | 1714 (10.8%) | 0.04 |
| Internal medicine/family medicine visits; n (%) | 1,920 (89.2%) | 1,911 (88.8%) | 0.01 | 4,445 (78.3%) | 4,436 (78.2%) | 0.00 | 7,824 (97.0%) | 7,851 (97.3%) | 14189 (89.3%) | 14198 (89.3%) | 0.00 |
| Internal medicine/family medicine visits (30 days<br>prior) v2; n (%) | 1,743 (81.0%) | 1,723 (80.0%) | 0.03 | 3,220 (56.7%) | 3,134 (55.2%) | 0.03 | 7,554 (93.7%) | 7,574 (93.9%) | 12517 (78.8%) | 12431 (78.2%) | 0.01 |
| Internal medicine/family medicine visits (31 to 180 | 1,743 (01.070) | 1,723 (00.070) | 0.03 | 3,220 (30.7/8) | 3,134 (33.270) | 0.03 | 7,554 (55.770) | (0.5.5) | 12317 (70.070) | 12431 (70.270) | 0.01 |
| days prior) v2; n (%) | 1,375 (63.9%) | 1,360 (63.2%) | 0.01 | 3,520 (62.0%) | 3,585 (63.2%) | -0.02 | 5,892 (73.1%) | 5,955 (73.8%) | 10787 (67.9%) | 10900 (68.6%) | -0.02 |
| Cardiologist visit; n (%) | 1,530 (71.1%) | 1,486 (69.0%) | 0.05 | 1,416 (25.0%) | 1,453 (25.6%) | -0.01 | 5,922 (73.4%) | 5,904 (73.2%) | 8868 (55.8%) | 8843 (55.6%) | 0.00 |
| Number of Cardiologist visits (30 days prior); n (%) | 1,393 (64.7%) | 1,361 (63.2%) | 0.03 | 1,000 (17.6%) | 1,011 (17.8%) | -0.01 | 5,390 (66.8%) | 5,362 (66.5%) | 7783 (49.0%) | 7734 (48.7%) | 0.01 |
| Number of Cardiologist visits (31 to 180 days prior); | | | | | | | | | | | |
| n (%) | 405 (18.8%)<br>1.793 (83.3%) | 404 (18.8%)<br>1.843 (85.6%) | 0.00<br>-0.06 | 619 (10.9%)<br>2,747 (48.4%) | 637 (11.2%)<br>2,750 (48.5%) | -0.01<br>0.00 | 2,029 (25.2%)<br>7,025 (87.1%) | 2,030 (25.2%)<br>7,025 (87.1%) | 3053 (19.2%)<br>11565 (72.8%) | 3071 (19.3%)<br>11618 (73.1%) | 0.00<br>-0.01 |
| Electrocardiogram v2; n (%) Use of glucose test strips; n (%) | 1,793 (83.3%)<br>28 (1.3%) | 1,843 (85.6%) | -0.06 | 2,747 (48.4%)<br>46 (0.8%) | 2,750 (48.5%)<br>46 (0.8%) | 0.00 | 7,025 (87.1%)<br>98 (1.2%) | 7,025 (87.1%)<br>98 (1.2%) | 11565 (72.8%) | 11618 (/3.1%) | -0.01<br>0.00 |
| Dialysis; n (%) | 28 (1.3%)<br>0 (0.0%) | 29 (1.3%)<br>0 (0.0%) | #DIV/0! | 46 (0.8%)<br>0 (0.0%) | 0 (0.0%) | #DIV/0! | 98 (1.2%)<br>** (0.0%) | 98 (1.2%)<br>** (0.0%) | 1/2 (1.1%)<br>#VALUE! | 1/3 (1.1%)<br>#VALUE! | #VALUE! |
| | - (/0) | - (/0) | , 0. | 2 (3.070) | - (0/0) | | \/ | (=.=/0) | | | |

| number of different/distinct medication | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| prescriptions | | | | | | | | | | | |
| mean (sd) | 9.05 (5.56) | 9.04 (5.50) | 0.00 | 8.49 (5.04) | 8.53 (5.59) | -0.01 | 9.74 (4.89) | 9.85 (4.98) | 9.20 (5.04) | 9.27 (5.28) | -0.01 |
| Number of Hospitalizations | 445 (0.53) | 1.17 (0.70) | -0.02 | 1.18 (0.52) | 1.17 (0.48) | 0.02 | 1.25 (0.72) | 1.26 (0.68) | 1.21 (0.64) | 1.22 (0.62) | -0.02 |
| mean (sd) Number of hospital days | 1.16 (0.62) | 1.17 (0.70) | -0.02 | 1.18 (0.52) | 1.17 (0.48) | 0.02 | 1.25 (0.72) | 1.26 (0.68) | 1.21 (0.64) | 1.22 (0.62) | -0.02 |
| mean (sd) | 5.88 (3.52) | 5.78 (5.88) | 0.02 | 5.05 (3.36) | 4.99 (4.88) | 0.01 | 6.38 (3.73) | 6.32 (6.02) | 5.84 (3.57) | 5.77 (5.62) | 0.01 |
| Number of Emergency Department (ED) visits v3 | 3.00 (3.32) | 3.70 (3.00) | 0.02 | 3.03 (3.30) | 4.55 (4.66) | 0.01 | 0.50 (5.75) | 0.52 (0.02) | 3.04 (3.37) | 3.77 (3.02) | 0.01 |
| mean (sd) | 1.58 (2.36) | 1.60 (2.03) | -0.01 | 3.00 (4.68) | 2.87 (4.74) | 0.03 | 1.67 (1.95) | 1.72 (2.10) | 2.13 (3.24) | 2.11 (3.29) | 0.01 |
| Number of Office visits | | | | | | | | | | | |
| mean (sd) | 5.23 (4.60) | 5.24 (4.55) | 0.00 | 4.86 (4.49) | 4.89 (4.50) | -0.01 | 13.55 (14.34) | 13.53 (13.73) | 9.32 (10.70) | 9.32 (10.28) | 0.00 |
| Number of internal medicine/family medicine visits | 44.40 (44.00) | 0.00 (4.2.20) | | 5 50 (0 40) | 5 56 (0 53) | 2.24 | 42.74 (40.02) | 44.04/40.57\ | 0.00 (40.04) | 0.35 (40.45) | 0.05 |
| mean (sd) Number of Cardiologist visits | 11.10 (14.06) | 9.98 (12.28) | 0.08 | 5.68 (9.10) | 5.56 (8.53) | 0.01 | 12.71 (10.92) | 11.84 (10.57) | 9.98 (10.81) | 9.35 (10.15) | 0.06 |
| mean (sd) | 2.39 (3.48) | 2.36 (3.42) | 0.01 | 0.64 (1.87) | 0.63 (2.02) | 0.01 | 2.81 (4.08) | 2.87 (4.25) | 1.98 (3.37) | 2.00 (3.49) | -0.01 |
| Number electrocardiograms received v2 | () | , | | | () | | () | (, | , | , | |
| mean (sd) | 1.98 (2.14) | 2.01 (2.00) | -0.01 | 0.83 (1.16) | 0.83 (1.22) | 0.00 | 2.02 (1.75) | 2.03 (1.70) | 1.59 (1.63) | 1.60 (1.59) | -0.01 |
| Number of HbA1c tests ordered | | | | | | | | | | | |
| mean (sd) | 0.32 (0.65) | 0.32 (0.64) | 0.00 | 0.20 (0.51) | 0.20 (0.50) | 0.00 | 0.35 (0.66) | 0.35 (0.65) | 0.29 (0.61) | 0.29 (0.60) | 0.00 |
| Number of glucose tests ordered | | | | | | | | | () | | |
| mean (sd) Number of lipid tests ordered | 0.21 (1.51) | 0.19 (0.99) | 0.02 | 0.10 (0.52) | 0.11 (0.78) | -0.02 | 0.14 (0.59) | 0.14 (0.54) | 0.14 (0.76) | 0.14 (0.71) | 0.00 |
| mean (sd) | 0.47 (0.72) | 0.50 (1.17) | -0.03 | 0.35 (0.72) | 0.35 (0.70) | 0.00 | 0.55 (0.71) | 0.55 (0.74) | 0.47 (0.71) | 0.47 (0.80) | 0.00 |
| Total N distinct ICD9/ICD10 diagnoses at the 3rd | 0.47 (0.72) | 0.30 (1.17) | -0.03 | 0.33 (0.72) | 0.55 (0.70) | 0.00 | 0.55 (0.71) | 0.55 (0.74) | 0.47 (0.71) | 0.47 (0.00) | 0.00 |
| digit level Copy | | | | | | | | | | | |
| mean (sd) | 11.03 (11.87) | 11.05 (12.50) | 0.00 | 7.05 (9.40) | 6.75 (9.53) | 0.03 | 13.29 (12.56) | 12.93 (13.09) | 10.76 (11.43) | 10.47 (11.86) | 0.02 |
| For PS | | | | | | | | | | | |
| Hemorrhagic stroke+Other cerebrovascular | 22 (4 50/) | 20 (4 20/) | 0.03 | 44 (0.00() | 20 (0 70() | 2.24 | 457 (4.00() | 472 (2.40() | 224/4 50/1 | 240 (4.50() | 2.22 |
| disease+Cerebrovascular procedure (for PS); n (%) Major trauma potentially causing prolonged immobili | 33 (1.5%)<br>173 (8.0%) | 29 (1.3%)<br>170 (7.9%) | 0.02<br>#DIV/0! | 44 (0.8%)<br>379 (6.7%) | 39 (0.7%)<br>349 (6.1%) | 0.01<br>#DIV/0! | 157 (1.9%)<br>559 (6.9%) | 172 (2.1%)<br>538 (6.7%) | 234 (1.5%)<br>379 (6.7%) | 240 (1.5%)<br>349 (6.1%) | 0.00 |
| Major trauma potentiany causing profonged minobin | 1/3 (8.0%) | 170 (7.5%) | #DIV/0: | 375 (0.7%) | 345 (0.1%) | #510/0: | 335 (0.5%) | 338 (0.7 %) | 379 (0.7%) | 345 (0.1%) | 0.02 |
| Occurrence of creatinine tests ordered (for PS); n (%) | 159 (7.4%) | 154 (7.2%) | 0.01 | 327 (5.8%) | 314 (5.5%) | 0.01 | 846 (10.5%) | 782 (9.7%) | 1332 (8.4%) | 1250 (7.9%) | 0.02 |
| Occurrence of BUN tests ordered (for PS); n (%) | 78 (3.6%) | 76 (3.5%) | 0.01 | 153 (2.7%) | 169 (3.0%) | -0.02 | 407 (5.0%) | 413 (5.1%) | 638 (4.0%) | 658 (4.1%) | -0.01 |
| Occurrence of chronic renal insufficiency w/o CKD | | | | | | | | | | | |
| (for PS) v2; n (%) | 118 (5.5%) | 122 (5.7%) | -0.01 | 142 (2.5%) | 136 (2.4%) | 0.01 | 464 (5.8%) | 515 (6.4%) | 724 (4.6%) | 773 (4.9%) | -0.01 |
| Chronic kidney disease Stage 1-2 (for PS); n (%)<br>Chronic kidney disease Stage 3-6 (for PS); n (%) | 52 (2.4%)<br>154 (7.2%) | 55 (2.6%)<br>158 (7.3%) | -0.01<br>0.00 | 43 (0.8%)<br>121 (2.1%) | 49 (0.9%)<br>139 (2.4%) | -0.01<br>-0.02 | 129 (1.6%)<br>595 (7.4%) | 133 (1.6%)<br>649 (8.0%) | 224 (1.4%)<br>870 (5.5%) | 237 (1.5%)<br>946 (6.0%) | -0.01<br>-0.02 |
| Acute kidney injury; n (%) | 238 (11.1%) | 231 (10.7%) | #DIV/0! | 350 (6.2%) | 363 (6.4%) | #DIV/0! | 824 (10.2%) | 887 (11.0%) | 350 (6.2%) | 363 (6.4%) | -0.02 |
| Bladder stones+Kidney stones (for PS); n (%) | 87 (4.0%) | 62 (2.9%) | 0.06 | 167 (2.9%) | 179 (3.2%) | -0.02 | 312 (3.9%) | 275 (3.4%) | 566 (3.6%) | 516 (3.2%) | 0.02 |
| Alcohol abuse or dependence+Drug abuse or | | , | | . , , | , | | , | , | , | , | |
| dependence (for PS); n (%) | 131 (6.1%) | 127 (5.9%) | 0.01 | 220 (3.9%) | 205 (3.6%) | 0.02 | 186 (2.3%) | 166 (2.1%) | 537 (3.4%) | 498 (3.1%) | 0.02 |
| Other atherosclerosis+Cardiac conduction | | | | | | | | | | | |
| disorders+Other CVD (for PS) v2 Copy; n (%) | 668 (31.0%) | 666 (30.9%) | 0.00 | 1,387 (24.4%) | 1,374 (24.2%) | 0.00 | 2,499 (31.0%) | 2,539 (31.5%) | 4554 (28.7%) | 4579 (28.8%) | 0.00 |
| Previous cardiac procedure (CABG or PTCA or Stent) +<br>History of CABG or PTCA (for PS) v3; n (%) | 94 (4.4%) | 92 (4.3%) | 0.00 | 85 (1.5%) | 77 (1.4%) | 0.01 | 698 (8.7%) | 736 (9.1%) | 877 (5.5%) | 905 (5.7%) | -0.01 |
| Diabetes with complication; n (%) | 194 (9.0%) | 192 (8.9%) | #DIV/0! | 246 (4.3%) | 251 (4.4%) | #DIV/0! | 611 (7.6%) | 661 (8.2%) | 246 (4.3%) | 251 (4.4%) | 0.00 |
| Delirium + Psychosis (for PS); n (%) | 112 (5.2%) | 133 (6.2%) | -0.04 | 153 (2.7%) | 137 (2.4%) | 0.02 | 469 (5.8%) | 463 (5.7%) | 734 (4.6%) | 733 (4.6%) | 0.00 |
| Any use of Meglitinides (for PS); n (%) | ** (0.2%) | ** (0.2%) | 0.00 | ** (0.2%) | ** (0.1%) | 0.03 | 29 (0.4%) | 24 (0.3%) | #VALUE! | #VALUE! | #VALUE! |
| Any use of AGIs (for PS); n (%) | ** (0.0%) | **(0.0%) | #DIV/0! | ** (0.0%) | ** (0.1%) | -0.04 | ** (0.0%) | ** (0.0%) | #VALUE! | #VALUE! | #VALUE! |
| CKD stage 3-6 + dialysis (for PS); n (%) | 154 (7.2%) | 159 (7.4%) | -0.01 | 121 (2.1%) | 139 (2.4%) | -0.02 | 598 (7.4%) | 651 (8.1%) | 873 (5.5%) | 949 (6.0%) | -0.02 |
| Use of thiazide; n (%) | 184 (8.5%)<br>517 (24.0%) | 197 (9.2%)<br>523 (24.3%) | -0.02<br>-0.01 | 388 (6.8%)<br>1,040 (18.3%) | 414 (7.3%)<br>1,072 (18.9%) | -0.02<br>-0.02 | 964 (12.0%)<br>2,759 (34.2%) | 1,010 (12.5%)<br>2,859 (35.4%) | 1536 (9.7%)<br>4316 (27.2%) | 1621 (10.2%)<br>4454 (28.0%) | -0.02<br>-0.02 |
| Use of beta blockers; n (%) Use of calcium channel blockers; n (%) | 392 (18.2%) | 406 (18.9%) | -0.01 | 1,040 (18.5%)<br>825 (14.5%) | 832 (14.7%) | -0.02 | 2,170 (26.9%) | 2,859 (35.4%) | 3387 (21.3%) | 3435 (21.6%) | -0.02 |
| All antidiabetic medications except Insulin; n (%) | 308 (14.3%) | 331 (15.4%) | -0.03 | 650 (11.5%) | 655 (11.5%) | 0.00 | 1.245 (15.4%) | 1,281 (15.9%) | 2203 (13.9%) | 2267 (14.3%) | -0.01 |
| DM Medications - Insulin Copy; n (%) | 109 (5.1%) | 104 (4.8%) | 0.01 | 219 (3.9%) | 224 (3.9%) | 0.00 | 276 (3.4%) | 297 (3.7%) | 604 (3.8%) | 625 (3.9%) | -0.01 |
| Use of Low Intensity Statins; n (%) | 433 (20.1%) | 458 (21.3%) | -0.03 | 804 (14.2%) | 874 (15.4%) | -0.03 | 2,351 (29.2%) | 2,398 (29.7%) | 3588 (22.6%) | 3730 (23.5%) | -0.02 |
| Use of High Intensity Statins; n (%) | 282 (13.1%) | 285 (13.2%) | 0.00 | 593 (10.4%) | 540 (9.5%) | 0.03 | 1,285 (15.9%) | 1,313 (16.3%) | 2160 (13.6%) | 2138 (13.5%) | 0.00 |
| Malignant hypertension; n (%) | 79 (3.7%) | 123 (5.7%) | -0.09 | 1,702 (30.0%) | 1,848 (32.6%) | -0.06 | 2,901 (36.0%) | 3,205 (39.7%) | 4682 (29.5%) | 5176 (32.6%) | -0.07 |
| Cardiovascular stress test; n (%) Echocardiogram; n (%) | 17 (0.8%)<br>1,240 (57.6%) | ** (0.3%)<br>1,203 (55.9%) | 0.07<br>0.03 | 41 (0.7%)<br>3,183 (56.1%) | 27 (0.5%)<br>3,236 (57.0%) | 0.03<br>-0.02 | 94 (1.2%)<br>4,635 (57.5%) | 97 (1.2%)<br>4,681 (58.0%) | 152 (1.0%)<br>9058 (57.0%) | #VALUE!<br>9120 (57.4%) | #VALUE!<br>-0.01 |
| Number of BNP tests | 1,240 (57.0%) | 1,203 (55.9%) | 0.03 | 3,183 (30.1%) | 3,230 (37.0%) | -0.02 | 4,033 (37.3%) | 4,081 (38.0%) | 9058 (57.0%) | 9120 (57.4%) | -0.01 |
| mean (sd) | 0.11 (0.39) | 0.12 (0.39) | -0.03 | 0.10 (0.36) | 0.10 (0.35) | 0.00 | 0.15 (0.41) | 0.16 (0.44) | 0.13 (0.39) | 0.13 (0.40) | 0.00 |
| • • | | , , | | | , , | | | | | , , | |
| Number of Cardiac biomarkers tests (tropnin, CK-MBs, My | | | | | | | | | | | |
| mean (sd) | 0.49 (1.92) | 0.49 (1.37) | 0.00 | 0.36 (1.04) | 0.38 (1.28) | -0.02 | 0.30 (0.62) | 0.32 (0.66) | 0.35 (1.04) | 0.36 (1.03) | 0.00 |
| Number of Ambulatory Blood pressure monitoring tests | | | | | | | | | | | |
| mean (sd) | 0.00 (0.00) | 0.00 (0.00) | #DIV/0! | 0.00 (0.02) | 0.00 (0.01) | 0.00 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.01) | 0.00 (0.01) | 0.00 |
| | 0.00 (0.00) | 3.00 (0.00) | 514/0: | 3.00 (0.02) | 3.00 (0.01) | 0.00 | 5.00 (0.00) | 5.00 (0.00) | 5.00 (0.01) | 3.00 (0.01) | 0.00 |
| N of days on antihypertensive medications during baseline | : | | | | | | | | | | |
| mean (sd) | 77.64 (79.51) | 81.69 (80.51) | -0.05 | 62.17 (77.97) | 63.02 (77.51) | -0.01 | 110.17 (77.59) | 112.91 (76.57) | 88.62 (77.99) | 90.87 (77.45) | 0.00 |
| N of days in database anytime prior | | | | | | | | | | | |
| mean (sd) | 1,744.50 (1,301.73) | 1,772.23 (1,328.01) | -0.02 | 1,984.17 (1,373.99) | 2,044.08 (1,376.43) | -0.04 | 638.67 (341.16) | 621.10 (306.74) | 1268.92 (981.16) | 1285.15 (981.38) | 0.00 |
| Mean Copay for per prescription cost (charges in U.S. \$) (1 | RO-1 day prior\ | | | | | | | | | | |
| mean (sd) | 22.68 (37.15) | 21.62 (36.53) | 0.03 | 14.31 (19.86) | 14.46 (36.77) | -0.01 | 109.17 (121.45) | 109.27 (115.41) | 63.58 (88.39) | 63.54 (86.16) | 0.00 |
| Missing; n (%) | 149 (6.9%) | 137 (6.4%) | 0.02 | 504 (8.9%) | 484 (8.5%) | 0.01 | 246 (3.1%) | 247 (3.1%) | 899 (5.7%) | 868 (5.5%) | 0.01 |
| - · · | | / | | () | - 17 | | / | 7 | | | |

| Colonoscopy; n (%) | 82 (3.8%) | 82 (3.8%) | 0.00 | 212 (3.7%) | 211 (3.7%) | 0.00 | 386 (4.8%) | 354 (4.4%) | 680 (4.3%) | 647 (4.1%) | 0.01 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Fecal occult blood (FOB) test; n (%) | 66 (3.1%) | 74 (3.4%) | -0.02 | 192 (3.4%) | 190 (3.3%) | 0.01 | 213 (2.6%) | 217 (2.7%) | 471 (3.0%) | 481 (3.0%) | 0.00 |
| Flu vaccine; n (%) | 329 (15.3%) | 332 (15.4%) | 0.00 | 576 (10.1%) | 577 (10.2%) | 0.00 | 2,499 (31.0%) | 2,520 (31.2%) | 3404 (21.4%) | 3429 (21.6%) | 0.00 |
| Mammogram; n (%) | 259 (12.0%) | 264 (12.3%) | -0.01 | 565 (10.0%) | 569 (10.0%) | 0.00 | 1,091 (13.5%) | 1,051 (13.0%) | 1915 (12.0%) | 1884 (11.9%) | 0.00 |
| Pap smear; n (%) | 105 (4.9%) | 116 (5.4%) | -0.02 | 447 (7.9%) | 442 (7.8%) | 0.00 | 235 (2.9%) | 231 (2.9%) | 787 (5.0%) | 789 (5.0%) | 0.00 |
| Pneumonia vaccine; n (%) | 332 (15.4%) | 312 (14.5%) | 0.03 | 385 (6.8%) | 370 (6.5%) | 0.01 | 1,839 (22.8%) | 1,696 (21.0%) | 2556 (16.1%) | 2378 (15.0%) | 0.03 |
| PSA test or Prostate exam for DRE; n (%) | 201 (9.3%) | 201 (9.3%) | 0.00 | 463 (8.2%) | 480 (8.5%) | -0.01 | 939 (11.6%) | 905 (11.2%) | 1603 (10.1%) | 1586 (10.0%) | 0.00 |
| Bone mineral density; n (%) | 71 (3.3%) | 73 (3.4%) | -0.01 | 93 (1.6%) | 95 (1.7%) | -0.01 | 399 (4.9%) | 389 (4.8%) | 563 (3.5%) | 557 (3.5%) | 0.00 |
| Use of CNS stimulants; n (%) | 18 (0.8%) | 18 (0.8%) | 0.00 | 65 (1.1%) | 93 (1.6%) | -0.04 | 37 (0.5%) | 39 (0.5%) | 120 (0.8%) | 150 (0.9%) | -0.01 |
| Use of estrogens, progestins, androgens; n (%) | 197 (9.2%) | 183 (8.5%) | 0.02 | 817 (14.4%) | 822 (14.5%) | 0.00 | 331 (4.1%) | 320 (4.0%) | 1345 (8.5%) | 1325 (8.3%) | 0.01 |
| Use of Angiogenesis inhibitors; n (%) | 0 (0.0%) | ** (0.0%) | #DIV/0! | ** (0.1%) | ** (0.0%) | 0.04 | ** (0.1%) | ** (0.0%) | #VALUE! | #VALUE! | #VALUE! |
| Use of Oral Immunosuppressants; n (%) | ** (0.2%) | ** (0.1%) | 0.03 | 15 (0.3%) | 13 (0.2%) | 0.02 | ** (0.0%) | ** (0.1%) | #VALUE! | #VALUE! | #VALUE! |
| Use of fondaparinux or Bivalirudin; n (%) | ** (0.3%) | ** (0.3%) | 0.00 | ** (0.2%) | 15 (0.3%) | -0.02 | ** (0.1%) | ** (0.1%) | #VALUE! | #VALUE! | #VALUE! |
| Use of other direct thrombin inhibitors (lepirudin, des | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Use of Ticagrelor ON CED; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | ** (0.0%) | #DIV/0! | 0 (0.0%) | ** (0.0%) | 0 (0.0%) | #VALUE! | #VALUE! |
| Use of Ticagrelor; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | ** (0.0%) | ** (0.0%) | #DIV/0! | ** (0.1%) | ** (0.1%) | #VALUE! | #VALUE! | #VALUE! |
| Number of D-dimer tests | , | , | | , | , | | ( / | | | | |
| mean (sd) | 0.13 (0.36) | 0.11 (0.36) | 0.06 | 0.14 (0.39) | 0.13 (0.38) | 0.03 | 0.13 (0.37) | 0.13 (0.36) | 0.13 (0.38) | 0.13 (0.37) | 0.00 |
| | 0.13 (0.30) | 0.11 (0.30) | 0.00 | 0.14 (0.33) | 0.13 (0.38) | 0.03 | 0.13 (0.37) | 0.13 (0.30) | 0.13 (0.38) | 0.13 (0.37) | 0.00 |
| Numbe of CRP, high-sensitivity CRP tests | | | | | | | | | | | |
| mean (sd) | 0.12 (0.49) | 0.11 (0.48) | 0.02 | 0.08 (0.46) | 0.08 (0.41) | 0.00 | 0.14 (0.55) | 0.14 (0.59) | 0.12 (0.51) | 0.11 (0.52) | 0.00 |
| Number of PT or aPTTt tests | | | | | | | | | | | |
| mean (sd) | 0.66 (1.64) | 0.64 (1.64) | 0.01 | 0.53 (1.27) | 0.50 (1.36) | 0.02 | 0.35 (0.78) | 0.35 (0.84) | 0.46 (1.12) | 0.44 (1.18) | 0.00 |
| Number of Bleeding time tests | | | | | | | | | | | |
| mean (sd) | 0.00 (0.00) | 0.00 (0.00) | #DIV/0! | 0.00 (0.00) | 0.00 (0.01) | 0.00 | 0.00 (0.03) | 0.00 (0.02) | 0.00 (0.02) | 0.00 (0.02) | 0.00 |
| HAS-BLED Score (ICD-9 and ICD-10), 180 days | 0.00 (0.00) | 0.00 (0.00) | 1151170. | 0.00 (0.00) | 0.00 (0.01) | 0.00 | 0.00 (0.03) | 0.00 (0.02) | 0.00 (0.02) | 0.00 (0.02) | 0.00 |
| | | | | / \ | | | | | / \ | / 1 | |
| mean (sd) | 2.77 (1.05) | 2.78 (1.01) | -0.01 | 2.25 (0.99) | 2.26 (0.96) | -0.01 | 3.45 (0.80) | 3.46 (0.79) | 2.93 (0.91) | 2.94 (0.89) | 0.00 |
| N of Generic name drugs | | | | | | | | | | | |
| mean (sd) | 15.55 (13.45) | 15.82 (15.34) | -0.02 | 12.64 (11.01) | 12.67 (12.69) | 0.00 | 17.54 (13.04) | 18.06 (15.69) | 15.52 (12.41) | 15.83 (14.64) | 0.00 |
| N of Brand name drugs | | | | | | | | | | | |
| mean (sd) | 3.36 (5.57) | 3.32 (3.34) | 0.01 | 3.47 (5.19) | 3.52 (3.38) | -0.01 | 3.69 (5.67) | 3.68 (3.75) | 3.57 (5.49) | 3.57 (3.57) | 0.00 |
| Use of clopidogrel ; n (%) | 55 (2.6%) | 65 (3.0%) | -0.02 | 101 (1.8%) | 97 (1.7%) | 0.01 | 398 (4.9%) | 418 (5.2%) | 554 (3.5%) | 580 (3.6%) | -0.01 |
| Systemic embolism; n (%) | 52 (2.4%) | 45 (2.1%) | 0.02 | 90 (1.6%) | 103 (1.8%) | -0.02 | 125 (1.5%) | 109 (1.4%) | 267 (1.7%) | 257 (1.6%) | 0.01 |
| DVT; n (%) | 1,045 (48.5%) | 1,024 (47.6%) | 0.02 | 2,760 (48.6%) | 2,714 (47.8%) | 0.02 | 3,571 (44.3%) | 3,541 (43.9%) | 7376 (46.4%) | 7279 (45.8%) | 0.01 |
| Post-thrombotic syndrome; n (%) | ** (0.1%) | ** (0.1%) | #DIV/0! | ** (0.1%) | ** (0.1%) | #DIV/0! | ** (0.1%) | ** (0.0%) | ** (0.1%) | ** (0.1%) | 0.00 |
| PE; n (%) | 2,153 (100.0%) | 2,153 (100.0%) | #DIV/0! | 5,673 (100.0%) | 5,670 (99.9%) | 0.04 | 8,060 (99.9%) | 8,061 (100.0%) | 15886 (100.0%) | 15884 (99.9%) | 0.04 |
| Coagulation defects; n (%) | 61 (2.8%) | 57 (2.6%) | #DIV/0! | 136 (2.4%) | 147 (2.6%) | #DIV/0! | 130 (1.6%) | 129 (1.6%) | 136 (2.4%) | 147 (2.6%) | -0.01 |
| * ' ' ' | | | | | | | | | | | |
| Diabetes: 1 inpatient or 2 outpatient claims within 18 | 462 (21.5%) | 486 (22.6%) | -0.03 | 879 (15.5%) | 890 (15.7%) | -0.01 | 1,976 (24.5%) | 2,034 (25.2%) | 3317 (20.9%) | 3410 (21.5%) | -0.01 |
| process of the contract of the | , , , | , | | , | | | , , | ,, | , , , , | | |
| | | **(0.0%) | #DIV/0! | ** (0.1%) | ** (0.0%) | 0.04 | ** (0.1%) | ** (0.1%) | #VALUE! | #VALUE! | #VALUE! |
| Internacial as established by bounded to a section | | | | | ··· (U.U%) | | | 2,786 (34.5%) | | | #VALUE!<br>0.00 |
| Intracranial or retroperitoneal hemorrhage: 1 inpatier | **(0.0%) | | | | | | | | | | |
| Peptic Ulcer Disease; n (%) | 639 (29.7%) | 621 (28.8%) | 0.02 | 1,051 (18.5%) | 1,072 (18.9%) | -0.01 | 2,798 (34.7%) | | 4488 (28.2%) | 4479 (28.2%) | |
| Peptic Ulcer Disease; n (%)<br>Major Surgery ; n (%) | 639 (29.7%)<br>181 (8.4%) | 621 (28.8%)<br>166 (7.7%) | 0.02<br>#DIV/0! | 1,051 (18.5%)<br>319 (5.6%) | 326 (5.7%) | #DIV/0! | 810 (10.0%) | 775 (9.6%) | 319 (5.6%) | 326 (5.7%) | 0.00 |
| Peptic Ulcer Disease; n (%) | 639 (29.7%) | 621 (28.8%) | 0.02 | 1,051 (18.5%) | | | | | | | |
| Peptic Ulcer Disease; n (%)<br>Major Surgery ; n (%) | 639 (29.7%)<br>181 (8.4%) | 621 (28.8%)<br>166 (7.7%) | 0.02<br>#DIV/0! | 1,051 (18.5%)<br>319 (5.6%) | 326 (5.7%) | #DIV/0! | 810 (10.0%) | 775 (9.6%) | 319 (5.6%) | 326 (5.7%) | 0.00 |
| Peptic Ulcer Disease; n (%)<br>Major Surgery ; n (%)<br>Upper Gi bleed; n (%)<br>Lower/ unspecified Gi bleed; n (%) | 639 (29.7%)<br>181 (8.4%)<br>0 (0.0%)<br>0 (0.0%) | 621 (28.8%)<br>166 (7.7%)<br>0 (0.0%) | 0.02<br>#DIV/0!<br>#DIV/0! | 1,051 (18.5%)<br>319 (5.6%)<br>0 (0.0%) | 326 (5.7%)<br>0 (0.0%) | #DIV/0!<br>#DIV/0! | 810 (10.0%)<br>0 (0.0%)<br>0 (0.0%) | 775 (9.6%)<br>0 (0.0%) | 319 (5.6%)<br>0 (0.0%) | 326 (5.7%)<br>0 (0.0%)<br>0 (0.0%) | 0.00<br>#DIV/0! |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gl bleed; n (%) Lower/ unspecified Gl bleed; n (%) Urogenital bleed; n (%) | 639 (29.7%)<br>181 (8.4%)<br>0 (0.0%)<br>0 (0.0%)<br>15 (0.7%) | 621 (28.8%)<br>166 (7.7%)<br>0 (0.0%)<br>0 (0.0%)<br>13 (0.6%) | 0.02<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>0.01 | 1,051 (18.5%)<br>319 (5.6%)<br>0 (0.0%)<br>0 (0.0%)<br>50 (0.9%) | 326 (5.7%)<br>0 (0.0%)<br>0 (0.0%)<br>48 (0.8%) | #DIV/0!<br>#DIV/0!<br>#DIV/0!<br>0.01 | 810 (10.0%)<br>0 (0.0%)<br>0 (0.0%)<br>** (0.0%) | 775 (9.6%)<br>0 (0.0%)<br>0 (0.0%)<br>0 (0.0%) | 319 (5.6%)<br>0 (0.0%)<br>0 (0.0%)<br>#VALUE! | 326 (5.7%)<br>0 (0.0%)<br>0 (0.0%)<br>61 (0.4%) | 0.00<br>#DIV/0!<br>#DIV/0!<br>#VALUE! |
| Peptic Ulcer Disease; n (%) Major Surgery ; n (%) Upper Gl bleed; n (%) Lower/ unspecified Gl bleed; n (%) Urogenital bleed; n (%) Other bleed; n (%) | 639 (29.7%)<br>181 (8.4%)<br>0 (0.0%)<br>0 (0.0%)<br>15 (0.7%)<br>113 (5.2%) | 621 (28.8%)<br>166 (7.7%)<br>0 (0.0%)<br>0 (0.0%)<br>13 (0.6%)<br>100 (4.6%) | 0.02<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>0.01<br>0.03 | 1,051 (18.5%)<br>319 (5.6%)<br>0 (0.0%)<br>0 (0.0%)<br>50 (0.9%)<br>201 (3.5%) | 326 (5.7%)<br>0 (0.0%)<br>0 (0.0%)<br>48 (0.8%)<br>201 (3.5%) | #DIV/0!<br>#DIV/0!<br>#DIV/0!<br>0.01<br>0.00 | 810 (10.0%)<br>0 (0.0%)<br>0 (0.0%)<br>** (0.0%)<br>393 (4.9%) | 775 (9.6%)<br>0 (0.0%)<br>0 (0.0%)<br>0 (0.0%)<br>390 (4.8%) | 319 (5.6%)<br>0 (0.0%)<br>0 (0.0%)<br>#VALUE!<br>707 (4.4%) | 326 (5.7%)<br>0 (0.0%)<br>0 (0.0%)<br>61 (0.4%)<br>691 (4.3%) | 0.00<br>#DIV/0!<br>#DIV/0!<br>#VALUE!<br>0.00 |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gl bled; n (%) Lower/unspecified Gl bleed; n (%) Urogenital bleed; n (%) Urogenital bleed; n (%) Prior cancer; n (%) | 639 (29.7%)<br>181 (8.4%)<br>0 (0.0%)<br>0 (0.0%)<br>15 (0.7%)<br>113 (5.2%)<br>353 (16.4%) | 621 (28.8%)<br>166 (7.7%)<br>0 (0.0%)<br>0 (0.0%)<br>13 (0.6%)<br>100 (4.6%)<br>337 (15.7%) | 0.02<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>0.01<br>0.03<br>0.02 | 1,051 (18.5%)<br>319 (5.6%)<br>0 (0.0%)<br>0 (0.0%)<br>50 (0.9%)<br>201 (3.5%)<br>593 (10.4%) | 326 (5.7%)<br>0 (0.0%)<br>0 (0.0%)<br>48 (0.8%)<br>201 (3.5%)<br>565 (10.0%) | #DIV/0!<br>#DIV/0!<br>#DIV/0!<br>0.01<br>0.00<br>0.01 | 810 (10.0%)<br>0 (0.0%)<br>0 (0.0%)<br>** (0.0%)<br>393 (4.9%)<br>1,581 (19.6%) | 775 (9.6%)<br>0 (0.0%)<br>0 (0.0%)<br>0 (0.0%)<br>390 (4.8%)<br>1,430 (17.7%) | 319 (5.6%)<br>0 (0.0%)<br>0 (0.0%)<br>#VALUE!<br>707 (4.4%)<br>2527 (15.9%) | 326 (5.7%)<br>0 (0.0%)<br>0 (0.0%)<br>61 (0.4%)<br>691 (4.3%)<br>2332 (14.7%) | 0.00<br>#DIV/0!<br>#DIV/0!<br>#VALUE!<br>0.00<br>0.03 |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gl bleed; n (%) Lower/unspecified Gl bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Antibiotics; n (%) | 639 (29.7%)<br>181 (8.4%)<br>0 (0.0%)<br>0 (0.0%)<br>15 (0.7%)<br>113 (5.2%)<br>353 (16.4%)<br>1,052 (48.9%) | 621 (28.8%) 166 (7.7%) 0 (0.0%) 0 (0.0%) 13 (0.6%) 100 (4.6%) 337 (15.7%) 1,088 (50.5%) | 0.02<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>0.01<br>0.03<br>0.02<br>#DIV/0! | 1,051 (18.5%)<br>319 (5.6%)<br>0 (0.0%)<br>0 (0.0%)<br>50 (0.9%)<br>201 (3.5%)<br>593 (10.4%)<br>2,823 (49.7%) | 326 (5.7%)<br>0 (0.0%)<br>0 (0.0%)<br>48 (0.8%)<br>201 (3.5%)<br>565 (10.0%)<br>2,803 (49.4%) | #DIV/0!<br>#DIV/0!<br>#DIV/0!<br>0.01<br>0.00<br>0.01<br>#DIV/0! | 810 (10.0%)<br>0 (0.0%)<br>0 (0.0%)<br>** (0.0%)<br>393 (4.9%)<br>1,581 (19.6%)<br>4,541 (56.3%) | 775 (9.6%)<br>0 (0.0%)<br>0 (0.0%)<br>0 (0.0%)<br>390 (4.8%)<br>1,430 (17.7%)<br>4,569 (56.7%) | 319 (5.6%)<br>0 (0.0%)<br>0 (0.0%)<br>#VALUE!<br>707 (4.4%)<br>2527 (15.9%)<br>2,823 (49.7%) | 326 (5.7%)<br>0 (0.0%)<br>0 (0.0%)<br>61 (0.4%)<br>691 (4.3%)<br>2332 (14.7%)<br>2,803 (49.4%) | 0.00<br>#DIV/0!<br>#DIV/0!<br>#VALUE!<br>0.00<br>0.03<br>0.01 |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gl bleed; n (%) Lower/ unspecified Gl bleed; n (%) Urogenital bleed; n (%) Other bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin, n (%) | 639 (29.7%)<br>181 (8.4%)<br>0 (0.0%)<br>0 (0.0%)<br>15 (0.7%)<br>113 (5.2%)<br>353 (16.4%)<br>1,052 (48.9%)<br>15 (0.7%) | 621 (28.8%) 166 (7.7%) 0 (0.0%) 0 (0.0%) 13 (0.6%) 100 (4.6%) 337 (15.7%) 1,088 (50.5%) 13 (0.6%) | 0.02<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>0.01<br>0.03<br>0.02<br>#DIV/0! | 1,051 (18.5%)<br>319 (5.6%)<br>0 (0.0%)<br>0 (0.0%)<br>50 (0.9%)<br>201 (3.5%)<br>593 (10.4%)<br>2,823 (49.7%)<br>74 (1.3%) | 326 (5.7%)<br>0 (0.0%)<br>0 (0.0%)<br>48 (0.8%)<br>201 (3.5%)<br>565 (10.0%)<br>2,803 (49.4%)<br>77 (1.4%) | #DIV/0!<br>#DIV/0!<br>#DIV/0!<br>0.01<br>0.00<br>0.01<br>#DIV/0!<br>-0.01 | 810 (10.0%)<br>0 (0.0%)<br>0 (0.0%)<br>** (0.0%)<br>393 (4.9%)<br>1,581 (19.6%)<br>4,541 (56.3%)<br>28 (0.3%) | 775 (9.6%)<br>0 (0.0%)<br>0 (0.0%)<br>0 (0.0%)<br>390 (4.8%)<br>1,430 (17.7%)<br>4,569 (56.7%)<br>34 (0.4%) | 319 (5.6%)<br>0 (0.0%)<br>0 (0.0%)<br>#VALUEI<br>707 (4.4%)<br>2527 (15.9%)<br>2,823 (49.7%)<br>117 (0.7%) | 326 (5.7%)<br>0 (0.0%)<br>0 (0.0%)<br>61 (0.4%)<br>691 (4.3%)<br>2332 (14.7%)<br>2,803 (49.4%)<br>124 (0.8%) | 0.00<br>#DIV/0!<br>#DIV/0!<br>#VALUE!<br>0.00<br>0.03<br>0.01 |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gl bleed; n (%) Lower/unspecified Gl bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Antibiotics; n (%) | 639 (29.7%) 181 (8.4%) 0 (0.0%) 0 (0.0%) 15 (0.7%) 113 (5.2%) 353 (16.4%) 1,052 (48.9%) 15 (0.7%) ** (0.1%) | 621 (28.8%) 166 (7.7%) 0 (0.0%) 0 (0.0%) 13 (0.6%) 100 (4.6%) 337 (15.7%) 1,088 (50.5%) 13 (0.6%) | 0.02<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>0.01<br>0.03<br>0.02<br>#DIV/0!<br>0.01 | 1,051 (18.5%)<br>319 (5.6%)<br>0 (0.0%)<br>0 (0.0%)<br>50 (0.9%)<br>201 (3.5%)<br>593 (10.4%)<br>2,823 (49.7%)<br>74 (1.3%)<br>** (0.1%) | 326 (5.7%)<br>0 (0.0%)<br>0 (0.0%)<br>48 (0.8%)<br>201 (3.5%)<br>565 (10.0%)<br>2,803 (49.4%)<br>77 (1.4%) | #DIV/0!<br>#DIV/0!<br>#DIV/0!<br>0.01<br>0.00<br>0.01<br>#DIV/0! | 810 (10.0%) 0 (0.0%) 0 (0.0%) ** (0.0%) ** (0.0%) 393 (4.9%) 1,581 (19.6%) 4,541 (56.3%) 28 (0.3%) 20 (0.2%) | 775 (9.6%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 390 (4.8%) 1,430 (17.7%) 4,569 (56.7%) 34 (0.4%) 24 (0.3%) | 319 (5.6%) 0 (0.0%) 0 (0.0%) 4 (0.0%) #VALUE! 707 (4.4%) 2527 (15.9%) 2,823 (49.7%) 117 (0.7%) #VALUE! | 326 (5.7%)<br>0 (0.0%)<br>0 (0.0%)<br>61 (0.4%)<br>691 (4.3%)<br>2332 (14.7%)<br>2,803 (49.4%)<br>124 (0.8%)<br>#VALUE! | 0.00<br>#DIV/0!<br>#DIV/0!<br>#VALUE!<br>0.00<br>0.03<br>0.01<br>-0.01<br>#VALUE! |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gl bleed; n (%) Lower/ unspecified Gl bleed; n (%) Urogenital bleed; n (%) Other bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin, n (%) | 639 (29.7%)<br>181 (8.4%)<br>0 (0.0%)<br>0 (0.0%)<br>15 (0.7%)<br>113 (5.2%)<br>353 (16.4%)<br>1,052 (48.9%)<br>15 (0.7%) | 621 (28.8%) 166 (7.7%) 0 (0.0%) 0 (0.0%) 13 (0.6%) 100 (4.6%) 337 (15.7%) 1,088 (50.5%) 13 (0.6%) | 0.02<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>0.01<br>0.03<br>0.02<br>#DIV/0! | 1,051 (18.5%)<br>319 (5.6%)<br>0 (0.0%)<br>0 (0.0%)<br>50 (0.9%)<br>201 (3.5%)<br>593 (10.4%)<br>2,823 (49.7%)<br>74 (1.3%) | 326 (5.7%)<br>0 (0.0%)<br>0 (0.0%)<br>48 (0.8%)<br>201 (3.5%)<br>565 (10.0%)<br>2,803 (49.4%)<br>77 (1.4%) | #DIV/0!<br>#DIV/0!<br>#DIV/0!<br>0.01<br>0.00<br>0.01<br>#DIV/0!<br>-0.01 | 810 (10.0%)<br>0 (0.0%)<br>0 (0.0%)<br>** (0.0%)<br>393 (4.9%)<br>1,581 (19.6%)<br>4,541 (56.3%)<br>28 (0.3%) | 775 (9.6%)<br>0 (0.0%)<br>0 (0.0%)<br>0 (0.0%)<br>390 (4.8%)<br>1,430 (17.7%)<br>4,569 (56.7%)<br>34 (0.4%) | 319 (5.6%)<br>0 (0.0%)<br>0 (0.0%)<br>#VALUEI<br>707 (4.4%)<br>2527 (15.9%)<br>2,823 (49.7%)<br>117 (0.7%) | 326 (5.7%)<br>0 (0.0%)<br>0 (0.0%)<br>61 (0.4%)<br>691 (4.3%)<br>2332 (14.7%)<br>2,803 (49.4%)<br>124 (0.8%) | 0.00<br>#DIV/0!<br>#DIV/0!<br>#VALUE!<br>0.00<br>0.03<br>0.01 |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gl bleed; n (%) Lower/unspecified Gl bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) | 639 (29.7%) 181 (8.4%) 0 (0.0%) 0 (0.0%) 15 (0.7%) 113 (5.2%) 353 (16.4%) 1,052 (48.9%) 15 (0.7%) ** (0.1%) | 621 (28.8%) 166 (7.7%) 0 (0.0%) 0 (0.0%) 13 (0.6%) 100 (4.6%) 337 (15.7%) 1,088 (50.5%) 13 (0.6%) | 0.02<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>0.01<br>0.03<br>0.02<br>#DIV/0!<br>0.01 | 1,051 (18.5%)<br>319 (5.6%)<br>0 (0.0%)<br>0 (0.0%)<br>50 (0.9%)<br>201 (3.5%)<br>593 (10.4%)<br>2,823 (49.7%)<br>74 (1.3%)<br>** (0.1%) | 326 (5.7%)<br>0 (0.0%)<br>0 (0.0%)<br>48 (0.8%)<br>201 (3.5%)<br>565 (10.0%)<br>2,803 (49.4%)<br>77 (1.4%) | #DIV/0!<br>#DIV/0!<br>#DIV/0!<br>0.01<br>0.00<br>0.01<br>#DIV/0!<br>-0.01<br>0.00 | 810 (10.0%) 0 (0.0%) 0 (0.0%) ** (0.0%) ** (0.0%) 393 (4.9%) 1,581 (19.6%) 4,541 (56.3%) 28 (0.3%) 20 (0.2%) | 775 (9.6%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 390 (4.8%) 1,430 (17.7%) 4,569 (56.7%) 34 (0.4%) 24 (0.3%) | 319 (5.6%)<br>0 (0.0%)<br>0 (0.0%)<br>#VALUE!<br>707 (4.4%)<br>2527 (15.9%)<br>2,823 (49.7%)<br>117 (0.7%)<br>#VALUE! | 326 (5.7%)<br>0 (0.0%)<br>0 (0.0%)<br>61 (0.4%)<br>691 (4.3%)<br>2332 (14.7%)<br>2,803 (49.4%)<br>124 (0.8%)<br>#VALUE! | 0.00<br>#DIV/0!<br>#DIV/0!<br>#VALUE!<br>0.00<br>0.03<br>0.01<br>-0.01<br>#VALUE! |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gl bleed; n (%) Lower/ unspecified Gl bleed; n (%) Urogenital bleed; n (%) Other bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) | 639 (29.7%) 181 (8.4%) 0 (0.0%) 0 (0.0%) 15 (0.7%) 113 (5.2%) 353 (16.4%) 1,052 (48.9%) 15 (0.7%) ** (0.1%) ** (0.2%) 484 (22.5%) | 621 (28.8%) 166 (7.7%) 0 (0.0%) 0 (0.0%) 13 (0.6%) 100 (4.6%) 337 (15.7%) 1,088 (50.5%) ** (0.1%) ** (0.2%) | 0.02<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>0.01<br>0.03<br>0.02<br>#DIV/0!<br>0.01<br>0.00 | 1,051 (18.5%) 319 (5.6%) 0 (0.0%) 0 (0.0%) 50 (0.9%) 201 (3.5%) 593 (10.4%) 2,823 (49.7%) 74 (1.3%) ** (0.1%) | 326 (5.7%)<br>0 (0.0%)<br>0 (0.0%)<br>48 (0.8%)<br>201 (3.5%)<br>565 (10.0%)<br>2,803 (49.4%)<br>77 (1.4%)<br>** (0.1%) | #DIV/0!<br>#DIV/0!<br>#DIV/0!<br>0.01<br>0.00<br>0.01<br>#DIV/0!<br>-0.01<br>0.00 | 810 (10.0%)<br>0 (0.0%)<br>0 (0.0%)<br>** (0.0%)<br>393 (4.9%)<br>1,581 (19.6%)<br>4,541 (56.3%)<br>28 (0.3%)<br>20 (0.2%)<br>29 (0.4%) | 775 (9.6%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 390 (4.8%) 1,430 (17.7%) 4,569 (56.7%) 34 (0.4%) 24 (0.3%) | 319 (5.6%) 0 (0.0%) 0 (0.0%) 4 VALUE! 707 (4.4%) 2527 (15.9%) 2,823 (49.7%) 117 (0.7%) #VALUE! #VALUE! | 326 (5.7%) 0 (0.0%) 0 (0.0%) 61 (0.4%) 691 (4.3%) 2332 (14.7%) 2,803 (49.4%) 124 (0.8%) #VALUE! #VALUE! | 0.00<br>#DIV/0!<br>#DIV/0!<br>#VALUE!<br>0.00<br>0.03<br>0.01<br>-0.01<br>#VALUE! |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gl bleed; n (%) Lower/unspecified Gl bleed; n (%) Urogenital bleed; n (%) Urogenital bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) | 639 (29.7%) 181 (8.4%) 0 (0.0%) 0 (0.0%) 15 (0.7%) 113 (5.2%) 353 (16.4%) 1,052 (48.9%) 15 (0.7%) ** (0.1%) ** (0.2%) | 621 (28.8%) 166 (7.7%) 0 (0.03%) 0 (0.03%) 13 (0.65%) 100 (4.65%) 337 (15.7%) 1,088 (50.5%) 13 (0.65%) ** (0.1%) ** (0.2%) 480 (22.3%) | 0.02<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>0.01<br>0.03<br>0.02<br>#DIV/0!<br>0.01<br>0.00<br>0.00 | 1,051 (18.5%) 319 (5.6%) 0 (0.0%) 0 (0.0%) 50 (0.9%) 201 (3.5%) 593 (10.4%) 2,823 (49.7%) 74 (1.3%) ** (0.1%) 1,254 (22.1%) | 326 (5.7%)<br>0 (0.0%)<br>48 (0.8%)<br>201 (3.5%)<br>565 (10.0%)<br>2,803 (49.4%)<br>77 (1.4%)<br>** (0.1%)<br>1,233 (21.7%) | #DIV/0!<br>#DIV/0!<br>#DIV/0!<br>0.01<br>0.00<br>0.01<br>#DIV/0!<br>-0.01<br>0.00<br>0.00 | 810 (10.0%) 0 (0.0%) 0 (0.0%) ** (0.0%) ** (0.0%) 393 (4.9%) 1,581 (19.6%) 4,541 (56.3%) 28 (0.3%) 20 (0.2%) 29 (0.4%) 2,139 (26.5%) | 775 (9.6%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 390 (4.8%) 1,430 (17.7%) 4,569 (56.7%) 34 (0.4%) 24 (0.3%) 2,148 (26.6%) | 319 (5.6%) 0 (0.0%) 0 (0.0%) 4 (0.0%) 3 (0.0%) 4 (0.0%) 4 (0.0%) 4 (0.0%) 5 | 326 (5.7%)<br>0 (0.0%)<br>0 (0.0%)<br>61 (0.4%)<br>691 (4.3%)<br>2332 (14.7%)<br>2,803 (49.4%)<br>124 (0.8%)<br>#VALUE!<br>3861 (24.3%) | 0.00<br>#DIV/0!<br>#DIV/0!<br>#VALUE!<br>0.00<br>0.03<br>0.01<br>-0.01<br>#VALUE!<br>#VALUE! |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gl bleed; n (%) Lower/unspecified Gl bleed; n (%) Urogenital bleed; n (%) Other bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests ordered | 639 (29.7%) 181 (8.4%) 0 (0.0%) 0 (0.0%) 15 (0.7%) 113 (5.2%) 353 (16.4%) 1,052 (48.9%) 15 (0.7%) ** (0.1%) ** (0.2%) 484 (22.5%) 32 (1.5%) | 621 (28.8%) 166 (7.7%) 0 (0.0%) 0 (0.0%) 13 (0.6%) 130 (4.6%) 337 (15.7%) 1,088 (50.5%) 1 (0.6%) ** (0.1%) 40 (22.3%) 29 (1.3%) | 0.02 #DIV/0! #DIV/0! #DIV/0! 0.01 0.03 0.02 #DIV/0! 0.01 0.00 0.00 0.00 | 1,051 (18.5%) 319 (5.6%) 0 (0.0%) 0 (0.0%) 50 (0.9%) 201 (3.5%) 593 (10.4%) 2,823 (49.7%) 74 (1.3%) ** (0.1%) 1,254 (22.1%) 71 (1.3%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 48 (0.8%) 201 (3.5%) 555 (10.0%) 77 (1.4%) ** (0.1%) ** (0.1%) 1,233 (21.7%) 71 (1.3%) | #DIV/0!<br>#DIV/0!<br>#DIV/0!<br>0.01<br>0.00<br>0.01<br>#DIV/0!<br>-0.01<br>0.00<br>0.00 | 810 (10.0%) 0 (0.0%) 0 (0.0%) ** (0.0%) 393 (4.9%) 1,581 (19.6%) 4,541 (56.3%) 28 (0.3%) 20 (0.2%) 29 (0.4%) 2,139 (26.5%) 148 (1.8%) | 775 (9.6%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 390 (4.8%) 1,430 (17.7%) 4,569 (56.7%) 34 (0.4%) 24 (0.3%) 28 (0.3%) 2,148 (26.6%) 162 (2.0%) | 319 (5.6%) 0 (0.0%) 0 (0.0%) 10 (0.0%) #VALUE! 707 (4.4%) 2527 (15.9%) 2,823 (49.7%) 117 (0.7%) #VALUE! #VALUE! 3877 (24.4%) 251 (1.6%) | 326 (5.7%)<br>0 (0.0%)<br>0 (0.0%)<br>61 (0.4%)<br>691 (4.3%)<br>2332 (14.7%)<br>2,803 (49.4%)<br>124 (0.8%)<br>#VALUE!<br>3861 (24.3%)<br>262 (1.6%) | #DIV/0!<br>#DIV/0!<br>#DIV/0!<br>#VALUE!<br>0.00<br>0.03<br>0.01<br>-0.01<br>#VALUE!<br>#VALUE!<br>0.00 |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Lower/unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (cd) | 639 (29.7%) 181 (8.4%) 0 (0.0%) 0 (0.0%) 15 (0.7%) 113 (5.2%) 353 (16.4%) 1,052 (48.9%) 15 (0.7%) ** (0.1%) ** (0.2%) 484 (22.5%) 32 (1.5%) | 621 (28.8%) 166 (7.7%) 0 (0.0%) 0 (0.0%) 13 (0.6%) 100 (4.6%) 337 (15.7%) 1,088 (50.5%) 13 (0.6%) ** (0.1%) ** (0.2%) 480 (22.3%) 29 (1.3%) 0.50 (1.17) | 0.02 #DIV/01 #DIV/01 #DIV/01 0.01 0.03 0.02 #DIV/01 0.01 0.00 0.00 0.00 0.00 0.00 | 1,051 (18.5%) 319 (5.6%) 0 (0.0%) 0 (0.0%) 50 (0.9%) 201 (3.5%) 593 (10.4%) 2,823 (49.7%) 74 (1.3%) ** (0.1%) \$ (0.1%) 1,254 (22.1%) 71 (1.3%) 0.35 (0.72) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 48 (0.8%) 201 (3.5%) 555 (10.0%) 7 (1.4%) ** (0.1%) 1,233 (21.7%) 71 (1.3%) 0.35 (0.70) | #DIV/0!<br>#DIV/0!<br>#DIV/0!<br>0.01<br>0.00<br>0.01<br>#DIV/0!<br>-0.01<br>0.00<br>0.00 | 810 (10.0%) 0 (0.0%) 0 (0.0%) ** (0.0%) ** (0.0%) 393 (4.9%) 1,581 (19.6%) 4,541 (56.3%) 28 (0.3%) 20 (0.2%) 29 (0.4%) 2,139 (26.5%) 148 (1.8%) 0.58 (0.79) | 775 (9.6%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 390 (4.8%) 1,430 (17.7%) 4,569 (56.7%) 34 (0.4%) 24 (0.3%) 28 (0.3%) 2,148 (26.6%) 162 (2.0%) | 319 (5.6%)<br>0 (0.0%)<br>0 (0.0%)<br>0 (0.0%)<br>#VALUE!<br>707 (4.4%)<br>2527 (15.9%)<br>2,823 (49.7%)<br>117 (0.7%)<br>#VALUE!<br>#VALUE!<br>3877 (24.4%)<br>251 (1.6%)<br>0.48 (0.76) | 326 (5.7%)<br>0 (0.0%)<br>0 (0.0%)<br>61 (0.4%)<br>691 (4.3%)<br>2332 (14.7%)<br>2,803 (49.4%)<br>124 (0.8%)<br>#VALUE!<br>#VALUE!<br>#VALUE!<br>\$65 (24.3%)<br>262 (1.6%) | 0.00 #DIV/01 #DIV/01 #VALUEI 0.00 0.03 0.01 -0.01 #VALUEI #VALUEI 0.00 0.00 |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gl bleed; n (%) Lower/unspecified Gl bleed; n (%) Urogenital bleed; n (%) Other bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin, n (%) Aspirin, n (%) Aspirin, n (%) Aspirin, blibiotics; n (%) Other antiplatelet agents; n (%) Other antiplatelet agents; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) | 639 (29.7%) 181 (8.4%) 0 (0.0%) 0 (0.0%) 15 (0.7%) 113 (5.2%) 353 (16.4%) 1,052 (48.9%) 15 (0.7%) 18 (0.2%) 484 (22.5%) 32 (1.5%) 0.47 (0.72) 528 (24.5%) | 621 (28.8%) 166 (7.7%) 0 (0.0%) 0 (0.0%) 13 (0.6%) 100 (4.6%) 337 (15.7%) 1,088 (50.5%) 13 (0.6%) ** (0.1%) ** (0.2%) 480 (22.3%) 29 (1.3%) 0.50 (1.17) 528 (24.5%) | 0.02 #DIV/01 #DIV/01 #DIV/01 0.01 0.03 0.02 #DIV/01 0.01 0.00 0.00 0.00 0.02 | 1,051 (18.5%) 319 (5.6%) 0 (0.0%) 0 (0.0%) 50 (0.9%) 201 (3.5%) 593 (10.4%) 2,823 (49.7%) 74 (1.3%) ** (0.1%) ** (0.1%) 1,254 (22.1%) 71 (1.3%) 0.35 (0.72) 1,233 (21.7%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 48 (0.8%) 201 (3.5%) 565 (10.0%) 2,803 (49.4%) 77 (1.4%) ** (0.1%) 1,233 (21.7%) 71 (1.3%) 0.35 (0.70) 1,226 (21.6%) | #DIV/0! #DIV/0! #DIV/0! #DIV/0! 0.01 0.00 0.01 #DIV/0! 0.00 0.01 #DIV/0! 0.00 0.00 0.00 0.00 0.00 0.00 0.00 0 | 810 (10.0%) 0 (0.0%) 0 (0.0%) ** (0.0%) 393 (4.9%) 1,581 (19.6%) 4,541 (56.3%) 28 (0.3%) 20 (0.2%) 29 (0.4%) 2,139 (26.5%) 148 (1.8%) 0.58 (0.79) 2,637 (32.7%) | 775 (9.6%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 390 (4.8%) 1,430 (17.7%) 4,569 (56.7%) 34 (0.4%) 28 (0.3%) 2,148 (26.6%) 162 (2.0%) 0.58 (0.83) 2,717 (33.7%) | 319 (5.6%) 0 (0.0%) 0 (0.0%) 10 (0.0%) #VALUE! 707 (4.4%) 2527 (15.9%) 2,823 (49.7%) 117 (0.7%) #VALUE! #VALUE! 3877 (24.4%) 251 (1.6%) 0.48 (0.75) 4398 (27.7%) | 326 (5.7%)<br>0 (0.0%)<br>0 (0.0%)<br>61 (0.4%)<br>691 (4.3%)<br>2332 (14.7%)<br>2,803 (49.4%)<br>124 (0.8%)<br>#VALUE!<br>#VALUE!<br>3861 (24.3%)<br>262 (1.6%)<br>0.49 (0.84)<br>4471 (28.1%) | 0.00 #DIV/0! #DIV/0! #VALUE! 0.00 0.03 0.01 -0.01 #VALUE! #VALUE! 0.00 0.00 -0.00 |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gl bleed; n (%) Lower/unspecified Gl bleed; n (%) Urogenital bleed; n (%) Other bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiblatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) | 639 (29.7%) 181 (8.4%) 0 (0.0%) 0 (0.0%) 15 (0.7%) 113 (5.2%) 353 (16.4%) 1,052 (48.9%) 15 (0.7%) ** (0.1%) ** (0.2%) 484 (22.5%) 32 (1.5%) 0.47 (0.72) 528 (24.5%) 75 (3.5%) | 621 (28.8%) 166 (7.7%) 0 (0.05%) 0 (0.05%) 13 (0.65%) 130 (4.65%) 337 (15.7%) 1,088 (50.5%) 13 (0.6%) ** (0.1%) ** (0.2%) 480 (22.3%) 29 (1.3%) 0.50 (1.17) 528 (24.5%) 89 (4.15%) | 0.02 #DIV/01 #DIV/01 #DIV/01 0.01 0.03 0.02 #DIV/01 0.01 0.00 0.00 0.00 0.00 0.00 0.00 0 | 1,051 (18.5%) 319 (5.6%) 0 (0.0%) 0 (0.0%) 50 (0.9%) 201 (3.5%) 593 (10.4%) 2,823 (49.7%) 74 (1.3%) ** (0.1%) 1,254 (22.1%) 71 (1.3%) 0.35 (0.72) 1,233 (21.7%) 186 (3.3%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 48 (0.8%) 201 (3.5%) 555 (10.0%) 2,803 (49.4%) 77 (1.4%) ** (0.1%) ** (0.1%) 71 (1.3%) 0.35 (0.70) 1,226 (21.6%) 199 (3.5%) | #DIV/0! #DIV/0! #DIV/0! 0.01 0.00 0.01 #DIV/0! -0.01 0.00 0.00 0.00 0.00 0.00 0.00 0.0 | 810 (10.0%) 0 (0.0%) 0 (0.0%) ** (0.0%) 393 (4.9%) 1,581 (19.6%) 4,541 (56.3%) 28 (0.3%) 20 (0.2%) 29 (0.4%) 2,139 (26.5%) 148 (1.8%) 0.58 (0.79) 2,637 (32.7%) 506 (6.3%) | 775 (9.6%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 390 (4.8%) 1,430 (17.7%) 4,569 (56.7%) 34 (0.4%) 24 (0.3%) 28 (0.3%) 2,148 (26.6%) 162 (2.0%) 0.58 (0.83) 2,717 (33.7%) 511 (6.3%) | 319 (5.6%) 0 (0.0%) 0 (0.0%) 10 (0.0%) #VALUE! 707 (4.4%) 2527 (15.9%) 2,823 (49.7%) 117 (0.7%) #VALUE! #VALUE! 3877 (24.4%) 251 (1.6%) 0.48 (0.76) 4398 (27.7%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 61 (0.4%) 691 (4.3%) 593 (14.7%) 2,803 (49.4%) 124 (0.8%) #VALUE! #VALUE! 3861 (24.3%) 262 (1.6%) 0.49 (0.84) 4471 (28.1%) 799 (5.0%) | 0.00 #DIV/01 #DIV/01 #VALUE! 0.00 0.03 0.01 -0.01 *VALUE! #VALUE! 0.00 0.00 -0.00 |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Lower/unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) Other antiplatelet agents; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) Hz receptor antagonist; n (%) Vitamin K therapy; n (%) | 639 (29.7%) 181 (8.4%) 0 (0.0%) 0 (0.0%) 15 (0.7%) 113 (5.2%) 353 (16.4%) 1,052 (48.9%) 15 (0.7%) 18 (0.2%) 484 (22.5%) 32 (1.5%) 0.47 (0.72) 528 (24.5%) | 621 (28.8%) 166 (7.7%) 0 (0.0%) 0 (0.0%) 13 (0.6%) 100 (4.6%) 337 (15.7%) 1,088 (50.5%) 13 (0.6%) ** (0.1%) ** (0.2%) 480 (22.3%) 29 (1.3%) 0.50 (1.17) 528 (24.5%) | 0.02 #DIV/01 #DIV/01 #DIV/01 0.01 0.03 0.02 #DIV/01 0.01 0.00 0.00 0.00 0.02 | 1,051 (18.5%) 319 (5.6%) 0 (0.0%) 0 (0.0%) 50 (0.9%) 201 (3.5%) 593 (10.4%) 2,823 (49.7%) 74 (1.3%) ** (0.1%) ** (0.1%) 1,254 (22.1%) 71 (1.3%) 0.35 (0.72) 1,233 (21.7%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 48 (0.8%) 201 (3.5%) 565 (10.0%) 2,803 (49.4%) 77 (1.4%) ** (0.1%) 1,233 (21.7%) 71 (1.3%) 0.35 (0.70) 1,226 (21.6%) | #DIV/0! #DIV/0! #DIV/0! #DIV/0! 0.01 0.00 0.01 #DIV/0! 0.00 0.01 #DIV/0! 0.00 0.00 0.00 0.00 0.00 0.00 0.00 0 | 810 (10.0%) 0 (0.0%) 0 (0.0%) ** (0.0%) 393 (4.9%) 1,581 (19.6%) 4,541 (56.3%) 28 (0.3%) 20 (0.2%) 29 (0.4%) 2,139 (26.5%) 148 (1.8%) 0.58 (0.79) 2,637 (32.7%) | 775 (9.6%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 390 (4.8%) 1,430 (17.7%) 4,569 (56.7%) 34 (0.4%) 28 (0.3%) 2,148 (26.6%) 162 (2.0%) 0.58 (0.83) 2,717 (33.7%) | 319 (5.6%) 0 (0.0%) 0 (0.0%) 10 (0.0%) #VALUE! 707 (4.4%) 2527 (15.9%) 2,823 (49.7%) 117 (0.7%) #VALUE! #VALUE! 3877 (24.4%) 251 (1.6%) 0.48 (0.75) 4398 (27.7%) | 326 (5.7%)<br>0 (0.0%)<br>0 (0.0%)<br>61 (0.4%)<br>691 (4.3%)<br>2332 (14.7%)<br>2,803 (49.4%)<br>124 (0.8%)<br>#VALUE!<br>#VALUE!<br>3861 (24.3%)<br>262 (1.6%)<br>0.49 (0.84)<br>4471 (28.1%) | 0.00 #DIV/0! #DIV/0! #VALUE! 0.00 0.03 0.01 -0.01 #VALUE! #VALUE! 0.00 0.00 -0.00 |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gl bleed; n (%) Lower/unspecified Gl bleed; n (%) Urogenital bleed; n (%) Other bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiblatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) | 639 (29.7%) 181 (8.4%) 0 (0.0%) 0 (0.0%) 15 (0.7%) 113 (5.2%) 353 (16.4%) 1,052 (48.9%) 15 (0.7%) ** (0.1%) ** (0.2%) 484 (22.5%) 32 (1.5%) 0.47 (0.72) 528 (24.5%) 75 (3.5%) | 621 (28.8%) 166 (7.7%) 0 (0.05%) 0 (0.05%) 13 (0.65%) 130 (4.65%) 337 (15.7%) 1,088 (50.5%) 13 (0.6%) ** (0.1%) ** (0.2%) 480 (22.3%) 29 (1.3%) 0.50 (1.17) 528 (24.5%) 89 (4.15%) | 0.02 #DIV/01 #DIV/01 #DIV/01 0.01 0.03 0.02 #DIV/01 0.01 0.00 0.00 0.00 0.00 0.00 0.00 0 | 1,051 (18.5%) 319 (5.6%) 0 (0.0%) 0 (0.0%) 50 (0.9%) 201 (3.5%) 593 (10.4%) 2,823 (49.7%) 74 (1.3%) ** (0.1%) 1,254 (22.1%) 71 (1.3%) 0.35 (0.72) 1,233 (21.7%) 186 (3.3%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 48 (0.8%) 201 (3.5%) 555 (10.0%) 2,803 (49.4%) 77 (1.4%) ** (0.1%) ** (0.1%) 71 (1.3%) 0.35 (0.70) 1,226 (21.6%) 199 (3.5%) | #DIV/0! #DIV/0! #DIV/0! 0.01 0.00 0.01 #DIV/0! -0.01 0.00 0.00 0.00 0.00 0.00 0.00 0.0 | 810 (10.0%) 0 (0.0%) 0 (0.0%) ** (0.0%) 393 (4.9%) 1,581 (19.6%) 4,541 (56.3%) 28 (0.3%) 20 (0.2%) 29 (0.4%) 2,139 (26.5%) 148 (1.8%) 0.58 (0.79) 2,637 (32.7%) 506 (6.3%) | 775 (9.6%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 390 (4.8%) 1,430 (17.7%) 4,569 (56.7%) 34 (0.4%) 24 (0.3%) 28 (0.3%) 2,148 (26.6%) 162 (2.0%) 0.58 (0.83) 2,717 (33.7%) 511 (6.3%) | 319 (5.6%) 0 (0.0%) 0 (0.0%) 10 (0.0%) #VALUE! 707 (4.4%) 2527 (15.9%) 2,823 (49.7%) 117 (0.7%) #VALUE! #VALUE! 3877 (24.4%) 251 (1.6%) 0.48 (0.76) 4398 (27.7%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 61 (0.4%) 691 (4.3%) 593 (14.7%) 2,803 (49.4%) 124 (0.8%) #VALUE! #VALUE! 3861 (24.3%) 262 (1.6%) 0.49 (0.84) 4471 (28.1%) 799 (5.0%) | 0.00 #DIV/01 #DIV/01 #VALUE! 0.00 0.03 0.01 -0.01 *VALUE! #VALUE! 0.00 0.00 -0.00 |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Lower/unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) Other antiplatelet agents; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) Hz receptor antagonist; n (%) Vitamin K therapy; n (%) | 639 (29.7%) 181 (8.4%) 0 (0.0%) 0 (0.0%) 15 (0.7%) 113 (5.2%) 353 (16.4%) 1,052 (48.9%) 15 (0.7%) ** (0.1%) ** (0.2%) 484 (22.5%) 32 (1.5%) 0.47 (0.72) 528 (24.5%) 75 (3.5%) | 621 (28.8%) 166 (7.7%) 0 (0.05%) 0 (0.05%) 13 (0.65%) 130 (4.65%) 337 (15.7%) 1,088 (50.5%) 13 (0.6%) ** (0.1%) ** (0.2%) 480 (22.3%) 29 (1.3%) 0.50 (1.17) 528 (24.5%) 89 (4.15%) | 0.02 #DIV/01 #DIV/01 #DIV/01 0.01 0.03 0.02 #DIV/01 0.01 0.00 0.00 0.00 0.00 0.00 0.00 0 | 1,051 (18.5%) 319 (5.6%) 0 (0.0%) 0 (0.0%) 50 (0.9%) 201 (3.5%) 593 (10.4%) 2,823 (49.7%) 74 (1.3%) ** (0.1%) 1,254 (22.1%) 71 (1.3%) 0.35 (0.72) 1,233 (21.7%) 186 (3.3%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 48 (0.8%) 201 (3.5%) 555 (10.0%) 2,803 (49.4%) 77 (1.4%) ** (0.1%) ** (0.1%) 71 (1.3%) 0.35 (0.70) 1,226 (21.6%) 199 (3.5%) | #DIV/0! #DIV/0! #DIV/0! 0.01 0.00 0.01 #DIV/0! -0.01 0.00 0.00 0.00 0.00 0.00 0.00 0.0 | 810 (10.0%) 0 (0.0%) 0 (0.0%) ** (0.0%) 393 (4.9%) 1,581 (19.6%) 4,541 (56.3%) 28 (0.3%) 20 (0.2%) 29 (0.4%) 2,139 (26.5%) 148 (1.8%) 0.58 (0.79) 2,637 (32.7%) 506 (6.3%) | 775 (9.6%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 390 (4.8%) 1,430 (17.7%) 4,569 (56.7%) 34 (0.4%) 24 (0.3%) 28 (0.3%) 2,148 (26.6%) 162 (2.0%) 0.58 (0.83) 2,717 (33.7%) 511 (6.3%) | 319 (5.6%) 0 (0.0%) 0 (0.0%) 10 (0.0%) #VALUE! 707 (4.4%) 2527 (15.9%) 2,823 (49.7%) 117 (0.7%) #VALUE! #VALUE! 3877 (24.4%) 251 (1.6%) 0.48 (0.76) 4398 (27.7%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 61 (0.4%) 691 (4.3%) 593 (14.7%) 2,803 (49.4%) 124 (0.8%) #VALUE! #VALUE! 3861 (24.3%) 262 (1.6%) 0.49 (0.84) 4471 (28.1%) 799 (5.0%) | 0.00 #DIV/01 #DIV/01 #VALUE! 0.00 0.03 0.01 -0.01 *VALUE! #VALUE! 0.00 0.00 -0.00 |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Lower/unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiblatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) Vitamin K therapy; n (%) Number of INR (prothrombin) tests orderedmean (sd) | 639 (29.7%) 181 (8.4%) 0 (0.0%) 0 (0.0%) 15 (0.7%) 113 (5.2%) 353 (16.4%) 1,052 (48.9%) 15 (0.7%) ** (0.1%) ** (0.1%) 484 (22.5%) 32 (1.5%) 0.47 (0.72) 528 (24.5%) 75 (3.5%) 0 (0.0%) | 621 (28.8%) 166 (7.7%) 0 (0.05%) 0 (0.05%) 13 (0.65%) 130 (4.65%) 337 (15.7%) 1,088 (50.5%) 13 (0.65%) ** (0.15%) ** (0.2%) 480 (22.3%) 29 (1.3%) 0.50 (1.17) 528 (24.5%) 89 (4.15%) 0 (0.0%) 0.37 (0.92) | 0.02 #DIV/01 #DIV/01 #DIV/01 0.01 0.03 0.02 #DIV/01 0.00 0.00 0.00 0.02 -0.03 0.00 -0.03 | 1,051 (18.5%) 319 (5.6%) 0 (0.0%) 0 (0.0%) 50 (0.9%) 201 (3.5%) 593 (10.4%) 2,823 (49.7%) 74 (1.3%) ** (0.1%) 1,254 (22.1%) 71 (1.3%) 0.35 (0.72) 1,233 (21.7%) 186 (3.3%) 0 (0.0%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 48 (0.8%) 201 (3.5%) 555 (10.0%) 2,803 (49.4%) 77 (1.4%) ** (0.1%) 1,233 (21.7%) 71 (1.3%) 0.35 (0.70) 1,226 (21.6%) 199 (3.5%) 0 (0.0%) | #DIV/0! #DIV/0! #DIV/0! 0.01 0.00 0.01 #DIV/0! -0.01 0.00 0.00 0.00 0.00 0.00 0.00 0.0 | 810 (10.0%) 0 (0.0%) 0 (0.0%) ** (0.0%) 393 (4.9%) 1,581 (19.6%) 4,541 (56.3%) 28 (0.3%) 20 (0.2%) 29 (0.4%) 2,139 (26.5%) 148 (1.8%) 0.58 (0.79) 2,637 (32.7%) 506 (6.3%) ** (0.0%) | 775 (9.6%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 390 (4.8%) 1,430 (17.7%) 4,569 (56.7%) 34 (0.4%) 24 (0.3%) 28 (0.3%) 2,148 (26.6%) 162 (2.0%) 0.58 (0.83) 2,717 (33.7%) 511 (6.3%) 0 (0.0%) | 319 (5.6%) 0 (0.0%) 0 (0.0%) 10 (0.0%) #VALUE! 707 (4.4%) 2527 (15.9%) 2,823 (49.7%) 117 (0.7%) #VALUE! #VALUE! 3877 (24.4%) 251 (1.6%) 0.48 (0.76) 4398 (27.7%) 767 (4.8%) #VALUE! | 326 (5.7%) 0 (0.0%) 0 (0.0%) 61 (0.4%) 691 (4.3%) 5932 (14.7%) 2,803 (49.4%) 124 (0.8%) #WALUE! #VALUE! 3861 (24.3%) 262 (1.6%) 0.49 (0.84) 4471 (28.1%) 799 (5.0%) 0 (0.0%) | 0.00 #DIV/01 #DIV/01 #VALUEI 0.00 0.03 0.01 -0.01 #VALUEI 0.00 0.00 0.00 -0.01 -0.01 #VALUEI |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Lower/unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of INR (prothrombin) tests orderedmean (sd) | 639 (29.7%) 181 (8.4%) 0 (0.0%) 0 (0.0%) 15 (0.7%) 113 (5.2%) 353 (16.4%) 1,052 (48.9%) 15 (0.7%) ** (0.1%) ** (0.2%) 484 (22.5%) 32 (1.5%) 0.47 (0.72) 528 (24.5%) 75 (3.5%) 0 (0.0%) 0.48 (1.24) 1,407 (65.4%) | 621 (28.8%) 166 (7.7%) 0 (0.0%) 0 (0.0%) 13 (0.65%) 100 (4.6%) 337 (15.7%) 1,088 (50.5%) 13 (0.6%) ** (0.1%) ** (0.2%) 480 (22.3%) 29 (1.3%) 0.50 (1.17) 528 (24.5%) 89 (4.1%) 0 (0.0%) | 0.02 #DIV/01 #DIV/01 #DIV/01 0.01 0.03 0.02 #DIV/01 0.00 0.00 0.00 0.00 0.00 0.00 #DIV/01 0.00 0.00 0.00 0.00 0.00 | 1,051 (18.5%) 319 (5.6%) 0 (0.0%) 50 (0.9%) 50 (0.9%) 201 (3.5%) 593 (10.4%) 2,823 (49.7%) 74 (1.3%) ** (0.1%) 1,254 (22.1%) 71 (1.3%) 0.35 (0.72) 1,233 (21.7%) 186 (3.3%) 0 (0.0%) 0.39 (0.95) 3,348 (59.0%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 48 (0.8%) 201 (3.5%) 555 (10.0%) 2,803 (49.4%) 77 (1.4%) ** (0.1%) 1,233 (21.7%) 71 (1.3%) 0.35 (0.70) 1,226 (21.6%) 199 (3.5%) 0 (0.0%) 0.33 (0.81) 3,290 (58.0%) | #DIV/O! #DIV/O! #DIV/O! #DIV/O! #DIV/O! 0.01 0.00 0.01 #DIV/O! 0.00 0.00 0.00 0.00 0.00 0.00 0.00 0. | 810 (10.0%) 0 (0.0%) 0 (0.0%) ** (0.0%) 393 (4.9%) 1,581 (19.6%) 4,541 (56.3%) 28 (0.3%) 20 (0.2%) 29 (0.4%) 2,139 (26.5%) 148 (1.8%) 0.58 (0.79) 2,637 (32.7%) 506 (6.3%) ** (0.0%) 0.33 (0.72) 5,390 (66.8%) | 775 (9.6%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 390 (4.8%) 1,430 (17.7%) 4,569 (56.7%) 34 (0.4%) 28 (0.3%) 28 (0.3%) 2,148 (26.6%) 162 (2.0%) 0.58 (0.83) 2,717 (33.7%) 511 (6.3%) 0 (0.0%) | 319 (5.6%) 0 (0.0%) 0 (0.0%) 10 (0.0%) #VALUE! 707 (4.4%) 2527 (15.9%) 2,823 (49.7%) 117 (0.7%) #VALUE! #VALUE! 3877 (24.4%) 251 (1.6%) 0.48 (0.76) 4398 (27.7%) 767 (4.8%) #VALUE! 0.37 (0.89) 10145 (63.8%) | 326 (5.7%)<br>0 (0.0%)<br>0 (0.0%)<br>61 (0.4%)<br>691 (4.3%)<br>2332 (14.7%)<br>2,803 (49.4%)<br>124 (0.8%)<br>#VALUE!<br>#VALUE!<br>#VALUE!<br>#VALUE!<br>#VALUE!<br>4471 (28.1%)<br>0.49 (0.84)<br>4471 (28.1%)<br>799 (5.0%)<br>0 (0.0%) | 0.00 #DIV/01 #DIV/01 #VALUEI 0.00 0.03 0.01 -0.01 #VALUEI #VALUEI #VALUEI -0.00 0.00 -0.01 -0.01 -0.01 -0.01 -0.01 |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Lower/unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin, n (%) Aspirin, n (%) Aspirin, n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (xd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of iNR (prothrombin) tests orderedmean (xd) Treating prescriber - Primary Care Physician; n (%) | 639 (29.7%) 181 (8.4%) 0 (0.0%) 0 (0.0%) 15 (0.7%) 113 (5.2%) 353 (16.4%) 1,052 (48.9%) 15 (0.7%) 18 (0.2%) 484 (22.5%) 32 (1.5%) 0.47 (0.72) 528 (24.5%) 75 (3.5%) 0 (0.0%) 0.48 (1.24) 1,407 (65.4%) 1,960 (91.0%) | 621 (28.8%) 166 (7.7%) 0 (0.0%) 0 (0.0%) 13 (0.6%) 100 (4.6%) 337 (15.7%) 1,088 (50.5%) 13 (0.6%) ** (0.1%) ** (0.2%) 480 (22.3%) 29 (1.3%) 0.50 (1.17) 528 (24.5%) 89 (4.1%) 0 (0.0%) 0.37 (0.92) 1,372 (63.7%) 1,950 (91.0%) | 0.02 #DIV/01 #DIV/01 #DIV/01 0.01 0.03 0.02 #DIV/01 0.00 0.00 0.00 0.00 0.02 -0.03 #DIV/01 0.01 0.00 0.00 0.00 0.00 | 1,051 (18.5%) 319 (5.6%) 0 (0.0%) 0 (0.0%) 50 (0.9%) 201 (3.5%) 593 (10.4%) 2,823 (49.7%) 74 (1.3%) ** (0.1%) 1,254 (22.1%) 71 (1.3%) 0.35 (0.72) 1,233 (21.7%) 186 (3.3%) 0 (0.0%) 0.39 (0.95) 3,348 (59.0%) 2,531 (44.6%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 48 (0.8%) 201 (3.5%) 555 (10.0%) 2,803 (49.4%) 77 (1.4%) ** (0.1%) \$** (0.1%) 1,233 (21.7%) 71 (1.3%) 0.35 (0.70) 1,226 (21.6%) 199 (3.5%) 0 (0.0%) 0.33 (0.81) 3,290 (58.0%) 2,528 (44.5%) | #DIV/0! #DIV/0! #DIV/0! #DIV/0! #DIV/0! 0.01 0.00 0.01 #DIV/0! 0.00 0.00 0.00 0.00 0.00 0.00 0.00 0 | 810 (10.0%) 0 (0.0%) 0 (0.0%) ** (0.0%) ** (0.0%) 393 (4.9%) 1,581 (19.5%) 4,541 (56.3%) 28 (0.3%) 20 (0.2%) 29 (0.4%) 2,139 (26.5%) 148 (1.8%) 0.58 (0.79) 2,637 (32.7%) 506 (6.3%) ** (0.0%) 0.33 (0.72) 5,390 (66.8%) 3,504 (43.4%) | 775 (9.6%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 390 (4.8%) 1,430 (17.7%) 4,569 (56.7%) 34 (0.4%) 24 (0.3%) 28 (0.3%) 2,148 (26.6%) 162 (2.0%) 0.58 (0.83) 2,717 (33.7%) 511 (6.3%) 0 (0.0%) 0.31 (0.68) 5,362 (66.5%) | 319 (5.6%) 0 (0.0%) 0 (0.0%) 10 (0.0%) 4WALUE! 707 (4.4%) 2527 (15.9%) 2,823 (49.7%) 117 (0.7%) 4WALUE! 4WALUE! 3877 (24.4%) 251 (1.6%) 0.48 (0.76) 4398 (27.7%) 767 (4.8%) 4WALUE! 0.37 (0.89) 10145 (63.8%) 7995 (50.3%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 61 (0.4%) 691 (4.3%) 2332 (14.7%) 2,803 (49.4%) 124 (0.8%) #VALUE! #VALUE! #VALUE! 3861 (24.3%) 262 (1.6%) 0.49 (0.84) 4477 (28.1%) 799 (5.0%) 0 (0.0%) 0.33 (0.76) 10024 (63.1%) 8034 (50.6%) | 0.00 #DIV/01 #DIV/01 #VALUEI 0.00 0.03 0.01 -0.01 #VALUEI 0.00 0.00 -0.01 -0.01 #VALUEI |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Lower/unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin, n (%) Aspirin, n (%) Aspirin/dipyridamole; n (%) Other antiblatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) Vitamin K therapy; n (%) Vitamin K therapy; n (%) Number of INR (prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Other; n (%) Treating prescriber - Other; n (%) | 639 (29.7%) 181 (8.4%) 0 (0.0%) 0 (0.0%) 15 (0.7%) 113 (5.2%) 353 (16.4%) 1,052 (48.9%) 15 (0.7%) ** (0.1%) ** (0.1%) ** (0.2%) 484 (22.5%) 32 (1.5%) 0.47 (0.72) 528 (24.5%) 75 (3.5%) 0 (0.0%) 0.48 (1.24) 1,407 (65.4%) 1,960 (91.0%) 2,143 (99.5%) | 621 (28.8%) 166 (7.7%) 0 (0.0%) 0 (0.0%) 13 (0.6%) 13 (0.6%) 337 (15.7%) 1,088 (50.5%) ** (0.1%) ** (0.2%) 480 (22.3%) 29 (1.3%) 0.50 (1.17) 528 (24.5%) 89 (4.1%) 0 (0.0%) 0.37 (0.92) 1,372 (63.7%) 1,960 (91.0%) 2,145 (99.6%) | 0.02 #DIV/01 #DIV/01 #DIV/01 0.01 0.03 0.02 #DIV/01 0.01 0.00 0.00 0.00 0.02 -0.03 #DIV/01 0.10 0.00 0.00 0.00 0.00 0.00 0.00 0 | 1,051 (18.5%) 319 (5.6%) 0 (0.0%) 50 (0.9%) 201 (3.5%) 593 (10.4%) 2,823 (49.7%) 74 (1.3%) ** (0.1%) 1,254 (22.1%) 71 (1.3%) 0.35 (0.72) 1,233 (21.7%) 186 (3.3%) 0 (0.0%) 0.39 (0.95) 3,348 (59.0%) 2,531 (44.6%) 5,286 (93.1%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 48 (0.8%) 201 (3.5%) 555 (10.0%) **(0.1%) **(0.1%) **(0.1%) 1,233 (21.7%) 71 (1.3%) 0.35 (0.70) 1,226 (21.6%) 199 (3.5%) 0 (0.0%) 0.33 (0.81) 3,290 (58.0%) 2,528 (44.5%) 5,228 (44.5%) 5,228 (44.5%) | #DIV/0! #DIV/0! #DIV/0! 0.01 0.00 0.01 #DIV/0! -0.01 0.00 0.00 0.00 0.00 0.01 #DIV/0! 0.00 0.00 0.00 0.00 0.00 0.00 0.00 0 | 810 (10.0%) 0 (0.0%) 0 (0.0%) 10 (0.0%) ** (0.0%) 393 (4.9%) 1,581 (19.6%) 4,541 (56.3%) 28 (0.3%) 20 (0.2%) 29 (0.4%) 2,139 (26.5%) 148 (1.8%) 0.58 (0.79) 2,637 (32.7%) 506 (6.3%) ** (0.0%) 0.33 (0.72) 5,390 (66.8%) 3,504 (43.4%) 8,058 (99.9%) | 775 (9.6%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 390 (4.8%) 1,430 (17.7%) 4,569 (56.7%) 34 (0.4%) 28 (0.3%) 2,148 (26.6%) 162 (2.0%) 0.58 (0.83) 2,717 (33.7%) 511 (6.3%) 0 (0.0%) 0.31 (0.68) 5,362 (66.5%) 3,546 (44.0%) 8,057 (99.9%) | 319 (5.6%) 0 (0.0%) 0 (0.0%) 10 (0.0%) #VALUE! 707 (4.4%) 2,823 (49.7%) 117 (0.7%) #VALUE! #VALUE! #VALUE! 3877 (24.4%) 251 (1.6%) 0.48 (0.76) 4398 (27.7%) 767 (4.8%) #VALUE! 0.37 (0.89) 10145 (63.8%) 7995 (50.3%) 15487 (97.4%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 61 (0.4%) 691 (4.3%) 2332 (14.7%) 2,803 (49.4%) 124 (0.8%) #VALUEI #VALUEI #VALUEI #VALUEI #VALUEI #VALUEI 0.49 (0.84) 4471 (28.1%) 799 (5.0%) 0 (0.0%) 0.33 (0.76) 10024 (63.1%) 8034 (50.6%) 15496 (97.5%) | 0.00 #DIV/01 #DIV/01 #VALUE! 0.00 0.03 0.01 -0.01 #VALUE! #VALUE! 0.00 0.00 -0.01 -0.01 #VALUE! |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Lower/unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipit dets or orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of lipit dets or deredmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Cardiologist; n (%) Treating prescriber - Cher; n (%) Alpha blockers; n (%) | 639 (29.7%) 181 (8.4%) 0 (0.0%) 0 (0.0%) 15 (0.7%) 113 (5.2%) 353 (16.4%) 1,052 (48.9%) 15 (0.7%) 18 (0.2%) 484 (22.5%) 32 (1.5%) 0.47 (0.72) 528 (24.5%) 75 (3.5%) 0 (0.0%) 0.48 (1.24) 1,407 (65.4%) 1,960 (91.0%) | 621 (28.8%) 166 (7.7%) 0 (0.0%) 0 (0.0%) 13 (0.6%) 100 (4.6%) 337 (15.7%) 1,088 (50.5%) 13 (0.6%) ** (0.1%) ** (0.2%) 480 (22.3%) 29 (1.3%) 0.50 (1.17) 528 (24.5%) 89 (4.1%) 0 (0.0%) 0.37 (0.92) 1,372 (63.7%) 1,950 (91.0%) | 0.02 #DIV/01 #DIV/01 #DIV/01 0.01 0.03 0.02 #DIV/01 0.00 0.00 0.00 0.00 0.02 -0.03 #DIV/01 0.01 0.00 0.00 0.00 0.00 | 1,051 (18.5%) 319 (5.6%) 0 (0.0%) 0 (0.0%) 50 (0.9%) 201 (3.5%) 593 (10.4%) 2,823 (49.7%) 74 (1.3%) ** (0.1%) 1,254 (22.1%) 71 (1.3%) 0.35 (0.72) 1,233 (21.7%) 186 (3.3%) 0 (0.0%) 0.39 (0.95) 3,348 (59.0%) 2,531 (44.6%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 48 (0.8%) 201 (3.5%) 555 (10.0%) 2,803 (49.4%) 77 (1.4%) ** (0.1%) \$** (0.1%) 1,233 (21.7%) 71 (1.3%) 0.35 (0.70) 1,226 (21.6%) 199 (3.5%) 0 (0.0%) 0.33 (0.81) 3,290 (58.0%) 2,528 (44.5%) | #DIV/0! #DIV/0! #DIV/0! #DIV/0! #DIV/0! 0.01 0.00 0.01 #DIV/0! 0.00 0.00 0.00 0.00 0.00 0.00 0.00 0 | 810 (10.0%) 0 (0.0%) 0 (0.0%) ** (0.0%) ** (0.0%) 393 (4.9%) 1,581 (19.5%) 4,541 (56.3%) 28 (0.3%) 20 (0.2%) 29 (0.4%) 2,139 (26.5%) 148 (1.8%) 0.58 (0.79) 2,637 (32.7%) 506 (6.3%) ** (0.0%) 0.33 (0.72) 5,390 (66.8%) 3,504 (43.4%) | 775 (9.6%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 390 (4.8%) 1,430 (17.7%) 4,569 (56.7%) 34 (0.4%) 24 (0.3%) 28 (0.3%) 2,148 (26.6%) 162 (2.0%) 0.58 (0.83) 2,717 (33.7%) 511 (6.3%) 0 (0.0%) 0.31 (0.68) 5,362 (66.5%) | 319 (5.6%) 0 (0.0%) 0 (0.0%) 10 (0.0%) 4WALUE! 707 (4.4%) 2527 (15.9%) 2,823 (49.7%) 117 (0.7%) 4WALUE! 4WALUE! 3877 (24.4%) 251 (1.6%) 0.48 (0.76) 4398 (27.7%) 767 (4.8%) 4WALUE! 0.37 (0.89) 10145 (63.8%) 7995 (50.3%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 61 (0.4%) 691 (4.3%) 2332 (14.7%) 2,803 (49.4%) 124 (0.8%) #VALUE! #VALUE! #VALUE! 3861 (24.3%) 262 (1.6%) 0.49 (0.84) 4477 (28.1%) 799 (5.0%) 0 (0.0%) 0.33 (0.76) 10024 (63.1%) 8034 (50.6%) | 0.00 #DIV/01 #DIV/01 #VALUEI 0.00 0.03 0.01 -0.01 #VALUEI 0.00 0.00 -0.01 -0.01 #VALUEI |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gl bleed; n (%) Lower/unspecified Gl bleed; n (%) Urogenital bleed; n (%) Urogenital bleed; n (%) Other bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) Vitamin K therapy; n (%) Number of link (prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Cardiologist; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) Alpha blockers; n (%) CHA2DS2 VASc score, 180 days, V | 639 (29.7%) 181 (8.4%) 0 (0.0%) 0 (0.0%) 15 (0.7%) 113 (5.2%) 353 (16.4%) 1,052 (48.9%) 15 (0.7%) ** (0.1%) ** (0.2%) 484 (22.5%) 32 (1.5%) 0.47 (0.72) 528 (24.5%) 75 (3.5%) 0 (0.0%) 0.48 (1.24) 1,407 (65.4%) 1,960 (91.0%) 2,143 (99.5%) 170 (7.9%) | 621 (28.8%) 166 (7.7%) 0 (0.0%) 0 (0.0%) 13 (0.6%) 13 (0.6%) 137 (15.7%) 1,088 (50.5%) 13 (0.6%) 14 (0.1%) 15 (0.2%) 480 (22.3%) 29 (1.3%) 0.50 (1.17) 528 (24.5%) 89 (4.1%) 0 (0.0%) 0.37 (0.92) 1,372 (63.7%) 1,960 (91.0%) 2,145 (99.6%) 164 (7.6%) | 0.02 #IDIV/01 #IDIV/01 #IDIV/01 0.01 0.03 0.02 #IDIV/01 0.01 0.00 0.00 0.00 0.02 -0.03 0.00 -0.03 #IDIV/01 0.10 0.04 0.04 0.05 | 1,051 (18.5%) 319 (5.6%) 0 (0.0%) 0 (0.0%) 50 (0.9%) 201 (3.5%) 593 (10.4%) 2,823 (49.7%) 74 (1.3%) ** (0.1%) 1,254 (22.1%) 71 (1.3%) 0.35 (0.72) 1,233 (21.7%) 186 (3.3%) 0 (0.0%) 0.39 (0.95) 3,348 (59.0%) 5,286 (93.1%) 281 (5.0%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 48 (0.8%) 201 (3.5%) 555 (10.0%) 2,803 (49.4%) 77 (1.4%) ** (0.1%) ** (0.1%) 1,233 (21.7%) 71 (1.3%) 0.35 (0.70) 1,226 (21.6%) 199 (3.5%) 0 (0.0%) 0.33 (0.81) 3,290 (58.0%) 2,528 (44.5%) 5,294 (93.3%) 291 (5.1%) | #DIV/0! #DIV/0! #DIV/0! 0.01 0.00 0.01 #DIV/0! -0.01 0.00 0.00 0.00 0.01 0.00 0.00 0.0 | 810 (10.0%) 0 (0.0%) 0 (0.0%) ** (0.0%) ** (0.0%) 393 (4.9%) 1,581 (19.5%) 4,541 (56.3%) 28 (0.3%) 20 (0.2%) 29 (0.4%) 2,139 (26.5%) 148 (1.8%) 0.58 (0.79) 2,637 (32.7%) 506 (6.3%) ** (0.0%) 0.33 (0.72) 5,390 (66.8%) 8,058 (99.9%) 827 (10.3%) | 775 (9.6%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 390 (4.8%) 1,430 (17.7%) 4,569 (56.7%) 34 (0.4%) 28 (0.3%) 2,148 (26.6%) 162 (2.0%) 0.58 (0.83) 2,717 (33.7%) 511 (6.3%) 0 (0.0%) 0.31 (0.68) 5,362 (66.5%) 3,546 (44.0%) 8,057 (99.9%) 807 (10.0%) | 319 (5.6%) 0 (0.0%) 0 (0.0%) 10 (0.0%) 4 WALUE! 707 (4.4%) 2527 (15.9%) 2,823 (49.7%) 117 (0.7%) 4 WALUE! 4 WALUE! 3877 (24.4%) 251 (1.6%) 0.48 (0.76) 4398 (27.7%) 767 (4.8%) 4 WALUE! 0.37 (0.89) 10145 (63.8%) 17995 (50.3%) 15487 (97.4%) 1278 (8.0%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 61 (0.4%) 691 (4.3%) 5932 (14.7%) 2.803 (49.4%) 124 (0.8%) #WALUEI #WALUEI #VALUEI 3861 (24.3%) 262 (1.6%) 0.49 (0.84) 4477 (28.1%) 799 (5.0%) 0 (0.0%) 0.33 (0.76) 10024 (63.1%) 8034 (50.6%) 15496 (97.5%) 1262 (7.9%) | 0.00 #DIV/01 #DIV/01 #VALUE! 0.00 0.03 0.01 -0.01 #VALUE! #VALUE! 0.00 0.00 -0.01 -0.01 -0.01 #VALUE! |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gl bleed; n (%) Lower/unspecified Gl bleed; n (%) Urogenital bleed; n (%) Other bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin, n (%) Aspirin, n (%) Aspirin, dipyridamole; n (%) Other antiplatel agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid ests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of liNR (prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHA2DS2 VASc score, 180 days, Vmean (sd) | 639 (29.7%) 181 (8.4%) 0 (0.0%) 0 (0.0%) 15 (0.7%) 113 (5.2%) 353 (16.4%) 1,052 (48.9%) 15 (0.7%) ** (0.1%) ** (0.1%) ** (0.2%) 32 (1.5%) 0.47 (0.72) 528 (24.5%) 75 (3.5%) 0 (0.0%) 0.48 (1.24) 1,407 (65.4%) 1,960 (91.0%) 2,143 (99.5%) 170 (7.9%) | 621 (28.8%) 166 (7.7%) 0 (0.0%) 0 (0.0%) 13 (0.6%) 130 (4.6%) 337 (15.7%) 1,088 (50.5%) ** (0.1%) ** (0.2%) 480 (22.3%) 29 (1.3%) 0.50 (1.17) 528 (24.5%) 89 (4.1%) 0 (0.0%) 0.37 (0.92) 1,372 (63.7%) 1,960 (91.0%) 2,145 (99.6%) 164 (7.6%) | 0.02 #DIV/0! #DIV/0! #DIV/0! 0.01 0.03 0.02 #DIV/0! 0.01 0.00 0.00 0.00 0.02 -0.03 0.00 0.00 0.00 0.00 0.01 0.01 0.01 | 1,051 (18.5%) 319 (5.6%) 0 (0.0%) 50 (0.9%) 50 (0.9%) 503 (10.4%) 2,823 (49.7%) 74 (1.3%) ** (0.1%) \$1,254 (22.1%) 71 (1.3%) 0.35 (0.72) 1,233 (21.7%) 186 (3.3%) 0 (0.0%) 0.39 (0.95) 3,348 (59.0%) 2,531 (44.6%) 5,286 (93.1%) 281 (5.0%) 2.80 (1.64) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 48 (0.8%) 201 (3.5%) 555 (10.0%) 7 (1.4%) ** (0.1%) ** (0.1%) 1,233 (21.7%) 71 (1.3%) 0.35 (0.70) 1,226 (21.6%) 199 (3.5%) 0 (0.0%) 0.33 (0.81) 3,290 (58.0%) 2,528 (44.5%) 5,294 (93.3%) 291 (5.1%) | #DIV/O! #DIV/O! #DIV/O! #DIV/O! #DIV/O! 0.01 0.00 0.01 #DIV/O! 0.00 0.00 0.00 0.00 0.00 0.00 0.00 0. | 810 (10.0%) 0 (0.0%) 0 (0.0%) ** (0.0%) 393 (4.9%) 1,581 (19.6%) 4,541 (56.3%) 28 (0.3%) 20 (0.2%) 29 (0.4%) 2,139 (26.5%) 148 (1.8%) 0.58 (0.79) 2,637 (32.7%) 506 (6.3%) ** (0.0%) 0.33 (0.72) 5,390 (66.8%) 3,504 (43.4%) 8,058 (9.99%) 827 (10.3%) | 775 (9.6%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 390 (4.8%) 1,430 (17.7%) 4,569 (56.7%) 34 (0.4%) 24 (0.3%) 28 (0.3%) 2,148 (26.6%) 162 (2.0%) 0.58 (0.83) 2,717 (33.7%) 511 (6.3%) 0 (0.0%) 0.31 (0.68) 5,362 (66.5%) 3,546 (44.0%) 8,057 (9.9-%) 807 (10.0%) | 319 (5.6%) 0 (0.0%) 0 (0.0%) 10 (0.0%) 4VALUE! 707 (4.4%) 2,527 (15.9%) 2,823 (49.7%) 117 (0.7%) 4VALUE! 4VALUE! 4VALUE! 3877 (24.4%) 251 (1.6%) 0.48 (0.76) 4398 (27.7%) 767 (4.8%) 4VALUE! 0.37 (0.89) 10145 (63.8%) 7995 (50.3%) 15487 (97.4%) 15487 (97.4%) 15487 (97.4%) 15488 (97.4%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 61 (0.4%) 691 (4.3%) 2332 (14.7%) 2,803 (49.4%) 124 (0.8%) #VALUE! #VALUE! #VALUE! #VALUE! #VALUE! #VALUE! #0.41 (28.1%) 799 (5.0%) 0 (0.0%) 0.33 (0.76) 10024 (63.1%) 8034 (50.6%) 1262 (7.9%) | 0.00 #DIV/01 #DIV/01 #VALUEI 0.00 0.03 0.01 -0.01 #VALUEI #VALUEI #VALUEI #VALUEI #VALUEI 0.00 0.00 -0.01 |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Glo bled; n (%) Lower/unspecified Glo bled; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of link (prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Cardiologist; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) Alpha blockers; n (%) Alpha blockers; n (%) Alpha blockers; n (%) | 639 (29.7%) 181 (8.4%) 0 (0.0%) 0 (0.0%) 15 (0.7%) 113 (5.2%) 353 (16.4%) 1,052 (48.9%) 15 (0.7%) ** (0.1%) ** (0.2%) 484 (22.5%) 32 (1.5%) 0.47 (0.72) 528 (24.5%) 75 (3.5%) 0 (0.0%) 0.48 (1.24) 1,407 (65.4%) 1,960 (91.0%) 2,143 (99.5%) 170 (7.9%) | 621 (28.8%) 166 (7.7%) 0 (0.0%) 0 (0.0%) 13 (0.6%) 13 (0.6%) 137 (15.7%) 1,088 (50.5%) 13 (0.6%) 14 (0.1%) 15 (0.2%) 480 (22.3%) 29 (1.3%) 0.50 (1.17) 528 (24.5%) 89 (4.1%) 0 (0.0%) 0.37 (0.92) 1,372 (63.7%) 1,960 (91.0%) 2,145 (99.6%) 164 (7.6%) | 0.02 #IDIV/01 #IDIV/01 #IDIV/01 0.01 0.03 0.02 #IDIV/01 0.01 0.00 0.00 0.00 0.02 -0.03 0.00 -0.03 #IDIV/01 0.10 0.04 0.04 0.05 | 1,051 (18.5%) 319 (5.6%) 0 (0.0%) 0 (0.0%) 50 (0.9%) 201 (3.5%) 593 (10.4%) 2,823 (49.7%) 74 (1.3%) ** (0.1%) 1,254 (22.1%) 71 (1.3%) 0.35 (0.72) 1,233 (21.7%) 186 (3.3%) 0 (0.0%) 0.39 (0.95) 3,348 (59.0%) 5,286 (93.1%) 281 (5.0%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 48 (0.8%) 201 (3.5%) 555 (10.0%) 2,803 (49.4%) 77 (1.4%) ** (0.1%) ** (0.1%) 1,233 (21.7%) 71 (1.3%) 0.35 (0.70) 1,226 (21.6%) 199 (3.5%) 0 (0.0%) 0.33 (0.81) 3,290 (58.0%) 2,528 (44.5%) 5,294 (93.3%) 291 (5.1%) | #DIV/0! #DIV/0! #DIV/0! 0.01 0.00 0.01 #DIV/0! -0.01 0.00 0.00 0.00 0.01 0.00 0.00 0.0 | 810 (10.0%) 0 (0.0%) 0 (0.0%) ** (0.0%) ** (0.0%) 393 (4.9%) 1,581 (19.5%) 4,541 (56.3%) 28 (0.3%) 20 (0.2%) 29 (0.4%) 2,139 (26.5%) 148 (1.8%) 0.58 (0.79) 2,637 (32.7%) 506 (6.3%) ** (0.0%) 0.33 (0.72) 5,390 (66.8%) 8,058 (99.9%) 827 (10.3%) | 775 (9.6%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 390 (4.8%) 1,430 (17.7%) 4,569 (56.7%) 34 (0.4%) 28 (0.3%) 2,148 (26.6%) 162 (2.0%) 0.58 (0.83) 2,717 (33.7%) 511 (6.3%) 0 (0.0%) 0.31 (0.68) 5,362 (66.5%) 3,546 (44.0%) 8,057 (99.9%) 807 (10.0%) | 319 (5.6%) 0 (0.0%) 0 (0.0%) 10 (0.0%) 4 WALUE! 707 (4.4%) 2527 (15.9%) 2,823 (49.7%) 117 (0.7%) 4 WALUE! 4 WALUE! 3877 (24.4%) 251 (1.6%) 0.48 (0.76) 4398 (27.7%) 767 (4.8%) 4 WALUE! 0.37 (0.89) 10145 (63.8%) 17995 (50.3%) 15487 (97.4%) 1278 (8.0%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 61 (0.4%) 691 (4.3%) 5932 (14.7%) 2.803 (49.4%) 124 (0.8%) #WALUEI #WALUEI #VALUEI 3861 (24.3%) 262 (1.6%) 0.49 (0.84) 4477 (28.1%) 799 (5.0%) 0 (0.0%) 0.33 (0.76) 10024 (63.1%) 8034 (50.6%) 15496 (97.5%) 1262 (7.9%) | 0.00 #DIV/01 #DIV/01 #VALUE! 0.00 0.03 0.01 -0.01 #VALUE! #VALUE! 0.00 0.00 -0.01 -0.01 -0.01 #VALUE! |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gl bleed; n (%) Lower/unspecified Gl bleed; n (%) Urogenital bleed; n (%) Other bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin, n (%) Aspirin, n (%) Aspirin, dipyridamole; n (%) Other antiplatel agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid ests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of liNR (prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHA2DS2 VASc score, 180 days, Vmean (sd) | 639 (29.7%) 181 (8.4%) 0 (0.0%) 0 (0.0%) 15 (0.7%) 113 (5.2%) 353 (16.4%) 1,052 (48.9%) 15 (0.7%) ** (0.1%) ** (0.1%) ** (0.2%) 32 (1.5%) 0.47 (0.72) 528 (24.5%) 75 (3.5%) 0 (0.0%) 0.48 (1.24) 1,407 (65.4%) 1,960 (91.0%) 2,143 (99.5%) 170 (7.9%) | 621 (28.8%) 166 (7.7%) 0 (0.0%) 0 (0.0%) 13 (0.6%) 130 (4.6%) 337 (15.7%) 1,088 (50.5%) ** (0.1%) ** (0.2%) 480 (22.3%) 29 (1.3%) 0.50 (1.17) 528 (24.5%) 89 (4.1%) 0 (0.0%) 0.37 (0.92) 1,372 (63.7%) 1,960 (91.0%) 2,145 (99.6%) 164 (7.6%) | 0.02 #DIV/0! #DIV/0! #DIV/0! 0.01 0.03 0.02 #DIV/0! 0.01 0.00 0.00 0.00 0.02 -0.03 0.00 0.00 0.00 0.00 0.01 0.01 0.01 | 1,051 (18.5%) 319 (5.6%) 0 (0.0%) 50 (0.9%) 50 (0.9%) 503 (10.4%) 2,823 (49.7%) 74 (1.3%) ** (0.1%) \$1,254 (22.1%) 71 (1.3%) 0.35 (0.72) 1,233 (21.7%) 186 (3.3%) 0 (0.0%) 0.39 (0.95) 3,348 (59.0%) 2,531 (44.6%) 5,286 (93.1%) 281 (5.0%) 2.80 (1.64) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 48 (0.8%) 201 (3.5%) 555 (10.0%) 7 (1.4%) ** (0.1%) ** (0.1%) 1,233 (21.7%) 71 (1.3%) 0.35 (0.70) 1,226 (21.6%) 199 (3.5%) 0 (0.0%) 0.33 (0.81) 3,290 (58.0%) 2,528 (44.5%) 5,294 (93.3%) 291 (5.1%) | #DIV/O! #DIV/O! #DIV/O! #DIV/O! #DIV/O! 0.01 0.00 0.01 #DIV/O! 0.00 0.00 0.00 0.00 0.00 0.00 0.00 0. | 810 (10.0%) 0 (0.0%) 0 (0.0%) ** (0.0%) 393 (4.9%) 1,581 (19.6%) 4,541 (56.3%) 28 (0.3%) 20 (0.2%) 29 (0.4%) 2,139 (26.5%) 148 (1.8%) 0.58 (0.79) 2,637 (32.7%) 506 (6.3%) ** (0.0%) 0.33 (0.72) 5,390 (66.8%) 3,504 (43.4%) 8,058 (9.99%) 827 (10.3%) | 775 (9.6%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 390 (4.8%) 1,430 (17.7%) 4,569 (56.7%) 34 (0.4%) 24 (0.3%) 28 (0.3%) 2,148 (26.6%) 162 (2.0%) 0.58 (0.83) 2,717 (33.7%) 511 (6.3%) 0 (0.0%) 0.31 (0.68) 5,362 (66.5%) 3,546 (44.0%) 8,057 (9.9-%) 807 (10.0%) | 319 (5.6%) 0 (0.0%) 0 (0.0%) 10 (0.0%) 4VALUE! 707 (4.4%) 2,527 (15.9%) 2,823 (49.7%) 117 (0.7%) 4VALUE! 4VALUE! 4VALUE! 3877 (24.4%) 251 (1.6%) 0.48 (0.76) 4398 (27.7%) 767 (4.8%) 4VALUE! 0.37 (0.89) 10145 (63.8%) 7995 (50.3%) 15487 (97.4%) 15487 (97.4%) 15487 (97.4%) 15488 (97.4%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 61 (0.4%) 691 (4.3%) 2332 (14.7%) 2,803 (49.4%) 124 (0.8%) #VALUE! #VALUE! #VALUE! #VALUE! #VALUE! #VALUE! #0.41 (28.1%) 799 (5.0%) 0 (0.0%) 0.33 (0.76) 10024 (63.1%) 8034 (50.6%) 1262 (7.9%) | 0.00 #DIV/01 #DIV/01 #VALUEI 0.00 0.03 0.01 -0.01 #VALUEI #VALUEI #VALUEI #VALUEI #VALUEI 0.00 0.00 -0.01 |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Lower/unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (xd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of link (prothrombin) tests orderedmean (xd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHA2DS2 VASc score, 180 days, Vmean (xd) Use of Prasugrel; n (%) | 639 (29.7%) 181 (8.4%) 0 (0.0%) 0 (0.0%) 15 (0.7%) 113 (5.2%) 353 (16.4%) 1,052 (48.9%) 15 (0.7%) ** (0.1%) ** (0.2%) 484 (22.5%) 32 (1.5%) 0.47 (0.72) 528 (24.5%) 75 (3.5%) 0 (0.0%) 0.48 (1.24) 1,407 (65.4%) 1,960 (91.0%) 2,143 (99.5%) 170 (7.7%) 3.05 (1.73) ** (0.1%) | 621 (28.8%) 166 (7.7%) 0 (0.0%) 0 (0.0%) 13 (0.6%) 13 (0.6%) 130 (4.6%) 337 (15.7%) 1,088 (50.5%) ** (0.1%) ** (0.2%) 480 (22.3%) 29 (1.3%) 0.50 (1.17) 528 (24.5%) 0 (0.0%) 0.37 (0.92) 1,372 (63.7%) 1,960 (91.0%) 2,145 (99.6%) 164 (7.6%) 3.21 (1.73) ** (0.1%) | 0.02 #DIV/01 #DIV/01 #DIV/01 0.01 0.03 0.02 #DIV/01 0.01 0.00 0.00 0.02 -0.03 0.00 -0.03 #DIV/01 0.10 0.04 0.04 0.00 -0.01 0.01 0.04 0.00 -0.01 0.01 | 1,051 (18.5%) 319 (5.6%) 0 (0.0%) 50 (0.9%) 50 (0.9%) 503 (10.4%) 2,823 (49.7%) 74 (1.3%) ** (0.1%) 1,254 (22.1%) 71 (1.3%) 0.35 (0.72) 1,233 (21.7%) 186 (3.3%) 0 (0.0%) 0.39 (0.95) 3,348 (59.0%) 2,531 (44.6%) 5,286 (93.1%) 281 (5.0%) 2.80 (1.64) ** (0.1%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 48 (0.8%) 201 (3.5%) 555 (10.0%) 2,803 (49.4%) 77 (1.4%) ** (0.1%) \$** (0.1%) 1,233 (21.7%) 71 (1.3%) 0.35 (0.70) 1,226 (21.6%) 199 (3.5%) 0 (0.0%) 0.33 (0.81) 3,290 (58.0%) 2,528 (44.5%) 5,294 (93.3%) 291 (5.1%) 2.93 (1.60) ** (0.1%) | #DIV/O! #DIV/O! #DIV/O! #DIV/O! #DIV/O! 0.01 0.00 0.01 #DIV/O! 0.00 0.00 0.00 0.00 0.00 0.00 0.00 0. | 810 (10.0%) 0 (0.0%) 0 (0.0%) 10 (0.0%) 393 (4.9%) 1,581 (19.5%) 4,541 (56.3%) 28 (0.3%) 20 (0.2%) 29 (0.4%) 2,139 (26.5%) 148 (1.8%) 0.58 (0.79) 2,637 (32.7%) 506 (6.3%) ** (0.0%) 0.33 (0.72) 5,390 (66.8%) 3,504 (43.4%) 8,058 (99.9%) 827 (10.3%) 3.97 (1.85) 0 (0.0%) | 775 (9.6%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 390 (4.8%) 1,430 (17.7%) 4,569 (56.7%) 34 (0.4%) 28 (0.3%) 2,148 (26.6%) 162 (2.0%) 0.58 (0.83) 2,717 (33.7%) 511 (6.3%) 0 (0.0%) 0.31 (0.68) 5,362 (66.5%) 3,546 (44.0%) 8,057 (99.9%) 807 (10.0%) | 319 (5.6%) 0 (0.0%) 0 (0.0%) 10 (0.0%) 4 VALUE! 707 (4.4%) 2527 (15.9%) 2,823 (49.7%) 117 (0.7%) 4 VALUE! 4 VALUE! 3877 (24.4%) 251 (1.6%) 0.48 (0.76) 4398 (27.7%) 767 (4.8%) 4 VALUE! 0.37 (0.89) 10145 (63.8%) 7995 (50.3%) 15487 (97.4%) 1278 (8.0%) 3.43 (1.76) #VALUE! | 326 (5.7%) 0 (0.0%) 0 (0.0%) 61 (0.4%) 691 (4.3%) 5932 (14.7%) 2.803 (49.4%) 124 (0.8%) #WALUEI #WALUEI \$861 (24.3%) 262 (1.6%) 0.49 (0.84) 4477 (28.1%) 799 (5.0%) 0 (0.0%) 0.33 (0.76) 10024 (63.1%) 8034 (50.6%) 15496 (97.5%) 1262 (7.9%) 3.60 (1.73) #WALUEI | 0.00 #DIV/01 #DIV/01 #VALUEI 0.00 0.03 0.01 -0.01 #VALUEI #VALUEI #VALUEI #VALUEI #VALUEI 0.00 0.00 -0.01 |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gl bleed; n (%) Lower/unspecified Gl bleed; n (%) Urogenital bleed; n (%) Other bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin, n (%) Aspirin, n (%) Aspirin, dipyridamole; n (%) Other antiplatel agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid ests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of liNR (prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHA2DS2 VASc score, 180 days, Vmean (sd) | 639 (29.7%) 181 (8.4%) 0 (0.0%) 0 (0.0%) 15 (0.7%) 113 (5.2%) 353 (16.4%) 1,052 (48.9%) 15 (0.7%) ** (0.1%) ** (0.1%) ** (0.2%) 32 (1.5%) 0.47 (0.72) 528 (24.5%) 75 (3.5%) 0 (0.0%) 0.48 (1.24) 1,407 (65.4%) 1,960 (91.0%) 2,143 (99.5%) 170 (7.9%) | 621 (28.8%) 166 (7.7%) 0 (0.0%) 0 (0.0%) 13 (0.6%) 130 (4.6%) 337 (15.7%) 1,088 (50.5%) ** (0.1%) ** (0.2%) 480 (22.3%) 29 (1.3%) 0.50 (1.17) 528 (24.5%) 89 (4.1%) 0 (0.0%) 0.37 (0.92) 1,372 (63.7%) 1,960 (91.0%) 2,145 (99.6%) 164 (7.6%) | 0.02 #DIV/0! #DIV/0! #DIV/0! 0.01 0.03 0.02 #DIV/0! 0.01 0.00 0.00 0.00 0.02 -0.03 0.00 0.00 0.00 0.00 0.01 0.01 0.01 | 1,051 (18.5%) 319 (5.6%) 0 (0.0%) 50 (0.9%) 50 (0.9%) 503 (10.4%) 2,823 (49.7%) 74 (1.3%) ** (0.1%) \$1,254 (22.1%) 71 (1.3%) 0.35 (0.72) 1,233 (21.7%) 186 (3.3%) 0 (0.0%) 0.39 (0.95) 3,348 (59.0%) 2,531 (44.6%) 5,286 (93.1%) 281 (5.0%) 2.80 (1.64) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 48 (0.8%) 201 (3.5%) 555 (10.0%) 7 (1.4%) ** (0.1%) ** (0.1%) 1,233 (21.7%) 71 (1.3%) 0.35 (0.70) 1,226 (21.6%) 199 (3.5%) 0 (0.0%) 0.33 (0.81) 3,290 (58.0%) 2,528 (44.5%) 5,294 (93.3%) 291 (5.1%) | #DIV/0! #DIV/0! #DIV/0! 0.01 0.00 0.01 #DIV/0! -0.01 0.00 0.00 0.01 0.00 0.01 0.00 0.00 | 810 (10.0%) 0 (0.0%) 0 (0.0%) ** (0.0%) 393 (4.9%) 1,581 (19.6%) 4,541 (56.3%) 28 (0.3%) 20 (0.2%) 29 (0.4%) 2,139 (26.5%) 148 (1.8%) 0.58 (0.79) 2,637 (32.7%) 506 (6.3%) ** (0.0%) 0.33 (0.72) 5,390 (66.8%) 3,504 (43.4%) 8,058 (9.99%) 827 (10.3%) | 775 (9.6%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 390 (4.8%) 1,430 (17.7%) 4,569 (56.7%) 34 (0.4%) 24 (0.3%) 28 (0.3%) 2,148 (26.6%) 162 (2.0%) 0.58 (0.83) 2,717 (33.7%) 511 (6.3%) 0 (0.0%) 0.31 (0.68) 5,362 (66.5%) 3,546 (44.0%) 8,057 (9.9-%) 807 (10.0%) | 319 (5.6%) 0 (0.0%) 0 (0.0%) 10 (0.0%) 4VALUE! 707 (4.4%) 2,527 (15.9%) 2,823 (49.7%) 117 (0.7%) 4VALUE! 4VALUE! 4VALUE! 3877 (24.4%) 251 (1.6%) 0.48 (0.76) 4398 (27.7%) 767 (4.8%) 4VALUE! 0.37 (0.89) 10145 (63.8%) 7995 (50.3%) 15487 (97.4%) 15487 (97.4%) 15487 (97.4%) 15488 (97.4%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 61 (0.4%) 691 (4.3%) 2332 (14.7%) 2,803 (49.4%) 124 (0.8%) #VALUE! #VALUE! #VALUE! #VALUE! #VALUE! #VALUE! #0.41 (28.1%) 799 (5.0%) 0 (0.0%) 0.33 (0.76) 10024 (63.1%) 8034 (50.6%) 1262 (7.9%) | 0.00 #DIV/01 #DIV/01 #VALUE! 0.00 0.03 0.01 -0.01 #VALUE! #VALUE! 0.00 0.00 -0.01 -0.01 -0.01 -0.01 -0.01 0.00 0.00 |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Lower/unspecified Gi bleed; n (%) Urogenital bleed; n (%) Orther bleeds; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Vitamin K therapy; n (%) Treating prescriber-Cardiologist; n (%) Treating prescriber-Other; n (%) Alpha blockers; n (%) CHA2DS2 VASc score, 180 days, Vmean (sd) Use of Prasugrel; n (%) Use of Loop Diuretics+other diuretics+other hyperten: | 639 (29.7%) 181 (8.4%) 0 (0.0%) 0 (0.0%) 15 (0.7%) 113 (5.2%) 353 (16.4%) 1,052 (48.9%) 15 (0.7%) ** (0.1%) ** (0.2%) 484 (22.5%) 32 (1.5%) 0.47 (0.72) 528 (24.5%) 75 (3.5%) 0 (0.0%) 0.48 (1.24) 1,407 (65.4%) 1,960 (91.0%) 2,143 (99.5%) 170 (7.9%) 3.05 (1.73) ** (0.1%) | 621 (28.8%) 166 (7.7%) 0 (0.0%) 0 (0.0%) 13 (0.6%) 13 (0.6%) 130 (4.6%) 337 (15.7%) 1,088 (50.5%) ** (0.1%) ** (0.2%) 480 (22.3%) 29 (1.3%) 0.50 (1.17) 528 (24.5%) 0 (0.0%) 0.37 (0.92) 1,372 (63.7%) 1,960 (91.0%) 2,145 (99.6%) 164 (7.6%) 3.21 (1.73) ** (0.1%) | 0.02 #DIV/01 #DIV/01 #DIV/01 0.01 0.03 0.02 #DIV/01 0.01 0.00 0.00 0.02 -0.03 0.00 -0.03 #DIV/01 0.10 0.04 0.04 0.00 -0.01 0.01 0.04 0.00 -0.01 0.01 | 1,051 (18.5%) 319 (5.6%) 0 (0.0%) 50 (0.9%) 50 (0.9%) 503 (10.4%) 2,823 (49.7%) 74 (1.3%) ** (0.1%) 1,254 (22.1%) 71 (1.3%) 0.35 (0.72) 1,233 (21.7%) 186 (3.3%) 0 (0.0%) 0.39 (0.95) 3,348 (59.0%) 2,531 (44.6%) 5,286 (93.1%) 281 (5.0%) 2.80 (1.64) ** (0.1%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 48 (0.8%) 201 (3.5%) 555 (10.0%) 2,803 (49.4%) 77 (1.4%) ** (0.1%) \$** (0.1%) 1,233 (21.7%) 71 (1.3%) 0.35 (0.70) 1,226 (21.6%) 199 (3.5%) 0 (0.0%) 0.33 (0.81) 3,290 (58.0%) 2,528 (44.5%) 5,294 (93.3%) 291 (5.1%) 2.93 (1.60) ** (0.1%) | #DIV/0! #DIV/0! #DIV/0! 0.01 0.00 0.01 #DIV/0! -0.01 0.00 0.00 0.01 0.00 0.01 0.00 0.00 | 810 (10.0%) 0 (0.0%) 0 (0.0%) ** (0.0%) 393 (4.9%) 1,581 (19.6%) 4,541 (56.3%) 28 (0.3%) 20 (0.2%) 29 (0.4%) 2,139 (26.5%) 148 (1.8%) 0.58 (0.79) 2,637 (32.7%) 506 (6.3%) ** (0.0%) 0.33 (0.72) 5,390 (66.8%) 3,504 (43.4%) 8,058 (99.9%) 827 (10.3%) 3.97 (1.85) 0 (0.0%) 1,414 (17.5%) | 775 (9.6%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 390 (4.8%) 1,430 (17.7%) 4,569 (56.7%) 34 (0.4%) 28 (0.3%) 2,148 (26.6%) 162 (2.0%) 0.58 (0.83) 2,717 (33.7%) 511 (6.3%) 0 (0.0%) 0.31 (0.68) 5,362 (66.5%) 3,546 (44.0%) 8,057 (99.9%) 807 (10.0%) 4.17 (1.82) 0 (0.0%) | 319 (5.6%) 0 (0.0%) 0 (0.0%) 10 (0.0%) 4 VALUE! 707 (4.4%) 2527 (15.9%) 2,823 (49.7%) 117 (0.7%) 4 VALUE! 4 VALUE! 3877 (24.4%) 251 (1.6%) 0.48 (0.76) 4398 (27.7%) 767 (4.8%) 4 VALUE! 0.37 (0.89) 10145 (63.8%) 7995 (50.3%) 15487 (97.4%) 1278 (8.0%) 3.43 (1.76) #VALUE! | 326 (5.7%) 0 (0.0%) 0 (0.0%) 61 (0.4%) 691 (4.3%) 5932 (14.7%) 2.803 (49.4%) 124 (0.8%) #WALUEI #WALUEI \$861 (24.3%) 262 (1.6%) 0.49 (0.84) 4477 (28.1%) 799 (5.0%) 0 (0.0%) 0.33 (0.76) 10024 (63.1%) 8034 (50.6%) 15496 (97.5%) 1262 (7.9%) 3.60 (1.73) #WALUEI | 0.00 #DIV/01 #DIV/01 #VALUE! 0.00 0.03 0.01 -0.01 #VALUE! #VALUE! 0.00 0.00 -0.01 -0.01 -0.01 -0.01 -0.01 0.00 0.00 |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Lower/unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin, n (%) Aspirin, n (%) Aspirin/dipyridamole; n (%) Other antiblatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) Vitamin K therapy; n (%) Number of INR (prothrombin) tests orderedmean (sd) Treating prescriber - Cheri; n (%) Treating prescriber - Cher; n (%) Treating prescriber - Other; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHA2DS2 VASC score, 180 days, Vmean (sd) Use of Prasugrel; n (%) Use of Loop Diuretics+other diuretics+other hyperten: Commercial vs Medicare Advantage- Business Type Code-CC | 639 (29.7%) 181 (8.4%) 0 (0.0%) 0 (0.0%) 15 (0.7%) 113 (5.2%) 353 (16.4%) 1,052 (48.9%) 15 (0.7%) ** (0.1%) ** (0.1%) ** (0.2%) 484 (22.5%) 32 (1.5%) 0,47 (0.72) 528 (24.5%) 75 (3.5%) 0 (0.0%) 0.48 (1.24) 1,407 (65.4%) 1,960 (91.0%) 2,143 (99.5%) 170 (7.9%) 3.05 (1.73) ** (0.1%) | 621 (28.8%) 166 (7.7%) 0 (0.05%) 0 (0.05%) 13 (0.65%) 130 (4.65%) 337 (15.7%) 1,088 (50.5%) 13 (0.65%) 14 (0.15%) 15 (0.25%) 480 (22.3%) 29 (1.3%) 0.50 (1.17) 528 (24.5%) 89 (4.15%) 0 (0.0%) 0.37 (0.92) 1,372 (63.7%) 1,960 (91.0%) 2,145 (99.6%) 164 (7.6%) 3.21 (1.73) ** (0.1%) | 0.02 #DIV/0! #DIV/0! #DIV/0! 0.01 0.03 0.02 #DIV/0! 0.01 0.00 0.00 0.02 -0.03 0.00 -0.03 #DIV/0! 0.10 0.04 0.04 0.00 -0.01 0.01 0.01 -0.01 -0.01 | 1,051 (18.5%) 319 (5.6%) 0 (0.0%) 50 (0.9%) 201 (3.5%) 593 (10.4%) 2,823 (49.7%) 74 (1.3%) ** (0.1%) 1,254 (22.1%) 71 (1.3%) 0.35 (0.72) 1,233 (21.7%) 186 (3.3%) 0 (0.0%) 0.39 (0.95) 3,348 (59.0%) 2,531 (44.6%) 5,286 (93.1%) 281 (5.0%) 2.80 (1.64) ** (0.1%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 48 (0.8%) 201 (3.5%) 555 (10.0%) 2,803 (49.4%) 77 (1.4%) ** (0.1%) 1,233 (21.7%) 71 (1.3%) 0.35 (0.70) 1,226 (21.6%) 199 (3.5%) 0 (0.0%) 0.33 (0.81) 3,290 (58.0%) 2,528 (44.5%) 5,294 (93.3%) 291 (5.1%) 2.93 (1.60) ** (0.1%) | #DIV/O! #DIV/O! #DIV/O! #DIV/O! #DIV/O! 0.01 0.00 0.01 #DIV/O! 0.00 0.00 0.00 0.00 0.00 0.00 0.00 0. | 810 (10.0%) 0 (0.0%) 0 (0.0%) 10 (0.0%) 393 (4.9%) 1,581 (19.5%) 4,541 (56.3%) 28 (0.3%) 20 (0.2%) 29 (0.4%) 2,139 (26.5%) 148 (1.8%) 0.58 (0.79) 2,637 (32.7%) 506 (6.3%) ** (0.0%) 0.33 (0.72) 5,390 (66.8%) 3,504 (43.4%) 8,058 (99.9%) 827 (10.3%) 3.97 (1.85) 0 (0.0%) | 775 (9.6%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 390 (4.8%) 1,430 (17.7%) 4,569 (56.7%) 34 (0.4%) 28 (0.3%) 2,148 (26.6%) 162 (2.0%) 0.58 (0.83) 2,717 (33.7%) 511 (6.3%) 0 (0.0%) 0.31 (0.68) 5,362 (66.5%) 3,546 (44.0%) 8,057 (99.9%) 807 (10.0%) | 319 (5.6%) 0 (0.0%) 0 (0.0%) 0 (0.0%) #VALUE! 707 (4.4%) 2,527 (15.9%) 2,823 (49.7%) 117 (0.7%) #VALUE! #VALUE! #VALUE! 3877 (24.4%) 251 (1.6%) 0.48 (0.76) 4398 (27.7%) 767 (4.8%) #VALUE! 0.37 (0.89) 10145 (63.8%) 7995 (50.3%) 15487 (97.4%) 15487 (97.4%) 15488 (97.4%) 3.43 (1.76) #VALUE! 2213 (13.9%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 61 (0.4%) 691 (4.3%) 2332 (14.7%) 2,803 (49.4%) 124 (0.8%) #VALUEI #VALUEI #VALUEI #VALUEI #VALUEI #VALUEI #0.4 (1.6%) 0.49 (0.84) 4471 (28.1%) 799 (5.0%) 0 (0.0%) 0.33 (0.76) 10024 (63.1%) 8034 (50.6%) 15496 (97.5%) 1262 (7.9%) 3.60 (1.73) #VALUEI | 0.00 #DIV/01 #DIV/01 #VALUEI 0.00 0.03 0.01 -0.01 #VALUEI #VALUEI 0.00 0.00 -0.01 -0.01 #VALUEI 0.00 0.01 -0.01 -0.01 #VALUEI 0.00 0.00 0.01 -0.01 -0.01 -0.01 -0.01 -0.01 -0.01 -0.01 |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Lower/unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleed; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) Por inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) Vitamin K therapy; n (%) Vitamin K therapy; n (%) Number of lipid rests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Cardiologist; n (%) Treating prescriber - Cardiologist; n (%) Treating prescriber - Cher; n (%) Alpha blockers; n (%) CHAZDSZ VASc score, 180 days, Vmean (sd) Use of Prasugrel; n (%) Use of Loop Diuretics+other diuretics+other hyperten: Commercial; n (%) | 639 (29.7%) 181 (8.4%) 0 (0.0%) 0 (0.0%) 15 (0.7%) 113 (5.2%) 353 (16.4%) 1,052 (48.9%) 15 (0.7%) ** (0.1%) ** (0.2%) 32 (1.5%) 0.47 (0.72) 528 (24.5%) 75 (3.5%) 0 (0.0%) 0.48 (1.24) 1,407 (65.4%) 1,960 (91.0%) 2,143 (99.5%) 170 (7.9%) 3.05 (1.73) ** (0.1%) | 621 (28.8%) 166 (7.7%) 0 (0.0%) 0 (0.0%) 13 (0.6%) 130 (6.6%) 100 (4.6%) 337 (15.7%) 1,088 (50.5%) 13 (0.6%) ** (0.1%) ** (0.2%) 29 (1.3%) 0.50 (1.17) 528 (24.5%) 89 (4.1%) 0 (0.0%) 0.37 (0.92) 1,372 (63.7%) 1,960 (91.0%) 2,145 (99.6%) 164 (7.6%) 3.21 (1.73) ** (0.1%) 289 (13.4%) 878 (40.8%) | 0.02 #DIV/0! #DIV/0! #DIV/0! 0.01 0.03 0.02 #DIV/0! 0.01 0.00 0.00 0.00 0.02 -0.03 #DIV/0! 0.10 0.04 0.00 0.00 -0.01 0.01 0.01 | 1,051 (18.5%) 319 (5.6%) 0 (0.0%) 50 (0.9%) 50 (0.9%) 501 (3.5%) 593 (10.4%) 2,823 (49.7%) 74 (1.3%) ** (0.1%) 1,254 (22.1%) 71 (1.3%) 0.35 (0.72) 1,233 (21.7%) 186 (3.3%) 0 (0.0%) 0.39 (0.95) 3,348 (59.0%) 2,531 (44.6%) 5,286 (93.1%) 281 (5.0%) 2.80 (1.64) ** (0.1%) 517 (9.1%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 48 (0.8%) 201 (3.5%) 555 (10.0%) 2,803 (49.4%) 77 (1.4%) ** (0.1%) 1,233 (21.7%) 71 (1.3%) 0.35 (0.70) 1,226 (21.6%) 199 (3.5%) 0 (0.0%) 0,33 (0.81) 3,290 (58.0%) 2,528 (44.5%) 5,294 (93.3%) 291 (5.1%) 2.93 (1.60) ** (0.1%) | #DIV/O! #DIV/O! #DIV/O! #DIV/O! #DIV/O! 0.01 0.00 0.01 #DIV/O! 0.00 0.00 0.00 0.00 0.00 0.00 0.00 0. | 810 (10.0%) 0 (0.0%) 0 (0.0%) ** (0.0%) 393 (4.9%) 1,581 (19.6%) 4,541 (56.3%) 28 (0.3%) 20 (0.2%) 29 (0.4%) 2,139 (26.5%) 148 (1.8%) 0.58 (0.79) 2,637 (32.7%) 506 (6.3%) ** (0.0%) 0.33 (0.72) 5,390 (66.8%) 3,504 (43.4%) 8,058 (99.9%) 827 (10.3%) 3.97 (1.85) 0 (0.0%) 1,414 (17.5%) | 775 (9.6%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 390 (4.8%) 1,430 (17.7%) 4,569 (56.7%) 34 (0.4%) 28 (0.3%) 2,148 (26.6%) 162 (2.0%) 0.58 (0.83) 2,717 (33.7%) 511 (6.3%) 0 (0.0%) 0.31 (0.68) 5,362 (66.5%) 3,546 (44.0%) 8,057 (99.9%) 807 (10.0%) 4.17 (1.82) 0 (0.0%) | 319 (5.6%) 0 (0.0%) 0 (0.0%) 10 (0.0%) 10 (0.0%) #VALUE! 707 (4.4%) 2527 (15.9%) 2,823 (49.7%) 117 (0.7%) #VALUE! 3877 (24.4%) 251 (1.6%) 0.48 (0.76) 4398 (27.7%) 767 (4.5%) #VALUE! 0.37 (0.89) 10145 (63.6%) 7995 (50.3%) 15487 (97.4%) 1278 (8.0%) 3.43 (1.76) #VALUE! 2213 (13.9%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 61 (0.4%) 691 (4.3%) 2332 (14.7%) 2,803 (49.4%) 124 (0.8%) #WALUE! #WALUE! #WALUE! 3661 (24.3%) 262 (1.6%) 0.49 (0.84) 4471 (28.1%) 799 (5.0%) 0 (0.0%) 0.33 (0.76) 10024 (63.1%) 8034 (50.6%) 15496 (97.5%) 1262 (7.9%) 3.60 (1.73) #WALUE! 2288 (14.4%) | 0.00 #DIV/01 #DIV/01 #VALUEI 0.00 0.03 0.01 -0.01 #VALUEI #VALUEI #VALUEI 0.00 0.00 -0.01 |
| Peptic Ulcer Disease; n (%) Major Surgery; n (%) Upper Gi bleed; n (%) Lower/unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Antibiotics; n (%) Aspirin, n (%) Aspirin, of (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) Vitamin K therapy; n (%) Number of INR (prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Other; n (%) Irreating prescriber - Other; n (%) Alpha blockers; n (%) CHA2DS2 VASC score, 180 days, Vmean (sd) Use of Prasugrel; n (%) Use of Loop Diuretics+other diuretics+other hyperten: Commercial vs Medicare Advantage- Business Type Code- CC | 639 (29.7%) 181 (8.4%) 0 (0.0%) 0 (0.0%) 15 (0.7%) 113 (5.2%) 353 (16.4%) 1,052 (48.9%) 15 (0.7%) ** (0.1%) ** (0.1%) ** (0.2%) 484 (22.5%) 32 (1.5%) 0,47 (0.72) 528 (24.5%) 75 (3.5%) 0 (0.0%) 0.48 (1.24) 1,407 (65.4%) 1,960 (91.0%) 2,143 (99.5%) 170 (7.9%) 3.05 (1.73) ** (0.1%) | 621 (28.8%) 166 (7.7%) 0 (0.05%) 0 (0.05%) 13 (0.65%) 130 (4.65%) 337 (15.7%) 1,088 (50.5%) 13 (0.65%) 14 (0.15%) 15 (0.25%) 480 (22.3%) 29 (1.3%) 0.50 (1.17) 528 (24.5%) 89 (4.15%) 0 (0.0%) 0.37 (0.92) 1,372 (63.7%) 1,960 (91.0%) 2,145 (99.6%) 164 (7.6%) 3.21 (1.73) ** (0.1%) | 0.02 #DIV/0! #DIV/0! #DIV/0! 0.01 0.03 0.02 #DIV/0! 0.01 0.00 0.00 0.02 -0.03 0.00 -0.03 #DIV/0! 0.10 0.04 0.04 0.00 -0.01 0.01 0.01 -0.01 -0.01 | 1,051 (18.5%) 319 (5.6%) 0 (0.0%) 50 (0.9%) 201 (3.5%) 593 (10.4%) 2,823 (49.7%) 74 (1.3%) ** (0.1%) 1,254 (22.1%) 71 (1.3%) 0.35 (0.72) 1,233 (21.7%) 186 (3.3%) 0 (0.0%) 0.39 (0.95) 3,348 (59.0%) 2,531 (44.6%) 5,286 (93.1%) 281 (5.0%) 2.80 (1.64) ** (0.1%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 48 (0.8%) 201 (3.5%) 555 (10.0%) 2,803 (49.4%) 77 (1.4%) ** (0.1%) 1,233 (21.7%) 71 (1.3%) 0.35 (0.70) 1,226 (21.6%) 199 (3.5%) 0 (0.0%) 0.33 (0.81) 3,290 (58.0%) 2,528 (44.5%) 5,294 (93.3%) 291 (5.1%) 2.93 (1.60) ** (0.1%) | #DIV/O! #DIV/O! #DIV/O! #DIV/O! #DIV/O! 0.01 0.00 0.01 #DIV/O! 0.00 0.00 0.00 0.00 0.00 0.00 0.00 0. | 810 (10.0%) 0 (0.0%) 0 (0.0%) ** (0.0%) 393 (4.9%) 1,581 (19.6%) 4,541 (56.3%) 28 (0.3%) 20 (0.2%) 29 (0.4%) 2,139 (26.5%) 148 (1.8%) 0.58 (0.79) 2,637 (32.7%) 506 (6.3%) ** (0.0%) 0.33 (0.72) 5,390 (66.8%) 3,504 (43.4%) 8,058 (99.9%) 827 (10.3%) 3.97 (1.85) 0 (0.0%) 1,414 (17.5%) | 775 (9.6%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 390 (4.8%) 1,430 (17.7%) 4,569 (56.7%) 34 (0.4%) 28 (0.3%) 2,148 (26.6%) 162 (2.0%) 0.58 (0.83) 2,717 (33.7%) 511 (6.3%) 0 (0.0%) 0.31 (0.68) 5,362 (66.5%) 3,546 (44.0%) 8,057 (99.9%) 807 (10.0%) 4.17 (1.82) 0 (0.0%) | 319 (5.6%) 0 (0.0%) 0 (0.0%) 0 (0.0%) #VALUE! 707 (4.4%) 2,527 (15.9%) 2,823 (49.7%) 117 (0.7%) #VALUE! #VALUE! #VALUE! 3877 (24.4%) 251 (1.6%) 0.48 (0.76) 4398 (27.7%) 767 (4.8%) #VALUE! 0.37 (0.89) 10145 (63.8%) 7995 (50.3%) 15487 (97.4%) 15487 (97.4%) 15488 (97.4%) 3.43 (1.76) #VALUE! 2213 (13.9%) | 326 (5.7%) 0 (0.0%) 0 (0.0%) 61 (0.4%) 691 (4.3%) 2332 (14.7%) 2,803 (49.4%) 124 (0.8%) #VALUEI #VALUEI #VALUEI #VALUEI #VALUEI #VALUEI #0.4 (1.6%) 0.49 (0.84) 4471 (28.1%) 799 (5.0%) 0 (0.0%) 0.33 (0.76) 10024 (63.1%) 8034 (50.6%) 15496 (97.5%) 1262 (7.9%) 3.60 (1.73) #VALUEI | 0.00 #DIV/01 #DIV/01 #VALUEI 0.00 0.03 0.01 -0.01 #VALUEI #VALUEI 0.00 0.00 -0.01 -0.01 #VALUEI 0.00 0.01 -0.01 -0.01 #VALUEI 0.00 0.00 0.01 -0.01 -0.01 -0.01 -0.01 -0.01 -0.01 -0.01 |

| Commercial vs Medicare Advantage- Business Type Code | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| COM = COMMERCIAL; n (%) | 950 (44.1%) | 878 (40.8%) | 0.07 | - | - | #VALUE! | - | - | 950 (44.1%) | 878 (40.8%) | 0.07 |
| MCR = MEDICARE; n (%) | 1,203 (55.9%) | 1,275 (59.2%) | -0.07 | - | - | #VALUE! | - | - | 1,203 (55.9%) | 1,275 (59.2%) | -0.07 |
| MCD = MEDICAID; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | - | - | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| NONE = NO BUSINESS LINE CODE (added in 2015); n ( | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | - | - | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| UNK = UNKNOWN (added in 2015); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | - | - | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Commercial vs Medicare Advantage- Data Type | - | - | | 0 | 0 | | - | - | | | |
| 1 - Fee For Service; n (%) | - | - | | 3,978 (70.1%) | 3,898 (68.7%) | | - | - | 3,978 (70.1%) | 3,898 (68.7%) | 0.00 |
| 2 - Encounter; n (%) | - | - | | 493 (8.7%) | 496 (8.7%) | | - | - | 493 (8.7%) | 496 (8.7%) | 0.00 |
| 3 - Medicare; n (%) | - | - | | 1,080 (19.0%) | 1,153 (20.3%) | | - | - | 1,080 (19.0%) | 1,153 (20.3%) | 0.00 |
| 4 - Medicare Encounter; n (%) | - | - | | 124 (2.2%) | 128 (2.3%) | | - | - | 124 (2.2%) | 128 (2.3%) | 0.00 |
| Metropolitan Statistical Area - Urban (any MSA) vs Rural (non-MSA) | | | | | | | | | 0 | 0.00 | |
| Urban; n (%) | - | - | | 4,248 (74.9%) | 4,262 (75.1%) | | - | - | 4,248 (74.9%) | 4,262 (75.1%) | |
| Rural; n (%) | - | - | | 226 (4.0%) | 198 (3.5%) | | - | - | 226 (4.0%) | 198 (3.5%) | |
| Unknown/Missing; n (%) | - | - | | 1,201 (21.2%) | 1,215 (21.4%) | | - | - | 1,201 (21.2%) | 1,215 (21.4%) | |